# **Protocol Amendment 4**

**Study ID: 207636** 

A prospective epidemiological study of women between 24-27 weeks of pregnancy to describe pregnancy outcomes and events of interest in the mother and neonate, as well as determine incidence in infants of RSV LRTI and RSV hospitalization

**Date of Document:** 29-May-2020

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final



Study Protocol Sponsor:

GlaxoSmithKline Biologicals SA

Rue de l'institut 89, 1330 Rixensart, Belgium

eTrack study number and Abbreviated Title 207636 (EPI-RSV-008 BOD)

**Date of protocol** Final Version 1: 11 July 2017

**Date of Amendment** Amendment 1 Final: 12 February 2018

Amendment 2 Final: 03 July 2018
Amendment 3 Final: 18 February 2019

Amendment 4 Final: 29 May 2020

**Title** A prospective epidemiological study of pregnancy

outcomes and of events of interest in pregnant women,

neonates and infants (PEPNI)

**Detailed Title** A prospective epidemiological study of women

between 24-27 weeks of pregnancy to describe pregnancy outcomes and events of interest in the mother and neonate, as well as determine incidence in

infants of RSV LRTI and RSV hospitalization.

Coordinating author

PPD

**Contributing authors** 

- PPD , Clinical & Epidemiological Project Lead
- PPD , Lead Epidemiologist
- PPD , Expert Biostatistician, PPD PPD Lead *Biostatistician*
- PPD , PPD , Study Delivery Leads
- PPD , Clinical Read-Out Team Leader
- PPD , Clinical Laboratory Sciences Study Manager, Business & Decision Life Sciences Contractor for GSK Biologicals
- PPD , Safety Physician
- PPD , Oversight Data Manager

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### eTrack study number and Abbreviated Title

207636 (EPI-RSV-008 BOD)

#### **Detailed Title**

A prospective epidemiological study of women between 24-27 weeks of pregnancy to describe pregnancy outcomes and events of interest in the mother and neonate, as well as determine incidence in infants of RSV LRTI and RSV hospitalization.

Authors who contributed to previous versions of the protocol:

- PPD Clinical & Epidemiological Project Leads
- PPD Epidemiologists ,
- PPD , PPD , Study Delivery Leads
- PPD , Clinical Research and Development Lead
- PPD , Clinical Research and Development Lead
- PPD , Lead Epi Statistician
- PPD , Study statistician
- PPD (Aixial for GSK Biologicals), Clinical Trial Supply manager
- PPD , Clinical Trial Supply manager
- PPD , Safety Physician
- PPD , Clinical Read-Out Team Leader
- PPD (Business & Decision Life Sciences for GSK Biologicals), Clinical Laboratory Sciences Study Manager
- PPD , Safety Physician
- PPD , Oversight Data Manager
- PPD , Study Data Manager (Tata Consultancy Services for GSK Biologicals)
- PPD , Regulatory Affairs Representative

GSK Biologicals' Protocol DS v15.0

©2017-2020 GSK group of companies or its licensor.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# **Protocol Amendment 4 Sponsor Signatory Approval**

| eTrack study number and<br>Abbreviated Title | 207636 (EPI-RSV-008 BOD) |
|---|---|
| Date of Amendment | Amendment 4 Final: 29 May 2020 |
| Detailed Title | A prospective epidemiological study of women between 24-27 weeks of pregnancy to describe pregnancy outcomes and events of interest in the mother and neonate, as well as determine incidence in infants of RSV LRTI and RSV hospitalization. |
| Sponsor signatory | Ouzama Henry, Clinical & Epidemiological Project<br>Lead |
| Signature | |
| Date | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

### **Protocol Amendment 4 Rationale**

**Amendment number:** Amendment 4

# Rationale/background for changes:

This amendment outlines measures that may be applicable during special circumstances (e.g., COVID-19 pandemic). The primary purpose of the amendment is to protect the subject's welfare, and as far as possible ensure the potential benefit to the subject and promote data integrity. Several additional modifications and clarifications have also been made.

Changes are outlined below.

#### • Globally:

- Intervals between study visits/contacts/observations: the window for the first infant subject visit has been extended from 0-10 to 0-21 days to provide site personnel with additional time to obtain and document post-delivery/birth informed consent (where this is required).
- References to Gestational Age Range at maternal Visits 2, 3 and 4 have been removed as their inclusion was only intended as a guide and was not intended to further restrict allowed intervals between study visits.
- Synopsis, Section 3.3, Tertiary Objectives, and Section 11.1.3, Tertiary Endpoints, have been updated to indicate that the incidence of LRTIs/ Severe LRTIs (using alternative case definitions) will also be evaluated.
- Synopsis and Section 11.1.3, Tertiary Endpoints, has been updated to clarify that
  further exploratory characterization of immune responses to RSV and/or other
  respiratory tract infections or infections of relevance to pregnant women and their
  newborns (based on maternal serum and cord blood) includes, for example, levels
  of RSV-B neutralizing antibodies.
- The List of Abbreviations has been updated to include a reference to COVID-19.
- Section 2.3, Overall Benefit: Risk Conclusion has been updated.
- Section 4, Figure 1: A note has been added to indicate that COVID-19 cases identified within the surveillance framework of the study will be captured to the eCRF.
- Section 5.4, Table 4, Alternative LRTI/Severe LRTI Case Definitions, has been added. All subsequent Table numbers therefore increase by one.
- Section 8.2.1, Study procedures during special circumstances, has been added.
- Section 8.3, Table 5 and Table 6, List of study procedures for maternal subjects, and List of study procedures for neonates/infants, have been clarified to indicate that COVID-19 cases are considered clinically significant events and will be recorded as such in the eCRF.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- Sections 8.5.8, 8.6.2, 8.6.7 have been modified to reference the collection of COVID-19 case information.
- Section 8.6.5.2 has been modified to clarify that RTI surveillance in infants cannot begin before additional consent for the infant's participation (where required) has been supplied.
- Section 8.7, Reporting COVID-19 cases, has been added.
- Section 11.3 has been modified to introduce definitions for the Enrolled set, and to clarify definitions for the Exposed, and Per Protocol sets for analysis.
- Section 11.6, 11.7, and 11.8 have been modified for consistency with the changes in Section 11.3.
- Section 11.11.1, Statistical considerations for interim analysis, has been modified to indicate that an interim analysis for RSV LRTIs may be performed if deemed necessary.
- Section 14 has been updated to include a reference to the WHO Guidance for surveillance of COVID-19.
- Additional editorial clarifications have been made and typographic errors have been corrected.
- A detailed summary of changes (including deletions) appears in APPENDIX E.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# **Protocol Amendment 4 Investigator Agreement**

### I agree:

- To conduct the study in compliance with this protocol, any mutually agreed future protocol amendments or protocol administrative changes, with the terms of the study agreement and with any other study conduct procedures and/or study conduct documents provided by GlaxoSmithKline (GSK) Biologicals.
- To assume responsibility for the proper conduct of the study at this site.
- That I am aware of, and will comply with, 'Good Clinical Practice' (GCP) and all applicable regulatory requirements.
- To ensure that all persons assisting me with the study are adequately informed about study-related duties and functions as described in the protocol.
- To acquire the reference ranges for laboratory tests performed locally and, if required by local regulations, obtain the laboratory's current certification or Quality Assurance procedure manual.
- To ensure that no samples (including serum samples) are retained onsite or elsewhere without the approval of GSK Biologicals and the express written informed consent of the subject and/or the subject's legally acceptable representative.
- To perform no other biological assays on the samples except those described in the protocol or its amendment(s).
- To co-operate with a representative of GSK Biologicals in the monitoring process of the study and in resolution of queries about the data.
- That I have been informed that certain regulatory authorities require the sponsor to obtain and supply, as necessary, details about the investigator's ownership interest in the sponsor, and more generally about his/her financial ties with the sponsor. GSK Biologicals will use and disclose the information solely for the purpose of complying with regulatory requirements.

# Hence I:

- Agree to supply GSK Biologicals with any necessary information regarding ownership interest and financial ties (including those of my spouse and dependent children).
- Agree to promptly update this information if any relevant changes occur during the course of the study and for one year following completion of the study.
- Agree that GSK Biologicals may disclose any information it has about such ownership interests and financial ties to regulatory authorities.
- Agree to provide GSK Biologicals with an updated Curriculum Vitae and other documents required by regulatory agencies for this study.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| | Frotocol Amendment 4 mila |
|---|---|
| eTrack study number and<br>Abbreviated Title | 207636 (EPI-RSV-008 BOD) |
| <b>Date of Amendment</b> | Amendment 4 Final: 29 May 2020 |
| Detailed Title | A prospective epidemiological study of women<br>between 24-27 weeks of pregnancy to describe<br>pregnancy outcomes and events of interest in the<br>mother and neonate, as well as determine incidence<br>in infants of RSV LRTI and RSV hospitalization. |
| Investigator name | |
| Signature | |
| _ | |
| Date | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# **Sponsor Information**

# 1. Sponsor

# **GlaxoSmithKline Biologicals**

Rue de l'institut 89,1330 Rixensart, Belgium

# 2. Sponsor Medical Expert for the Study

Refer to the local study contact information document.

# 3. Sponsor Study Monitor

Refer to the local study contact information document.

# 4. Study Contact for Reporting of a Serious Adverse Event (SAE)

GSK Biologicals Central Back-up Study Contact for Reporting SAEs: refer to protocol Section 9.4.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### SYNOPSIS

**Detailed Title** A prospective epidemiological study of women between 24-27 weeks of pregnancy to describe pregnancy outcomes and events of interest in the mother and neonate, as well as determine incidence in infants of RSV LRTI and RSV hospitalization.

# **Objectives** (Amended 29-MAY-2020)

### **Primary**

In healthy pregnant women with uncomplicated pregnancies:

- To determine the frequencies of pregnancy outcomes.
- To determine the frequencies of pregnancy related events of interest from enrollment (Visit 1) through 42 days after delivery (Visit 6).

(Although pregnancy related events of interest occur within the first 42 days after delivery they may only be detected later, and are to be reported throughout the study.)

In all neonates live-born to women enrolled in the study:

To determine the frequencies of neonatal events of interest.

Neonatal events of interest occur within the first 28 days after birth but may only be detected later, and are to be reported throughout the study.

# **Secondary**

In healthy pregnant women with uncomplicated pregnancies

- To determine frequencies of pregnancy related events of interest according to GAIA levels of diagnostic certainty (where these are specified) from enrollment (Visit 1) through 42 days after delivery (Visit 6). (Although pregnancy related events of interest occur within the first 42 days after delivery they may only be detected later, and are to be reported throughout the study.)
- To describe the distribution of RSV-A antibody titers in maternal blood at delivery.

In all neonates live-born to women enrolled in the study:

- To determine frequencies of neonatal events of interest according to GAIA levels of diagnostic certainty (where these are specified). Neonatal events of interest occur within the first 28 days after birth (but may only be detected later and are to be reported throughout the study).
- To describe the distribution of RSV-A antibody titers in cord blood at delivery.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

In all neonates/infants live-born to women enrolled in the study, from birth through 1 year of age:

- To determine the incidence of all, of severe, and of very severe RSV-lower respiratory tract illnesses (LRTIs).
- To determine the incidence of RSV hospitalization.

#### **Tertiary**

- To describe co-infections of RSV-LRTI with other respiratory viruses in infants.
- To estimate the association of RSV-LRTI in neonates/infants and the level of RSV neutralizing antibodies in cord blood.
- To determine the incidence of LRTIs/Severe LRTIs (using alternative case definitions)
- To determine risk factors for pregnancy-related and neonatal events of interest
- If deemed necessary, to further characterize the immune responses to RSV and other infections in maternal subjects and infants (based on maternal serum and cord blood).

Rationale for the study and study design Maternal immunization aims to prevent diseases in neonates and infants via transplacental antibody transfer from the mother to the fetus following vaccination of the pregnant woman. Several marketed vaccines are already recommended for and routinely administered to pregnant women, including influenza, tetanus, and Tdap vaccines (CDC 2013a, CDC 2013b). There are also a number of maternal vaccines in development that aim to protect neonates and infants from pathogens in addition to respiratory syncytial virus (RSV). GlaxoSmithKline (GSK) is developing an investigational vaccine for use in pregnant women against RSV disease. Of note this vaccine is developed solely for immunization in pregnancy.

Maternal immunization is implemented worldwide and has the potential to make a major contribution to reducing RSV lower respiratory tract illnesses (LRTI) and the burden of other diseases in infants globally. Therefore, it is imperative that clinical trials are conducted across different countries in different settings. GSK is proactively addressing potential challenges of conducting clinical trials in pregnant women in low- and middle income countries (LMIC).

Before conducting clinical trials it is important to understand the frequency of pregnancy outcomes and the maternal and neonatal events of interest (i.e. clinically significant events that may be considered adverse events if they occur after vaccination) in each setting where clinical trials may be conducted for better interpretation of safety data. Also, to ensure safety of the participating women, and to characterize the safety profile of the product, adverse events (AEs)

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

in pregnancy should be appropriately detected and managed. This study addresses gaps in understanding of anticipated rates of pregnancy outcomes as well as events of interest in pregnant women and neonates. Furthermore, this study will be conducted at potential sites for future maternal immunization trials and will help assure the capacity of sites to detect and manage clinically significant events of interest in pregnant women and their neonates.

Secondarily, the study will establish surveillance mechanisms for RSV associated illnesses in the neonate/infant (through the first 12 months of life. Whilst there is good documentation of the global burden of RSV disease, incidence of RSV-LRTI according to the World Health Organization (WHO) 2015 case definitions [Modjarrad, 2016] is limited in the literature, particularly in many LMIC settings. Hence, this study will also estimate the incidence of infant RSV-LRTI using WHO case definitions across geographically distinct locations to support incidence rate assumptions for planning of future efficacy trials.

To achieve these goals, GSK will be guided by the WHO recommendations on antenatal care for a positive pregnancy experience [WHO, 2016] and the Global Alignment of Immunization Safety Assessment in pregnancy (GAIA) case definitions [Bonhoeffer, 2016; Bauwens, 2016; Kochhar, 2017]. Standardization of surveillance methodology and case definitions (applicable to maternal immunization AEs) may support comparison of data across different countries [Jones, 2016].

This multi-country study will enroll pregnant women  $\geq 24^{0/7}$  weeks and  $\leq 27^{6/7}$  weeks gestational age (GA). Study procedures in this protocol are defined to ensure that maternal and neonatal events of interest are captured. They are not intended to replace procedures performed by local healthcare providers as part of standard care. Prenatal screening and care will be provided by local healthcare providers (in accordance with local standards).

#### Study design

- Type of design: Prospective, epidemiological, interventional (without administration of medicinal products as described in a research protocol), multi-country, cohort study.
- Study population: The study will be conducted in multiple countries, in pregnant women and their infants.
- Type of study: self-contained.
- Data collection: Electronic Case Report Form (eCRF).

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### Synopsis Table 1 Sampling schedule for maternal subjects

| | | | | | Visit | |
|---|---|---|---|---|---|---|
| Sample | Parameter(s) evaluated | 1 | 2 | 3 | 4 | Delivery |
| Maternal<br>Blood | Hematology/<br>biochemistry <sup>1, 4</sup> | Х | | <b>X</b> <sup>3</sup> | | |
| | Antibody titer (RSV-A) | | | | | ≤ 72 hours after<br>delivery⁵ |
| Cord Blood | Antibody titer (RSV-A) | | | | | Х |
| Urine | Protein, glucose, RBC, WBC <sup>2, 4</sup> | Х | Х | Х | Х | |

<sup>&</sup>lt;sup>1</sup> To be performed preferentially by local healthcare providers, as per local practice. To be performed by the investigator/study staff ONLY if not done by the local healthcare provider within 2 weeks before the study visit.

# Sampling schedule for neonates/infants

Surveillance for RSV LRTI will be conducted in infants through the 12 month study period. During this 1-year post-birth surveillance period, for each RTI with suspicion of difficulty in breathing, or wheezing, or with parental concern, a nasal swab will be collected at a visit to assess potential RSV associated RTIs/LRTIs

# Primary Completion Date (PCD)

42 days post-delivery/birth (i.e. Visit 6 for the mother and Visit 2-NB for the infant) or last visit of Epoch 2.

# End of Study (EoS)

Last testing results released of samples collected up to Visit 4-NB (assays related to primary and secondary endpoints)

# **Duration of the study**

Approximately 4.5 to 6 months for participating pregnant women; approximately 1 year for participating infants.

- Epoch 001: Screening
- Epoch 002: Primary starting at Visit 1 and ending 42 days post-delivery/birth (Visit 6 for the mothers and Visit 2-NB for the infants).\*
- Epoch 003: Follow-up of infants starting 43 days post-delivery/birth and ending at Visit 4-NB (1 year post-birth).

#### Synopsis Table 2 Study groups and epochs foreseen in the study

| Study Groups | Number of | Age (Min/Max) | Epochs | | |
|---|---|---|---|---|---|
| | subjects enrolled | | Epoch 001 | Epoch 002 | Epoch 003 |
| Maternal subjects | Up to ~ 2300 | 18 years - 45 | Х | Х | |
| | | years | | | |
| Infants | Up to ~ 2300 | NA | | Х | Х |

Approximately 200 to 300 subjects per country. To achieve the enrollment targets noted above, the number of pregnant women SCREENED in each country may exceed the country-specific enrollment target.

<sup>&</sup>lt;sup>2</sup>The investigator/site staff will perform a urine dipstick test using supplies provided by GSK.

<sup>&</sup>lt;sup>3</sup> Hemoglobin only

<sup>&</sup>lt;sup>4</sup> If results are abnormal, subjects will be referred per local standard of care.

<sup>&</sup>lt;sup>5</sup> This sample may be collected from start of labor (e.g. when the mother arrives at the hospital to deliver and an intravenous line is inserted) through 72 hours after delivery.

<sup>\*</sup>Any safety and disease surveillance data collected after Visit 2-NB will be collected in Epoch 003.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- Surveillance for pregnancy outcomes and pregnancyrelated events of interest that occur from Visit 1 up to 42 days after delivery (Visit 6).
- Surveillance for neonatal events of interest that occur from birth up to 28 days of age
- Surveillance for RSV LRTI and RSV hospitalization in infants: from birth up to 1 year of age

#### **Number of subjects**

• Approximately 2300 pregnant women. Neonates of enrolled pregnant women who consent to the infant's continued study participation will also be enrolled.

# Endpoints (Amended 29-MAY-2020)

### **Primary**

- Pregnancy outcomes. Of note, fetal death/stillbirth has multiple subcategories. For example, fetal death/stillbirth with no congenital anomalies is an outcome with two subcategories that include: 1) antepartum stillbirth; 2) intrapartum stillbirth. For each outcome, the investigator should select the applicable sub-category.
  - Live birth with no congenital anomalies,
  - Live birth with congenital anomalies,
  - Fetal death/stillbirth (loss at or after 22 weeks of gestation) with no congenital anomalies:
    - Antepartum stillbirth
    - o Intrapartum stillbirth
  - Fetal death/still birth (loss at or after 22 weeks of gestation) with congenital anomalies:
    - o Antepartum stillbirth
    - o Intrapartum stillbirth
  - Elective/therapeutic termination with no congenital anomalies,
  - Elective/therapeutic termination with congenital anomalies.
- Pregnancy related events of interest from Visit 1 through Visit 6. Although pregnancy related events of interest occur within the first 42 days after delivery they may only be detected later, and are to be reported throughout the study. They are listed below. Of note, some events of interest fall under a single category but have multiple subcategories. For example, hypertensive disorders of pregnancy is an event with three subcategories that include: 1) gestational hypertension; 2) pre-eclampsia; and

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- 3) pre-eclampsia with severe features (including eclampsia). For each event, the investigator should identify the event and select the applicable sub-category.
- Maternal death
- Hypertensive disorders of pregnancy:
  - Gestational hypertension,
  - o Pre-eclampsia,
  - Pre-eclampsia with severe features (including eclampsia)
- Antenatal bleeding:
  - Morbidly adherent placenta
  - o Placental abruption
  - Cesarean Scar Pregnancy
  - Uterine rupture
- Postpartum hemorrhage
- Fetal growth restriction
- Dysfunctional labor
  - o first stage of labor
  - second stage of labor
- Gestational diabetes mellitus,
- Non reassuring fetal status
- Pathways to preterm birth:
  - o Premature preterm rupture of membranes,
  - Preterm labor,
  - o Provider-initiated preterm birth.
- Chorioamnionitis
- Oligohydramnios
- Polyhydramnios
- Gestational Liver Disease:
  - o Intrahepatic Cholestasis of Pregnancy (ICP)
  - Acute Fatty Liver of Pregnancy
- Maternal Sepsis
- Any other pregnancy related event considered by the investigator to be of concern (specify)

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- Neonatal events of interest from birth through 28 days of age. Neonatal events of interest occur within the first 28 days after birth, but may only be detected later and are to be reported throughout the study. They include:
  - Small for gestational age,
  - Low birth weight including very low birth weight,
  - Neonatal encephalopathy,
  - Congenital microcephaly,
    - Postnatally diagnosed
    - o Prenatally diagnosed
  - Congenital anomalies,
    - Major external structural defects
    - o Internal structural defects
    - Functional defects
  - Neonatal death,
    - Neonatal death in a preterm live birth (gestational age>=28 to < 37 weeks)</li>
    - Neonatal death in a term live birth
  - Neonatal infections,
    - o Blood stream infections
    - Meningitis
    - Respiratory infection
  - Respiratory distress in the neonate,
  - Preterm birth,
  - Failure to thrive,
  - Large for gestational age,
  - Macrosomia,
  - Any other neonatal event considered by the investigator to be of concern (specify, e.g. neurodevelopment delay)

#### Secondary

 Pregnancy related events of interest from Visit 1 through Visit 6 (as defined in primary endpoints) for each GAIA level of diagnostic certainty (where applicable and feasible)

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

• Neonatal events of interest from birth through 28 days of age (as defined in primary endpoints) for each GAIA level of diagnostic certainty (where applicable and feasible)

Of note, some events of interest fall under a single category but have multiple subcategories. For each event, the investigator should identify the event and select the applicable sub-category and the GAIA level of diagnostic certainty.

- RSV-A neutralizing antibody titers in maternal blood at delivery.
- RSV-A neutralizing antibody titers in cord blood at delivery.
- Episode(s) of RSV-LRTI from birth up to 1 year of age.
- Episode(s) of RSV hospitalization from birth up to 1 year of age.

## **Tertiary**

- Co-infections of RSV-LRTI with other respiratory viruses in infants, confirmed by PCR of nasal swabs in infants from birth up to 1 year of age:
  - Influenza A virus (Flu A)
  - Influenza B virus (Flu B)
  - Human Influenza A virus subtype H1 (Flu A-H1)
  - Human Influenza A virus subtype H3 (Flu A-H3)
  - Human Influenza A virus subtype H1pdm09 (Flu A-H1pdm09)
  - Human adenovirus (AdV)
  - Human metapneumovirus (MPV)
  - Human enterovirus (HEV)
  - Human parainfluenza virus 1 (PIV1)
  - Human parainfluenza virus 2 (PIV2)
  - Human parainfluenza virus 3 (PIV3)
  - Human parainfluenza virus 4 (PIV4)
  - Human bocavirus 1/2/3/4 (HBoV)
  - Human rhinovirus A/B/C (HRV)
  - Human coronavirus 229E (229E)
  - Human coronavirus NL63 (NL63)
  - Human coronavirus OC43 (OC43)
- Episodes of LRTIs/Severe LRTIs up to one year of age using alternative case definitions

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- Potential risk factors for pregnancy related and neonatal events of interest.
- Any further exploratory characterization of immune responses to RSV and/or other respiratory tract infections or infections of relevance to pregnant women and their newborns (based on maternal serum and cord blood). (For example, levels of RSV-B neutralizing antibodies).

References

Bauwens J, Bonhoeffer J, Chen RT, editors. Harmonising Immunisation Safety Assessment in Pregnancy. Vaccine. 2016. 34 (49): 5991 – 6110.

Bonhoeffer J, Kochhar S, Hirschfeld S, et al. Global alignment of immunization safety assessment in pregnancy - The GAIA project. Vaccine. 2016;34(49):5993-5997. doi: 10.1016/j.vaccine.2016.07.006.

Centers for Disease Control and Prevention (CDC). Updated recommendations for use of tetanus toxoid, reduced diphtheria toxoid, and acellular pertussis vaccine (Tdap) in pregnant women. Advisory Committee on Immunization Practices (ACIP) - 2012. MMWR. 2013a; 62 (7):131-135.

Centers for Disease Control and Prevention (CDC). Influenza Vaccination Coerage Among Pregnant Women — United States, 2012–13 Influenza Season. MMWR. \_2013b; 62 (38): 787–792.

Jones CE, Munoz FM, Kochhar S et al. Guidance for the collection of case report form variables to assess safety in clinical trials of vaccines in pregnancy. Vaccine. 2016; 34(49):6007-6014.

Kochhar S, Bauwens J, Bonhoeffer J, editors. Harmonising Immunization Safety Assessment in Pregnancy – Part II. Vaccine. 2017. 35 (48): 6469-6582.

Modjarrad K, Giersing B, Kaslow DC, Smith PG, Moorthy VS; WHO RSV Vaccine Consultation Expert Group. WHO consultation on Respiratory Syncytial Virus Vaccine Development Report from a World Health Organization Meeting held on 23-24 March 2015. Vaccine. 2016;34(2):190-7.

World Health Organization (WHO). WHO recommendations on antenatal care for a positive pregnancy experience. Published in 2016.

http://www.who.int/reproductivehealth/publications/maternal\_perinatal\_health/anc-positive-pregnancy-experience/en. Last accessed on 09 February 2017.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| SP | ONSO | R INFORMATION | 8 |
| SY | NOPS | S | 9 |
| LIS | T OF / | ABBREVIATIONS (AMENDED 29-MAY-2020) | 26 |
| GL | OSSAI | RY OF TERMS | 28 |
| 1. | INITD | ODUCTION | 32 |
| 1. | 1.1. | Background and rationale for the study | |
| | 1.2. | Rationale for the study population | |
| | 1.3. | Rationale for the surveillance of pregnancy related events of interest | |
| | 1.4. | Rationale for the use of Global Alignment of Immunization safety | |
| | 1.4. | Assessment in pregnancy (GAIA) case definitions | 34 |
| | 1.5. | Rationale for the active and passive surveillance for RSV | |
| | 1.0. | associated respiratory tract illnesses (RTI) with suspicion of | |
| | | difficulty in breathing/wheezing or with parental concern in | |
| | | neonates/ infants | 34 |
| 2. | BENE | FIT: RISK ASSESSMENT | 35 |
| | 2.1. | Risk Assessment | |
| | 2.2. | Benefit Assessment | |
| | 2.3. | Overall Benefit:Risk Conclusion (Amended 29-MAY-2020) | |
| 3. | OBJE | CTIVES | 36 |
| | 3.1. | Primary objectives | 36 |
| | 3.2. | Secondary objectives | |
| | 3.3. | Tertiary objectives (Amended 29-MAY2020) | 37 |
| 4. | STU | DY DESIGN OVERVIEW (AMENDED 29-MAY-2020) | 38 |
| 5. | CASE | DEFINITIONS | 40 |
| | 5.1. | | |
| | 5.2. | Neonatal events of interest | |
| | 5.3. | Respiratory tract illness (RTI) / Lower respiratory tract illness (LRTI) | |
| | 5.4. | RSV infection (Amended 29-MAY-2020) | 40 |
| 6. | STUE | DY POPULATION | |
| | 6.1. | Number of subjects/ centers (Amended 29-MAY-2020) | |
| | 6.2. | Inclusion criteria for enrollment | |
| | | 6.2.1. Maternal subjects: | |
| | | 6.2.2. Infants (Amended 29-MAY-2020): | |
| | 6.3. | Exclusion criteria for enrollment | |
| | | 6.3.1. Maternal subjects: | |
| | | 6.3.2. Infants: | 45 |
| 7 | CONI | DUCT OF THE STUDY | 15 |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| | 7.1. | | ory and ethical considerations process | , including the informed | 45 |
|---|---|---|---|---|---|
| 8. | DETA | ILED ST | IDY PROCEDURES | | 46 |
| | 8.1. | | | | |
| | 8.2. | • | | | |
| | J | 8.2.1. | | ecial circumstances (Amended | |
| | | 0.2 | | | 47 |
| | 8.3. | Outline | of study procedures (Amende | d 29-MAY-2020) | 48 |
| | 8.4. | Interval | between study visits (Amend | led 29-MAY-2020) | 54 |
| | 8.5. | | | aternal subjects | |
| | | 8.5.1. | | mation | |
| | | 8.5.2. | | S | |
| | | 8.5.3. | | ıbjects | |
| | | 8.5.4. | | | |
| | | 8.5.5. | Biological Specimens / Labo | | |
| | | | | | 56 |
| | | 8.5.6. | | | |
| | | 8.5.7. | | and supplements administered | |
| | | | | standard of care | 57 |
| | | 8.5.8. | Outcomes and Events of Int | | |
| | | | | | 57 |
| | | 8.5.9. | Additional Antenatal / medic | | |
| | | | study visits / procedures | | 58 |
| | 8.6. | Descrip | ion of study procedures for Ne | eonates / Infants (Amended | |
| | | | | | 58 |
| | | 8.6.1. | Eligibility Review and Confirm | mation for Neonates | 58 |
| | | 8.6.2. | History and Examinations fo | | |
| | | | | | 59 |
| | | 8.6.3. | | | |
| | | 8.6.4. | Surveillance for Neonatal ev | ents of interest | 60 |
| | | 8.6.5. | Surveillance for potential Lo | wer Respiratory Tract Illness | |
| | | | (LRTI) | | 60 |
| | | | 8.6.5.1. Definitions | | 60 |
| | | | 8.6.5.2. Overview (Amend | ded 29-MAY-2020) | 61 |
| | | | 8.6.5.3. Active surveilland | ce | 63 |
| | | | | nce | |
| | | 8.6.6. | | o assess a potential LRTI | |
| | | 8.6.7. | | RTI | |
| | | | | ded 29-MAY-2020) | |
| | | | 8.6.7.2. Clinical evaluatio | n (Amended 29-MAY-2020) | 64 |
| | | | | ent visit | 65 |
| | | 8.6.8. | • | ent visit to evaluate a potential | |
| | | 8.6.9. | • | | 66 |
| | 8.7. | | g Covid-19 Cases – Maternal | | |
| | 8.8. | | | | |
| | 8.9. | | | | |
| | 8.10. | Screen | ng failures | | 67 |
| | 8.11. | Biologic | al sample handling and analys | sis | 67 |

| | | | 207636 (EPI-RSV-008<br>Protocol Amendment | |
|---|---|---|---|---|
| | | 8.11.1. | Use of specified study materials | |
| | | 8.11.2. | Biological samples | |
| | | 8.11.3. | Laboratory assays | |
| | | | 8.11.3.1. Antibody determination (Amended 29-MAY- | |
| | | | 2020) | 69 |
| | | | 8.11.3.2. Molecular biology | |
| | | | 8.11.3.3. Hematology, biochemistry and urinalysis | |
| | | | 8.11.3.4. Additional tests | |
| | | 8.11.4. | Biological samples evaluation | |
| | | | 8.11.4.1. Immunological read-outs | |
| | | | 8.11.4.2. Molecular biology | 72 |
| | | | 8.11.4.3. Hematology/blood chemistry | 73 |
| 9. | SERIC | OUS ADV | ERSE EVENTS RELATED TO STUDY PARTICIPATION | 73 |
| | 9.1. | Definitio | n | 73 |
| | 9.2. | Event Id | lentification | 74 |
| | 9.3. | Subject | cards | 74 |
| | 9.4. | | ontact information, GSK Reporting Timeframes, and | |
| | | | ory reporting requirements | |
| | 9.5. | | tion to be reported | |
| | 9.6. | | port Completion and transmission to GSK | 76 |
| | | 9.6.1. | 1 7 | 76 |
| | | 0.6.2 | | 76 |
| | | 9.6.2. | Updating of SAE information after removal of write access to the subject's eCRF | 76 |
| | 9.7. | Follow- | up of SAEs related to study participation (Amended 29-MAY- | 70 |
| | 3.1. | | ip of OALS related to study participation (Amerided 29-MAT- | 77 |
| | | 9.7.1. | | |
| | | 9.7.2. | | |
| | | | (Amended 29-MAY-2020) | 77 |
| 10. | | | MPLETION AND WITHDRAWAL | |
| | 10.1. | | completion | |
| | 10.2. | Subject | withdrawal | // |
| 11. | STATI | ISTICAL I | METHODS | 79 |
| | 11.1. | | ts | |
| | | 11.1.1. | Primary endpoints | |
| | | | 11.1.1.1. Pregnancy outcomes | |
| | | | 11.1.1.2. Pregnancy related events of interest from Visit | |
| | | | 1 through Visit 6. | 79 |
| | | | 11.1.1.3. Neonatal events of interest from birth through | |
| | | | 28 days of age | |
| | | 11.1.2. | Secondary endpoints | |
| | 44.0 | 11.1.3. | Tertiary endpoints (Amended 29-MAY-2020) | |
| | 11.2. | Determi | nation of sample size | 83 |
| | 11.3. | 11.3.1. | for Analyses (Amended 29-MAY-2020)<br>Exposed Sets (ES) | |
| | | 11.3.1. | 11.3.1.1. Pregnant women (mothers) | 04 |
| | | | 11.3.1.2. Neonates/Infants | |
| | | 11.3.2. | Enrolled sets | |
| | | | 11.3.2.1. Pregnant women (mothers) | |

| | | | | | endment 4 Final |
|---|---|---|---|---|---|
| | | | 11.3.2.2. | Neonates/Infants | 84 |
| | | 11.3.3. | Per Proto | ocol Sets (PPS) (Amended 29-MAY-2020) | 84 |
| | | | 11.3.3.1. | Pregnant women (mothers) | 84 |
| | | | 11.3.3.2. | Neonates/Infants | 84 |
| | 11.4. | | | ormed data | |
| | | | | of missing values/censoring/discontinuation | |
| | 11.5. | | | raphic and baseline characteristics | |
| | 11.6. | | | objectives (Amended 29 May 2020) | |
| | 11.7. | | | ary objectives (Amended 29-MAY-2020) | |
| | 11.8. | | | objectives (Amended 29-MAY-2020) | |
| | 11.9. | | | alyses | |
| | | • | • | | |
| | 11.11. | | | es | |
| | | 11.11.1. | | I considerations for interim analyses (Amen | |
| | | | 29-MAY-2 | 2020) | 89 |
| 2. | ADMIN | NISTRATI | IVE MATTE | ERS | 90 |
| | 12.1. | Electron | ic Case Re | eport Form instructions | 90 |
| | 12.2. | Study m | onitoring by | y GSK Biologicals | 90 |
| | 12.3. | | | ure | |
| | 12.4. | Record | retention | | 91 |
| | 12.5. | Quality a | assurance. | | 92 |
| | 12.6. | Posting | of informati | ion on publicly available registers and public | cation |
| | 12.7. | Provision | n of study r | results to investigators | 92 |
| | 12.8. | Data Sh | aring | | 92 |
| 13. | COUN | TRY SPE | ECIFIC REC | QUIREMENTS | 92 |
| 4 | REFF | RENCES | (AMENDE | D 29-MAY-2020) | 93 |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# **LIST OF TABLES**

| | | PAGE |
|---|---|---|
| Table 1 | Sampling schedule for maternal subjects | 39 |
| Table 2 | Study groups and epochs foreseen in the study | 40 |
| Table 3 | RTI/LRTI case definitions for data analysis | 41 |
| Table 4 | Alternative LRTI / Severe LRTI Case Definitions (Amended 29-MAY-2020) | 42 |
| Table 5 | List of study procedures for maternal subjects (Amended 29-MAY-2020) | 48 |
| Table 6 | List of study procedures for neonates/ infants (Amended 29-MAY-2020) | 52 |
| Table 7 | Intervals between study visits/contacts/observations* (Amended 29-MAY-2020) | 54 |
| Table 8 | Biological samples | 69 |
| Table 9 | Humoral immunity (Antibody determination) (Amended 29-MAY-2020) | 69 |
| Table 10 | Molecular biology | 70 |
| Table 11 | Hematology, biochemistry, urine tests | 71 |
| Table 12 | Immunological read-outs | 72 |
| Table 13 | Molecular biology for nasal swab specimen analysis | 72 |
| Table 14 | Hematology/blood chemistry tests | 73 |
| Table 15 | Contact information for reporting SAEs related to study participation to GSK | 75 |
| Table 16 | Timeframes for submitting SAEs related to study participation to GSK | 75 |
| Table 17 | Precision (exact 95% confidence interval) on the percentage of subjects with maternal, fetal and neonatal events of interest for sample size of 270, 180 and 100 subjects | 83 |
| Table 18 | GSK Biologicals' laboratories | 96 |
| Table 19 | Outsourced laboratories | 96 |
| Table 20 | Fetal death / Stillbirth | 100 |

| | | 7636 (EPI-RSV-008 BOD)<br>otocol Amendment 4 Final |
|---|---|---|
| Table 21 | Maternal Death | 103 |
| Table 22 | Hypertensive disorders of pregnancy (Gestational Pre-eclampsia, Pre-eclampsia with severe features eclampsia) | sincluding |
| Table 23 | Antenatal Bleeding | 106 |
| Table 24 | Postpartum hemorrhage | 108 |
| Table 25 | Fetal growth restriction | 108 |
| Table 26 | Dysfunctional labor | 109 |
| Table 27 | Gestational diabetes mellitus (pregnancy induced hyperglycemia) | 110 |
| Table 28 | Non-reassuring fetal status | 111 |
| Table 29 | Pathways to preterm birth | 112 |
| Table 30 | Standard Definitions for Maternal Events of interes as events in GAIA | |
| Table 31 | Small for Gestational Age | 116 |
| Table 32 | Low Birth Weight (LBW) | 117 |
| Table 33 | Neonatal encephalopathy | 118 |
| Table 34 | Congenital Microcephaly | 119 |
| Table 35 | Major Congenital anomalies | 122 |
| Table 36 | Neonatal Death | 125 |
| Table 37 | Neonatal Infections | 127 |
| Table 38 | Respiratory Distress in the Neonate | 130 |
| Table 39 | Preterm Birth | 131 |
| Table 40 | Failure to Thrive | 132 |
| Table 41 | Standard Definitions for Neonatal Events of interes as events in GAIA | |

# 207636 | Protocol Amendment 4 03 Jun 2020 | TMF-1793653 | 1.0

# CONFIDENTIAL

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# **LIST OF FIGURES**

| | | PAGE |
|----------|-----------------------------------------------|------|
| Figure 1 | Study design (Amended 29-MAY-2020) | 38 |
| Figure 2 | Active and Passive Surveillance Decision Tree | 62 |

# 207636 | Protocol Amendment 4 03 Jun 2020 | TMF-1793653 | 1.0

# CONFIDENTIAL

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# LIST OF APPENDICES

| | PAGE |
|---|---|
| APPENDIX A LABORATORY ASSAYS | 95 |
| APPENDIX B CLINICAL LABORATORIES | 96 |
| APPENDIX C GAIA GESTATIONAL AGE ASSESSMENT FORM | 97 |
| APPENDIX D DEFINITIONS OF MATERNAL, FETAL AND NEONATAL EVENTS OF INTEREST AS PER GAIA | 99 |
| APPENDIX E AMENDMENTS AND ADMINISTRATIVE CHANGES TO THE PROTOCOL | 134 |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# **LIST OF ABBREVIATIONS (Amended 29-MAY-2020)**

AE Adverse Event

BMI Body mass index

CI Confidence Interval

CLS Clinical Laboratory Sciences

COVID-19 Corona Virus Disease 2019

eCRF electronic Case Report Form

EoS End of Study

FU Follow-Up

GAIA Global Alignment of Immunization Safety Assessment in

pregnancy

GCP Good Clinical Practice

GMC Geometric Mean Concentration

GMT Geometric Mean Titer

GSK GlaxoSmithKline

HIV Human Immunodeficiency Virus

ICF Informed Consent Form

ICH International Council for Harmonisation

IEC Independent Ethics Committee

IRB Institutional Review Board

LAR Legally Acceptable Representative

LLOQ Lower Limit of Quantification

LMP Last Menstrual Period

LRTI Lower Respiratory Tract Illness

LSLV Last Subject Last Visit

NB Newborn

# 207636 | Protocol Amendment 4 03 Jun 2020 | TMF-1793653 | 1.0

#### CONFIDENTIAL

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

PCD Primary Completion Date

PCR Polymerase Chain Reaction

RBC Red Blood Cell

RR Respiratory Rate

RSV Respiratory Syncytial Virus

RTI Respiratory Tract Illness

SAE Serious Adverse Event

SPM Study Procedures Manual

SpO2 Blood oxygen saturation as measured by pulse oximetry

WBC White Blood Cell

WHO World Health Organization

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### **GLOSSARY OF TERMS**

Adverse event:

Any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product, or temporally associated with a study procedure.

An adverse event (AE) can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse or misuse.

**Body Mass Index** 

A key index for relating weight to height. Calculated as follows: Weight  $(kg) / (Height (m))^2$ 

Child

A young human being below the legal age of majority (generally < 18 years of age).

Child in care:

A child who has been placed under the control or protection of an agency, organisation, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation. The definition of a child in care can include a child cared for by foster parents or living in a care home or institution, provided that the arrangement falls within the definition above. The definition of a child in care does not include a child who is adopted or has an appointed legal guardian.

Cohort study:

A form of epidemiological study where subjects in a study population are classified according to their exposure status/disease and followed over time (prospective/ retrospective) to ascertain the outcome(s).

Eligible:

Qualified for enrollment into the study based upon strict adherence to inclusion/exclusion criteria.

Enrollment

Pregnant woman who meet all eligibility criteria at the Screening visit and return to the study site for Visit 1 are considered enrolled. Live born neonates who meet all eligibility criteria and complete Visit 1-NB are considered enrolled.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Epidemiological study: An observational or interventional study without

administration of medicinal product(s) as described in a

research protocol.

End of Study (Synonym of

End of Trial)

For studies with collection of Human Biological Samples or imaging data, EoS is defined as the date of the last testing/reading released of the Human Biological Samples or imaging data, related to primary and secondary endpoints. EoS must be achieved no later than 8 months

after LSLV

An epoch is a set of consecutive timepoints or a single Epoch:

> timepoint from a single protocol. Epochs are defined to support a main purpose which either to draw conclusions on subject participation or to draw a complete conclusion to define or precise the targeted label of the product. Supporting means that data collected at the timepoints included in an epoch must be sufficient to fulfill the

purpose of the epoch.

Typical examples of epochs are screening,

immunogenicity follow-up, safety follow-up, ESFU,

follow-up.

GSK Biologicals' tracking tool for clinical/ eTrack:

epidemiological trials.

Evaluable: Meeting all eligibility criteria, complying with the

procedures defined in the protocol, and, therefore,

included in the per-protocol analysis (see Section 11.3 for

details on criteria for evaluability).

**GAIA** Global Alignment of Immunization Safety Assessment in

> pregnancy. A project that aims to improve the quality of outcome data from clinical vaccine trials in pregnant women with a specific focus on the needs and

requirements for safety monitoring in low to middle

income countries.

A measure of the age of a pregnancy where the origin is Gestational age:

> the first day of the woman's last normal menstrual period, or the corresponding age as estimated by other methods. Gestational age will be described in weeks of pregnancy completed + number of days completed of the following week. For example: 28 0/7 means completed 28 weeks of pregnancy + 0 days of the 29th week and 28 6/7 means completed 28 weeks of pregnancy + 6 days of the 29th

week.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Infant A child younger than 1 year of age

Interventional Human Subject Research:

Studies in which participants are administered medical care, medicinal products and/or medical/scientific procedures as described in a research protocol.

Legally acceptable representative (LAR)

An individual or juridical or other body authorized under applicable law to consent, on behalf of a prospective subject, to the subject's participation in the trial. (The terms legal representative or legally authorized representative are used in some settings.)

Level 2 ultrasound (or fetal morphology ultrasound)

Comprehensive, detailed evaluation of fetal anatomy and development that is usually performed at approximately 20 weeks of gestational age. In addition to standard ultrasound parameters such as fetal heart activity and gestational age estimation, a Level 2 ultrasound usually includes assessment of amniotic fluid levels; assessment of the condition of the placenta, cervix, and uterus; and detection of fetal anomalies. May also be referred to as a fetal anomaly scan or fetal morphology assessment.

Local healthcare provider

A healthcare provider who provides subjects with medical care per local standards. This individual may or may not be a member of the study staff.

Neonate (or Newborn)

An infant  $\leq$  28 days old.

Neonatal events of interest

Clinically significant events that occur from birth through 28 days of age and may be considered adverse events if they occur after vaccination. They are listed in Section 11.1 and described in detail in APPENDIX D

Parental concern

The parent(s) / Legally Acceptable Representative(s) or their designates are concerned about the infant's respiratory tract illness, or general health in the context of the respiratory tract illness, and intend to seek medical care

Pregnancy related events of interest

Clinically significant events that occur up to 42 days after delivery and may be considered adverse events if they occur after vaccination. They are listed in Section 11.1 and described in detail in APPENDIX D

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Primary completion date: The date that the final subject was examined or received

an intervention for the purpose of final collection of data for all primary outcomes, whether the clinical trial/pharmaco-epidemiological study was concluded

according to the pre-specified protocol or was terminated.

Prospective study: A study in which the subjects/cases are identified and

then followed forward in time in order to address one or

more study objectives.

Protocol amendment: The International Council for Harmonisation (ICH)

defines a protocol amendment as: 'A written description of a change(s) to or formal clarification of a protocol.' GSK Biologicals further details this to include a change to an approved protocol that affects the safety of subjects, scope of the investigation, study design, or scientific

integrity of the study.

Research protocol: A document that describes the objective(s), design,

methodology, statistical considerations, and organisation

of a study. The protocol usually also gives the

background and rationale for the study, but these could be

provided in other protocol referenced documents.

Self-contained study: Study with objectives not linked to the data of another

study.

Serious Adverse Event (SAE) related to study

participation

Any untoward medical occurrence related to study participation (e.g., protocol mandated procedures, invasive tests) that:

- Results in death,
- Is life-threatening,
- Requires hospitalization or prolongation of an existing hospitalization,
- Results in disability /incapacity (i.e., a substantial disruption of a person's ability to conduct normal life functions)

Site Monitor: An individual assigned by the sponsor who is responsible

for assuring the proper conduct of epidemiological studies

at one or more investigational sites.

Study population: Sample of population of interest.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# 1. INTRODUCTION

# 1.1. Background and rationale for the study

Maternal immunization aims to prevent diseases in neonates and infants via transplacental antibody transfer from the mother to the fetus following vaccination of the pregnant woman. Several marketed vaccines are already recommended for and routinely administered to pregnant women, including influenza, tetanus and Tdap vaccines [CDC, 2013a, CDC, 2013b]. There are also a number of maternal vaccines in development that aim to protect neonates and infants from pathogens in addition to, respiratory syncytial virus (RSV). GlaxoSmithKline (GSK) is developing an investigational vaccine for use in pregnant women, against RSV disease. Of note this vaccine is developed solely for immunization in pregnancy.

Maternal immunization is implemented worldwide and has the potential to make a major contribution to reducing RSV lower respiratory tract illnesses (LRTI) and the burden of other diseases in infants globally. Therefore, it is imperative that clinical trials are conducted across different countries in different settings. GSK is proactively addressing potential challenges of conducting clinical trials in pregnant women in low- and middle income countries (LMIC).

Before conducting clinical trials it is important to understand the frequency of pregnancy outcomes and the maternal and neonatal events of interest (i.e. clinically significant events that may be considered adverse events if they occur after vaccination) in each setting where clinical trials may be conducted for better interpretation of safety data. Also, to ensure safety of the participating women, and to characterize the safety profile of the product, adverse events (AEs) in pregnancy should be appropriately detected and managed. This study addresses gaps in understanding of anticipated rates of pregnancy outcomes as well as events of interest in pregnant women and neonates. Furthermore, this study will be conducted at potential sites for future maternal immunization trials and will help assure the capacity of sites to detect and manage clinically significant events of interest in pregnant women and their neonates.

Secondarily, the study will establish surveillance mechanisms for RSV associated illnesses in the neonate/infant (through the first 12 months of life. Whilst there is good documentation of the global burden of RSV disease, incidence of RSV-LRTI according to the World Health Organization (WHO) 2015 case definitions [Modjarrad, 2016] is limited in the literature, particularly in many LMIC settings. Hence, this study will also estimate the incidence of infant RSV-LRTI using WHO case definitions across geographically distinct locations to support incidence rate assumptions for planning of future efficacy trials.

To achieve these goals, GSK will be guided by the WHO recommendations on antenatal care for a positive pregnancy experience [WHO, 2016] and the Global Alignment of Immunization Safety Assessment in pregnancy (GAIA) case definitions [Bonhoeffer, 2016; Bauwens, 2016; Kochhar, 2017]. Standardization of surveillance methodology and case definitions (applicable to maternal immunization AEs) may support comparison of data across different countries [Jones, 2016].

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# 1.2. Rationale for the study population

The intention of this epidemiological study is to obtain an estimate of the background rate of adverse pregnancy outcomes and events that may be seen in future vaccine trial populations and, separately, to assess whether sites are suitable for Phase II/III vaccine trials. The study aims to enroll healthy women with normal uncomplicated pregnancies so that event rates for pregnancy and neonatal events of interest are applicable to the intended population for future vaccine trials. Regardless of enrollment location, healthy pregnant women aged 18 to 45 years with normal, uncomplicated, singleton pregnancies, who have had a level 2 (fetal morphology) ultrasound without any significant findings will be eligible for possible study participation. Inclusion / exclusion criteria have been structured in a way that resembles those of Phase II/III criteria to ensure good comparability between the current study population and that of anticipated future vaccine trials.

Pregnant women  $24^{0/7}$  up to and including  $27^{6/7}$  weeks of gestation will be enrolled, to ensure that they are followed as of the time of potential vaccination in a clinical trial.

Women who do not meet the enrollment criteria will be referred for appropriate local standard of care.

# 1.3. Rationale for the surveillance of pregnancy related events of interest

There are particular challenges in conducting clinical trials in pregnant women, among them limited data on background rates of pregnancy outcomes as well as what may be observed in clinical trials as maternal and neonatal adverse events. A large number of countries aim to strengthen their ability to provide comprehensive antenatal care for all and to enable a positive pregnancy experience. The WHO 2016 recommendations on antenatal care for a positive pregnancy experience [WHO, 2016] give guidance on the frequency of clinic visits, examination procedures and screening tests.

To achieve these goals, GSK will be guided by the WHO recommendations on antenatal care for a positive pregnancy experience [WHO, 2016] and the Global Alignment of Immunization Safety Assessment in pregnancy (GAIA) case definitions [Bonhoeffer, 2016; Bauwens, 2016; Kochhar, 2017]. Standardization of surveillance methodology and case definitions (applicable to maternal immunization AEs) may support comparison of data across different countries [Jones, 2016].

The number and timing of study visits was informed by WHO recommendations on antenatal care [WHO, 2016]. However, local standards of care differ from country-to country. Women should follow the local standard of care. Study data will be collected, in part, from records of the data obtained during the locally recommended antenatal care visits.

In this study, best efforts will be made to work with local healthcare providers to collect the key data on maternal, fetal, neonatal and infant health from routine health records to avoid duplication and an undue burden on the trial subjects.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# 1.4. Rationale for the use of Global Alignment of Immunization safety Assessment in pregnancy (GAIA) case definitions

GAIA, a Brighton collaboration project, aims to develop standardized case definitions and criteria for diagnostic certainty of maternal outcomes and events of interest and neonatal events of interest in the context of immunization trials [Bauwens, 2016; Bonhoeffer, 2016; Kochhar, 2017].

GAIA was established in response to a WHO request to work on a globally aligned approach to monitor safety of maternal immunization clinical trials. The application of these case definitions (APPENDIX D) aims to improve the quality of data generated and to support safety assessment. The goal is to pilot these case definitions prior to the initiation of large maternal immunization trials. To achieve this, the level of diagnostic certainty (APPENDIX D) will be collected for all of the events of interest for which GAIA criteria have been developed.

# 1.5. Rationale for the active and passive surveillance for RSV associated respiratory tract illnesses (RTI) with suspicion of difficulty in breathing/wheezing or with parental concern in neonates/ infants

RSV infects 50-70% of infants in their first year of life, and practically all children have experienced RSV infection and / or illness by their third birthday [Hall, 2009]. In industrialized countries, approximately 2% of infants under one year of age are hospitalized as a consequence of RSV-induced lower respiratory tract illnesses (LRTI) each year. Infants younger than six months have the highest risk of developing severe RSV-induced LRTI. Approximately half of all pediatric LRTI occur in the first six months of life, and LRTI is the leading cause of hospitalization in this age group [Boyce, 2000; Deshpande, 2003; Hall, 2009; Holman, 2004; Iwane, 2004; Nair, 2010; Vicente, 2003].

The implementation of surveillance will also assist in establishing robust infrastructure and processes for RSV-LRTI and RSV hospitalization detection in future vaccine trials.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### 2. BENEFIT: RISK ASSESSMENT

The following section outlines the risk assessment and mitigation strategy for this study protocol:

#### 2.1. Risk Assessment

| Important Potential/Identified Risk | Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Study Procedures | | |
| Blood sample collection- While giving blood the subject may feel faint, or locally experience mild pain, bruising, irritation or redness. | Spontaneous data | Sample collection will only be performed by appropriately trained study personnel. All subjects will remain under observation, post venipuncture, through completion of the applicable study visit. Subjects will be notified of this risk in the informed consent form. |
| Nasal swab collection from infant subjects may cause discomfort | Spontaneous data | Sample collection will only be performed by appropriately trained personnel. Subjects' parent(s)/LAR(s) will be notified of this risk in the informed consent form. |

### 2.2. Benefit Assessment

Study participation may have limited or no benefit for the study subjects themselves.

Study procedures aim to ensure surveillance for maternal outcomes and events of interest and neonatal events of interest. The attention to surveillance may enhance the ability to detect these safety events and to refer subjects for management according to local standard of care. The protocol also includes procedures that may enhance surveillance for RSV, and possibly other lower respiratory tract illnesses, in neonates and infants. Thus, the procedures described in this protocol may enhance the ability to detect these events or illnesses and to refer subjects for management according to local standard of care.

Data collected during the study may enhance understanding of the frequency of maternal events of interest in women with low risk pregnancies, neonatal events of interest, and RSV-associated lower respiratory tract illnesses in neonates and infants.

Surveillance methods explored and data collected during this study may inform future care and prevention efforts and will be used to design robust monitoring systems for future clinical trials of maternal immunization.

# 2.3. Overall Benefit:Risk Conclusion (Amended 29-MAY-2020)

This is an epidemiologic study that describes the prevalence of pregnancy outcomes and maternal/neonatal events of interest. The study does not include the administration of any investigational vaccine. It is not expected that the participation of pregnant women and their babies in the study would create any further risk to study participants. The study includes the establishment of a surveillance system for lower respiratory tract infections (LRTI) which may facilitate detection of respiratory tract infections, including COVID-19 cases, that might be diagnosed in children enrolled in the study.
207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Potential risks to subjects participating in this study are limited to those associated with the collection of biological specimens. Taking into account the measures to minimize these potential risks for subjects participating in this study, the potential or identified risks are justified by the potential benefits of enhanced surveillance for the subjects, and by the knowledge gained about the frequency of events of interest.

## 3. OBJECTIVES

## 3.1. Primary objectives

In healthy pregnant women with uncomplicated pregnancies:

- To determine the frequencies of pregnancy outcomes.
- To determine the frequencies of pregnancy related events of interest from enrollment (Visit 1) through 42 days after delivery (Visit 6). (Although pregnancy related events of interest occur within the first 42 days after delivery they may only be detected later, and are to be reported throughout the study.)

In all neonates live-born to women enrolled in the study:

• To determine the frequencies of neonatal events of interest.

Neonatal events of interest occur within the first 28 days after birth, but may only be detected later and are to be reported throughout the study.

Refer to Section 11.1.1 for the definition of the primary endpoints.

# 3.2. Secondary objectives

*In healthy pregnant women with uncomplicated pregnancies at enrollment:* 

- To determine frequencies of pregnancy related events of interest according to GAIA levels of diagnostic certainty (where these are specified) (APPENDIX D) from enrollment (Visit 1) through 42 days after delivery (Visit 6). (Although pregnancy related events of interest occur within the first 42 days after delivery they may only be detected later, and are to be reported throughout the study.)
- To describe the distribution of RSV-A antibody titers in maternal blood at delivery.

In all neonates live-born to women enrolled in the study:

- To determine frequencies of neonatal events of interest according to GAIA levels of diagnostic certainty (where these are specified). (APPENDIX D). Neonatal events of interest occur within the first 28 days after birth, but may only be detected later and are to be reported throughout the study.
- To describe the distribution of RSV-A antibody titers in cord blood at delivery.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

In all neonates/infants live-born to women enrolled in the study, from birth through 1 year of age:

- To determine the incidence of all, of severe, and of very severe RSV-lower respiratory tract illnesses (LRTIs).
- To determine the incidence of RSV hospitalization.
- Refer to Section 11.1.2 for the definition of the secondary endpoints.

Refer to the GLOSSARY OF TERMS for the definition of enrollment.

# 3.3. Tertiary objectives (Amended 29-MAY--2020)

- To describe co-infections of RSV-LRTI with other respiratory viruses in infants.
- To estimate the association of RSV-LRTI in neonates/infants and the level of RSV neutralizing antibodies in cord blood.
- To determine the incidence of LRTIs/Severe LRTIs (using alternative case definitions)
- To determine risk factors for pregnancy-related and neonatal events of interest.
- If deemed necessary, to further characterize the immune responses to RSV and other infections in maternal subjects and infants (based on maternal serum and cord blood).

Refer to Section 11.1.3 for the definition of the tertiary endpoints.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# 4. STUDY DESIGN OVERVIEW (AMENDED 29-MAY-2020)

Figure 1 Study design (Amended 29-MAY-2020)



D = day; M = month; V = visit; W = week; Y = year. NB = newborn; GA = Gestational age; BS = blood sample; US = urine sample for dipstick testing; IMM = immune response; HB = hematology/biochemistry; RBC = red blood cell(s); WBC = white blood cell(s); RSV = respiratory syncytial virus; RTI = respiratory tract illness; LRTI = lower respiratory tract illness;

Refer to Section 11.11 for additional information about the analyses indicated above.

- <sup>1</sup> If delivery occurs prematurely, skip to Visit 5 ("at delivery").
- <sup>2</sup> At Delivery, RSV-A antibody titers for all women
- <sup>3</sup> At V3, only hemoglobin testing.
- <sup>4</sup> Allowed interval for blood sample collection begins with start of labor (e.g. when the mother arrives at the hospital to deliver and an intravenous line is inserted) and ends 72 hours after delivery.
- <sup>5</sup> RSV-A antibodies in cord blood

NOTE: Covid-19 cases identified within the surveillance framework of the study in maternal and infant subjects will also be recorded.

Protocol waivers or exemptions are not allowed unless necessary for the management of immediate safety concerns. Therefore, adherence to the study design requirements, including those specified in the outline of study procedures (Section 8.3), are essential and required for study conduct.

<sup>&</sup>lt;sup>6</sup>Neonatal events of interest occur (by definition) between 0 and 28 days after birth. They will be reported once site staff become aware of them (whether this occurs during the first 28 days after birth, or at a later time).

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- Type of design: Prospective, epidemiological, interventional (without administration of medicinal products as described in a research protocol), multi-country, cohort study.
- Study population: The study will be conducted in multiple countries, in pregnant women and their infants.
- Type of study: self-contained.
- Data collection: Electronic Case Report Form (eCRF).

Table 1 Sampling schedule for maternal subjects

| | | | | | Visit | |
|---|---|---|---|---|---|---|
| Sample | Parameter(s) evaluated | 1 | 2 | 3 | 4 | Delivery |
| Maternal Blood | Hematology/ | | | | | |
| | biochemistry <sup>1, 4</sup> | Х | | <b>x</b> <sup>3</sup> | | |
| | | | | | | ≤ 72 hours after |
| | Antibody titer (RSV-A) | | | | | delivery <sup>5</sup> |
| Cord Blood | Antibody titer (RSV-A) | | | | | Х |
| Urine | Protein, glucose, RBC, WBC <sup>2, 4</sup> | Х | Χ | Х | Х | |

<sup>&</sup>lt;sup>1</sup> To be performed preferentially by local healthcare providers, as per local practice. To be performed by the investigator/study staff ONLY if not done by the local healthcare provider within 2 weeks before the study visit.

- Sampling schedule for **neonates/infants**: Surveillance for RSV LRTI will be conducted in infants through the 12 month study period. During this 1-year post-birth surveillance period, for each RTI with suspicion of difficulty in breathing, or wheezing, or with parental concern, a nasal swab will be collected at a visit to assess potential RSV associated RTIs/LRTIs.
- Primary Completion Date (PCD): 42 days post-delivery/birth (i.e. Visit 6 for maternal subjects and Visit 2-NB for infant subjects) or last visit of Epoch 002.
- End of Study (EoS): Last testing results released of samples collected up to Visit 4-NB (assays related to primary and secondary endpoints).
- Duration of the study: Approximately 4.5 to 6 months for maternal subjects; approximately 1 year for infant subjects.
  - Epoch 001: Screening
  - Epoch 002: Primary starting at Visit 1 and ending 42 days post-delivery/birth (Visit 6 for maternal subjects and Visit 2-NB for infant subjects).\*
  - Epoch 003: Follow-up of infants starting 43 days post-delivery/birth and ending at Visit 4-NB (1 year post-birth).

<sup>&</sup>lt;sup>2</sup>The investigator/site staff will perform a urine dipstick test using supplies provided by GSK.

<sup>&</sup>lt;sup>3</sup> Hemoglobin only

<sup>&</sup>lt;sup>4</sup> If results are abnormal, subjects will be referred per local standard of care.

<sup>&</sup>lt;sup>5</sup> This sample may be collected from start of labor (e.g. when the mother arrives at the hospital to deliver and an intravenous line is inserted) through 72 hours after delivery.

<sup>\*</sup>Any safety and disease surveillance data collected after Visit 2-NB will be collected in Epoch 003.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Table 2 Study groups and epochs foreseen in the study

| Study Groups | Number of | Age (Min/Max) | Epochs | | |
|---|---|---|---|---|---|
| | subjects enrolled | | Epoch 001 | Epoch 002 | Epoch 003 |
| Maternal subjects | Up to ~ 2300 | 18 years - 45 | Х | Х | |
| | | years | | | |
| Infants | Up to ~ 2300 | NA | | Х | Х |

Approximately 200 to 300 per country. To achieve the enrollment targets noted above, the number of pregnant women SCREENED in each country may exceed the country-specific enrollment goal.

- Surveillance for pregnancy outcomes and pregnancy-related events of interest (Section 8.5.8) that occur from Visit 1 up to 42 days after delivery (Visit 6).
- Surveillance for neonatal events of interest(Section 8.6.3) that occur from birth up to 28 days of age.
- Surveillance for RSV LRTI and RSV hospitalization (refer to Section 8.6.8) in infants, from birth up to 1 year of age.

### 5. CASE DEFINITIONS

# 5.1. Pregnancy related events of interest

Pregnancy related events of interest are briefly defined in the GLOSSARY OF TERMS, listed in Section 11.1 and described in detail in APPENDIX D.

## 5.2. Neonatal events of interest

Neonatal events of interest are briefly defined in the GLOSSARY OF TERMS, listed in Section 11.1 and described in detail in APPENDIX D.

# 5.3. Respiratory tract illness (RTI) / Lower respiratory tract illness (LRTI)

During data analysis, cases of respiratory tract illness (RTI) identified from birth up to 1 year of age will be classified according to the case definitions in Table 3.

# 5.4. RSV infection (Amended 29-MAY-2020)

Nasal swabs will be analyzed by the sponsor for the presence of RSV A/B. A positive test result constitutes a case of RSV infection. Refer to Section 8.6.7.3.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## Table 3 RTI/LRTI case definitions for data analysis

| RSV-RTI | Runny nose, OR Blocked nose, OR Cough |
|---|---|
| KOV-KII | AND |
| | · " · = |
| | Confirmed RSV infection <sup>4</sup> |
| RSV-LRTI | History of cough OR difficulty in breathing <sup>1</sup> |
| | AND |
| | SpO <sub>2</sub> < 95% <sup>2</sup> , OR RR increase <sup>3</sup> |
| | AND |
| | Confirmed RSV infection <sup>4</sup> |
| RSV-severe LRTI | Meeting the case definition of RSV-LRTI |
| | AND |
| | SpO <sub>2</sub> < 93%, OR lower chest wall in-drawing |
| RSV-very severe LRTI | Meeting the case definition of RSV-LRTI |
| _ | AND |
| | SpO2 < 90%, OR inability to feed OR failure to respond / unconscious |
| RSV hospitalization | Confirmed RSV infection 5 |
| | AND |
| | Hospitalized for acute medical condition <sup>6</sup> |
| All-cause RTI | Runny nose, OR Blocked nose, OR Cough |
| All-cause LRTI | History of cough OR difficulty in breathing <sup>1</sup> |
| | AND |
| | SpO2 < 95% 2, OR RR increase <sup>3</sup> |

Definitions based on [Modjarrad, 2016]

RTI = respiratory tract illness; LRTI = lower respiratory tract illness; RR = respiratory rate;  $SpO_2$  = blood oxygen saturation by pulse oximetry.

- > 60/minute (< 2 months of age)
- > 50/minute (2 to < 12 months of age)
- > 40/minute (12 to 24 months of age)

<sup>&</sup>lt;sup>1</sup> Based on history reported by parents/LARs and includes difficulty in breathing (e.g. showing signs of wheezing or stridor, tachypnoea, flaring [of nostrils], chest in-drawing, apnoea).

<sup>&</sup>lt;sup>2</sup> For blood oxygen saturation (SpO<sub>2</sub>), the lowest value monitored will be used. In high altitudes (>2500m), SpO<sub>2</sub> <92% for LRTI, <90% for severe LRTI, <87% for very severe LRTI.

<sup>&</sup>lt;sup>3</sup> RR increase defined as:

<sup>&</sup>lt;sup>4</sup> RSV infection confirmed on nasal swab positive for RSV A or B by quantitative reverse transcription polymerase chain reaction (gRT-PCR).

<sup>&</sup>lt;sup>5</sup> RSV sampling and testing is described in Sections 8.6.7, 8.6.8 and 8.6.9.

<sup>&</sup>lt;sup>6</sup> Hospitalization is defined as admission for observation or treatment based on the judgement of a health care provider

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# Table 4 Alternative LRTI / Severe LRTI Case Definitions (Amended 29-MAY-2020)

| | | Documented physical examination (PE) findings indicating lower | |
|---|---|---|---|
| | RSV | , , | Objective measures of clinical severity (at |
| | confirmed | one symptom) | least one symptom) |
| LRTI | Confirmed | Rhonchi <sup>1</sup> | Increased respiratory rate (bpm) |
| | RSV infection | Rales <sup>1</sup> | ≥ 60 for < 2 mo |
| | | Crackles | ≥ 50 for 2-6 mo |
| | | Wheeze | Hypoxemia: |
| | | | SpO2 <95% at ≤1800 meters |
| | | | SpO2 <92% at > 1800 meters |
| | | | New onset apnea |
| | | | Nasal flaring |
| | | | Retractions <sup>2</sup> |
| | | | Grunting |
| Severe<br>LRTI | Confirmed<br>RSV infection | Rhonchi <sup>1</sup> | Нурохетіа |
| | | Rales <sup>1</sup> | SpO2 <93% at ≤1800 meters |
| | | Crackles | SpO2 <90% at > 1800 meters |
| | | Wheeze | Acute hypoxic or ventilatory failure <sup>3</sup> |
| | | | Dehydration due to respiratory distress |
| | | | requiring IV hydration⁴ |
| | | | Failure to respond or unconscious |

<sup>&</sup>lt;sup>1</sup>Term not listed in the eCRF page in this study.

## 6. STUDY POPULATION

# 6.1. Number of subjects/ centers (Amended 29-MAY-2020)

The study will be conducted at multiple centers in multiple countries. The total enrolled study population will consist of up to (approximately) 2,300 pregnant women and their neonates.

In each participating country, approximately 200 to 300 pregnant women  $\geq 24^{0/7}$  and  $\leq 27^{6/7}$  weeks of gestation will be enrolled. Neonates of enrolled pregnant women who consent to their child's study participation will also be enrolled.

<sup>&</sup>lt;sup>2</sup> Intercostal recession or chest wall indrawing are considered synonymous with and will be used as alternatives to the term "retractions," which is not listed in the eCRF page for this study.

<sup>&</sup>lt;sup>3</sup> Acute hypoxic or ventilatory failure is not listed in the eCRF page for this study. Instead, the presence of either respiratory support excluding mechanical ventilation OR requirement for mechanical ventilation or both will be used.

<sup>&</sup>lt;sup>4</sup> Dehydration due to respiratory distress requiring IV hydration is not listed in the eCRF page for this study. Skin turgor > 2 seconds or administration of IV fluid therapy will be used instead.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

### 6.2. Inclusion criteria for enrollment

Deviations from inclusion criteria are not allowed because they can potentially jeopardise the scientific integrity and regulatory acceptability of the study or subject safety. Therefore, adherence to the criteria as specified in the protocol is essential.

All subjects must satisfy ALL the following criteria at study entry:

## 6.2.1. Maternal subjects:

- Healthy pregnant women 18-45 years of age who are  $\geq$  24 0/7 weeks GA at screening and  $\leq$  27 6/7 weeks GA at Visit 1, as established by ultrasound examination and/or last menstrual period (LMP) date\*
- \* The level of diagnostic certainty of the gestational age should be established by using the GAIA gestational age assessment form (provided in APPENDIX C).
- Women with pre-pregnancy body mass index (BMI)  $\geq$ 18.5 and  $\leq$  39.9 kg/m<sup>2</sup>.
- Women whose pregnancy is considered low risk, based on medical history, obstetric history, and clinical findings during the current pregnancy.
- Women who had no significant findings (such as abnormal fetal morphology, amniotic fluid levels, placenta, or umbilical cord) observed during a Level 2 ultrasound (fetal morphology assessment).
- HIV uninfected women who have been tested within the past year and have documented HIV negative test results.
- Individuals who give written or witnessed/thumb printed informed consent after the study has been explained according to local regulatory requirements.
  - The informed consent given at screening should either include consent for both the mother's participation and participation of the infant after the infant's birth (if consistent with local regulations/guidelines), or consent for the mother's participation and expressed willingness to consider permitting the infant to take part after the infant has been born (if local regulations/guidelines require parent(s) to provide an additional informed consent after the infant's birth).
  - Both mother and father should consent if local regulations/guidelines require it.
- Individuals who consent to have cord blood collected at delivery for the purpose of the study;
- Individuals who plan to reside in the study area for at least one year after delivery.
- Individuals who are in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator;
- Individuals who, in the opinion of the investigator can and will comprehend and comply with all study procedures (e.g., return for study follow-up visits, be contactable and available on a regular basis for surveillance).

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## 6.2.2. Infants (Amended 29-MAY-2020):

- Infants who were in utero at the time maternal (and paternal, if required) informed consent was given, and who are live-born.
- If local law requires it: Written or witnessed/thumb printed informed consent for study participation of the infant obtained from parent(s)/LAR(s) within 21 days of birth.

## 6.3. Exclusion criteria for enrollment

Deviations from exclusion criteria are not allowed because they can potentially jeopardise the scientific integrity and regulatory acceptability of the study or subject safety. Therefore, adherence to the criteria as specified in the protocol is essential.

The following criteria should be checked at the screening visit and at Visit 1. If ANY exclusion criterion applies, the subject must not be included in the study:

## 6.3.1. Maternal subjects:

- Individuals determined to have one of the following conditions associated with increased risk for a serious obstetrical complication (specify any/all that apply in the eCRF)
  - Gestational hypertension;
  - Gestational diabetes uncontrolled by diet and exercise;
  - Pre-eclampsia or eclampsia;
  - Multiple pregnancy;
  - Intrauterine growth restriction;
  - Placenta previa;
  - Polyhydramnios;
  - Oligohydramnios.
- Individuals determined to have (during the current pregnancy) one of the following infections or conditions associated with risk of adverse outcome (specify any/all that apply in the eCRF):
  - Known or suspected:
    - Syphilis infection,
    - o Parvovirus B19,
    - Rubella infection,
    - o primary genital herpes simplex infection,
    - o primary cytomegalovirus infection,
    - o varicella infection,

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- o Zika infection,
- o Active tuberculosis infection,
- Incompetent cervix or cerclage
- Individuals who have any underlying condition or infection that would predispose them to increased risk for a serious obstetrical complication that is not mentioned above.
- Individuals who have behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, could interfere with the subject's ability to participate in the study.
- Individuals who have known or suspected impairment of the immune system, an active autoimmune disorder that is not well-controlled, or who are receiving systemic immunosuppressive therapy.
- Individuals participating in any concurrent clinical trial during the current pregnancy.
- Individuals pregnant with a fetus with a confirmed or suspected major congenital anomaly at the time of enrollment.

#### **6.3.2.** Infants:

Child in care

Please refer to the GLOSSARY OF TERMS for the definition of child in care.

## 7. CONDUCT OF THE STUDY

# 7.1. Regulatory and ethical considerations, including the informed consent process

The study will be conducted in accordance with the ICH Guideline for Good Clinical Practice (GCP), all applicable subject privacy requirements and the guiding principles of the Declaration of Helsinki.

The study has been designed and will be conducted in accordance with the ICH Harmonised Tripartite Guideline for clinical investigation of medicinal products in the pediatric population (ICH E11) and all other applicable ethical guidelines.

GSK will obtain favourable opinion/approval to conduct the study prior to a site initiating the study in that country or will document that neither a favourable opinion nor an approval to conduct the study is needed

Conduct of the study includes, but is not limited to, the following:

- Institutional Review Board (IRB)/Independent Ethics Committee (IEC) review and favourable opinion/approval of study protocol and any subsequent amendments.
- Subject/ subject's parent(s)/LAR(s) informed consent, as appropriate.
- Investigator reporting requirements as stated in the protocol.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

GSK Biologicals will provide full details of the above procedures to the investigator, either verbally, in writing, or both.

Freely given and written or witnessed/thumb printed informed consent must be obtained from each subject and/or each subject's parent(s)/LAR(s) or the impartial witnesses appropriate, prior to participation in the study.

GSK Biologicals will prepare a model Informed Consent Form (ICF) which will embody the applicable ICH GCP, and GSK Biologicals required elements. While it is strongly recommended that this model ICF be followed as closely as possible, the informed consent requirements given in this document are not intended to pre-empt any local regulations which require additional information to be disclosed for informed consent to be legally effective. Clinical judgement, local regulations and requirements should guide the final structure and content of the local version of the ICF.

The investigator has the final responsibility for the final presentation of the ICF, respecting the mandatory requirements of local regulations. The ICF generated by the investigator with the assistance of the sponsor's representative must be acceptable to GSK Biologicals and be approved (along with the protocol, and any other necessary documentation) by the IRB/IEC.

## 8. DETAILED STUDY PROCEDURES

# 8.1. Subject identification

Subject numbers for pregnant women (mothers) who consent to participate in the study will be assigned at screening. Subject numbers for their (yet to be born) neonates will be assigned at Visit 1. Subject numbers will be assigned sequentially according to the range of numbers allocated to each study centre. Subject numbers of mother –infant pairs will be clearly linked.

# 8.2. General study aspects

Critical study conduct information not mandated to be present in this protocol is provided in the Study Procedures Manual (SPM). As such, the SPM should be viewed as a companion document that should be read carefully to fully understand the study protocol. The SPM provides the investigator and the site personnel with detailed operational information that is essential for correct study execution and does not impact the safety of the subjects.

Study visits and procedures in this protocol are defined to ensure that maternal and neonatal events of interest, as well as RSV-associated LRTIs and RSV hospitalization in infants, are captured. Prenatal screening and care will be provided by local healthcare providers (in accordance with local standards).

Study visits are not intended to replace local standard of care antenatal visits. If local standard of care recommends additional visits/medical evaluations during pregnancy, women participating in this study should comply with their regular antenatal care visit schedules, per local recommendations.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Study procedures are not intended to replace procedures performed by local healthcare providers as part of standard care.

# 8.2.1. Study procedures during special circumstances (Amended 29-MAY-2020)

During special circumstances (e.g., the COVID-19 pandemic), the specific guidance from local public health and other competent authorities regarding the protection of individuals' welfare must be applied.

For the duration of such special circumstances, the following measures may be implemented for enrolled subjects if deemed feasible by the investigator.

- If it is not possible to conduct a protocol-specified, scheduled or event-driven (e.g., LRTI assessment) visit as described in Section 8.3, the visit may be replaced with a contact conducted by telephone, videotelephony or telemedicine. SMS and email are not allowed.
- Biological samples may be collected at a different location\* other than the study site, or at the subject's home. Biological samples should not be collected if they cannot be obtained within the visit interval (Section 8.4), processed in a timely manner or appropriately stored until the intended use.
  - Nasal swabs should only be collected using centrally provided supplies.
  - Cord Blood for assessment of immune response may be collected locally but must be retrieved, processed and stored in accordance with the Investigator Laboratory Manual.
  - Additional blood samples for assessment of immune response should only be collected using centrally provided supplies.
- Diary cards may be transmitted from and to the site by electronic mail, and / or conventional mail.

Impact on the per protocol sets for analysis will be determined on a case by case basis.

Any impact of the above mentioned measures on the study results will be described in the clinical study report.

\* It is the investigator's responsibility to identify an alternate location. The investigator should ensure that this alternate location meets ICH GCP requirements, such as adequate facilities to perform study procedures, appropriate training of the staff and documented delegation of responsibilities in this location. This alternate location should be covered by proper insurance for the conduct of study on participants by investigator and staff at a site other than the designated study site. Refer to EMA Guidance on the Management of Clinical Trials during the COVID-19 (Coronavirus) pandemic (version 2, 27 March, 2020) for more details.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# 8.3. Outline of study procedures (Amended 29-MAY-2020)

Potential study participants (pregnant women) are to be screened at  $\geq$  24  $^{0/7}$  weeks gestational age. Pregnant women for whom eligibility has been confirmed are to complete Visit 1 not later than at 27  $^{6/7}$  weeks gestational age.

Table 5 List of study procedures for maternal subjects (Amended 29-MAY-2020)

| Gestational age | 24 <sup>0/7</sup> –<br>27 <sup>6/7</sup> | 24 <sup>0/7</sup> –<br>27 <sup>6/7</sup> | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Epoch | Epoch 001 | ch 001 Epoch 002 | | | | | | |
| Type of contact | Screening | Visit 1 | Visit 2 <sup>2</sup> | Visit 3 <sup>2</sup> | Visit 4 <sup>2</sup> | Visit 5 | Visit 6 <sup>3</sup> ,4 | Additional<br>antenatal/medical<br>evaluations <sup>5</sup> |
| Timepoints | | Day 1 | Day 28 | Day 56 | Day 84 | At<br>Delivery | Post-Delivery<br>Day 42 | |
| Eligibility Review and Confirmation | | | | | | | | |
| Informed consent 1 | • | | | | | | | |
| Check inclusion/exclusion criteria | • | 0 | | | | | | |
| Assign subject study number (mother) | • | | | | | | | |
| Assign subject study number (child) | | 0 | | | | | | |
| Ensure that site study physicians (both obstetrician(s) and pediatrician(s)) are informed | | 0 | | | | 0 | | |
| Medical History / Examinations | | | | | | | | |
| Distribute Maternal Subject Card | | 0 | | | | | | |
| Distribute maternal diary card | | 0 | 0 | 0 | 0 | 0 | | |
| Review and collect maternal diary card | | | 0 | 0 | 0 | 0 | 0 | |
| Transcribe applicable diary card data to the eCRF | | | • | • | • | • | • | |
| Record demographic data | • | | | | | | | |
| Record lifestyle characteristics | | • | | | | | | |
| Record outcome of Level 2 ultrasound (fetal morphology scan) <sup>9</sup> | • | | | | | | | |
| Record outcome(s) of subsequent ultrasounds if clinically significant 5 | | O <sup>5</sup> | O 5 | O 5 | O 5 | O 5 | | • 5 |
| Review and collect medical history | 0 | • | | | | | | |
| Review and collect obstetric history from past pregnancies | • | | | | | | | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| | 24 0/7 - | <b>24</b> <sup>0/7</sup> – | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Gestational age | 27 <sup>6/7</sup> | 27 <sup>6/7</sup> | | | | | | |
| Epoch | Epoch 001 | 21 | 1 | | | poch 002 | | |
| Type of contact | Screening | Visit 1 | Visit 2 <sup>2</sup> | Visit 3 <sup>2</sup> | Visit 4 <sup>2</sup> | Visit 5 | Visit 6 <sup>3</sup> ,4 | Additional<br>antenatal/medical<br>evaluations <sup>5</sup> |
| Timepoints | | Day 1 | Day 28 | Day 56 | Day 84 | At<br>Delivery | Post-Delivery<br>Day 42 | |
| Review and collect obstetric history from current pregnancy, including: gestational age, expected date of delivery and method of EDD estimation including pre-pregnancy weight | • | | | | | | | |
| Travel history to, or living in, countries/regions with Zika virus transmission (during the current pregnancy) | 0 | • | 0 | 0 | 0 | 0 | | • |
| Where authorized by the local Ethics Committee, inquire whether mother would have agreed to take part in the study if an investigational vaccine were given | | • | | | | | | |
| Record outcome of HIV test 10 | • | | | | | | | |
| Record results of General and Obstetric examination 11 | • | • | • | • | • | | • | • 14 |
| Check and record prescription medications, vaccinations, folate and/or iron (independently or included in a multivitamin) 13 | • | • | • | • | • | • | • | • |
| Biological Specimens / Laboratory Test Results | | | | | | | | |
| Collect blood sample for antibody assessment by sponsor (~5 ml) | | | | | | • | | |
| Collect cord blood for antibody assessment by sponsor (~5 to 10 ml) | | | | | | • | | |
| Record results of local hematology/ biochemical analysis (Visit 1~5.5 ml; Visit 3~2 ml – hemoglobin only) <sup>6</sup> | | • | | • | | | | • 14 |
| Record results of urine dipstick to check for presence of proteins, glucose, RBC, WBC 8 | | • | • | • | • | | | • 14 |
| Record results of oral glucose challenge / tolerance test(s) if performed by local healthcare provider and available <sup>7</sup> | • | O 5 | O 5 | O 5 | O <sup>5</sup> | | | <b>●</b> 5 |
| Record results of any clinically significant abnormal laboratory tests (including positive urine culture) if performed by local healthcare provider and available <sup>5</sup> | | O 5 | O 5 | O 5 | O 5 | O 5 | O 5 | • 5 |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Gestational age | 24 <sup>0/7</sup> –<br>27 <sup>6/7</sup> | 24 <sup>0/7</sup> –<br>27 <sup>6/7</sup> | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Epoch | Epoch 001 | | • | | | poch 002 | | |
| Type of contact | Screening | Visit 1 | Visit 2 <sup>2</sup> | Visit 3 <sup>2</sup> | Visit 4 <sup>2</sup> | Visit 5 | Visit 6 <sup>3</sup> ,4 | Additional<br>antenatal/medical<br>evaluations <sup>5</sup> |
| Timepoints | | Day 1 | Day 28 | Day 56 | Day 84 | At<br>Delivery | Post-Delivery<br>Day 42 | |
| Labor / Delivery | | | | | | | | |
| Collect and record labor and delivery information 12 | | | | | | • | | |
| Outcomes and Events of Interest | | | | | | | | |
| Record Pregnancy/Delivery outcome(s) | | | | | | • | | |
| Record pregnancy-related events of interest. Record | | | | | | | | |
| other clinically significant events or diagnoses <sup>15</sup> | | | | • | | | • | |
| Record all hospitalizations (except hospitalization for | | | | | | | | |
| delivery), and all extensions of hospitalizations (including | | • | • | • | • | • | • | • |
| extension of hospitalization for delivery) 5 | | | | | | | | |
| Serious Adverse Events | | | 1 | I | | 1 | | |
| Record SAEs related to study participation | • | • | • | • | • | • | • | |
| Screening/Study Conclusion | | | 1 | | | ı | | |
| Screening conclusion | • | | | | | | | |
| Study conclusion | | | | | | | • | |
| Investigator sign-off on eCRF before analysis | • | | | | | | • | |

**SAE** = serious adverse event; • is used to indicate a study procedure that requires documentation in the individual electronic case report form (eCRF)

- o is used to indicate a study procedure that does not require documentation in the individual eCRF.
- <sup>1</sup> Refer to Section 6.2.1, sixth bullet.
- <sup>2</sup> If delivery occurs prematurely, skip to Visit 5 ("at delivery").
- <sup>3</sup> Visit 6 (Day 42) may take place in the subject's home or at the investigator's clinical facility as appropriate to the circumstances in the judgment of the investigator
- <sup>4</sup> To coincide with Visit 2-NB (Day 42) for infants
- <sup>5</sup> Information from additional antenatal / medical evaluations (external to study visits/procedures) may be collected during, before or after a scheduled study visit but should only be recorded in the additional antenatal/medical evaluations eCRF
- <sup>6</sup> To be performed preferentially by local healthcare providers as per local practice. To be performed by the investigator/site staff ONLY if not done by the local healthcare provider within 2 weeks before the study visit. If results are abnormal, subjects will be referred per local standard of care.
- <sup>7</sup> If results of an oral glucose challenge / tolerance test are not available to confirm that the subject does not have Gestational Diabetes at screening, then fasting blood glucose or hemoglobin A1C test results (if performed by local healthcare provider and available) may be used as described in Table 27.
- 8 The Investigator/ site staff will perform a urine dipstick test to detect the presence of proteins, glucose, RBC and WBC.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- 9 If ultrasound results are not available at time of screening, the ultrasound can be performed as a study procedure under certain conditions. Refer to SPM for further details. If abnormal, subjects will be referred per local standard of care.
- <sup>10</sup> **Where** HIV testing is not part of the standard of care for pregnant women, the screening HIV test can be performed locally as a study procedure. Refer to SPM for further details. If results are positive, subject will be referred per local standard of care.
- Height at screening. Weight, temperature, systolic/diastolic blood pressure, heart rate and respiratory rate after at least 10 minutes of rest, blood oxygen saturation by pulse oximetry, fetal heart tones, fetal movement, and fundal height at Screening and Visits 1 4. Temperature, systolic/diastolic blood pressure, heart rate and respiratory rate after at least 10 minutes of rest, and blood oxygen saturation by pulse oximetry at Visit 6.
- 12 Includes date and time of rupture of membranes, date and time of delivery, type of delivery, and other delivery information related to the health and safety of the mother and fetus.
- <sup>13</sup> Beginning the month before the estimated date of conception and while on study. (Routine medications administered during labor and delivery need not be collected.)
- <sup>14</sup> Record clinically significant abnormal results

<sup>&</sup>lt;sup>15</sup>Includes events or diagnoses that could impact the pregnancy including COVID-19 cases

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## Table 6 List of study procedures for neonates/ infants (Amended 29-MAY-2020)

| Epoch | Epo | ch 002 | Epoc | h 003 | Epoch 002 and Epoch 003 | |
|---|---|---|---|---|---|---|
| Age | 0- <i>21</i> days | 42 Days | 6 Months | 12 months | 0-12 months | |
| Type of contact | Visit 1-NB | Visit 2-NB b | Visit 3-NB b | Visit 4-NB b | Contact for<br>active/ passive<br>surveillance | Visit to assess<br>potential LRTI b |
| Timepoints | Birth | Day 42 | М6 | Y1 | | |
| Check inclusion/exclusion criteria | • | | | | | |
| Obtain post-delivery informed consent from parent(s)/LAR(s) if | <ul><li>a</li></ul> | | | | | |
| required per local regulations | | | | | | |
| Record infant's subject number | • | | | | | |
| Record Apgar assessment | • | | | | | |
| Record demographic data | • | | | | | |
| Record lifestyle characteristics | | • | | | | |
| Distribute Infant's Subject Card | 0 | | | | | |
| Distribute infant diary card <sup>d</sup> | 0 | 0 | 0 | | | 0 |
| Review infant diary card | | 0 | 0 | 0 | | 0 |
| Collect infant diary card e f | | 0 | 0 | 0 | | 0 |
| Transcribe applicable infant diary card data to eCRF | | • | • | • | | • |
| Weight, length, head circumference, results of targeted medical history, and results of physical examination | • | • | • | • | | |
| Record prescription medications / vaccinations | • | • | • | • | • | • |
| Record neonatal events of interest | • | • | • | • | | |
| Clinical evaluation of potential LRTI | | | | | | • |
| Nasal swab <sup>b</sup> | | | | | | • c |
| Record all hospitalizations and clinically significant events <sup>h</sup> | • | • | • | • | • | • |
| Record SAEs related to study participation | • | • | • | • | • | • |
| Study conclusion | | | | • | | |
| Investigator sign-off on eCRF before analysis | | • | <b>●</b> 9 | • | | |

LAR = legally acceptable representative; LRTI = lower respiratory tract illness; NB = newborn; RTI = respiratory tract illness; SAE = serious adverse event; M=month; Y = year. Grey shaded columns represent study procedures to be performed for active/passive surveillance of RTIs/LRTIs which are applicable throughout the entire study period (from birth up to study end). Note: The double-line borders indicate primary analyses.

<sup>•</sup> is used to indicate a study procedure that requires documentation in the individual electronic case report form (eCRF).

o is used to indicate a study procedure that does not require documentation in the individual eCRF.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- <sup>a</sup> If local regulations require that written consent / confirmation of consent for the infant's participation be obtained at birth.
- b Visits 2-, 3-, and 4-NB and LRTI assessment visits may take place in the subject's home (if the standard of care allows for home visits), at the investigator's clinical facility or at another facility per the investigator's judgment.
- c If more than one assessment visit is conducted to evaluate a potential LRTI, additional nasal swabs may be collected at the discretion of the Investigator.
- d Distribute at V1-NB: Distribute additional diary cards at subsequent visits as needed.
- e Collect diary cards that are fully filled out and / or document (L)RTI symptoms that have ended. Provide new diary cards as needed.
- f Collect all diary cards for potential RTIs that are considered resolved. Collect the diary card for the current potential LRTI once the LRTI symptoms have ended.
- 9 When approximately 50% of infants have completed up to Visit 3-NB, an interim analysis may be conducted to assess the accumulated RSV LRTI cases and the distribution of maternal and cord blood serum RSV Ab.

h Includes COVID-19 cases

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## 8.4. Intervals between study visits (Amended 29-MAY-2020)

Whenever possible, the investigator should arrange study visits within the interval described in Table 7.

Table 7 Intervals between study visits/contacts/observations\* (Amended 29-MAY-2020)

| Interval | Optimal interval | Allowed interval** |
|---|---|---|
| Screening → Visit 1 | 1 days | 0 - 28 days |
| Visit 1 → Visit 2** | 28 days | 21 –35 days |
| Visit 1 → Visit 3** | 56 days | 49 – 63 days |
| Visit 1 → Visit 4** | 84 days | 77 – 91 days |
| Maternal blood sample collection "at" Visit 5 | 0 days | 0 (Start of labor) - 3 days (i.e., 72 hours |
| (delivery) | | post-delivery) |
| Visit 5 → Visit 6 | 42 days | 35 – 49 days |
| Birth → Visit 1-NB | 0 days | 0 - <b>21</b> days |
| Birth → Visit 2-NB | 42 days | 35 - 49 days |
| Birth → Visit 3-NB | 180 days | 166 -194 days |
| Birth → Visit 4-NB | 365 days | 351 - 379 days |

<sup>\*</sup>If other visits and medical evaluations are performed (outside of study visits/procedures), data should be collected in the electronic case report forms (eCRFs) (see Section 8.5.7).

Investigators should make at least 3 documented attempts (through telephone call(s) or any other convenient procedure) to contact (as relevant) the pregnant woman/mother or the child's parents/ LAR(s) (or their designates) if they do not return for scheduled visits or follow-up. Additional details can be found in the SPM.

# 8.5. Description of study procedures for maternal subjects

This section lists procedures to be performed / data to be recorded during the study and presents additional details where relevant. For the study procedures schedule, refer to Table 5.

# 8.5.1. Eligibility Review and Confirmation

- Obtain Informed consent as described in Sections 6.2.1 and 7.1.
- Check all applicable inclusion and exclusion criteria as described in Sections 6.2 and 6.3 before enrollment and record results.
- Assign / record subject study number (pregnant woman)
- Assign subject study number (infant) for eligible pregnant women who complete Visit 1.
- For eligible pregnant women who complete visit 1 (are enrolled): ensure that site study physicians (both obstetrician(s) and pediatrician(s)) are informed. In particular, the study pediatrician and/or staff should be notified as soon as possible after a pregnant woman's enrolment to ensure the study pediatrician is informed of the approximate date of delivery and potential enrolment of the neonate.

<sup>\*\*</sup>If a subject returns for the visit outside the allowed time interval, he/she may still be considered for analysis.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## 8.5.2. History for maternal subjects

- Distribute the Maternal Subject Card (Section 9.3).
- Distribute the Maternal Diary Card to the subject (Section 8.5.4).
- Record demographic data, which may include (but are not limited to) information such as geographic ancestry (race), month and year of birth, and ethnicity.
- Record information about lifestyle characteristics (exposures), which may include (but are not limited to) data on highest level of education, factors such as smoking status/exposures, household environment, and other factors that could place subjects at risk of study outcomes.
- Record information about whether (during the current pregnancy) the subject has travelled to / is living in countries / regions with Zika virus transmission.
- Where authorized by the local Ethics Committee, inquire whether mother would have agreed to take part in the study if an investigational vaccine were given and record the answer.
- Record outcome of Level 2 ultrasound (fetal morphology assessment). Please see GLOSSARY OF TERMS for description. If Level 2 ultrasound results are not available at screening, then the ultrasound can be performed as a study procedure under certain conditions. Refer to the SPM for further details.
- ONLY record outcome(s) of any subsequent ultrasound(s) if clinically significant.
- Record the subject's pre-pregnancy weight (i.e., weight during the months before the subject became pregnant) in the subject's eCRF. This information can be obtained either via medical record review or subject interview.
- Confirm that the subject's pre-pregnancy BMI is within the range specified in Section 6.2.1. This information can be obtained from the medical record, or, if unavailable, may be calculated based on the subject's height and reported pre-pregnancy weight.
- Obtain the subject's medical and obstetric history by interview and/or review of her medical records. Record any pre-existing conditions or signs and/or symptoms present before participation in the study
  - For past pregnancies, record:
    - Number of past pregnancies and their outcome(s),
    - o Presence of caesarian section scars (if any).
  - For the current pregnancy, record:
    - Gestational age, along with GAIA level of certainty, using priorities defined in APPENDIX C.
    - o Expected date of delivery (EDD) and method of estimation
    - Number of prenatal visits attended up to the date of the study Screening visit,

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- o Approximate date of first prenatal visit,
- Results of any clinically significant, abnormal pregnancy screening laboratory tests,
- o Results of any procedures intended to screen for congenital anomalies.

## 8.5.3. Examinations of maternal subjects

### Record results of General and Obstetric examinations.

- Record height at screening. Height measurements should be performed preferentially by local healthcare providers, in which case the information will be collected and recorded in the mother's eCRF. If not done by the local healthcare provider as per local practice, the investigator/study staff should perform the measurement.
- Unless the study visit is performed concurrently with a routine care visit at which the below data are collected, the investigator/study staff should perform General and Obstetric examinations as follows:
  - Screening and Visits 1 4 should include assessment of weight, fetal heart tones, fetal movement, and fundal height;
  - Screening, Visits 1 to 4, and Visit 6 should include assessment of temperature, systolic/diastolic blood pressure, heart rate and respiratory rate after at least 10 minutes of rest) and blood oxygen saturation by pulse oximetry.
  - If the Screening Visit and Visit 1 occur on the same day, only one General and Obstetric examination will be performed.

# 8.5.4. Maternal Diary Card

A maternal diary card will be provided to each subject at visit 1, then collected and replenished throughout the study as needed. It will document any prescription medications, folate and/or iron (independently or included in a multivitamin) taken, any vaccinations received during pregnancy and after delivery, and any additional visits the subject may make to a healthcare provider not affiliated with the study.

The diary card will be reviewed with the subject during study visits. If review indicates that the subject visited a healthcare provider not affiliated with the study, study staff should (if permitted by local regulation) contact that healthcare provider to obtain the medical record(s) for the visit.

Refer to the SPM for additional details.

## 8.5.5. Biological Specimens / Laboratory Data for maternal subjects

- The Investigator/site staff will arrange for collection of maternal blood and cord blood samples at delivery.
- The Investigator/site staff will perform urine dipstick tests using supplies provided by GSK.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- If HIV test results are not available at time of screening, the HIV test can be performed as a study procedure under certain conditions. Refer to the SPM for further details. If results are positive, the subject will be referred per local standard of care.
- It is preferred that local healthcare providers perform hematology and biochemistry tests per local practice; the investigator/site staff will then collect and record the results. The investigator/site staff will only perform hematology/biochemistry tests if not done by the local healthcare provider within 2 weeks before a study visit.
- If performed by local healthcare provider and results are available, the investigator/site staff will also:
  - Record oral glucose challenge / oral glucose tolerance test results
  - Record any positive urine bacterial culture results
  - Record abnormal and clinically significant laboratory test results
  - Record results of Group B Streptococcus screening test(s).

## 8.5.6. Labor / Delivery

Record information related to labor and delivery, including:

- Any medications administered during labor and delivery as per standard of care if not considered routine
- Date and time of rupture of membranes
- Date and time of delivery
- Type of delivery
- Other delivery related information relevant to the health and safety of the mother and fetus

# 8.5.7. Medications, vaccinations, and supplements administered to maternal subjects as per standard of care

Record medications / vaccinations / folate and iron supplements beginning the month before the estimated date of conception and while on study. Folic acid and/or iron supplements should be reported when taken independently and/or when included in a multivitamin mineral supplement.

# 8.5.8. Outcomes and Events of Interest in maternal subjects (Amended 29-MAY-2020)

• Record delivery and pregnancy outcomes. Of note, fetal death/stillbirth has multiple subcategories. For example, fetal death/stillbirth with no congenital anomalies is an outcome with two subcategories that include: 1) antepartum stillbirth; 2) intrapartum stillbirth. For each outcome, the investigator should select the applicable subcategory.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- If there is no live birth, all study visits and procedures related to the maternal subject should still be followed up to study end.
- Record pregnancy related events of interest.
  - The investigator will review all medical records pertaining to prenatal care based on GAIA definitions (APPENDIX D) when applicable.
  - Maternal events of interest (including, but not limited to, those described in Section 11.1.1) occurring up to Visit 6 (Post-delivery Day 42) should be recorded in the eCRF along with additional details pertinent to the diagnosis, GAIA assessment and level of diagnostic certainty (APPENDIX D), when applicable. Of note, some events of interest fall under a single category but have multiple subcategories. For example, hypertensive disorders of pregnancy is an event with three subcategories that include: 1) gestational hypertension; 2) pre-eclampsia; and 3) pre-eclampsia with severe features (including eclampsia). For each event, the investigator should identify the event and select the applicable sub-category.
  - Information about maternal hospitalizations, clinically significant events, and diagnoses that could impact the pregnancy will be recorded.
  - Any events of interest in mother or fetus will be referred to and managed by the routine health services as locally appropriate.
- Record all hospitalizations and/or clinically significant events, *including COVID-19* cases.
- Record all study participation related SAEs as specified in Section 9.

# 8.5.9. Additional Antenatal / medical evaluations external to study visits / procedures

For any additional antenatal / medical evaluations at which a pregnancy related event of interest is identified, record information that supports the diagnosis of the event, if available.

# 8.6. Description of study procedures for Neonates / Infants (Amended 29-MAY-2020)

This section lists procedures to be performed / data to be recorded during the study and presents additional details where relevant. For the study procedures *schedule*, refer to Table 6. Note that the investigator or study staff will perform (if not performed by local healthcare provider) a minimum of 2 clinical examinations: one at birth (or up to 21 days after birth), and another at approximately 42 days of age.

## 8.6.1. Eligibility Review and Confirmation for Neonates

- Check all applicable inclusion and exclusion criteria as described in Sections 6.2.2 and 6.3.2.
- Record subject study number.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# 8.6.2. History and Examinations for Neonates / Infants (Amended 29-MAY-2020)

- Record demographic data including month and year of birth, gender, geographic ancestry (race) and ethnicity.
- Record Appar scores at 1, 5, 10 min after birth (when available).
- Record lifestyle characteristics. Data may include (but are not limited to) passive smoking and contact with young children under 6 years of age.
- Record weight, length, head circumference, results of targeted medical history, and results of physical examinations.
- Record prescription medications/ vaccinations.
- Distribute the Infant Subject Card to the parent(s)/LAR(s)/designate(s). (Section 9.3).
- Distribute the Infant Diary Card to the parent(s)/LAR(s)/designate(s) (Section 8.6.3).
- Record all hospitalizations and/or clinically significant events, *including COVID-19 cases.* For hospitalizations where an RSV infection is suspected, refer to Section 8.6.8.
- Record all study participation related SAEs (Section 9).

# 8.6.3. Infant Diary Cards

Infant diary cards will be provided at the infant Visit 1 NB. They should be completed by the Parent(s)/LAR(s)/designate(s) of the infant subject.

The infant diary cards will be used to document:

- RTI symptoms experienced by the infant, including start and end dates for those symptoms, and
- Additional visits to a pediatric healthcare provider not affiliated with the study, as well as prescription medications (including those taken to treat an RTI) and vaccinations administered to the infant. (If the infant subject was taken to a healthcare provider not affiliated with the study, the study staff should (if permitted by local regulation) contact that healthcare provider to obtain the medical record(s) for the visit.)

At each study visit (including any assessment visits), RTI symptoms may have ended or may be ongoing.

If blocked nose, cough and symptoms of difficulty in breathing (including wheezing) have ended by the time of a study visit:

 Study staff should collect the Diary card(s), and replenish the parent(s)/LAR(s)/designate(s) supply of blank cards as needed.

If blocked nose, cough or symptoms of difficulty in breathing (including wheezing) are ongoing at the time of a study visit (including any assessment visit):

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- Study staff should review the diary card, make a photocopy of it, and return it to the parent(s)/LAR(s)/designate(s) so information can continue to be collected until the symptoms have ended.
- As soon as possible after these symptoms have ended, study staff must collect the completed diary card by a site visit, home visit, or postal mail, whichever is most effective based on local practice. The site should make every effort to collect completed diary cards as soon after the symptoms have ended as possible. If diary card collection occurs during a visit to the study site or to the subject's home, a brief clinical evaluation may be performed to confirm that the symptoms have ended.

Refer to the SPM for additional details.

### 8.6.4. Surveillance for Neonatal events of interest

To detect events of interest in neonates, the investigator will collect a medical history and review all medical records pertaining to medical events in the neonatal period (birth -28 days), including assessment of congenital anomalies.

## 8.6.5. Surveillance for potential Lower Respiratory Tract Illness (LRTI)

#### 8.6.5.1. Definitions

Symptoms of Respiratory Tract Illness (RTI) include:

- Regular bursts of cough,
- Nasal discharge running freely out of the infant's nose (runny nose), or
- Breathing through the mouth because the infant's nose is blocked (blocked nose).

A potential lower respiratory tract illness (LRTI) is one in which the infant has one or more of the RTI symptoms listed above AND at least one of the following:

- Difficulty in breathing (fast breathing, poor feeding, working hard to breathe, or making unusual sounds when breathing);
- Wheezing (a whistling sound when the infant breathes out) (another sign of difficulty in breathing);
- Parental concern (the parent(s)/LAR(s) or their designate(s) are concerned about the infant's respiratory tract illness, or general health in the context of the respiratory tract illness, and intend to seek medical care).

Worsening means any clinically observed/diagnosed symptoms and signs that are reported during the same respiratory tract illness and reflect a deterioration in the child's respiratory tract functions.

Start and stop dates will be collected in the diary card for cough, runny nose, blocked nose, wheezing and difficulty in breathing.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Start dates for all symptoms will also be recorded in the eCRF.

Only stop dates for cough and difficulty in breathing will be recorded in the eCRF so that GSK may later define the end of each LRTI episode (Section 5.4)

## 8.6.5.2. Overview (Amended 29-MAY-2020)

Surveillance for potential LRTIs begins at birth (or after additional consent, has been provided for the infant's participation in the study, if required,) and ends with the Year 1 study visit.

It will be accomplished via two types of contact. Both may be made with/ by either the Parent(s)/ LAR(s), or a person designated by the parent(s)/LAR(s), such as grandparents or a nanny (as long as the parent(s)/LAR(s) have given approval).

- In an Active contact, site personnel contact the subject's parent(s) / LAR(s) or their designate(s). Active contacts will occur at regular intervals and will be scripted.
- In a Passive contact, the subject's parent(s) / LAR(s) or their designate(s) contact site personnel. Site personnel will use a script to guide data collection once a passive contact has been made.

Site staff will use information gathered during each active or passive surveillance contact to determine whether a visit to assess a potential LRTI (Sections 8.6.6 and 8.6.7) should be scheduled.

For all interactions between parent(s)/LAR(s)/designates and study staff, the safety of the infant is paramount. For any reported illness, the investigator/study staff should assess the need for any intervention and advise the parent(s) / LAR(s) to seek care as necessary. This study is not intended to replace local standards of care.

A decision tree for active and passive surveillance is provided in Figure 2, which is presented on the next page.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Figure 2 Active and Passive Surveillance Decision Tree



RR: Respiratory rate: SpO<sub>2</sub>: Blood oxygen saturation by pulse oximetry.

<sup>&</sup>lt;sup>1</sup>Details regarding Active and Passive Surveillance are provided in Sections 8.6.5.3, 8.6.5.4, and the SPM.

<sup>&</sup>lt;sup>2</sup>Cough, runny nose, blocked nose, difficulty in breathing, wheezing and parental concern are defined in Section 8.6.5.1.

<sup>&</sup>lt;sup>3</sup>Details regarding the assessment visit to evaluate a potential LRTI are provided in Sections 8.6.6 and 8.6.7 and the SPM.

<sup>&</sup>lt;sup>4</sup> Post-visit follow up is described in Section 8.6.8 and in the SPM. Worsening is defined in Section 8.6.5.1

<sup>&</sup>lt;sup>5</sup>If a follow-up assessment visit is conducted, collection of additional nasal swabs are at the Investigator's discretion.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### 8.6.5.3. Active surveillance

*In countries where RSV transmission is seasonal:* The study staff will contact the infant's parents/ LAR(s) (or their designates) (phone call, SMS or by other means, depending on local best practice) approximately every week during the RSV season and approximately every month outside the RSV season, up to study end.

In countries with year-round RSV transmission: The study staff will contact the infant's parents/ LAR(s) (or their designates) (phone call, SMS or by other means, depending on local best practice) approximately every 2 weeks, up to study end.

Three attempts should be made to contact the infant's parents/ LAR(s) (or their designates) within the week of a scheduled contact. If these attempts are unsuccessful, that active contact is considered a missed contact. The next active contact will be made according to schedule.

The purpose of the contact is to check with the infant's parent(s)/LAR(s) or their designate(s) if, as defined in Section 8.6.5.1:

- the infant has developed (new) symptoms of RTI, difficulty in breathing, or wheezing;
- there is parental concern as defined in Section 8.6.5.1.

#### 8.6.5.4. Passive surveillance

Infants' parents/LAR(s) or their designate(s) will be instructed to contact the site whenever:

- the infant has developed (new) symptoms of RTI, difficulty in breathing, or wheezing as defined in Section 8.6.5.1,
- the infant's symptoms worsen as defined in Section 8.6.5.1,
- there is parental concern as defined in Section 8.6.5.1.

Contact may be via phone call, SMS or other means, depending on local best practice. If the study site is the primary treating facility for the child, Parent(s)/LAR(s) or their designate(s) may also make "contact" by taking the child directly to the study site.

## 8.6.6. Decision to conduct a Visit to assess a potential LRTI

**If there is <u>NO</u>** suspicion of difficulty in breathing, nor wheezing, nor parental concern in the context of the RTI:

- No assessment visit will be conducted.
- The study staff will remind the infant's parent(s)/LAR(s) to report any worsening of symptoms.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

**If there** <u>IS</u> difficulty in breathing, or wheezing (both based on parental assessment), or there is parental concern in the context of the RTI:

An assessment visit will be conducted as soon as possible, ideally within 3 calendar days after learning of the potential LRTI case. Note that the visit may be conducted, and a nasal swab collected, even if beyond the ideal 3-day window as long as symptoms are ongoing.

## 8.6.7. Visit to assess a potential LRTI

## 8.6.7.1. Overview (Amended 29-MAY-2020)

The purpose of the visit is to objectively document signs and symptoms by an appropriately qualified person (i.e. medical or nursing), provide medical advice, and take a nasal swab for detection of RSV infection.

The appropriately qualified person will also evaluate whether the LRTI might be related to COVID19. The appropriately qualified person must follow the local standard of care regarding the reporting, and management of COVID-19 cases (suspected, probable or confirmed COVID-10 case), and complete both the COVID-19 form and LRTI form in the CRF. Refer to Section 8.7.

The visit may take place in the subject's home (if allowed per standard of care), the investigator's clinical facility or another medical facility, as appropriate per the judgment of the investigator.

Note that if the reported symptoms are severe enough to warrant urgent care, the parent(s)/LAR(s)/designates should be advised to seek such care (e.g. Emergency Room).

## 8.6.7.2. Clinical evaluation (Amended 29-MAY-2020)

The investigator/study staff will evaluate the clinical signs and symptoms of the RTI. Data to be collected and recorded include (but are not limited to):

- Temperature
- Respiratory rate
- Blood oxygen saturation (measured by pulse oximetry in room air, if feasible)
- Signs of difficulty in breathing (including wheezing, tachypnoea, nasal flaring, chest in-drawing and apnoea)
- Possible presence of COVID-19 infection (Section 8.7). As noted above, both the LRTI and COVID-19 eCRFs are to be completed (whether or not the investigator/study staff consider the LRTI to be due to COVID-19.

Refer to the Study Procedures Manual (SPM) for additional details.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### 8.6.7.3. Nasal swab

A nasal swab will be collected using sponsor-provided supplies and sent to the sponsor (or sponsor-designated) laboratory for detection of RSV-A/B using quantitative RT-qPCR.

Each nasal swab positive for RSV by quantitative RT-qPCR will also be assessed using a multiplex PCR for detection of a panel of respiratory viruses (Allplex<sup>TM</sup> Respiratory Panel or similar). Further assessment of RSV-A/B negative samples with multiplex PCR may be performed if deemed necessary.

If more than one assessment visit is conducted to evaluate a potential LRTI, additional nasal swabs may be collected (using sponsor-provided supplies and sent to the sponsor laboratory) at the discretion of the Investigator.

Note: Only the results generated by the sponsor (or sponsor-designated) laboratory (analyzing nasal swabs collected using sponsor-provided supplies) will be used when applying the case definitions for data analysis in Table 3. If other nasal swabs are collected and tested locally as per routine standard of care, results will be required to be entered into the eCRF however this will not form part of the sponsor's application of case definitions for data analysis.

Therefore where mandated by the protocol every effort should please be made to obtain samples for analysis by the sponsor (or sponsor-designated) laboratory.

### 8.6.7.4. Missed assessment visit

If the criteria for an assessment visit have been met, but the visit cannot take place while symptoms are ongoing, it is a missed assessment visit.

If it is truly not possible to perform an assessment visit (for example, if the child develops a potential LRTI while the family is travelling, and all symptoms have resolved by the time the family returns), then the LRTI assessment visit page of the eCRF should be filled in as completely as possible using available medical history and medical records.

## 8.6.8. Follow-up after an assessment visit to evaluate a potential LRTI

After an assessment visit (Section 8.6.7) the child will be followed with at least weekly active surveillance contacts, until the RTI/LRTI has resolved. During these active contacts, worsening of symptoms (clinically observed/diagnosed symptoms and signs that are reported during the same respiratory tract illness and reflect a deterioration in the child's respiratory tract functions; for example, onset of additional symptoms or an increase in the intensity of a previously reported symptom) will be assessed. Parent(s) / LAR(s) / designate(s) will be reminded to call/contact/visit the site if symptoms worsen.

If parent(s)/LAR(s)/designates report during an active or passive contact that symptoms have worsened, the site should perform a follow-up visit.

During the follow-up visit, collection of a nasal swab is at the Investigator's discretion.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

After symptoms that resulted in one or more assessment visits have ended (Section 8.6.5.1), site staff will ensure that the diary card for those symptoms is returned to the site via site visit, home visit, or postal mail (depending on the most effective local best practice for prompt retrieval of the completed infant diary card following the end of the symptoms).

Important details are provided in the SPM.

## 8.6.9. RSV Hospitalization

If the child is admitted to hospital for an acute medical event and RSV infection is suspected, during the surveillance period:

- The event will be documented in the eCRF.
- If possible, a nasal swab will be collected from any subject who is hospitalized with a RTI (or soon after release, as long as symptoms are ongoing, per SPM specifications). The nasal swab should be collected using sponsor-provided supplies, for transmission to and testing by the sponsor laboratory.
- If other specimens are collected and tested locally as per routine standard of care, results will be entered into the eCRF. However, only the sponsor laboratory results will be used when applying the case definitions for data analysis in Table 3.

# 8.7. Reporting Covid-19 Cases – Maternal and Infant subjects (Amended 29-MAY-2020)

In addition to satisfying local reporting requirements for COVID-19 cases, maternal and infant COVID-19 cases identified within the existing framework of the study will be captured and reported on the COVID-19 eCRF for the study.

COVID-19 cases should be reported in the eCRF according to the WHO Case Definition [WHO, 2020] using one of the following terms:

- Suspected COVID-19 infection
- Probable COVID-19 infection
- Confirmed COVID-19 infection

# 8.8. SAEs related to study participation

The subjects will be instructed to contact the investigator immediately should they (or their neonates/infants) manifest any signs or symptoms they perceive as serious.

Refer to Section 9 for procedures for the investigator to record SAEs, and for guidelines on how to submit SAE reports to GSK Biologicals.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## 8.9. Study Conclusion

The investigator will review data collected to ensure accuracy and completeness and complete the Study Conclusion screen in the pregnant woman's (mother's) and infant's eCRFs

## 8.10. Screening failures

Screening failures are defined as subjects who withdraw or are withdrawn from the study after giving informed consent, but before study eligibility (presence of all inclusion and absence of all exclusion criteria) is confirmed.

Discovery during screening of any pregnancy related-event of interest or other condition that violates the requirements for study eligibility should be considered a screening failure.

Discovery during Visit 1 of any condition that violates the requirements for study eligibility should also be considered a screening failure.

The development of such conditions (after Visit 1) does not constitute screening failure and should be captured on the eCRF, as applicable.

Limited data for screening failures will be reported to the eCRF. This limited data set is specified in the eCRF.

# 8.11. Biological sample handling and analysis

Please refer to the SPM for details of biospecimen management (handling, storage and shipment).

Samples will not be labeled with information that directly identifies the subjects but will be coded with the identification number for the subject (subject number).

Collected samples will be used for protocol mandated research. In addition, these samples may be used to perform research related to the improvement, development and quality assurance of the laboratory tests described in this protocol. This may include the management of the quality of these tests, the maintenance or improvement of these tests, the development of new test methods, as well as making sure that new tests are comparable to previous methods and work reliably.

It is also possible that future findings may make it desirable to use the samples acquired in this study for future research, not described in this protocol. Therefore, all subjects in countries where this is allowed will be invited to give another specific consent to allow GSK or a contracted partner use of the samples for future research including development of tests and their quality assurance. Future research will be subject to the laws and regulations in the respective countries and will only be performed once an independent Ethics Committee or Review Board has approved this research.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Information on further investigations and their rationale can be obtained from GSK Biologicals.

If additional testing is performed, the priority ranking given in Section 8.11.4.1 may be changed.

Any sample testing will be done in line with the consent of the individual subject/subject's parent(s)/LAR(s).

Refer also to the Investigator Agreement, where it is noted that the investigator cannot perform any other biological assays except those described in the protocol or its amendment(s).

Collected samples will be stored for a maximum of 20 years (counting from when the last subject performed the last study visit, unless local rules, regulations or guidelines require different timeframes or different procedures, which will then be in line with the subject consent. These extra requirements need to be communicated formally to and discussed and agreed with GSK Biologicals.

## 8.11.1. Use of specified study materials

When materials are provided by GSK Biologicals, it is MANDATORY that all samples (including serum samples) be collected and stored exclusively using those materials in the appropriate manner. The use of other materials could result in the exclusion of the subject from the per-protocol analysis (See Section 11.3 for the definition of study cohorts/data sets to be analyzed). The investigator must ensure that his/her personnel and the laboratory(ies) under his/her supervision comply with this requirement. However, when GSK Biologicals does not provide material for collecting and storing samples, appropriate materials from the investigator's site must be used. Refer to the Module on Clinical Trial Supplies in the SPM.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## 8.11.2. Biological samples

Table 8 Biological samples

| Sample Type <sup>†</sup> | Quantity | Unit | Timepoint | Group |
|---|---|---|---|---|
| Samples collected by Investigator / site staff | | | | |
| Maternal Blood for antibody titers | ~ 5 | ml | Visit 5 (Delivery) | All Maternal subjects |
| Cord blood | ~ 5 up to<br>10 | ml | Visit 5 (Delivery) | All Maternal subjects |
| Urine (dipstick) | - | - | Visit 1 (Day 1)<br>Visit 2 (Day 28)<br>Visit 3 (Day 56)<br>Visit 4 (Day 84) | All Maternal subjects |
| Nasal swab | - | - | Visit to assess potential LRTI | All Infants event-driven |
| Samples preferen | tially collected | by local h | ealth care provider per loc | al practice1 |
| Maternal Blood for hematology/<br>biochemistry <sup>1</sup> | Up to 5.5 | ml | Visit 1 (Day 1) | All Maternal subjects |
| Maternal Blood for Hemoglobin | Up to 2 | ml | Visit 3 (Day 56) | |

<sup>&</sup>lt;sup>1</sup>To be performed preferentially by local healthcare providers, as per local practice. To be performed by the investigator/study staff ONLY if not done by the local healthcare provider within 2 weeks before the study visit.

## 8.11.3. Laboratory assays

Please refer to APPENDIX A for a detailed description of the assays performed in the study. Please refer to APPENDIX B for the addresses of the clinical laboratories used for sample analysis.

The GSK Biologicals' clinical laboratories have established a Quality System supported by procedures. The activities of GSK Biologicals' clinical laboratories are audited regularly for quality assessment by an internal (sponsor-dependent) but laboratory-independent Quality Department.

### 8.11.3.1. Antibody determination (Amended 29-MAY-2020)

• Functional (neutralizing) antibody titers against RSV-A will be measured by neutralization assay on serum samples (Table 9).

Table 9 Humoral immunity (Antibody determination) (Amended 29-MAY-2020)

| System | Component | Method | Kit / Manu-<br>facturer | Unit | Cut-off | Laboratory* |
|---|---|---|---|---|---|---|
| SERUM | Respiratory<br>Syncytial<br>Virus A Ab | NEUTRALISATION | In house | ED60<br>and/or<br>IU/ML | ED60: 18;<br>IU/ml: 56 | GSK Biologicals** or<br>GSK designated<br>lab*** |

Ab = antibody; ED60 = serum dilution inducing 60% inhibition in plaque forming units; *IU/mL: International Unit/milliliter* 

<sup>\*</sup> Refer to APPENDIX B for the laboratory addresses.

<sup>\*\*</sup> GSK Biologicals laboratory refers to the Clinical Laboratory Sciences (CLS) in Rixensart, Belgium; Wavre, Belgium. Marburg, Germany

<sup>\*\*\*</sup> Testing may possibly be outsourced to a laboratory designated by GSK. In this case, the method and unit may be different than the one indicated in this table.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## 8.11.3.2. Molecular biology

Table 10 Molecular biology

| System | Component**** | Kit /<br>Manufacturer | Method | Unit | Laboratory |
|---|---|---|---|---|---|
| Nasal | RSV A RNA | In-house | QRTPCR* | Copies/ml | GSK Biologicals |
| swab | RSV B RNA | | | | or GSK |
| | | | | | designated lab** |
| Nasal | Influenza A virus (Flu A) | Allplex™ | Multiplex | Qualitative | GSK Biologicals |
| swab | Human Influenza A virus subtype H1 | Respiratory | real-time | assay | or GSK |
| | (FLU A-H1) | Panel | PCR | (positive | designated lab** |
| | Human Influenza A virus subtype H3 | (Seegene) or | | /negative) | |
| | (FLU A-H3) | equivalent*** | | | |
| | Human Influenza A virus subtype | | | | |
| | H1pdm09 (FLU A-H1pdm09) | | | | |
| | Influenza B virus (Flu B) | | | | |
| | Human respiratory syncytial virus A (RSV A) | | | | |
| | Human respiratory syncytial virus B | | | | |
| | (RSV B) | | | | |
| | Human adenovirus (AdV) | | | | |
| | Human metapneumovirus (MPV) | | | | |
| | Human enterovirus (HEV) | | | | |
| | Human parainfluenza virus 1 (PIV1) | | | | |
| | Human parainfluenza virus 2 (PIV2) | | | | |
| | Human parainfluenza virus 3 (PIV3) | | | | |
| | Human parainfluenza virus 4 (PIV4) | | | | |
| | Human bocavirus 1/2/3/4 (HBoV) | | | | |
| | Human rhinovirus A/B/C (HRV) | | | | |
| | Human coronavirus 229E (229E) | | | | |
| | Human coronavirus NL63 (NL63) | | | | |
| | Human coronavirus OC43 (OC43) | | | | |

<sup>\*</sup>RSV-A/B quantitative reverse transcription PCR will be performed on all specimens of <u>infants</u> with RTI with suspicion of difficulty in breathing/wheezing or parental concern, reported during active or passive surveillance.

## 8.11.3.3. Hematology, biochemistry and urinalysis

Hematology and biochemistry tests are to be performed preferentially by local healthcare providers, as per local practice. They are to be performed by the investigator/study staff ONLY if not done by the local healthcare provider within 2 weeks before the study visit.

The investigator will perform urine dipstick tests to detect the presence of proteins, glucose, RBCs and/or WBCs. These tests do not replace those performed by local healthcare practitioners, per local practice, for clinical management of study subjects.

<sup>\*\*</sup> GSK Biologicals laboratory refers to the Clinical Laboratory Sciences (CLS) in Rixensart, Belgium; Wavre, Belgium.

Marburg Germany

<sup>\*\*\*</sup> Respiratory Viruses Panel (Allplex PCR) will be performed for all specimens RSV A/B-positive and if deemed necessary for RSV A/B-negative samples.

<sup>\*\*\*\*</sup>The list of components might be subject to change in case equivalent kit is used for multiplex RVP testing.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Table 11 Hematology, biochemistry, urine tests

| System | Discipline | Component | Time<br>Point | Method | Scale | Laboratory |
|---|---|---|---|---|---|---|
| Whole<br>blood | Hematology | Hemoglobin | Visit 1 | As per local | As per local Quantitative practice | Local |
| | | | Visit 3 | | | laboratory |
| | | Leukocytes (White Blood<br>Cells) | Visit 1 | | | |
| | | Neutrophils | Visit 1 | | | |
| | | Lymphocytes | Visit 1 | | | |
| | | Monocytes | Visit 1 | | | |
| | | Basophils | Visit 1 | | | |
| | | Eosinophils | Visit 1 | 1 | | |
| | | Platelets | Visit 1 | | | |
| Serum | Biochemistry | Alanine Aminotransferase (ALT) | Visit 1 | As per local practice | Quantitative | Local<br>laboratory |
| | | Aspartate Aminotransferase (AST) | Visit 1 | | | |
| | | Creatinine | Visit 1 | | | |
| | | Urea Nitrogen | Visit 1 | 1 | | |
| Urine | - | Protein | Visit 1<br>Visit 2<br>Visit 3<br>Visit 4 | As per local<br>practice,<br>dipsticks<br>provided by<br>GSK | Ordinal | Local<br>laboratory |
| | | Glucose | Visit 1 | | | |
| | | | Visit 2 | Biologicals | | |
| | | | Visit 3 | | | |
| | | | Visit 4 | | | |
| | | Hemoglobin | Visit 1 | | | |
| | | (RBC) | Visit 2 | | | |
| | | | Visit 3 | | | |
| | | | Visit 4 | | | |
| | | Leukocyte esterase | Visit 1 | 1 | | |
| | | (WBC) | Visit 2 | | | |
| | | ` ' | Visit 3 | | | |
| | | | Visit 4 | | | |

## 8.11.3.4. Additional tests

Additional exploratory testing on the disease under study and/or other respiratory tract infections or infections of relevance to pregnant women and their newborns may be performed within the framework of the study if deemed necessary for accurate interpretation of the data/ should such assay(s) become available at GSK. These assays may not be represented in the objectives/ endpoints of the study protocol.
207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## 8.11.4. Biological samples evaluation

## 8.11.4.1. Immunological read-outs

Table 12 Immunological read-outs

| Blood sampling timepoint Type of contact and time point | Group | No. subjects | Component | Component priority rank |
|---|---|---|---|---|
| • | | Maternal Bloo | d | |
| Visit 5 (Delivery) | All Maternal subjects | cts ~2300 Respiratory Syncytial Virus A Ab (RSV-A neutralising antibody) | | 1 |
| | | Cord Blood | | |
| Visit 5 (Delivery) | All Maternal subjects<br>(provides infant<br>antibody levels) | ~2300 | Respiratory Syncytial Virus A Ab (RSV-A neutralising antibody) | 1 |

## 8.11.4.2. Molecular biology

Table 13 Molecular biology for nasal swab specimen analysis

| Nasal swab sampling timepoint | | | No. | 0 |
|---|---|---|---|---|
| Type of contact (timepoint) | Sampling timepoint | Group | subjects | Component |
| Visit to assess potential LRTI | Unscheduled | All<br>Infants * | Event-<br>driven** | QRTPCR (quantitative reverse transcription PCR): RSV A RNA and RSV B RNA |
| Visit to assess potential LRTI | Unscheduled | All infants* | Event-<br>driven*** | Multiplex PCR including: Influenza A virus (Flu A) Influenza B virus (Flu B) Human respiratory syncytial virus A (RSV A) Human respiratory syncytial virus B (RSV B) Human Influenza A virus subtype H1 (Flu A-H1) Human Influenza A virus subtype H3 (Flu A-H3) Human Influenza A virus subtype H1pdm09 (Flu A-H1pdm09) Human adenovirus (AdV) Human metapneumovirus (MPV) Human enterovirus (HEV) Human parainfluenza virus 1 (PIV1) Human parainfluenza virus 2 (PIV2) Human parainfluenza virus 3 (PIV3) Human parainfluenza virus 4 (PIV4) Human bocavirus 1/2/3/4 (HBoV) Human rhinovirus A/B/C (HRV) Human coronavirus NL63 (NL63) Human coronavirus OC43 (OC43) |

<sup>\*</sup> Refer to Section 8.6.7.

<sup>\*\*</sup> RSV-A/B quantitative PCR (RSV-A/B RNA) will be performed on all specimens.

<sup>\*\*\*</sup> Respiratory Viruses Panel (Multiplex PCR) will be performed for all specimens RSV-A/B positive and if deemed necessary for RSV-A/B-negative sample.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### 8.11.4.3. Hematology/blood chemistry

Table 14 Hematology/blood chemistry tests

| Blood sampling timepoint Type of contact (timepoint) | Group | No.<br>subjects | Component |
|---|---|---|---|
| Visit 1 (Day 1) | All maternal subjects | ~2300* | Hematology (Leukocytes, Hemoglobin, Platelets)<br>Biochemistry (ALT, AST, Creatinine, blood urea<br>nitrogen) |
| Visit 3 (Day 56) | All maternal subjects | ~2300 | Hematology (Hemoglobin) |

<sup>\* 200</sup> to 300 subjects per country. Tests to be performed preferentially by local healthcare providers and information will be collected and recorded in the eCRF. The investigator/study staff will collect biological samples for the specified testing if not done by the local healthcare provider as per local practice.

## 9. SERIOUS ADVERSE EVENTS RELATED TO STUDY PARTICIPATION

The investigator or site staff is/are responsible for the detection, documentation and reporting of events meeting the SAE definition.

Treatment of any SAE **related to study participation** (e.g., protocol-mandated procedures, invasive tests) is at the sole discretion of the investigator and according to current good medical practice.

#### 9.1. Definition

An SAE **related to study participation** (e.g., protocol-mandated procedures, invasive tests) is any untoward medical occurrence related to study participation that:

- Results in death,
- Is life-threatening,

Note: The term 'life-threatening' in the definition of 'serious' refers to an event in which the subject was at risk of death at the time of the event. It does not refer to an event, which hypothetically might have caused death, had it been more severe.

• Requires hospitalization or prolongation of an existing hospitalization,

Note: In general, hospitalization signifies that the subject has been admitted at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or in an out-patient setting.

Complications that occur during hospitalization are also considered AEs. If a complication prolongs hospitalization or fulfils any other serious criteria, the event will also be considered serious. When in doubt as to whether 'hospitalization' occurred or was necessary, the AE should be considered serious.

Hospitalization for elective treatment of a pre-existing condition (known or diagnosed prior to informed consent signature) that did not worsen from baseline is NOT considered an SAE.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

• Results in disability/incapacity,

Note: The term disability means a substantial disruption of a person's ability to conduct normal life functions. This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhoea, influenza like illness, and accidental trauma (e.g., sprained ankle) which may interfere or prevent everyday life functions but do not constitute a substantial disruption.

Medical or scientific judgement should be exercised in deciding whether reporting is appropriate in other situations, such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardise the subject or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition. These should also be considered serious. Examples of such events are invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization.

#### 9.2. Event Identification

Blood and urine samples will be collected from pregnant women enrolled in the study. Nasal swabs will be collected from neonates/ infants enrolled in the study. Serious adverse events (SAEs) associated with collection of these biological specimens or any other study procedures will be documented and reported from the time the pregnant woman (mother) consents to participate / consents to her infant's participation until the pregnant woman (mother) / her infant is discharged from the study.

Each subject/ subject's parent(s)/ LAR(s) will be instructed to contact the investigator immediately should they/the subject manifest any signs or symptoms they perceive as serious/ of concern or indicating a change in their health status.

## 9.3. Subject cards

Study subjects/parents/LARs must be provided with the address and telephone number of the main contact for information about the clinical study. The investigator (or designate) must therefore provide subjects/parents/LARs with a "subject card."

For this study, a subject card will be provided to each pregnant woman who enrolls. A second subject card will be provided for each infant who is enrolled.

In an emergency situation these cards serve to inform the responsible attending physician(s) that the subject is in a clinical study and that relevant information may be obtained by contacting the investigator.

In a non-emergency situation, if subjects visit a local healthcare provider not affiliated with the study, these cards serve to inform the responsible local healthcare provider that the subject is in a clinical study and that relevant information may be obtained by contacting the investigator. Further, subject will have information on the card to contact the study site at any time.

Subjects/parents/LARs must be instructed to keep the subject cards in their possession at all times during the study.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## 9.4. GSK Contact information, GSK Reporting Timeframes, and Regulatory reporting requirements

Procedure related SAEs that occur during the study will be reported to the GSK representatives specified in Table 15, within the timeframes described in Table 16 once the investigator determines that the event meets the protocol definition provided in the Glossary of Terms.

The investigator will promptly report all SAEs related to study participation to GSK Biologicals as detailed in Table 15 and Table 16. GSK Biologicals has a legal responsibility to promptly notify, as appropriate, both the local regulatory authority and other regulatory agencies (as applicable, per country) about the event. Prompt notification of SAEs by the investigator to the Study Contact for Reporting SAEs is essential so that legal obligations and ethical responsibilities towards the safety of other subjects are met.

Table 15 Contact information for reporting SAEs related to study participation to GSK



Table 16 Timeframes for submitting SAEs related to study participation to GSK

| Type of event | Initial reports | | Follow-up of relevant information on a previous report | |
|---|---|---|---|---|
| | Timeframe | Documents | Timeframe | Documents |
| SAEs related to study | 24 hours**‡ | electronic | 24 hours* | electronic |
| participation | | Expedited Adverse | | Expedited Adverse Event |
| , | | Event Report | | Report |

<sup>\*</sup> Timeframe allowed after receipt or awareness of the information.

## 9.5. Information to be reported

The nature of the SAE, date and time of onset, outcome, intensity and possible relationship to the study procedure(s) should be established and recorded in the eCRF.

Any medication administered for the treatment of the SAE should be recorded in Expedited Adverse Event Report of the subject's eCRF.

<sup>\*\*</sup> Timeframe allowed after the diagnosis is established and known to the investigator.

<sup>&</sup>lt;sup>‡</sup>The investigator will be required to confirm review of the procedure related SAE causality by ticking the 'reviewed' box in the electronic Expedited Adverse Event Report within 72 hours of submission of the procedure related SAE

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

The outcome of the SAE related to study participation should be assessed, as follows:

- Recovered/ resolved.
- Recovering/ resolving.
- Not recovered/ not resolved.
- Recovered with sequelae/ resolved with sequelae.
- Fatal.

## 9.6. SAE Report Completion and transmission to GSK

Once an investigator becomes aware that a study-related SAE has occurred in a study subject, the investigator (or designee) must complete the information in the electronic Expedited Adverse Event Report WITHIN 24 HOURS. The report will always be completed as thoroughly as possible with all available details of the event. Even if the investigator does not have all information regarding an SAE, the report should still be completed within 24 hours. Once additional information is received, the report should be updated WITHIN 24 HOURS.

The investigator will always provide an assessment of causality at the time of the initial report.

## 9.6.1. Back-up system in case the electronic reporting system does not work

If the electronic reporting system does not work, the investigator (or designee) must complete, then date and sign a paper Expedited Adverse Event Report and fax it to the Study Contact for Reporting SAEs (refer to the Sponsor Information) or to the GSK Biologicals Clinical Safety and Pharmacovigilance department within 24 hours.

This back-up system should only be used if the electronic reporting system is not working and NOT if the system is slow. As soon as the electronic reporting system is working again, the investigator (or designee) must complete the electronic Expedited Adverse Event Report within 24 hours. The final valid information for regulatory reporting will be the information reported through the electronic reporting system.

## 9.6.2. Updating of SAE information after removal of write access to the subject's eCRF

When additional SAE information is received after removal of write access to the subject's eCRF, new or updated information should be recorded on a paper Expedited Adverse Event Report, with all changes signed and dated by the investigator. The updated report should be faxed to the GSK Biologicals Clinical Safety and Pharmacovigilance department or to the Study Contact for Reporting SAEs (see the Sponsor Information) within the designated reporting time frames specified in Table 16.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## 9.7. Follow-up of SAEs related to study participation (Amended 29-MAY-2020)

The investigator will follow-up subjects with SAEs related to study participation until the event has resolved, subsided, *stabilized*, disappeared, or until the event is otherwise explained, or the subject is lost to follow-up.

## 9.7.1. Follow-up during the study

After the initial SAE report, the investigator is required to proactively follow each subject and provide further relevant information on the subject's condition to GSK Biologicals (within 24 hours for SAEs, refer to Table 16).

All SAEs documented at a previous visit/ contact and recorded as not recovered/ not resolved or recovering/ resolving will be reviewed at subsequent visits/ contacts until the last visit of the subject.

## 9.7.2. Follow-up after the subject is discharged from the study (Amended 29-MAY-2020)

If the investigator receives additional relevant information on a previously reported SAE, he/ she will provide this information to GSK Biologicals using a paper Expedited Adverse Event Report.

GSK Biologicals may request that the investigator performs or arranges for the conduct of additional clinical examinations/ tests and/ or evaluations to elucidate as fully as possible the nature and/ or causality of the SAE. The investigator is obliged to assist. If a subject dies during participation in the study or during a *recognized* follow-up period, GSK Biologicals will be provided with any available post-mortem findings, including histopathology.

#### 10. SUBJECT COMPLETION AND WITHDRAWAL

## 10.1. Subject completion

A subject who returns for the concluding visit foreseen in the protocol is considered to have completed the study.

## 10.2. Subject withdrawal

Subjects who are withdrawn because of an event of interest or SAEs related to study participation must be clearly distinguished from subjects who are withdrawn for other reasons. The investigator will follow subjects who are withdrawn as the result of an SAE related to study participation until resolution of the event (see Section 9.7.2).

Withdrawals will not be replaced.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

From an analysis perspective, a 'withdrawal' from the study refers to any subject who did not come back for the concluding visit in the protocol.

All data collected until the date of withdrawal/last contact of the subject will be used for the analysis.

A subject is considered a 'withdrawal' from the study when no study procedure has occurred, no follow-up has been performed and no further information has been collected for this subject from the date of withdrawal/last contact.

Investigators will make at least 3 attempts to contact a subject who does not return for a scheduled visit as described in Section 8.4 and in the SPM.

A subject will be defined as lost to follow-up if there is no contact with the subject /subject's parent(s) / LAR(s) over a period of at least 3 months after a planned visit (see SPM for details). Efforts to contact the subject/subject's parents should be recorded in the source documents. The subject's data will be censored at the time of last contact once this definition is met.

Information relevant to the withdrawal will be documented in the eCRF. The investigator will document whether the decision to withdraw a subject from the study was made by the subject herself, by the subject's parent(s) or LAR(s), or by the investigator, as well as which of the following possible reasons was responsible for withdrawal:

- Study participation related SAE.
- Pregnancy related event of interest(specify). Note: includes maternal deaths.
- Maternal deaths not related to pregnancy/delivery (specify cause).
- Neonatal event of interest(specify). Note: includes death in infants from birth 28 days old
- Death in infants > 28 days old (specify cause). Note that death in neonates from birth
   28 days old is captured as a neonatal event of interest).
- Protocol violation (specify).
- Consent withdrawal\*.
- Moved from the study area.
- Lost to follow-up.
- Other (specify).

\*In case a subject is withdrawn from the study because she/the subject's parent(s)/ LAR(s) has withdrawn consent, the investigator will document the reason for withdrawal of consent, if specified by the subject/ the subject's parent(s)/LAR(s), in the CRF.

Subjects who are withdrawn from the study because of study participation related SAEs must be clearly distinguished from subjects who are withdrawn for other reasons. Investigators will follow subjects who are withdrawn from the study as result of a study participation related SAE until resolution of the event (see Section 9.7.2).

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## 11. STATISTICAL METHODS

The primary analysis will be performed by country and possibly by region or other relevant grouping if standard of antenatal care is similar in the different sites. This will be determined during site selection when more information is available.

## 11.1. Endpoints

## 11.1.1. Primary endpoints

## 11.1.1.1. Pregnancy outcomes.

These include:

- Live birth with no congenital anomalies,
- Live birth with congenital anomalies,
- Fetal death/stillbirth (loss at or after 22 weeks of gestation) with no congenital anomalies.
  - Antepartum stillbirth
  - Intrapartum stillbirth
- Fetal death/still birth (loss at or after 22 weeks of gestation) with congenital anomalies.
  - Antepartum stillbirth
  - Intrapartum stillbirth
- Elective/therapeutic termination with no congenital anomalies,
- Elective/therapeutic termination with congenital anomalies.
- Of note, fetal death/stillbirth has multiple subcategories. For example, fetal death/stillbirth with no congenital anomalies is an outcome with two subcategories that include: 1) antepartum stillbirth; 2) intrapartum stillbirth. For each outcome, the investigator should select the applicable sub-category.

#### 11.1.1.2. Pregnancy related events of interest from Visit 1 through Visit 6.

Although pregnancy related events of interest occur within the first 42 days after delivery they may only be detected later, and are to be reported throughout the study. They are listed below. Of note, some events of interest fall under a single category but have multiple subcategories. For example, hypertensive disorders of pregnancy is an event with three subcategories that include: 1) gestational hypertension; 2) pre-eclampsia; and 3) pre-eclampsia with severe features (including eclampsia). For each event, the investigator should select the event and the applicable sub-category.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- Maternal death
- Hypertensive disorders of pregnancy:
  - Gestational hypertension,
  - Pre-eclampsia,
  - Pre-eclampsia with severe features (including eclampsia)
- Antenatal bleeding:
  - Morbidly adherent placenta
  - Placental abruption
  - Cesarean Scar Pregnancy
  - Uterine rupture
- Postpartum hemorrhage
- Fetal growth restriction
- Dysfunctional labor
  - first stage of labor
  - second stage of labor
- Gestational diabetes mellitus,
- Non reassuring fetal status
- Pathways to preterm birth:
  - Premature preterm rupture of membranes,
  - Preterm labor,
  - Provider-initiated preterm birth.
- Chorioamnionitis
- Oligohydramnios
- Polyhydramnios
- Gestational Liver Disease:
  - Intrahepatic Cholestasis of Pregnancy (ICP)
  - Acute Fatty Liver of Pregnancy
- Maternal Sepsis
- Any other pregnancy related event considered by the investigator to be of concern (specify)

For events of interest that include subcategories, the frequency of the main event of interest and of each event subcategory will be included in the analysis. The overall frequency will include mothers who present with at least one of the subcategory events.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## 11.1.1.3. Neonatal events of interest from birth through 28 days of age

Neonatal events of interest occur within the first 28 days after birth, but may only be detected later and are to be reported throughout the study. They include:

- Small for gestational age,
- Low birth weight including very low birth weight,
- Neonatal encephalopathy,
- Congenital microcephaly,
  - Postnatally diagnosed
  - Prenatally diagnosed
- Congenital anomalies,
  - Major external structural defects
  - Internal structural defects
  - Functional defects
- Neonatal death,
  - Neonatal death in a preterm live birth (gestational age>=28 to < 37 weeks)</li>
  - Neonatal death in a term live birth
- Neonatal infections,
  - Blood stream infections
  - Meningitis
  - Respiratory infection
- Respiratory distress in the neonate,
- Preterm birth,
- Failure to thrive,
- Large for gestational age,
- Macrosomia,
- Any other neonatal event considered by the investigator to be of concern (specify, e.g. neurodevelopment delay)

For events of interest that include subcategories, the frequency of the main event of interest and of each event subcategory will be included in the analysis. The overall frequency will include infants who present at least one of the subcategory events.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

### 11.1.2. Secondary endpoints

- Pregnancy related events of interest from Visit 1 through Visit 6 (as defined in primary endpoints) for each GAIA level of diagnostic certainty (where applicable and feasible).
- Neonatal events of interest from birth through 28 days of age (as defined in primary endpoints) for each GAIA level of diagnostic certainty (where applicable and feasible).

Of note, some events of interest fall under a single category but have multiple subcategories. For each event, the investigator should identify the event and select the applicable sub-category and the GAIA level of diagnostic certainty.

- RSV-A neutralizing antibody titers in maternal blood at delivery
- RSV-A neutralizing antibody titers in cord blood at delivery.
- Episode(s) of RSV-LRTI from birth up to 1 year of age.
- Episode(s) of RSV hospitalization from birth up to 1 year of age.

### 11.1.3. Tertiary endpoints (Amended 29-MAY-2020)

- Co-infections of RSV-LRTI with other respiratory viruses in infants, confirmed by PCR of nasal swabs in infants from birth up to 1 year of age:
  - Influenza A virus (Flu A)
  - Influenza B virus (Flu B)
  - Human Influenza A virus subtype H1 (Flu A-H1)
  - Human Influenza A virus subtype H3 (Flu A-H3)
  - Human Influenza A virus subtype H1pdm09 (Flu A-H1pdm09)
  - Human adenovirus (AdV)
  - Human metapneumovirus (MPV)
  - Human enterovirus (HEV)
  - Human parainfluenza virus 1 (PIV1)
  - Human parainfluenza virus 2 (PIV2)
  - Human parainfluenza virus 3 (PIV3)
  - Human parainfluenza virus 4 (PIV4)
  - Human bocavirus 1/2/3/4 (HBoV)
  - Human rhinovirus A/B/C (HRV)
  - Human coronavirus 229E (229E)
  - Human coronavirus NL63 (NL63)
  - Human coronavirus OC43 (OC43)

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- Potential risk factors for pregnancy related and neonatal events of interest.
- Any further exploratory characterization of immune responses to RSV and/or other respiratory tract infections or infections of relevance to pregnant women and their newborns (based on maternal serum and cord blood) (For example, levels of RSV-B neutralizing antibodies.)
- Episode(s) of RSV-LRTI/severe LRTI based on alternative case definitions, from birth up to 1 year of age.

## 11.2. Determination of sample size

The target will be to enroll up to approximately 200 to 300 eligible subjects (pregnant women) by country. Subjects may drop-out from the study due to a variety of reasons, e.g. migration from the study area. Assuming a drop-out rate of about 10% during the course of follow-up, there will be up to approximately 180 to 270 evaluable subjects by country.

Considering a sample size of up to approximately 180 to 270 evaluable subjects by country, Table 17 illustrates the precision (exact 95% confidence interval [CI]) one can get on the percentage of subjects with maternal, fetal and neonatal events of interest. Precision (exact 95% CI) has also been computed for a sample size of 270, 180 and 100 evaluable subjects for estimate by study site.

The percentages of subjects with maternal, fetal and neonatal events of interest for the primary objectives are expected to range from 0 to 35%.

Table 17 Precision (exact 95% confidence interval) on the percentage of subjects with maternal, fetal and neonatal events of interest for sample size of 270, 180 and 100 subjects

| | 270 subje | ects | | 180 subje | ects | | 100 subje | cts | |
|---|---|---|---|---|---|---|---|---|---|
| % | N | Lower | Upper | N | Lower | Upper | N | Lower | Upper |
| | | limit | limit | | limit | limit | | limit | limit |
| 35 | 94.5 | 29.3 | 41 | 63 | 28.1 | 42.4 | 35 | 25.7 | 45.2 |
| 30 | 81 | 24.6 | 35.8 | 54 | 23.4 | 37.3 | 30 | 21.2 | 40 |
| 25 | 67.5 | 19.9 | 30.6 | 45 | 18.9 | 32 | 25 | 16.9 | 34.7 |
| 20 | 54 | 15.4 | 25.3 | 36 | 14.4 | 26.6 | 20 | 12.7 | 29.2 |
| 15 | 40.5 | 11 | 19.8 | 27 | 10.1 | 21.1 | 15 | 8.6 | 23.5 |
| 10 | 27 | 6.7 | 14.2 | 18 | 6 | 15.3 | 10 | 4.9 | 17.6 |
| 5 | 13.5 | 2.7 | 8.3 | 9 | 2.3 | 9.3 | 5 | 1.6 | 11.3 |
| 3 | 8.1 | 1.3 | 5.8 | 5.4 | 1 | 6.8 | 3 | 0.6 | 8.5 |
| 1 | 2.7 | 0.2 | 3.1 | 1.8 | 0.1 | 3.9 | 1 | 0 | 5.4 |
| 0 | 0 | 0 | 1.4 | 0 | 0 | 2 | 0 | 0 | 3.6 |

%= Percentage of subjects with maternal, fetal and neonatal events of interest

N= Number of subjects with maternal, fetal and neonatal events of interest

Lower and upper limits are exact 95% confidence intervals

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## 11.3. Cohorts for Analyses (Amended 29-MAY-2020)

### 11.3.1. Exposed Sets (ES)

#### 11.3.1.1. Pregnant women (mothers)

The ES will include all pregnant women (mothers) who signed a valid informed consent form.

#### 11.3.1.2. Neonates/Infants

Not applicable.

#### 11.3.2. Enrolled sets

#### 11.3.2.1. Pregnant women (mothers)

The enrolled set will include all pregnant women (mothers) with a valid informed consent who completed Visit 1.

#### 11.3.2.2. Neonates/Infants

#### The Enrolled Set will include all neonates/infants

- born to pregnant women in the enrolled set, and
- Who have a valid ICF signed by the mother/ parent(s) /LAR(s) (as appropriate per local regulations).

## 11.3.3. Per Protocol Sets (PPS) (Amended 29-MAY-2020)

#### 11.3.3.1. Pregnant women (mothers)

The maternal PPS will include all pregnant women (mothers) *in the enrolled set who* meet all eligibility criteria up to the time of their censoring, either at study completion or prematurely as drop-out (e.g. withdrawn consent, lost-to-follow-up).

#### 11.3.3.2. Neonates/Infants

The infant PPS will include all neonates / infants

- born to pregnant women in the PPS and
- **who** meet all eligibility criteria up to the time of their censoring, either at study completion or prematurely as drop-out (e.g. withdrawn consent, lost-to-follow-up) who have at least one time point evaluation (see Table 5).

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### 11.4. Derived and transformed data

Age of the infant subject at time of the LRTI case will be expressed in months and will be computed as the difference between the start date of the LRTI case and the date of birth.

Age of the mother at the time of childbirth will be expressed in years and will be computed as the difference between the birth date of the subject and the birth date of the mother.

Duration of the study for each subject will be computed as the difference between the date of last contact (i.e., active or passive surveillance contact or the date of the censoring) and the date when ICF was first signed by the subject / subject's parent[s]/LAR[s]).

All potential LRTI cases identified during the surveillance period will be classified as RTI, LRTI or severe LRTI according to the LRTI case definition and severity scale (refer to Table 3). The cases will also be classified according to the classification of WHO [Modjarrad, 2016].

### 11.4.1. Handling of missing values/censoring/discontinuations

For a given subject and a given demographic variable, missing measurements will not be replaced.

The number of missing values per variable may be provided for selected variables of interest as a separate category. Missing values will be examined to help determine if it is necessary to use multiple imputation or other techniques to deal with missing data.

## 11.5. Analysis of demographic and baseline characteristics

For the maternal PPS cohort, analyses of demographic and baseline characteristics at Visit 1 will be described.

For the infant PPS cohort, analyses of demographic characteristics at Visit 1-NB will be described. Analyses of lifestyle characteristics will be described at Visit 2 NB.

For Screening Failures, reasons for non-eligibility will be described.

Continuous variables will be summarized by providing the number of observations, mean, 95% confidence interval (CI), standard deviation (SD), median, and range. Categorical variables will be summarized by tabulating counts (N) and the percentage (%) of total subjects having the given characteristics, with missing data considered a separate category.

## 11.6. Analysis of primary objectives (Amended 29 May 2020)

The primary objectives analyses will be performed on the PPS cohorts overall and possibly by region or other relevant grouping. If there is a difference of 5% or more between the number of participants in the enrolled set and the PPS, primary objectives analyses on the enrolled set will also be performed.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### In healthy pregnant women with uncomplicated pregnancies at time of enrollment:

• To determine the frequencies of pregnancy outcomes.

The number and percentage (with exact 95% CI) of women presenting the following outcomes: live birth, fetal death/stillbirth (antepartum or intrapartum), and elective/therapeutic termination will be reported for each event by presence or absence of congenital anomalies.

• To determine the frequencies of pregnancy related events of interest as specified in Section 11.1.1.2.

The number and percentage (with exact 95% CI) of pregnant women presenting with the events of interest specified in Section 11.1.1.2 will be tabulated for each event within appropriate time windows to be specified in the statistical analysis plan (SAP). Missing data may be considered a separate category.

#### In all neonates live-born to women enrolled in the study:

• To determine the frequencies of neonatal events of interest. as specified in Section 11.1.1.3.

The number and percentage (with exact 95% CI) of neonates presenting the events of interest specified in Section 11.1.1.3 will be tabulated for each event. Missing data may be considered a separate category.

## 11.7. Analysis of secondary objectives (Amended 29-MAY-2020)

The secondary objectives analyses will be performed on the PPS cohorts (maternal or infant as applicable) overall and possibly by region or other relevant grouping. *If there is a difference of 5% or more between the number of participants in the enrolled set and the PPS, secondary objectives analyses on the enrolled set will also be performed.* 

#### In healthy pregnant women with uncomplicated pregnancies at time of enrollment:

- To determine frequencies of pregnancy related events of interest according to GAIA levels of diagnostic certainty (where these are specified) (APPENDIX D)
  - Considering all pregnant women followed from enrollment through Visit 6, the number and percentage of subjects with at least one maternal event of interest will be computed by GAIA levels of diagnostic certainty, with exact 95% CI.
- To describe the distribution of RSV-A antibody titers in maternal blood at delivery.
  - Geometric mean titers (GMTs) will be tabulated with 95% CI.
  - Percentage of subjects above thresholds will be tabulated.

#### In all neonates live-born to women enrolled in the study:

- To determine frequencies of neonatal events of interest according to GAIA levels of diagnostic certainty (where these are specified). (APPENDIX D)
  - Considering all neonates the number and percentage of subjects with at least one neonatal event of interest will be computed by GAIA levels of diagnostic certainty, with exact 95% CI.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- To describe the distribution of RSV-A antibody titers in cord blood at delivery.
  - Geometric mean titers (GMTs) will be tabulated with 95% CI.
  - Percentage of subjects above thresholds will be tabulated.

## In all neonates/infants live-born to women enrolled in the study:

- To determine the incidence of all, of severe, and of very severe RSV-lower respiratory tract illnesses (LRTIs).
  - Considering all infants followed from visit 1-NB to visit 4-NB, the percentage of subjects with at least one LRTI illness, exact 95% CI will be presented.
  - Incidence rates of LRTI illnesses will be calculated, with exact 95% CI.
  - Frequencies of repeat occurrences of LRTI will be tabulated.
- To determine the incidence of RSV hospitalization.
  - Considering all infants followed from visit 1-NB to visit 4-NB, the percentage of subjects with at least one RSV hospitalization, with exact 95% CI.
  - Incidence rates of RSV hospitalizations will be calculated, with exact 95% CI.
  - Frequencies of repeat occurrences of RSV hospitalization will be tabulated.

Continuous variables will be summarized by providing the number of observations, mean, 95% CI, SD, median, and range. Categorical variables will be summarized by tabulating N and % of total subjects having the given characteristics, with missing data considered a separate category.

## 11.8. Analysis of tertiary objectives (Amended 29-MAY-2020)

The following tertiary objectives analyses will be performed on infants within the PPS cohort, overall and possibly by region or other relevant grouping. *If there is difference of 5% or more between the number of participants in the enrolled set and the PPS, tertiary objectives analyses on the enrolled set will also be performed.* 

- To describe co-infections of RSV-LRTI with other respiratory viruses in infants.
  - Considering all infants followed from visit 1-NB to visit 4-NB, the percentage
    of subjects with the occurrence of RSV-LRTI and having other respiratory viral
    co- infection identified by multiplex PCR, with exact 95% CI; classified by
    respiratory viruses.
- To estimate the association of RSV-LRTI in neonates/infants and the level of RSV neutralizing antibodies in cord blood.
  - Correlation analysis will be done comparing the levels of RSV antibodies
    present in cord blood and the presence or absence of RSV-associated LRTI,
    RSV-associated severe LRTI, and RSV-associated very severe LRTI in infants.
    Details will be described in the SAP.

The following tertiary objectives analyses will be performed on the PPS cohorts (maternal or infant as applicable) by country, region, or other relevant grouping:

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- To determine risk factors for pregnancy-related and neonatal events of interest.
  - Risk factors will be described in the SAP.
  - The maternal events of interest will be described according to variables collected in the mother's clinical examination and obstetric risk factors.
     Frequency tables will be generated for categorical variables.
  - The neonatal events of interest will be described according to variables collected in the mother's clinical examination and obstetric risk factors. Frequency tables will be generated for categorical variables.
  - Furthermore, multiple variable analyses (such as multiple logistic regression for binary outcomes and multiple Poisson/negative binomial and/or other appropriate models for count outcomes) will be conducted to adjust for covariates of interest, provided there are sufficient numbers of events of interest.
- To determine the incidence of LRTIs/Severe LRTIs (using alternative case definitions)
- If deemed necessary, to further characterize the immune responses to RSV and other infections in maternal subjects and infants (based on maternal serum and cord blood).
  - For example, for levels of neutralizing antibodies to RSV-B:
    - o GMTs/ GMCs may be tabulated with 95% CI.
    - Percentage of subjects above various thresholds, depending on the antibody tested, may be tabulated with exact 95% CI.
    - Other relevant exploratory analyses may be defined in the SAP.

## 11.9. Interpretation of analyses

Analyses will be descriptive with the aim to characterize different sub-groups of women. These sub-groups will be defined prior to analyses and will be related to e.g. risk factors for maternal and neonatal events of interest and endemic disease. These descriptive analyses should be interpreted with caution considering that there is no adjustment for multiplicity for these comparisons.

Further details will be provided in the SAP.

## 11.10. Analysis of safety

Serious adverse events (SAEs) related to study participation will be recorded throughout the study period. In case of occurrence of SAE(s) related to study participation, a listing of SAEs will be provided.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## 11.11. Conduct of analyses

All analyses will be done on cleaned data.

Analyses will be performed in a stepwise manner after all subjects in all countries have completed all study visits in Epoch 002 and again after completion of all study visits in Epoch 003.

Analyses of pregnancy outcomes, pregnancy related events of interest, and neonatal events of interest will be performed when all data up to 42 days post-delivery are available (Epoch 002). For these analyses a statistical report but no CSR will be prepared.

Final analyses will be performed when all data up to study end are available (Epoch 002 and Epoch 003). An integrated *CSR* including all available data will be written and made available to the investigator(s).

If the data for tertiary endpoints become available at a later stage, additional analysis/analyses will be performed. These data will be documented in annex(es) to the study report and made available to the investigators.

Additional analyses may be performed if deemed necessary to inform the design or implementation of future clinical trials.

Analyses, and the sequence in which they will occur, will be described in detail in the SAP.

Any deviation(s) or change(s) from the original statistical plan outlined in this protocol will be described and justified in the final study report.

## 11.11.1. Statistical considerations for interim analyses (Amended 29-MAY-2020)

### **Interim analysis for RSV LRTIs**

If deemed necessary, an interim analysis may be performed on RSV surveillance data as part of the secondary objective of determining incidence of RSV LRTI. This interim analysis may be performed to obtain preliminary information on the performance of the case definitions used for RSV LRTI, severe LRTI, and very severe LRTI (Table 3) and to assess levels of RSV neutralising antibody in maternal and cord blood at delivery. The interim analysis may occur after the database freeze at the time point when approximately 50% of infants will have completed up to 6 months of follow up during the surveillance period following birth (up to Visit 3-NB). If an interim analysis is performed, data cleaning plans will be scheduled as needed to supply data for interim analyses in a timely manner. This interim analysis may be performed on data that is as clean as possible. Preliminary results will be made available in a timely manner for use in the potential adjustment of the RSV LRTI case definitions to be used in pivotal clinical trials scheduled to begin shortly thereafter. The results pertaining to this analysis (if performed) will be purely descriptive, with no adjustment of type I error, and will be reported in an interim statistical report. No CSR will be prepared.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### 12. ADMINISTRATIVE MATTERS

To comply with ICH GCP administrative obligations relating to data collection, monitoring, archiving data, audits, confidentiality, ownership, public disclosure requirements and publications must be met.

## 12.1. Electronic Case Report Form instructions

A validated GSK defined electronic data collection tool will be used as the method for data collection.

In all cases, subject initials will not be collected nor transmitted to GSK. Subject data necessary for analysis and reporting will be entered/transmitted into a validated database or data system. Clinical data management will be performed in accordance with applicable GSK standards and data cleaning procedures.

While completed eCRFs are reviewed by a GSK Biologicals' Site Monitor at the study site, omissions or inconsistencies detected by subsequent eCRF review may necessitate clarification or correction of omissions or inconsistencies with documentation and approval by the investigator or appropriately qualified designee. In all cases, the investigator remains accountable for the study data.

## 12.2. Study monitoring by GSK Biologicals

GSK will monitor the study to verify that, amongst other items, the:

- Data are authentic, accurate, and complete.
- Safety and rights of subjects are being protected.
- Study is conducted in accordance with the currently approved protocol, any other study agreements, GCP and all applicable regulatory requirements.

The investigator and the head of the medical institution (where applicable) agrees to allow the monitor direct access to all relevant documents.

The investigator must ensure provision of reasonable time, space and qualified personnel for monitoring visits.

Direct access to all study-site related and source data is mandatory for the purpose of monitoring review. The monitor will perform an eCRF review and a Source Document Verification (SDV). By SDV we understand verifying eCRF entries by comparing them with the source data that will be made available by the investigator for this purpose.

The Source Documentation Agreement Form describes the source data for the different data in the eCRF. This document should be completed and signed by the site monitor and investigator and should be filed in the investigator's study file. Any data item for which the eCRF will serve as the source must be identified, agreed and documented in the source documentation agreement form.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Upon completion or premature discontinuation of the study, the monitor will conduct site closure activities with the investigator or site staff, as appropriate, in accordance with applicable regulations, GCP, and GSK procedures.

## 12.3. Study and site closure

GSK or its designee reserves the right to close the study site or terminate the study at any time for any reason at the sole discretion of GSK, provided there is sufficient notice given to account for patient's safe exit from study participation. Study sites regular closure will be upon study completion. A study site is considered closed when all required data/documents and study supplies have been collected and a study-site closure visit has been performed.

The investigator may initiate study-site closure at any time, provided there is reasonable cause and sufficient notice is given in advance of the intended termination.

Reasons for the early closure of a study site by the sponsor or investigator may include but are not limited to:

- Failure of the investigator to comply with the protocol, the requirements of the IRB/IEC or local health authorities, the sponsor's procedures, or GCP guidelines
- Inadequate recruitment of subjects by the investigator
- Discontinuation of further study treatment development

#### 12.4. Record retention

Following closure of the study, the investigator must maintain all site study records (except for those required by local regulations to be maintained elsewhere) in a safe and secure location. The records must be easily accessible, when needed (e.g., audit or inspection), and must be available for review in conjunction with assessment of the facility, supporting systems, and staff. Where permitted by applicable laws/regulations or institutional policy, some or all of these records can be maintained in a validated format other than hard copy (e.g., microfiche, scanned, electronic); however, caution needs to be exercised before such action is taken. The investigator must ensure that all reproductions are legible and are a true and accurate copy of the original and meet accessibility and retrieval standards, including re-generating a hard copy, if required. Furthermore, the investigator must ensure that an acceptable back-up of the reproductions exists and that there is an acceptable quality control procedure in place for making these reproductions.

GSK will inform the investigator/institution of the time period for retaining these records to comply with all applicable regulatory requirements. The minimum retention time will meet the strictest standard applicable to a particular site, as dictated by ICH GCP any institutional requirements or applicable laws or regulations, or GSK standards/procedures otherwise, the minimum retention period will default to 25 years after completion of the study report.

The investigator/institution must notify GSK of any changes in the archival arrangements, including, but not limited to, archival at an off-site facility and transfer of ownership of the records in the event the investigator leaves the site.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## 12.5. Quality assurance

To ensure compliance with GCP and all applicable regulatory requirements, GSK may conduct a quality assurance audit. Regulatory agencies may also conduct a regulatory inspection of this study. Such audits/inspections can occur at any time during or after completion of the study. If an audit or inspection occurs, the investigator and institution agree to allow the auditor/inspector direct access to all relevant documents and to allocate his/her time and the time of his/her staff to the auditor/inspector to discuss findings and any relevant issues.

## 12.6. Posting of information on publicly available registers and publication policy

GSK assures that the key design elements of this protocol will be posted on the GSK website and in publicly accessible database(s) such as clinicaltrials.gov, in compliance with the current regulations.

GSK also assures that results of this study will be posted on the GSK website and in publicly accessible regulatory registry(ies) within the required time-frame, in compliance with the current regulations.

Studies that do not evaluate vaccines/products are progressed for publication in the scientific literature when the results provide important scientific or medical knowledge or are relevant for patient care, and will be considered for disclosure on the GSK website and in publicly accessible regulatory registry(ies).

## 12.7. Provision of study results to investigators

Where required by applicable regulatory requirements, an investigator signatory will be identified for the approval of the study report. The investigator will be provided reasonable access to statistical tables, figures, and relevant reports and will have the opportunity to review the complete study results at a GSK Biologicals site or other mutually-agreed location.

GSK Biologicals will also provide the investigator with the full summary of the study results. The investigator is encouraged to share the summary results with the study subjects, as appropriate.

## 12.8. Data Sharing

Under the framework of the SHARE initiative, results of GSK studies may be combined with non- GSK studies, to investigate further about the study product(s) and other product(s), and /or the disease/condition under investigation and related diseases and conditions.

### 13. COUNTRY SPECIFIC REQUIREMENTS

Not applicable.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## 14. REFERENCES (AMENDED 29-MAY-2020)

Barbas CF, Crowe JE, Cababa D, et al. Human monoclonal Fab fragments derived from a combinatorial library bind to respiratory syncytial virus F glycoprotein and neutralize infectivity. Proc Natl Acad Sci U S A. 1992;89(21):10164-8.

Bates JT, Keefer CJ, Slaughter JC, et al. Escape from neutralization by the respiratory syncytial virus-specific neutralizing monoclonal antibody palivizumab is driven by changes in on-rate of binding to the fusion protein. Virology. 2014; 454-455:139-144.

Bauwens J, Bonhoeffer J, Chen RT, editors. Harmonising Immunisation Safety Assessment in Pregnancy. Vaccine. 2016. 34 (49): 5991 – 6110.

Bonhoeffer J, Kochhar S, Hirschfeld S, et al. Global alignment of immunization safety assessment in pregnancy - The GAIA project. Vaccine. 2016;34(49):5993-5997. doi: 10.1016/j.vaccine.2016.07.006.

Boyce TG, Mellen BG, Mitchel EF Jr *et al.* Rates of hospitalization for respiratory syncytial virus infection among children in medicaid. *J. Pediatr.* 2000; 137: 865-70.

Centers for Disease Control and Prevention (CDC). Updated recommendations for use of tetanus toxoid, reduced diphtheria toxoid, and acellular pertussis vaccine (Tdap) in pregnant women. Advisory Committee on Immunization Practices (ACIP) - 2012. MMWR. 2013a; 62 (7):131-135.

Centers for Disease Control and Prevention (CDC). Influenza Vaccination Coverage Among Pregnant Women — United States, 2012–13 Influenza Season. MMWR. \_2013b; 62 (38): 787–792.

Deshpande SA and Northern V. The clinical and health economic burden of respiratory syncytial virus disease among children under 2 years of age in a defined geographical area. *Arch. Dis. Child.* 2003; 88: 1065-9.

Hall CB, Weinberg GA, Iwane MK, et al. The Burden of Respiratory Syncytial Virus Infection in Young Children. N Engl J Med. 2009; 360:588-98.

Holman RC, Curns AT, Cheek JE *et al*. Respiratory syncytial virus hospitalizations among American Indian and Alaska Native infants and the general United States infant population. *Pediatrics*. 2004; 114: e437-44.

Iwane MK, Edwards KM, Szilagyi PG *et al.* Population-based surveillance for hospitalizations associated with respiratory syncytial virus, influenza virus, and parainfluenza viruses among young children. *Pediatrics*. 2004; 113: 1758-64.

Jones CE, Munoz FM, Kochhar S et al. Guidance for the collection of case report form variables to assess safety in clinical trials of vaccines in pregnancy. Vaccine. 2016; 34(49):6007-6014.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Kochhar S, Bauwens J, Bonhoeffer J, editors. Harmonising Immunization Safety Assessment in Pregnancy – Part II. Vaccine. 2017. 35 (48): 6469-6582.

Modjarrad K, Giersing B, Kaslow DC, Smith PG, Moorthy VS; WHO RSV Vaccine Consultation Expert Group. WHO consultation on Respiratory Syncytial Virus Vaccine Development Report from a World Health Organization Meeting held on 23-24 March 2015. Vaccine. 2016;34(2):190-7.

Nair H, Nokes JD, Gessner BD, *et al*. Global burden of acute lower respiratory infections due to respiratory syncytial virus in young children: a systematic review and meta-analysis. *Lancet*. 2010; 375:1545-55.

Vicente D, Montes M, Cilla G et al. Hospitalization for respiratory syncytial virus in the paediatric population in Spain. *Epidemiol. Infect.* 2003; 131: 867-72.

World Health Organization (WHO). WHO recommendations on antenatal care for a positive pregnancy experience. Published in 2016. http://www.who.int/reproductivehealth/publications/maternal\_perinatal\_health/anc-positive-pregnancy-experience/en. Last accessed on 09 February 2017.

World Health Organization [WHO]. Global Surveillance for COVID-19 caused by human infection with COVID-19 virus: Interim Guidance. March 2020. Available at: https://apps.who.int/iris/rest/bitstreams/1272502/retrieve. Accessed 8 May 2020.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## APPENDIX A LABORATORY ASSAYS

Assay descriptions could be subjects to change, due to assay re-development and/or qualification.

### **Neutralization assay**

The serum neutralization assay is a functional assay that measures the ability of serum antibodies to neutralize RSV entry and replication in a host cell line.

Virus neutralization is performed by incubating a fixed amount of RSV-A strain (Long, ATCC No. VR-26) or RSV-B strain (18537, ATCC No. VR-1580) with serial dilutions of the test serum. The serum-virus mixture is then transferred onto a monolayer of Vero cells (African Green Monkey, kidney, Cercopitheus aethiops, ATCC CCL-81) and incubated for three days to allow infection of the Vero cells by non-neutralized virus and the formation of plaques in the cell monolayer. Following a fixation step, RSV-infected cells are detected using a primary antibody directed against RSV (anti-RSV IgG) and a secondary antibody conjugated to horse-radish peroxidase (HRP), allowing the visualization of plagues by immunofluorescence after coloration with TrueBlueTM peroxidase substrate. Viral plaques are counted using an automated microscope coupled to an image analyzer (Scanlab system with Axiovision software). For each serum dilution, a ratio, expressed as a percentage, is calculated between the number of plaques at that dilution and the number of plagues in the virus control wells (no serum added). The serum neutralizing antibody titer is expressed in ED60 (Estimated Dilution 60) and corresponds to the inverse of the interpolated serum dilution that yields a 60% reduction in the number of plagues compared to the virus control wells, as described by others [Barbas, 1992; Bates, 2014].

#### **PCR**

• Quantitative RT-PCR able to discriminate RSV-A and RSV-B subtypes:

Briefly, RSV A and RSV B RNAs extracted from the nasal swabs are detected in a duplex PCR format using specific amplification primers and fluorescent probes designed in the RSV N gene, encoding the RSV nucleocapsid protein. The process involves nucleic acids extraction, conversion of RNA to complementary deoxyribonucleic acid by reverse transcription and detection by real- time PCR reaction using a calibration curve (absolute quantitation). The RSV viral load is reported as copies of RSV RNA per mL of sample.

• Oualitative multiplex RT-PCR for detection of a panel of viruses.

A qualitative RT-PCR multiplex assay is used for the detection and identification of multiple respiratory virus nucleic acids in nasal swabs from individuals suspected of respiratory tract infections. The following virus types and subtypes can be identified in the assay:

- Influenza A virus (Flu A)
- Influenza B virus (Flu B)

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- Human Influenza A virus subtype H1 (Flu A-H1)
- Human Influenza A virus subtype H3 (Flu A-H3)
- Human Influenza A virus subtype H1pdm09 (Flu A-H1pdm09)
- Human respiratory syncytial virus A (RSV A)
- Human respiratory syncytial virus B (RSV B)
- Human adenovirus (AdV)
- Human metapneumovirus (MPV)
- Human enterovirus (HEV)
- Human parainfluenza virus 1 (PIV1)
- Human parainfluenza virus 2 (PIV2)
- Human parainfluenza virus 3 (PIV3)
- Human parainfluenza virus 4 (PIV4)
- Human bocavirus 1/2/3/4 (HBoV)
- Human rhinovirus A/B/C (HRV)
- Human coronavirus 229E (229E)
- Human coronavirus NL63 (NL63)
- Human coronavirus OC43 (OC43)

Following total nucleic acids extraction, viruses are detected by multiplex real-time RT-PCR assays targeting the above mentioned viruses. A comparative analysis of the fluorescence intensities of each target is performed to detect the viruses present in the sample.

## APPENDIX B CLINICAL LABORATORIES

Table 18 GSK Biologicals' laboratories

| Laboratory | Address |
|---|---|
| GSK Biologicals Clinical Laboratory | Biospecimen Reception - B7/44 |
| Sciences, Rixensart | Rue de l'Institut, 89 - B-1330 Rixensart – Belgium |
| | Avenue Fleming, 20 - B-1300 Wavre - Belgium |
| Sciences, Wavre-Nord Noir Epine | |
| GSK Vaccines GmbH | Emil-von-Behring-Str. 76 |
| Clinical Laboratory Sciences, | 35041 Marburg |
| Marburg, Germany | Germany |

#### Table 19 Outsourced laboratories

| Laboratory | Address |
|--------------------------------|-----------------------|
| DDL Diagnostic Laboratory B.V. | Headquarters |
| | Visseringlaan, 25 |
| | 2288 ER Rijswijk - NL |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## APPENDIX C GAIA GESTATIONAL AGE ASSESSMENT FORM

This gestational age (GA) assessment tool is based on the maternal immunization guideline matrix prepared by Jones, 2016 (March GAIA Meeting Washington, DC, 29 March 2016).

#### LEVELS OF CERTAINTY OF GESTATIONAL AGE ASSESSMENT

| Level | Description |
|---|---|
| Level 1 | <ul> <li>Certain LMP or IUI date or ET <u>WITH</u> confirmatory 1st trimester U/S,</li> </ul> |
| Highest level of | or |
| <u>certainty</u> | 1st trimester U/S |
| Level 2A | <ul> <li>Certain LMP <u>WITH</u> 2<sup>nd</sup> trimester U/S*,</li> </ul> |
| | or |
| | <ul> <li>Certain LMP <u>WITH</u> 1st trimester physical examination**</li> </ul> |
| Level 2B | <ul> <li>Uncertain LMP <u>WITH</u> 2<sup>nd</sup> trimester U/S</li> </ul> |
| Level 3A | <ul> <li>Certain LMP <u>WITH</u> 3<sup>rd</sup> trimester U/S***,</li> </ul> |
| | or |
| | <ul> <li>Certain LMP <u>WITH</u> confirmatory 2<sup>nd</sup> trimester FH,</li> </ul> |
| | or |
| | <ul> <li>Certain LMP <u>WITH</u> birth weight,</li> </ul> |
| | or |
| | <ul> <li>Uncertain LMP <u>WITH</u> 1st trimester physical examination</li> </ul> |
| Level 3B | <ul> <li>Uncertain LMP <u>WITH</u> FH,</li> </ul> |
| Lowest level of | or |
| <u>certainty</u> | <ul> <li>Uncertain LMP <u>WITH</u> neonatal physical assessment (New Ballard</li> </ul> |
| | score), |
| | or |
| | Uncertain LMP <u>WITH</u> birth weight |

grey highlights: applicable for enrollment in this study.

<sup>1</sup>st trimester U/S: ≤136/7 weeks, 2nd trimester U/S: 140/7 to 276/7 weeks, 3nd trimester U/S: ≥280/7 weeks.

GA: gestational age; U/S: ultrasound examination; LMP: last menstrual period; IUI: intrauterine insemination; ET: embryo transfer, FH: fundal height;

<sup>\*</sup> If LMP and U/S do not correlate, default to U/S GA assessment

<sup>\*\*</sup> For singleton pregnancies only. Unreliable if obesity, or uterine anomalies.

<sup>\*\*\*</sup> Depending on gestational age at Screening Visit/ Visit 1 and depending on the local standard of care, this will be applicable for inclusion in the study.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### METHODS OF GESTATIONAL AGE ASSESSMENT

Adapted from [ACOG, 2014]: The American College of Obstetricians and Gynecologists (ACOG) Committee on Obstetric Practice, American Institute of Ultrasound in Medicine and Society for Maternal-Fetal. Committee Opinions: Method for estimating Due Date. Number 611, October 2014 (accessed on-line on 13/Oct/2014 at:

http://www.acog.org/Resources-And-Publications/Committee-Opinions/Committee-on-Obstetric-Practice/Method-for-Estimating-Due-Date).

| Gestational age range | Method of measurement | Discrepancy between U/S dating and LMP dating |
|---|---|---|
| | 1st trimester ≤1 | 3 <sup>6/7</sup> weeks |
| ≤8 <sup>6/7</sup> weeks | CRL | > 5 days |
| 9 <sup>0/7</sup> to 13 <sup>6/7</sup> weeks | | > 7 days |
| | 2 <sup>nd</sup> trimester 14 <sup>0/7</sup> t | o 27 <sup>6/7</sup> weeks |
| 14 <sup>0/7</sup> to 15 <sup>6/7</sup> weeks | | > 7 days |
| 16 <sup>0/7</sup> to 21 <sup>6/7</sup> weeks | BPD, HC, AC, FL | > 10 days |
| 22 <sup>0/7</sup> to 27 <sup>6/7</sup> weeks | | > 14 days |

U/S: ultrasound examination; LMP: last menstrual period; CRL: crown-rump length; BPD: biparietal diameter; HC: head circumference; AC: abdominal circumference; FL: femur length

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## APPENDIX D DEFINITIONS OF MATERNAL, FETAL AND NEONATAL EVENTS OF INTEREST AS PER GAIA

The articles explaining the events of interest in detail and all corresponding information can be found in the following issues of Vaccine:

Bauwens J, Bonhoeffer J, Chen RT, editors. Harmonising Immunisation Safety Assessment in Pregnancy. Vaccine. 2016. 34 (49): 5991 – 6110.

Kochhar S, Bauwens J, Bonhoeffer J, editors. Harmonising Immunization Safety Assessment in Pregnancy – Part II. Vaccine. 2017. 35 (48): 6469-6582.

References specific to each event of interest are given at the end of the relevant Table.

Definitions and Levels of Diagnostic Certainty are presented in the following Tables.

| Pregnancy Outcomes | |
|---|---|
| Stillbirth | Table 20 |
| Maternal Events of Interest | |
| Maternal Death | Table 21 |
| Hypertensive Disorders of Pregnancy | Table 22 |
| Antenatal bleeding | Table 23 |
| Postpartum hemorrhage | Table 24 |
| Fetal Growth restriction | Table 25 |
| Dysfunctional Labor | Table 26 |
| Gestational Diabetes Mellitus | Table 27 |
| Non-reassuring fetal status | Table 28 |
| Pathways to Preterm Birth | Table 29 |
| Standard definitions for events of interest not defined as such in GAIA (Chorioamnionitis, Oligohydramnios, Polyhydramnios, Intrahepatic Cholestasis of Pregnancy (ICP), Acute Fatty Liver of Pregnancy, Maternal Sepsis) | Table 30 |
| Neonatal Events of Interest | |
| Small for Gestational Age | Table 31 |
| Low Birth Weight | Table 32 |
| Neonatal encephalopathy | Table 33 |
| Congenital Microcephaly | Table 34 |
| Congenital Anomalies | Table 35 |
| Neonatal Death | Table 36 |
| Neonatal Infections | Table 37 |
| Respiratory Distress in the Neonate | Table 38 |
| Preterm Birth | Table 39 |
| Failure to thrive | Table 40 |
| Standard definitions for events of interest not defined as such in GAIA (large for gestational age, macrosomia) | Table 41 |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### Table 20 Fetal death / Stillbirth

Fetal death occurring before birth after 20 to 28 weeks of gestation (variation due to country definitions). Descriptions are provided for reference in selecting the appropriate subcategory (antepartum or intrapartum). GAIA levels of diagnostic certainty will not be assessed in this protocol.

| | Antepartum Stillbirth (Fetal death occurs prior to the evidence of labor.) |
|---|---|
| Level | Description |
| 1 | Delivery of an infant with no of signs of life at birth (No spontaneous movements, no umbilical cord pulse, no heartbeat, no respirations, Apgar score of 0 at 1 and 5 min) determined by physical examination after delivery (with or without electronic monitoring of heart rate, respiratory rate, and pulse oximetry). AND |
| | Prenatal ultrasound examination documenting lack of fetal cardiac activity or movement before the onset of labor. OR |
| | Auscultation for fetal heart tones (using electronic devices or non-electronic devices) documenting lack of fetal heartbeat. AND |
| | Maternal report of lack of fetal movement for 24 h or more. OR |
| | Maternal physical examination confirming lack of fetal movement. OR |
| | Radiology findings consistent with intrauterine fetal death. AND |
| | Attended delivery followed by fetal physical examination afterbirth consistent with antepartum death, by obstetrician, neonatologist, pediatrician, maternal-fetal medicine specialist, or pathologist. In the setting where access to a specialist is not feasible, diagnosis by a health care provider trained or experienced to make the diagnosis is acceptable (e.g. general practice physician, mid-wife, nurse practitioner, a physician's assistant or other qualified trained practitioner). OR |
| | Fetal/placental pathology report consistent with antepartum death. AND |
| | •Gestational age within pre-defined range for selected stillbirth definition as assessed by maternal and/or fetal parameters (Level1 or 2 in GA assessment algorithm). |
| 2 | Delivery of an infant with no of signs of life at birth (No spontaneous movements, no umbilical cord pulse, no heartbeat, no respirations, Apgar score of 0 at 1 and 5 min) determined physical examination after delivery. AND |
| | Maternal report of lack of fetal movement for 24 h or more. OR |
| | Maternal physical examination confirming lack of fetal movement. OR |
| | Auscultation for fetal heart tones (using electronic or non-electronic devices) documenting lack of fetal heartbeat. AND |
| | Attended delivery followed by physical examination after birth consistent with antepartum death, by specialist or qualified trained practitioner appropriate to the health care setting. OR |
| | Fetal/placental pathology report consistent with antepartum death. AND |
| | •Gestational age within pre-defined range for selected stillbirth definition as assessed by maternal and/or fetal parameters (Level1–2 in GA assessment algorithm). |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| | Antepartum Stillbirth (Fetal death occurs prior to the evidence of labor.) (continued) |
|---|---|
| Lavel | |
| Level | Description Circ Hill (N) |
| 3 | Delivery of an infant reported to have no of signs of life at birth(No spontaneous movements, no umbilical cord pulse, no heart-beat, no cry or spontaneous respirations, no chest movement, and whole body cyanosis). AND |
| | Maternal report of lack of fetal movement for 24 h or more prior to delivery. OR |
| | Report of auscultation for fetal heart tones (using electronic or non-electronic devices) documenting lack of fetal heartbeat. AND |
| | Non-attended delivery followed by physical examination of the fetus after birth consistent with antepartum death by a healthcare professional appropriate to the level of standard of care in the health care setting. OR |
| | Verbal history by a trained health care provider, non-medical witness or the mother of a fetus born with no signs of life or unresponsive to resuscitation efforts immediately after birth and with physical features consistent with antepartum death. AND |
| | •Gestational age within pre-defined range for selected stillbirth definition as assessed by maternal and/or fetal parameters (Level2–3 in GA assessment algorithm). |
| 4 | Report of stillbirth but fetus is not available for physical examination after birth (no objective assessment can be made) •Maternal information insufficient to assess gestational age |
| Intrapart | um stillbirth (Fetal death occurs during labor and before delivery) |
| Level | Description |
| 1 | Delivery of an infant with no of signs of life at birth, including: No spontaneous movements, no umbilical cord pulse, no heartbeat, no respirations, and Apgar score of 0 at 1 and 5 min Determination of the absence of signs of life is made by physical examination after delivery, with or without electronic monitoring of heart rate, respiratory rate, and pulse oximetry. AND |
| | Evidence of live fetus prior to onset of labor (documentation of fetal movement and of fetal heart tones by ultrasound prior to onset of labor) (Note: in the absence of evidence of a live fetus prior to the onset of labor, the fetal death should be reported as a stillbirth or an antepartum stillbirth). AND |
| | Attended delivery followed by physical examination afterbirth consistent with intrapartum death by obstetrician, neonatologist, pediatrician, maternal-fetal medicine specialist, pathologist. In the setting where access to a specialist is not feasible, diagnosis by a health care provider trained or experienced to make the diagnosis is acceptable (e.g. general practice physician, midwife, or other qualified trained practitioner). AND |
| | Gestational age within pre-defined range for selected stillbirth definition as assessed by maternal and/or fetal-neonatal parameters (Level 1 in GA assessment algorithm) |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Intrapar | Intrapartum stillbirth (Fetal death occurs during labor and before delivery) (continued) |
|---|---|
| Level | Description |
| 2 | Delivery of an infant with no of signs of life at birth, including: No spontaneous movements, no umbilical cord pulse, no heartbeat, no respirations, and Apgar score of 0 at 1 and 5 min. Determination of the absence of signs of life is made by physical examination after delivery, with or without electronic monitoring of heart rate, respiratory rate, and pulse oximetry OR documentation of lack of response to resuscitation efforts. AND |
| | Evidence of live fetus prior to onset of labor (maternal report of fetal movement prior to onset of labor and documentation of fetal heart tones by auscultation or hand held Doppler) (Note: in the absence of evidence of a live fetus prior to the onset of labor, the fetal death should be reported as a stillbirth or an antepartum stillbirth). AND |
| | Attended delivery followed by physical examination after birth consistent with intrapartum death by a health care professional appropriate to the level of standard of care in the health care setting. AND |
| | Gestational age within pre-defined range for selected stillbirth definition as assessed by maternal and/or fetal parameters (Level1–2 in GA assessment algorithm). |
| 3 | Delivery of an infant reported to have no of signs of life at birth, including: No spontaneous movements, no umbilical cord pulse, no heartbeat, no cry, no spontaneous respirations or chest movement, and whole body cyanosis. AND |
| | Evidence of live fetus prior to onset of labor (maternal report of fetal movement prior to onset of labor OR auscultation of fetal heart tones) (Note: in the absence of evidence of a live fetus prior to the onset of labor, the fetal death should be reported as a stillbirth or an antepartum stillbirth). AND |
| | (Non-attended delivery followed by physical examination of the fetus after birth consistent with intrapartum death by a healthcare professional appropriate to the level of standard of care in the health care setting OR |
| | Verbal history by a trained health care provider, non-medical witness or the mother of a fetus born with no signs of life or unresponsive to resuscitation efforts immediately after birth.) AND |
| | Gestational age within pre-defined range for selected stillbirth definition as assessed by maternal and/or fetal parameters (Level2–3 in GA assessment algorithm). |
| 4 | Report of stillbirth but fetus is not available for physical examination after birth (no objective assessment can be made). |
| | Maternal information insufficient to assess gestational age. |

Reference: DaSilva FT, Gonik B, McMillan M, et al. Stillbirth: Case definition and guidelines for data collection, analysis, and presentation of maternal immunization safety data. Vaccine. 2016; 34(49):6057-6068.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### Table 21 Maternal Death

The death of a woman while pregnant or within 42 days of termination of pregnancy, irrespective of the duration and site of the pregnancy, from any cause related to or aggravated by the pregnancy or its management but not from accidental or incidental causes. (As ICD-10 terminology).

In the context of immunization: "Death of a woman during pregnancy, childbirth and the puerperium that is closely related temporally to an immunization event of the mother which is likely the single or contributory cause

| Levels of Diagnostic Certainty | |
|---|---|
| (Highest level (1) to lowest level of certainty) | |
| Level | Description |
| 1 | Diagnosis of pregnancy established by any of the following documented criteria: |
| | a. Ultrasound examination |
| | b. Fetal heart tones |
| | c. Positive serum or urine human chorionic gonadotropin pregnancy test |
| | d. Delivery of a neonate or other products of conception (abortus, stillborn) |
| | AND Dooth of the mether while prognent or within 42 days of termination of prognency irrespective of the |
| | Death of the mother while pregnant or within 42 days of termination of pregnancy, irrespective of the duration and site of the pregnancy AND |
| | Documentation of Cause of death as: |
| | a. Direct: abortive outcome, hypertensive disorder, obstetric hemorrhage, pregnancy related infection, |
| | other obstetric complications, unanticipated complications |
| | b. Indirect: non obstetric complications |
| | c. Death during pregnancy, childbirth and the puerperium: other or coincidental |
| 2 | Diagnosis of pregnancy established by any of the following criteria in the absence of Level 1 criteria: |
| | a. LMP date |
| | b. Serial Symphysio Fundal Height examinations |
| | AND |
| | Death of the mother while pregnant or within 42 days of termination of pregnancy, irrespective of the |
| | duration and site of the pregnancy And |
| | Documentation of Cause of death as: |
| | a. Direct: abortive outcome, hypertensive disorder, obstetric hemorrhage, pregnancy related infection, |
| | other obstetric complications, unanticipated complications b. Indirect: non-obstetric complications |
| | c. Death during pregnancy, childbirth and the puerperium: other or coincidental |
| | d. Unspecified: unknown or undetermined |
| 3 | Absence of Level 1 or 2 criteria for establishing diagnosis of pregnancy and: |
| | a. Unsure LMP |
| | b. No clinical examination <b>documented</b> |
| | AND |
| | Death of the mother temporal to pregnancy, childbirth or the postpartum period when exact timing of |
| | death is unknown |
| | AND |
| | Documentation of cause of death as: |
| | a. Direct: abortive outcome, hypertensive disorder, obstetric hemorrhage, pregnancy related infection, |
| | other obstetric com-plications, unanticipated complications |
| | b. Indirect: non-obstetric complications c. Death during pregnancy, childbirth and the puerperium: other or coincidental |
| | d. Unspecified: unknown or undetermined. |
| | o. Onspecified, unknown or undetermined. |

Reference: Patwardhan M, Eckert LO, Spiegel H, et al. Maternal death: Case definition and guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2016;34(49):6077-6083.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# Table 22 Hypertensive disorders of pregnancy (Gestational hypertension, Pre-eclampsia, Pre-eclampsia with severe features including eclampsia)

| | Levels of Diagnostic Certainty (Highest level (1) to lowest level of certainty) |
|---|---|
| Gestational Hypertension | |
| Level | Description |
| All | Clinical syndrome characterized by pregnancy ≥20 weeks AND New onset hypertension (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg) |
| | sustained on two measurements over a minimum of 1 h WITHOUT severe features (see preeclampsia with severe features category) and WITHOUT proteinuria |
| 1 | No proteinuria (as defined by 24 h urine collection < 300 mg, spot protein:creatinine ratio <0.3) |
| 2 | No proteinuria (as defined by urine dipstick negative or trace) |
| In Ev | Blood pressure cannot be measured OR No proteinuria evaluation is available |
| Preeclampsia has conventionally been defined as the development of gestational hypertension and proteinuria after 20 weeks gestation. Proteinuria can be quantified by: - 24 h urine collection, - a spot protein:creatinine ratio, or - with urinary dipstick. Proteinuria of ≥300 mg in a 24 h urine specimen (the gold standard for measurement of proteinuria), or ≥0.30 on a spot protein:creatinine ratio, or ≥1+ on a dipstick meets the criteria for preeclampsia. | |
| Level | Description |
| All | Clinical syndrome characterized by pregnancy ≥20 weeks AND New onset hypertension (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg) |
| | sustained on two measurements over a minimum of 1 h AND New onset proteinuria |
| 1 | Proteinuria diagnosed with ≥300 mg of protein on 24 h urine collection OR ≥0.3 on spot protein:creatinine ratio |
| 2 | Proteinuria diagnosed with ≥1+ protein on urine dipstick |
| In Ev. | Blood pressure cannot be measured OR |
| | no proteinuria evaluation is available (note diagnosis of preeclampsia with severe features does not require proteinuria, see definition below) |

In Ev = Insufficient Evidence

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### **Hypertensive Disorders of Pregnancy Continued**

**Preeclampsia with severe features** *NOTE* :can be diagnosed in the presence or absence of proteinuria.

#### •Vascular:

- Severely elevated blood pressures, with systolic blood pressure≥160 mmHg and/or diastolic blood pressure≥110 mmHg, which is confirmed after only minutes (to facilitate timely anti-hypertensive treatment)
   Neurologic:
- Development of a severe headache (which can be diffuse, frontal, temporal or occipital) that generally does not improve with over the counter pain medications (such as acetaminophen/paracetamol)
- Eclampsia
- Development of visual changes (including photopsia, scotomata, cortical blindness)

### •Hematologic:

• New onset thrombocytopenia, with platelet count <100,000/L

#### •Gastrointestinal:

- New onset of nausea, vomiting, epigastric pain
- Transaminitis (AST and ALT elevated to twice the upper limit of normal)
- · Liver capsular hemorrhage or liver rupture

#### •Renal:

- Worsening renal function, as evidenced by serum creatinine level greater than 1.1 mg/dL or a doubling of the serum creatinine(absent other renal disease)
- Oliguria (urine output <500 mL/24 h)</li>

#### •Respiratory:

Pulmonary edema (confirmed on clinical exam or imaging)

| Level | Description |
|---|---|
| All | Clinical syndrome characterized by pregnancy ≥20 weeks |
| | AND |
| | New onset hypertension (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg) |
| | sustained on two measurements over a minimum of 1 h |
| | AND |
| | At least one of the criteria for severe disease: |
| 1 | At least one of the following: |
| | Systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥110mmHg, which is |
| | confirmed after only minutes OR |
| | Development of severe, persistent headache OR |
| | Development of visual changes OR |
| | Eclampsia* OR |
| | New onset thrombocytopenia (platelets <100,000/L) OR |
| | New onset unremitting epigastric pain OR |
| | AST and ALT elevated to twice upper limit of normal OR |
| | <ul> <li>Evidence of liver capsular hematoma or liver rupture (diagnosed on clinical exam or with imaging)</li> <li>OR</li> </ul> |
| | Worsening renal function, as evidenced by serum creatinine level greater than 1.1 mg/dL or a |
| | doubling of the serum creatinine (absent other renal disease) or oliguria (<500 cc/24 h) OR |
| | Pulmonary edema (confirmed on imaging with chest X-ray, or on clinical exam) |
| 2 | New onset nausea and vomiting |
| In Ev | Blood pressure cannot be measured |

<sup>•\*</sup> ECLAMPSIA, or new-onset grand mal seizures in a patient with pre-eclampsia, without other provoking factors (such as evidence of cerebral malaria or preexisting seizure disorder). Seizures are often preceded by headaches, visual changes or altered mental status:

In Ev = Insufficient Evidence

Reference: Rouse CE, Eckert LO, Wylie BJ, et al. Hypertensive disorders of pregnancy: Case definitions & guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2016;34(49):6069-6076

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## Table 23 Antenatal Bleeding

Antenatal bleeding is a clinical syndrome characterized by bleeding in the second or third trimester of pregnancy. Pathologic etiologies attributable to the pregnant state include placenta previa, vasa previa and intra-abdominal pregnancy (categories that are not applicable in this study, as women with these conditions are ineligible), and morbidly adherent placentation, placental abruption, cesarean scar pregnancy and uterine rupture.

For both levels of diagnostic certainty for each etiology of antenatal bleeding:

Bleeding is either documented vaginally or suspected to be occurring intrauterine, intraperitoneally, or (rarely) retroperitoneally, based on clinical signs and symptoms.

In the case of ultrasound-based diagnosis, transvaginal ultrasound is more specific than transabdominal ultrasound, and transvaginal ultrasound is recommended where available.

| | Levels of Diagnostic Certainty (Highest level (1) to lowest level of certainty) |
|---|---|
| Morbidly adherent placenta | |
| Level | Description |
| 1 | There are two definitions of equal specificity. |
| | Second- or third-trimester ultrasound or MRI evidence of placenta previa, |
| | AND |
| | One of the following ultrasound features: |
| | Greyscale: loss of the retroplacental sonolucent zone, irregular retroplacental sonolucent zone, thinning or disruption of the hyperechoic serosa–bladder interface, presence of focal exophytic masses invading the urinary bladder, abnormal placental lacunae |
| | <ul> <li><u>Color Doppler:</u> diffuse or focal lacunar flow, vascular lakes with turbulent flow (peak systolic velocity<br/>over 15 cm/s), hypervascularity of serosa–bladder interface, markedly dilated vessels over<br/>peripheral subplacental zone</li> </ul> |
| | 3D Power Doppler: numerous coherent vessels involving the whole uterine serosa–bladder junction (basal view), hypervascularity (lateral view), inseparable cotyledonal and intervillous circulations, chaotic branching, detour vessels (lateral view) AND |
| | One of the risk factors: prior cesarean delivery, prior uterine surgery (including endometrial ablation or dilation and curettage) or cesarean scar pregnancy OR |
| | Morbidly adherent placentation found on histology in a hysterectomy or partial wedge resection specimen. |
| 2 | There are two definitions of equal specificity. |
| | 1. Ultrasound evidence of placenta previa, |
| | AND hypervascularity at the site of the uteroplacental interface,, diagnosed at laparotomy. OR |
| | Difficulty with placental separation after delivery of the infant, at either a vaginal or cesarean delivery with resultant hemorrhage due to partial separation. |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| | Automatal Blanding a sufficient |
|---|---|
| | Antenatal Bleeding continued |
| Placental abruption | |
| Level | Description |
| 1 | There are two definitions of equal specificity. |
| | 1. In the absence of placenta previa on ultrasound, vaginal bleeding in the second or third trimester, |
| | AND one of the following: |
| | Either uterine irritability or labor, |
| | Or |
| | clinical signs of hypovolemic shock or coagulopathy. |
| | OR |
| | Placental pathology with histologic findings of a chronic abruption. |
| 2 | There are two definitions of equal specificity. |
| | Vaginal bleeding in the second or third trimester, |
| | AND |
| | uterine irritability or labor, without clinical signs of hypovolemic shock or coagulopathy |
| | OR |
| | Vaginal bleeding in the second or third trimester, |
| | AND |
| | Clinical evidence of retroplacental clot or visually evident placental infarcts at the time of delivery. |
| | Cesarean Scar Pregnancy |
| Level | Description |
| 1 | There are two definitions of equal specificity. |
| | Transvaginal ultrasound with the following characteristics: empty uterine cavity, |
| | AND |
| | Empty cervical canal, without contact with the gestational sac, AND |
| | Presence of gestational sac, +/- fetal pole, +/- cardiac activity, in the anterior uterine segment adjacent to |
| | the cesarean scar, AND |
| | Absence or defect in myometrium between bladder and gestational sac, |
| | AND |
| | Gestational sac well perfused on Doppler ultrasound (to differentiate from an expulsing, avascular |
| | gestational sac). |
| | OR |
| | Hysterectomy specimen with evidence of pregnancy implanted into the cesarean scar. |
| 2 | There is no Level 2 definition for this event. |
| <u>Uterine Rupture</u> | |
| Level | Description |
| 1 | Complete uterine disruption at the time of laparotomy in the context of vaginal or intra-abdominal bleeding. |
| 2 | There is no Level 2 definition for this event. |

Reference: Prabhu M, Eckert LO, Belfort M et al. Antenatal bleeding: Case definition and guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2017; 35: 6529-6537.
207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## Table 24 Postpartum hemorrhage

Genital tract bleeding after delivery (up to 42 days) of a foetus or infant that leads to an adverse clinical outcome, such as hypovolemia or anaemia e.g. exertional dyspnoea, postural presyncope, tiredness or reduced consciousness. At the furthest extreme uncorrected hypovolaemic shock can lead to organ-dysfunction and maternal death.

ICD-10 definition: "heamorrhage after delivery of a foetus or infant"

| | Levels of Diagnostic Certainty (Highest level (1) to lowest level of certainty) |
|---|---|
| Level | Description |
| 1 | Genital bleeding after delivery leading to severe maternal out-come (maternal death or maternal near |
| | miss) as defined by WHO <sup>1</sup> . |
| 2 | Genital bleeding after delivery with at least one of the following: measured abnormal bleeding (1000 ml or |
| | more), or any bleeding leading to hypotension or blood transfusion. |
| 3 | Genital bleeding after delivery estimated at 1000 ml or more |

Reference: Kerr R, Eckert LO, Winikoff B, et al. Postpartum haemorrhage: Case definition and guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2016;34(49):6102-6109.

¹ Can be found in Kerr (op cit), Table 1.

## Table 25 Fetal growth restriction

A fetus with a sonographic estimation of fetal weight below the tenth percentile for a given gestational age with increasing specificity for adverse perinatal outcomes below the third percentile.

| | Levels of Diagnostic Certainty (Highest level (1) to lowest level of certainty) |
|---|---|
| Level | Description |
| | Fetal growth restriction is a sonographic finding characterized by: |
| 1a | Level 1* evidence of pregnancy dating |
| | AND |
| | Estimated fetal weight below 3% using locally-accepted growth curve |
| | OR This is the state of the sta |
| | Estimated fetal weight below 10% using locally-accepted growth curve AND |
| | Absent or reversed end-diastolic flow of the umbilical artery Doppler |
| | OR |
| | Oligohydramnios as defined as amniotic fluid index (AFI) < 8 cm or deepest vertical pocket (DVP) < |
| | 2 cm in the presence of intact membranes without concern for fetal anomalies contributing to its |
| | etiology |
| 1b | Level 1* evidence of pregnancy dating |
| | AND |
| | Estimated fetal weight below 10%ile using locally-accepted growth curve |
| | Lack of absent or reversed end-diastolic flow of the umbilical artery or oligohydramnios (as defined above, |
| | cfr. Level 1a) |
| 2a | Level 2 evidence of pregnancy dating |
| | AND |
| | Estimated fetal weight below 3% using locally-accepted growth curve |
| | OR |
| | Estimated fetal below 10% using locally-accepted growth curve |
| | AND |
| | Absent or reversed end-diastolic flow of the umbilical artery Doppler. |
| | OR Oligohydramnios (as defined above, cfr. Level 1a). |
| | Ongorrydrammos (as defined above, on. Lever ra). |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| | Fetal Growth Restriction continued |
|---|---|
| Level | Description |
| 2b | Level 2 evidence of pregnancy dating AND |
| | Estimated fetal weight below 10%ile using locally-accepted growth curve AND |
| | No findings of absent or reversed end-diastolic flow of the umbilical artery or oligohydramnios (as defined above, cfr Level 1a). |
| | OR |
| | Level 1* evidence of pregnancy dating |
| | AND |
| | Estimated fetal weight below 10% using locally-accepted growth curve with no findings of |
| | oligohydramnios (as defined abopve, cfr. Level 1a) with inability to assess umbilical artery Doppler. |
| In Ev | Absence of ultrasound for use in assessment of estimated fetal weight. |

<sup>\*</sup>Level 1 evidence of pregnancy dating as defined by the Preterm Birth Working Group of the Brighton Collaboration.

Level 1 pregnancy dating depends on a confirmatory ultrasound performed ≤13 <sup>6/7</sup> weeks gestation

In Ev = Insufficient Evidence

Reference: Easter SR, Eckert LO, Boghossian N, et al. Fetal growth restriction: Case definition & guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2017; 35: 6546-6554.

#### 

This is defined as prolonged labor at or after 37 weeks and before 42 weeks of gestational age in singleton pregnancies.

| Levels of Diagnostic Certainty (Highest level (1) to lowest level of certainty) | |
|---|---|
| First stage of labor | |
| | For both levels of diagnostic certainty the woman is in established labor defined by regular contractions and cervical |
| dilation of | dilation of at least 4cm. |
| Level | · |
| 1 | Progress of less than 0.5 cm cervical dilation per hour, for at least 4 hours, in women in established labor (i.e. have regular contractions and cervical dilation of at least 4cm) and with confirmed ruptured membranes. |
| 2 | Progress of less than 0.5cm cervical dilation per hour in women, for at least 4 hours, with established labor, (i.e. that is, regular contractions and cervical dilation of at least 4cm) without certainty of ruptured membranes. |
| Second | stage of labor |
| The defin | nitions below are applicable in cases with or without regional analgesia. |
| Level | Description |
| 1 | Full dilation of the cervix |
| | AND |
| | onset of the active stage (active maternal effort (i.e. pushing) or visible baby) |
| | AND |
| | In nulliparous women:> 2h of pushing |
| | In multiparous women: > 1h of pushing |
| | OR |
| | Use of instrument delivery (forceps vacuum/ventouse) for the indication of dystocia |
| | OR |
| | Caesarean delivery for the indication of dystocia. |
| 2 | Full dilation of the cervix in any phase of the second stage |
| | AND |
| | no delivery within 3 hours of full dilation OR |
| | use of instrument for the indication of dystocia |
| | OR |
| | caesarean delivery for the indication of dystocia. |
| l | Lacourtain delivery for the indication of dystocia. |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Reference: Boatin AA, Eckert LO, Boulvain M, et al. Dysfunctional labor: Case definition & guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2017; 35:6538-6545.

## Table 27 Gestational diabetes mellitus (pregnancy induced hyperglycemia)

Gestational diabetes mellitus (GDM) is a clinical syndrome characterized by the absence of pre-gestational diabetes diagnosis, defined by

- Previous diagnosis of diabetes while not pregnant OR
- First trimester hemoglobin A1c level of ≥ 6.5% (47.5 mmol/mol)
   OR
- First trimester fasting blood glucose 126 mg/dL / ≥ 7mmol/L
   AND

Identification of sustained hyperglycemia during pregnancy not due to other known causes (i.e. corticosteroids, beta-mimetics, etc.)

| Levels of Diagnostic Certainty (Highest level (1) to lowest level of certainty) | |
|---|---|
| Level | Description |
| 1 | Absence of pre-gestational diabetes mellitus diagnosis in the first trimester as defined above with level 1-2 certainty for gestational age using GAIA definition for gestational age (APPENDIX C) AND |
| | Diagnosis of gestational diabetes based on a positive internationally recognized oral glucose tolerance test ("major criteria" 1.2) using venous blood sample/samples |
| 2 | Absence of pre-gestational diabetes mellitus diagnosis in the first trimester as defined above with at least level 1-2 certainty for gestational age using GAIA definition for gestational age (APPENDIX C) AND |
| | Diagnosis of gestational diabetes based on positive internationally recognized oral glucose tolerance test ("major criteria" 1.2) using capillary blood sample/samples |

| Gestatio | Gestational Diabetes Mellitus continued |
|---|---|
| Level | Description |
| 3 | Absence of pre-gestational diabetes mellitus diagnosis in the first trimester as defined above with at least level 3 certainty for gestational age using GAIA definition for gestational age AND |
| | Diagnosis of gestational diabetes based on positive internationallyrecognized oral glucose tolerance test (see below "major criteria" <sup>1,2</sup> )using venous blood or capillary blood sample/samples OR |
| | Diagnosis of gestational diabetes based on fasting plasma glucose of 5.1-6.9 mmol/l (92-125 mg/dL) using venous or capillary blood samples. |
| In Ev | Blood glucose cannot be measured OR |
| | Elevated postprandial blood glucose level without confirmatory |
| | fasting venous blood or capillary glucose level OR |
| | Use of Hemoglobin A1c alone for the diagnosis of GDM without a diagnostic oral glucose tolerance test (OGTT) or elevated fasting plasma glucose level. OR |
| | Clinical and laboratory findings such as glucosuria, fundal height greater than dates, obesity, prior history of GDM or family history for the diagnosis of gestational diabetes mellitus without a diagnostic test. |

In Ev = Insufficient Evidence

Reference(s): Kachikis A, Eckert LO, Walker C, et al. Gestational diabetes mellitus: Case definition & guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2017; 35:6555-6562.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

### <sup>1</sup> Major criteria (presented in Kachikis op cit)

| Major criteria | |
|------------------------------|---------------------------|
| Endocrine | |
| Oral glucose | 75 g OGTT |
| Tolerance tests | IADPSG |
| | WHO |
| | NICE |
| | 100 g OGTT |
| | Carpenter-coustan |
| | NDDG |
| Fasting plasma glucose level | Based on WHO criteria (1) |
| [Absence of] pregestational | See above |
| diabetes mellitus criteria | |

<sup>&</sup>lt;sup>2</sup> Further details regarding oral glucose tolerance tests presented in footnote 1 (Major Criteria); also presented in Kachikis (op cit)

 Table 1

 Diagnostic oral glucose tolerance tests based on organization or country guidelines.

| Test | Guidelines | Number of abnormal values necessary for diagnosis | Fasting plasma glucose<br>mmol/l (mg/dl) | 1-h plasma glucose<br>mmol/l (mg/dl) | 2-h plasma glucose<br>mmol/l (mg/dl) | 3-h plasma glucose<br>mmol/l (mg/dl) | Timing |
|---|---|---|---|---|---|---|---|
| 75 g ( | OGTT | | | | | | |
| | WHO 2013 [1] | 1 | ≥5.1-6.9 (92-125) | ≥ 10.0 (180) | ≥8.5-11.0 (153-199) | N/A | 24–<br>28 wks |
| | IADPSG [25] | 1 | ≥5.1 (92) | ≥ 10.0 (180) | ≥8.5 (153) | N/A | |
| | NICE (UK)<br>[26] | 1 | ≥5.6 (101) | Not required | ≥7.8 (140) | N/A | 24–<br>28 wks |
| 100 g | OGTT | | | | | | |
| | Carpenter<br>Coustan [27] | 2 | ≥5.3 (95) | ≥ 10.0 (180) | ≥8.6 (155) | ≥7.8 (140) | 24–<br>28 wks |
| | NDDG [27] | 2 | ≥5.8 (105) | ≥ 10.6 (190) | ≥9.2 (165) | ≥ 8.0 (145) | |

OGTT (Oral glucose tolerance test); IADPSG (International Association of Diabetes and Pregnancy Study Groups); WHO (World Health Organization); NICE (The National Institute for Health and Care Excellence, UK); NDDG (National Diabetes Data Group).

## Table 28 Non-reassuring fetal status

Indicator of underlying event resulting in temporary or permanent oxygen deprivation to the fetus which may lead to fetal hypoxia and metabolic acidosis

| Levels o | Levels of Diagnostic Certainty (Highest level (1) to lowest level of certainty) |
|---|---|
| Level | Description |
| 1 | Category III fetal heart rate tracings detected via continuous cardiotocography as defined by NICHD Absent baseline fetal heart rate variability AND any of the following: - recurrent late decelerations - recurrent variable deceleration - bradycardia (<110 bpm) OR Sinusoidal pattern AND |
| | Umbilical cord blood analysis consistent with metabolic acidosis (pH < 7.0 and Base deficit >12 mmol/L) |
| 2 | Category III fetal heart rate tracings detected via continuous cardiotocography as defined by NICHD Absent baseline fetal heart rate variability AND any of the following: - recurrent late decelerations - recurrent variable deceleration - bradycardia (<110 bpm) OR Sinusoidal pattern |
| 3 | Fetal heart pattern detected via intermittent auscultation suggestive of fetal hypoxia Baseline Fetal Heart rate (FHR) <110 bpm or >160 bpm Presence of repetitive or prolonged (>3 min) decelerations More than 5 contractions in a 10 min period |

Reference: Gravett C, Eckert LO, Gravett MG, et al. Non-reassuring fetal status: Case definition & guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2016;34(49):6084-6092.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## Table 29 Pathways to preterm birth

Premature preterm rupture of membranes; Preterm labor; Insufficient cervix (not applicable to this study, as women with insufficient cervix are ineligible); Provider-initiated preterm birth

Preterm = Birth at less than 37 gestation-completed weeks (less than 259 days).

| Levels | of Diagnostic Certainty (Highest level (1) to lowest level of certainty) |
|---|---|
| Premate | ure Preterm rupture of membranes |
| Level | Description |
| All | Patient is determined to be preterm as defined above. On presentation, patient is determined to not be in preterm labor, having ≤4 contractions per hour documented clinically or on tocodynometer, with <2 cm cervical dilation (greater than 4 contractions per hour would qualify the patient as having preterm labor) Fluid can be noted to be clear, blood-tinged, meconium-tinged (fetal stool), purulent-tinged (yellowish, suggesting infection) |
| 1 | Clinical history of rupture of membranes AND Visible leakage of fluid on vaginal speculum exam AND Visible arborization (ferning) on microscopy of amniotic fluid OR Ultrasound with oligohydramnios (AFI <5 or MVP <2) AND Documented membrane rupture by a diagnostic test (one of the below options): Positive intra-amniotic dye-injection method Positive result on amniotic fluid alpha-fetoprotein test kit Amniotic fluid pH measurement (nitrazine paper test) Amniotic fluid placental alpha macroglobulin-1 protein assay (PAMG-1) test (AmniSure test) Amniotic fluid insulin-like growth factor binding protein(IGFBP-1) test (Actim PROM test) |
| 2 | Clinical history of rupture of membranes AND Visible leakage of fluid on vaginal speculum examination AND Visible arborization (ferning) on microscopy of amniotic fluid OR Documented membrane rupture by a diagnostic test (one of those listed above) OR Ultrasound with oligohydramnios (AFI <5 or MVP <2) |
| 3 | Clinical history of rupture of membranes AND Visible leakage of presumed amniotic fluid; this may be on vaginal speculum examination (pooling in vagina), on inspection of the perineum (wet perineum due to leakage of fluid from the vagina), or fluid soaked cloth/clothes/sanitary pad. |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Preterm | labor |
|---|---|
| Level | Description |
| All | Patient is determined to be have delivered preterm (at less than 37 gestation-completed weeks (less than |
| | 259 days)). |
| 1 | On presentation, >4 documented uterine contractions per hour as determined by a tocodynometer AND |
| | Documented change in length or dilation of cervix by physical examination or transvaginal ultrasound |
| | over a two hour period, with clinical criteria for documenting cervical change by exam including: |
| | a. Cervical dilation 2 cm or greater at the internal os by digital examination |
| | b. Cervical length of 1 cm or less by digital examination |
| 0 | c. 50% or greater effacement by digital examination |
| 2 | Greater than 4 uterine contractions per hour as determined by a tocodynometer or clinical assessment AND |
| | Documented change in length or dilation of cervix by physical examination, with clinical criteria including: |
| | a. Cervical dilation 2 cm or greater at the internal os by digital examination |
| | b. Cervical length of 1 cm or less by digital examination |
| • | c. 50% or greater effacement by digital examination |
| 3 | Greater than 4 documented uterine contractions per hour determined by clinical assessment |
| | AND Documented change in cervical examination (change in dilation or effacement) over a two hour period |
| Drovido | r-initiated preterm birth |
| Level | Description |
| All | Patient is determined to be preterm (birth at less than 37 gestation-completed weeks (less than 259 |
| ΛII | days). |
| 1 | Documentation in the healthcare record by a patient's delivering provider that there were no signs or symptoms of the spontaneous onset of preterm labor |
| | AND |
| | Documentation in the healthcare record by a patient's delivering provider that the patient needed to |
| | undergo induction of labor or cesarean delivery which led to the preterm delivery |
| 2 | From recall, delivering provider confirms that there was an absence of any signs or symptoms of the |
| | spontaneous onset of preterm labor |
| | AND |
| | Delivering provider reports from recall that he or she decided that the patient needed to undergo induction |
| • | of labor or cesarean delivery |
| 3 | From recall, patient confirms that there was an absence of any signs or symptoms of the spontaneous |
| | onset of preterm labor |
| | AND Retient reports from recall that the healthcare provider indicated that she needed to undergo industion of |
| | Patient reports from recall that the healthcare provider indicated that she needed to undergo induction of labor or cesarean delivery |
| | labol of cesareal delivery |

labor or cesarean delivery

Reference: Harrison MS, Eckert LO, Cutland C, et al. Pathways to preterm birth: Case definition and guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2016;34(49):6093-6101.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# Table 30 Standard Definitions for Maternal Events of interest not defined as events in GAIA

| Event of<br>Interest | Definition |
|---|---|
| Chorioamnionitis | Chorioamnionitis also known as intra-amniotic infection is an inflammation of the fetal membranes due to a bacterial infection. Clinical signs and symptoms of chorioamnionitis include the following: Fever (an intrapartum temperature >100.4°F or >37.8°C) Significant maternal tachycardia (>120 beats per minute [bpm]) Fetal tachycardia (>160-180 bpm) Purulent or foul-smelling amniotic fluid or vaginal discharge Uterine tenderness Maternal leukocytosis (total blood leukocyte count >15,000-18,000 cells/µL) Of these criteria, intrapartum maternal fever appears to be the most frequent. When at least 2 of the aforementioned criteria are present, the risk of neonatal sepsis is increased. Each clinical sign and symptom of chorioamnionitis, however, is by itself of low predictive value |
| Oligohydramnios | Amniotic fluid index (AFI) < 8 cm or deepest vertical pocket (DVP) < 2 cm in the presence of intact membranes without concern for fetal anomalies contributing to its etiology |
| Polyhydramnios | Polyhydramnios is the presence of excess amniotic fluid in the uterus. By definition, polyhydramnios is diagnosed if the deepest vertical pool is more than 8 cm or amniotic fluid index (AFI) is more than 95th percentile for the corresponding gestational age |
| Gestational liver<br>disease<br>(Intrahepatic<br>Cholestasis of<br>Pregnancy or<br>ICP) <sup>1</sup> | Intrahepatic cholestasis also called obstetric cholestasis should be suspected when pruritis develops during pregnancy in the absence of a rash. Lab evidence of cholestasis includes elevated bile acids (Glyco and Taurochenodeoxycholic Acid )(> 10 umol/L). Up to 60% of patients will have elevated transaminases and 20% of patients will have increased direct bilirubin levels. Jaundice may or may not be present. ICP typically is transient and resolves after delivery. Women that had ICP in previous pregnancy have higher risk to developing ICP in the following pregnancies or other hepatobiliary disorders in later life. ICP is associated with adverse fetal outcome like meconium-stained liquor, fetal asphyxia, spontaneous preterm delivery and intrauterine death. |
| Gestational liver<br>disease (Acute<br>Fatty Liver of<br>Pregnancy) <sup>2</sup> | Acute fatty liver of pregnancy (AFLP) is a rare, potentially fatal complication that occurs in the third trimester or early postpartum period. AFLP is characterized by microvesicular fatty infiltration of hepatocytes without any inflammation or necrosis. Most frequent signs and symptoms are the following: • Jaundice • Abdominal Pain (usually right upper quadrat, midepigastric or radiating to back) • Central nervous system (altered sensorium, confusion, disorientation, psychosis, restlessness, seizures or even coma) • Disseminated intravascular coagulation • Nausea and vomiting • Gastrointestinal bleeding • Acute renal failure • Oliguria • Tachycardia • Late onset pyrexia • Hypoglycemia • ALT<500 U/L • Hyperbilirubinemia, elevated ammonia, leukocytosis, hypofibrinogenemia Ultrasound examination and computed tomography may demonstrate fatty infiltration of the liver but are not sufficient for diagnosis |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| nterest | Definition | | | | | |
|---|---|---|---|---|---|---|
| Maternal Sepsis <sup>3</sup> | infection during Organ dysfunct consequent to t The baseline So organ dysfuncti A SOFA score a population with deteriorate furth | pregnancy, c<br>ion can be ide<br>the infection.<br>OFA score ca<br>on.<br>≥2 reflects an<br>suspected inf<br>ner, emphasiz | atening condition of<br>hild-birth, post-ab<br>entified as an acut<br>in be assumed to<br>overall mortality if<br>fection. Even pation<br>of the seriousness<br>of already being in | ortion, or post-pa<br>e change in total<br>be zero in patien<br>risk of approxima<br>ents presenting w<br>ss of this condition | artum period. I SOFA score ≥2 ts not known to stely 10% in a ge vith modest dysf | 2 points have preexisting eneral hospital unction can |
| | Table 1. Sequential [Sep: | sis-Related] Organ Fai | ilure Assessment Score <sup>a</sup> | | | |
| | | Score | | | | |
| | System<br>Respiration | 0 | 1 | 2 | 3 | 4 |
| | Pao <sub>2</sub> /Fio <sub>2</sub> , mm Hg<br>(kPa) | ≥400 (53.3) | <400 (53.3) | <300 (40) | <200 (26.7) with respiratory support | <100 (13.3) with respiratory support |
| | Coagulation | | | | | |
| | Platelets, ×10³/μL | ≥150 | <150 | <100 | <50 | <20 |
| | Liver | | | | | |
| | Bilirubin, mg/dL<br>(μmol/L) | <1.2 (20) | 1.2-1.9 (20-32) | 2.0-5.9 (33-101) | 6.0-11.9 (102-204) | >12.0 (204) |
| | Cardiovascular | MAP ≥70 mm Hg | MAP < 70 mm Hg | Dopamine <5 or<br>dobutamine (any dose) <sup>b</sup> | Dopamine 5.1-15<br>or epinephrine ≤0.1<br>or norepinephrine ≤0.1 <sup>b</sup> | Dopamine >15 or<br>epinephrine >0.1<br>or norepinephrine >0.1 <sup>b</sup> |
| | Central nervous system | | | | | |
| | Glasgow Coma Scale<br>score <sup>c</sup> | 15 | 13-14 | 10-12 | 6-9 | <6 |
| | Renal | | | | | () |
| | Creatinine, mg/dL<br>(µmol/L) | <1.2 (110) | 1.2-1.9 (110-170) | 2.0-3.4 (171-299) | 3.5-4.9 (300-440) | >5.0 (440) |
| | Urine output, mL/d | | | | <500 | <200 |
| | | | IAP, mean arterial pressure; | <sup>b</sup> Catecholamine doses a | ire given as μg/kg/min for at | least 1 hour. |
| | Pao <sub>2</sub> , partial pressure of or<br><sup>a</sup> Adapted from Vincent et | ,, | | <sup>c</sup> Glasgow Coma Scale so<br>neurological function. | cores range from 3-15; highe | r score indicates better |

References:

- 1 Geenes V et al . Intrahepatic cholestasis of pregnancy 2 Can J Gastroenterol Vol 20 26 No 1 January 2006 3 Bonet et al. Reproductive Health (2017) 14:67

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# Table 31 Small for Gestational Age

Weight below 10<sup>th</sup> percentile for gestational age as assessed against a validated global, regional or local standard.

| | | Levels of Diagnostic Certainty (1 highest level to 4 lowest level of certainty |
|---|---|---|
| Level | Desc | cription |
| 1 | • | Weight below 10th percentile for gestational age |
| | AND | |
| | • | The following used in assessment of weight: |
| | | <ul> <li>Newborn weighed within 24 hours of birth</li> </ul> |
| | | <ul> <li>Weight assessed using a calibrated electronic scale with 10 g resolution</li> </ul> |
| | AND | <del>-</del> 1 6 11 1 6 1 1 1 1 1 1 1 1 1 1 1 1 1 1 |
| | • | The following for assessment of gestational age: |
| | ΔD | Certain LMP or IUI or embryo transfer date AND confirmatory ultrasound in first trimester |
| | OR | First trimester ultrasound |
| 2a | • | Weight below 10th percentile for gestational age |
| | AND | The second secon |
| | • | The following used in assessment of weight: |
| | | <ul> <li>Newborn weighed within 24 hours of birth on any scale with a &lt; 50 g resolution, tared to zero</li> </ul> |
| | | and calibrated |
| | AND | |
| | • | The following for assessment of gestational age: |
| | ΩD | Certain LMP with first or second trimester ultrasound |
| | OR | Cortain LMD with first trimoster physical even |
| 2b | • | <ul> <li>Certain LMP with first trimester physical exam</li> <li>Weight below 10th percentile for gestational age</li> </ul> |
| 20 | AND | Weight below rour percentile for gestational age |
| | • | The following used in assessment of weight: |
| | | <ul> <li>Newborn weighed within 24 hours of birth on any scale with a &lt; 50 g resolution, tared to zero</li> </ul> |
| | | and calibrated |
| | AND | |
| | • | The following assessment of gestational age: |
| | | Uncertain LMP with second trimester ultrasound |
| 3a | • | Weight below 10th percentile for gestational age |
| | AND | The following wood in accompant of weights |
| | • | The following used in assessment of weight: o Infant weighed within the first 48 hours of life |
| | | Newborn weighed on any scale with a < 50 g resolution, tared to zero and calibrated |
| | AND | 140Wbbitt Weighted off arry social with a 100 g resolution, tarea to 2010 and cambrated |
| | • | The following assessment of gestational age: |
| | | Certain LMP with third trimester ultrasound |
| | OR | |
| | | <ul> <li>Certain LMP with confirmatory 2nd trimester fundal height</li> </ul> |
| | OR | 0 |
| | ΔD | Certain LMP with birthweight |
| | OR | LineCortain LMD with first trimester physical axem |
| | | <ul> <li>UncCertain LMP with first trimester physical exam</li> </ul> |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Small for Gestational Age (continued) | |
|---|---|
| Level | Description |
| 3b | Weight below 10th percentile for gestational age |
| | AND |
| | The following used in assessment of weight: |
| | <ul> <li>Infant weighed within the first 48 hours of life</li> </ul> |
| | <ul> <li>Newborn weight assessed by measuring the difference between an adult holding the infant</li> </ul> |
| | and the adult being weighed alone on any scale |
| | AND |
| | The following assessment of gestational age: |
| | <ul> <li>Uncertain LMP with fundal height</li> </ul> |
| | OR |
| | <ul> <li>Uncertain LMP with newborn physical assessment</li> </ul> |
| | OR |
| | Uncertain LMP with birthweight |
| 4 | Baby noted to be small, but no actual weight |
| | Baby with GA assessed only by infant examination |
| | Diagnosis extracted from billing codes or chart, with no documentation of actual birth weight or GA |

Reference: Schlaudecker EP, Munoz FM, Bardají A, et al. Small for gestational age: Case definition & guidelines for data collection, analysis, and presentation of maternal immunisation safety data. Vaccine. 2017; 35:6518-6528.

# Table 32 Low Birth Weight (LBW)

Regardless of gestational age:

- Low birth weight (LBW): <2500 grams.
- Very low birth weight (VLBW): <1500 grams
- Extremely low birth weight (ELBW): <1000grams

| | Levels of Diagnostic Certainty (1 highest level to 4 lowest level of certainty |
|---|---|
| Level | Description |
| 1 | 1.Newborn infant weighed within 24 hours of birth |
| | AND |
| | 2. Use electronic scale which is graduated to 10 grams |
| | AND |
| | 3. Scale is calibrated at least once a year |
| | AND |
| | 4. Scale placed on level, hard surface |
| | AND |
| | 5. Scale tared to zero grams |
| | AND |
| | 6. Weight recorded as <2500 grams |
| | OR |
| | 1.Birth weight recorded as <2500 grams |
| | AND |
| | 2. Birth weight assessed as per health care facility's standard operating procedure, which fulfills criteria 1 |
| | to 5 above. |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Low Birth Weight (continued) | |
|---|---|
| Level | Description |
| 2 | 1. Newborn infant weighed within 24 hours of birth |
| | AND |
| | 2. Scale (electronic/spring) is graduated to at least 50 grams |
| | AND |
| | 3. Scale is calibrated at least once a year, or more often if moved |
| | AND |
| | 4. Scale tared to zero grams or 0.00kg |
| | AND |
| | 5. Weight recorded as <2500 grams OR |
| | <ol> <li>Birth weight recorded as &lt;2500 grams AND</li> <li>Birth weight assessed as per health care facility's standard operating procedure, which fulfills criteria 1</li> </ol> |
| | to 4 above. |
| | (Scale used could be electronic or spring scale, including colour-coded scale) |
| 3 | Newborn infant weighed on day 1 or 2 of life (first 48 hours of life) |
| | AND |
| | Weight measured using dial/spring/colour-coded scale |
| | AND |
| | 3. Weight assessed as <2500 grams |
| 4 | 1. Newborn weight assessed between day 1 and 2 of life (first 48 hours) |
| | AND |
| | 2 Proxy measure (newborn foot length, chest circumference, mid upper arm circumference) of birth |
| | weight used |
| | AND |
| | 3. Weight CATEGORY assessed as <2500 grams |

Reference: Cutland CL, Lackritz EM, Mallett-Moore T, et al. Low birth weight: Case definition & guidelines for data collection, analysis, and presentation of maternal immunization safety data. Vaccine. 2017; 35:6492-6500.

## Table 33 Neonatal encephalopathy

Disease, malfunction of damage of the brain in a newborn (1–28 days) born at or beyond 35 weeks of gestation, that may be due to a variety of etiologies including but not limited to hypoxia/ischemia, metabolic disturbance, infection and traumatic processes

| Levels | Levels of Diagnostic Certainty (1 highest level to 4 lowest level of certainty |
|---|---|
| Level | Description |
| 1 | (Definite) |
| | Abnormal level of alertness or seizures AND |
| | Difficulty with initiating and maintaining respiration AND |
| | Depression of tone |
| 2 | (Probable) |
| | Abnormal level of alertness or seizures |
| | AND |
| | Difficulty with initiating and maintaining respiration OR Depression of tone |
| 3 | (Possible) |
| | Abnormal level of alertness or seizures without difficulty with initiating and maintaining respiration nor |
| | depression of tone |

Reference: Sell E, Munoz FM, Soe A, et al. Neonatal encephalopathy: Case definition & guidelines for data collection, analysis, and presentation of maternal immunisation safety data. Vaccine. 2017; 35: 6501-6505.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# Table 34 Congenital Microcephaly

Congenital microcephaly, also referred to as primary microcephaly due to its presence in utero or at birth, is a descriptive term for a structural defect in which a fetus or infant's head (cranium) circumference is smaller than expected when compared to other fetuses or infants of the same gestational age, sex and ethnic background

| | Levels of Diagnostic Certainty (1 highest level to 4 lowest level of certainty |
|---|---|
| | Postnatally Diagnosed Microcephaly |
| Level | Description |
| 1 | Live birth, stillbirth, or spontaneous or therapeutic abortion of at least 24 weeks of Gestational Age (GA)~ AND |
| | Head Circumference (HC) 2 Standard Deviations (SD) below mean or <3rd percentile according to GA and gender, using appropriate standardized reference charts for the population (e.g., WHO growth reference charts if GA ≥37 weeks and Intergrowth-21st reference charts for GA 24–36 weeks) AND |
| | Measured between 24–36 hours after birth or end of pregnancy. |
| | ~GA assessed based on certain Last Menstrual Period (LMP) with confirmatory 1st trimesteror 2nd trimester ultrasound (US) scan, intrauterine insemination (IUI), or embryo transfer date |
| 2a | Live birth, stillbirth, or spontaneous or therapeutic abortion of at least 24 weeks of GA~ AND |
| | HC 2 SD below mean or <3rd percentile according to GA and gender, using appropriate standardized reference charts for the population (e.g., WHO growth reference charts if GA ≥37 weeks and Intergrowth-21st reference charts for GA 24–36 weeks) AND |
| | Measured within the first 24 hours§ |
| | >36 hours and up to 6 weeks after birth or end of pregnancy with no apparent post-natal insult resulting in microcephaly |
| | ~GA assessed based on certain LMP with confirmatory 1st trimester or 2nd trimester US scan, IUI, or embryo transfer date |
| | §Take into account the variability in this period based on molding of the head |
| 2b | Live birth, stillbirth, or spontaneous or therapeutic abortion of at least 24 weeks of GA~ AND |
| | HC 2 SD below mean or <3rd percentile according to GA and gender, using appropriate standardized reference charts for the population (e.g., WHO growth reference charts if GA ≥37 weeks and Intergrowth-21st reference charts for GA 24–36 weeks) AND |
| | - within the first 24 hours§ |
| | >36 hours and up to 6 weeks after birth or end of pregnancy with no apparent post-natal insult resulting in microcephaly |
| | ~GA assessed based on uncertain LMP with 2nd trimester US scan<br>§Take into account the variability in this period based on molding of the head |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| | Protocol Amendment 4 Final |
|---|---|
| _ | Postnatally Diagnosed Microcephaly (continued) |
| Level | Description |
| 3a | Live birth, stillbirth, or spontaneous or therapeutic abortion of at least 24 weeks of GA~_ AND |
| | HC 2 SD below mean or <3rd percentile according to GA and gender, using appropriate standardized reference charts for the population (e.g., WHO growth reference charts if GA P37 weeks and Intergrowth-21st reference charts for GA 24–36 weeks) AND |
| | Measured up to 6 weeks after birth or end of pregnancy with no apparent post-natal insult resulting in microcephaly |
| | ~GA based on LMP without confirmatory 1st or 2nd trimester Ultrasound |
| 3b | Live birth, stillbirth, or spontaneous or therapeutic abortion AND |
| | Case meets criteria for microcephaly using a validated algorithm: 1 inpatient diagnosis OR 2 outpatient diagnoses OR 1 outpatient diagnosis AND death in first year using the following diagnostic codes ICD-9-CM code 742.1 or ICD-10-CM code Q02 |
| 4 | Live birth, stillbirth, or spontaneous or therapeutic abortion |
| | AND |
| | Diagnosis of congenital microcephaly based on: |
| | physical inspection without HC measurement |
| | OR |
| | ICD-9-CM or ICD-10-CM code that does not meet validated algorithm criteria above. |
| | Prenatally Diagnosed Microcephaly |
| Level | Description |
| 1a | Fetus of at least 24 weeks GA based on certain LMP with confirmatory 1st trimester (<14 weeks) or 2nd trimester US scan IUI, or embryo transfer date AND |
| | HC 2 SD below mean or <3rd percentile according to fetal ultrasound (US) examination using appropriate standardized reference charts according to GA and gender for the population (eg. WHO growth reference charts if GA ≥37 weeks and Intergrowth-21st reference charts for GA 24–36 weeks) AND |
| | Confirmation of microcephaly (i.e., HC 2 SD below mean or <3rd percentile) by: – at least one additional US after 24 weeks and at least one week after first US OR |
| | HC measurement with standard tape measure at birth or autopsy |
| 1b | Fetus of at least 24 weeks GA based on uncertain LMP with 2nd trimester US AND |
| | HC 2 SD below mean or <3rd percentile according to fetal ultrasound (US) examination using appropriate standardized reference charts according to GA and gender for the population (eg. WHO growth reference charts if GA ≥37 weeks and Intergrowth-21st reference charts for GA 24–36 weeks) AND |
| | Confirmation of microcephaly (i.e., HC 2 SD below mean or <3%) by: — at least one additional US after 24 weeks and at least one week after first US OR |
| | HC measurement with standard tape measure at birth or autopsy |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| | Pronotelly Diagnosed Missesenhely (continued) |
|---|---|
| | Prenatally Diagnosed Microcephaly (continued) |
| Level | Description |
| 2 | Fetus of at least 24 weeks GA based on certain or uncertain LMP with fundal height and no confirmatory 1st or 2nd trimester US scan AND |
| | HC 2 SD below mean or <3rd percentile according to fetal US scan using appropriate standardized reference charts according to GA and gender for the population (eg. WHO growth reference charts if GA ≥37 weeks and Intergrowth-21st reference charts for GA 24–36 weeks) with femur length and abdominal circumference concordant with GA assessment AND |
| | Confirmation of microcephaly (i.e., HC 2 SD below mean or <3%) by: at least one additional US scan after 24 weeks and at least one week after first US OR |
| | HC measurement with standard tape measure at birth or autopsy |
| 3a | Fetus of at least 24 weeks GA based on certain LMP with confirmatory 1st trimester or 2nd trimester US scan, uncertain LMP with 2nd trimester US, IUI, or embryo transfer date AND |
| | HC 2 SD below mean or <3rd percentile according to fetal US scan using appropriate standardized reference charts according to GA and gender for the population (eg. WHO growth reference charts if GA ≥37 weeks and Intergrowth-21st reference charts for GA 24–36 weeks) with femur length and abdominal circumference concordant with GA assessment AND |
| | No additional data to confirm microcephaly (i.e., No additional prenatal US scan or confirmation of microcephaly with any additional US or by HC measurement at birth or autopsy at birth or autopsy) |
| 3b | Fetus of at least 24 weeks GA based on certain or uncertain LMP with fundal height and no confirmatory 1st or 2nd trimester US AND |
| | HC 2 SD below mean or <3 percentile according to fetal US scan using appropriate standardized reference charts according to GA and gender for the population (e.g., WHO growth reference charts if GA P37 weeks and Intergrowth-21st reference charts for GA 24–36 weeks) with femur length and abdominal circumference concordant with GA assessment AND |
| | No additional data to confirm microcephaly (i.e., No additional prenatal US scan or confirmation of microcephaly by HC measurementat birth or autopsy) |
| 4 | Fetus of at least 24 weeks GA based on certain LMP with confirmatory 1st trimester or 2nd trimester US scan, uncertain LMP with 2nd trimester US, IUI, embryo transfer date, or certain or uncertain LMP with fundal height and no confirmatory 1st or 2nd trimester US scan AND |
| | HC 2 SD below mean or <3% according to fetal US examination using appropriate standardized reference charts according to GA and gender for the population (eg. WHO growth reference charts if GA ≥37 weeks and Intergrowth-21st reference charts for GA 24–36 weeks) AND |
| | HC at birth or autopsy is in the normal range using appropriate standardized reference charts according to GA and gender for the population, which means that this is NOT a case of prenatally diagnosed congenital microcephaly |

Reference: DeSilva M, Munoz FM, Sell E, et al. Congenital microcephaly: Case definition & guidelines for data collection, analysis, and presentation of safety data after maternal immunisation. Vaccine. 35; 6472 – 6482.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# Table 35 Major Congenital anomalies

Congenital anomalies, also commonly referred to as birth defects, congenital disorders, congenital malformations, or con-genital abnormalities. Major congenital anomalies are events of prenatal origin that a represent at birth, potentially impacting an infant's health, development and/or survival.

| | Levels of Diagnostic Certainty (1 highest level to 4 lowest level of certainty |
|---|---|
| | Major External Structural Defects |
| Level | Description |
| 1 | Alterations in external anatomy visible: |
| | at the time of <u>live birth</u> and persistent beyond the immediate peripartum period unless surgically |
| | repaired OR |
| | in a <u>stillbirth</u> or in the products of conception of a <u>spontaneous or therapeutic abortion</u> |
| | AND |
| | Confirmed by documentation of a diagnosis made by a clinician experienced in diagnosing congenital |
| | anomalies and with the highest level of morphology training for the specific setting |
| 2 | Alterations in external anatomy visible: |
| | at the time of live birth and persistent beyond the immediate peripartum period unless surgically |
| | repaired |
| | OR |
| | in a <u>stillbirth</u> or in the products of conception of a <u>spontaneous or therapeutic abortion</u> AND |
| | Confirmed by documentation of a diagnosis made by a clinician with some experience diagnosing |
| | congenital anomalies |
| 3 | Alterations in external anatomy visible: |
| | <ul> <li>at the time of <u>live birth</u> and persistent beyond the immediate peripartum period unless surgically</li> </ul> |
| | repaired |
| | OR - in a stillbirth or in the products of conception of a spontaneous or therapeutic abortion |
| | In a <u>stillbirth</u> or in the products of conception of a <u>spontaneous or therapeutic abortion</u> AND |
| | Confirmed: |
| | by documentation of a diagnosis made by a trained maternal or child health care provider with at least |
| | minimal experience diagnosing congenital anomalies |
| | OR |
| | <ul> <li>For <u>live births</u>, by using individual (ICD-9/ICD-10) codes or as part of an ICD-9/ICD-10 code based<br/>algorithm, where the outcome (individual code or algorithm) has been validated</li> </ul> |
| 4 | (Insufficient evidence to confirm) |
| 7 | Alterations in external anatomy visible: |
| | at the time of <u>live birth</u> and persistent beyond the immediate peripartum period unless surgically |
| | repaired |
| | OR |
| | in a <u>stillbirth</u> or in the products of conception of a <u>spontaneous or therapeutic abortion</u> |
| | AND<br>Confirmed: |
| | Confirmed: - by medical record review |
| | OR |
| | in claims data (ICD-9/ICD-10 diagnoses) |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| | Internal Structural Defects |
|---|---|
| Level | Description |
| 1 | Alterations in internal anatomy present at the time of <u>live birth</u> and persistent beyond the immediate |
| ' | peripartum period unless surgically repaired |
| | AND |
| | Confirmed by definitive imaging study or intraoperative diagnosis |
| | OR |
| | •Alterations in internal anatomy detected during autopsy for a <u>stillbirth, spontaneous or therapeutic</u> |
| | abortion confirmed by documentation by a pathologist or other relevant subspecialist |
| 2 | Alterations in internal anatomy present at the time of live birth and persistent beyond the immediate |
| | peripartum period unless surgically repaired |
| | AND |
| | •Confirmed by documentation of a diagnosis made by a clinician experienced in diagnosing congenital |
| | anomalies and with the highest level of morphology training for the specific setting without definitive |
| | imaging or intraoperative evaluation |
| | OR |
| | •For stillbirth, spontaneous or therapeutic abortion, internal structural defect is visible by ultrasound or |
| | other imaging modality prenatally |
| 3 | •Alterations in internal anatomy present at the time of <u>live birth</u> and persistent beyond the immediate |
| | peripartum period unless surgically repaired |
| | AND |
| | •Confirmed: |
| | by documentation of a diagnosis made by a clinician with some experience diagnosing congenital |
| | anomalies |
| | OR |
| | using individual (ICD-9/ICD-10) codes or as part of an ICD-9/ICD-10 code based algorithm, where the |
| | outcome (individual code or algorithm) has been validated |
| 4 | (Insufficient evidence to confirm) |
| | Alterations in internal anatomy present: |
| | at the time of live birth and persistent beyond the immediate peripartum period unless surgically repaired |
| | OR |
| | at time of stillbirth, spontaneous abortion, or induced abortion AND |
| | •Confirmed: |
| | through medical record review, with the medical record demonstrating that the anomaly was present at |
| | the time of live birth or time of fetal demise, and that the anomaly was diagnosed by a trained maternal or |
| | child health care provider with minimal experience diagnosing congenital anomalies |
| | OR |
| | by claims data (ICD-9/ICD-10 diagnoses) |
| | ay statute data (1.22 st. 22 st. 23 statute data) |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| | Protocol Amendment 4 Final |
|---|---|
| | Functional Defects |
| Level | Description |
| 1 | For live births, alterations in functioning of one or more organs or body parts not due to a structural defect, present at the time of birth (or propensity to develop alteration present at live birth), and persistent beyond the immediate peripartum period, unless treated through gene therapy or stem cell transplantation OR |
| | •For stillbirths, spontaneous or therapeutic abortions, alterations in functioning of one or more organs or body parts, not due to a structural defect AND |
| | Confirmed by definitive diagnostic study |
| 2 | For live births, alterations in functioning of one or more organs or body parts not due to a structural defect, present at livebirth (or propensity to develop alteration present at live birth), and persistent beyond the immediate peripartum period, unless treated through gene therapy or stem cell transplantation OR |
| | •For stillbirths, spontaneous or therapeutic abortions, alterations in functioning of one or more organs or body parts, not due to a structural defect AND |
| | •Confirmed by documentation of a diagnosis made by a clinician experienced in diagnosing congenital anomalies and with the highest level of training in the diagnosis of functional defects for the specific setting |
| 3 | For live births, alterations in functioning of one or more organs or body parts not due to a structural defect, present at livebirth (or propensity to develop alteration present at live birth), and persistent beyond the immediate peripartum period, unless treated through gene therapy or stem cell transplantation OR •For stillbirths, spontaneous or therapeutic abortions, alterations in functioning of one or more organs or body parts, not due to a structural defect AND •Confirmed: — by documentation of a diagnosis made by a clinician with some experience diagnosing functional defects OR — using individual (ICD-9/ICD-10) codes or as part of an ICD-9/ICD-10 code based algorithm, where |
| 4 | the outcome(individual code or algorithm) has been validated (Insufficient evidence to confirm) |
| 4 | For live births, alterations in functioning of one or more organs or body parts not due to a structural defect, present at the time of live birth (or propensity to develop alteration present at livebirth), and persistent beyond the immediate peripartum period, unless treated through gene therapy or stem cell transplantation OR |
| | •For stillbirths, spontaneous or therapeutic abortions, alterations in functioning of one or more organs or body parts, not due to a structural defect AND •Confirmed: |
| | <ul> <li>through medical record review, with the medical record demonstrating that the anomaly was present at the time of live birth or time of fetal demise, and that the anomaly was diagnosed by a trained maternal or child healthcare provider who is not a qualified geneticist, neonatologist, pathologist, subspecialist, pediatrician, obstetrician, or family medicine practitioner</li> <li>OR</li> </ul> |
| | by claims data (ICD-9/ICD-10 diagnoses) |

by claims data (ICD-9/ICD-10 diagnoses)

Reference: DeSilva M, Munoz FM, Mcmillan M, et al. Congenital anomalies: Case definition and guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2016;34(49):6015-6026.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# Table 36 Neonatal Death

Death of a live born infant regardless of gestational age at birth, within the first 28 completed days of life

| | Lovale of Diagnostic Cortainty (1 highest level to 4 lovest level of sectainty |
|---|---|
| | Levels of Diagnostic Certainty (1 highest level to 4 lowest level of certainty Neonatal death in a non-viable live birth |
| Laval | |
| Level 1 | Description 1. Live born infant |
| ' | AND |
| | 2. Gestational age <22 weeks (GA level of certainty = 1) OR |
| | 3. Birth weight <500 g |
| | AND |
| | 4. Death of infant in first 28 days of life |
| | AND |
| | 5. Medically-confirmed death |
| 2 | 1. Live born infant |
| _ | AND |
| | 2. Gestational age/size of newborn assessed as at least one of: |
| | a. Gestational age <22 weeks (GA Level of Certainty = 1 OR 2) |
| | b. Birth weight <500 g |
| | AND |
| | 3. Death of infant in first 28 days of life |
| | AND |
| | Medically-confirmed death OR non-medically-confirmed death |
| 3 | 1. Live born infant |
| | AND |
| | 2. Gestational age <5 months according to parent/family member/delivery attendant (GA Level of |
| | Certainty = 2 OR 3) |
| | AND |
| | 3. Death of infant in first 28 days of life |
| | AND |
| | 4. Medically-confirmed death OR non-medically-confirmed death |
| Level | Neonatal death in an extremely preterm live birth Description |
| 1 | 1. Live born infant |
| ' | AND |
| | 2. Gestational age ≥22 and <28 weeks (GA Level of Certainty = 1) |
| | OR |
| | 3. Birth weight ≥500 g but <1000 g |
| | AND |
| | 4. Death of infant in first 28 days of life |
| | AND |
| | 5. Medically-confirmed death |
| 2 | 1. Live born infant |
| | AND |
| | 2. Gestational age/size of newborn assesses as one or more of: |
| | a. Gestational age ≥22 and <28 weeks (GA Level of Certainty = 1 OR 2) |
| | b. Birth weight ≥500 g but <1000 g |
| | AND |
| | 3. Death of infant in first 28 days of life |
| | AND |
| | 4. Medically-confirmed death OR non-medically-confirmed death |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| | Protocol Amendment 4 Fin |
|---|---|
| | Neonatal death in an extremely preterm live birth (continued) |
| Level | Description |
| 3 | 1. Live born infant |
| | AND |
| | 2. Gestational age ≥5 months but <7 months according to neonate's parent (mother/father)/family |
| | member/delivery attendant (GA Level of Certainty = 2 OR 3) |
| | AND |
| | 3. Death of infant in first 28 days of life |
| | AND |
| | 4. Medically-confirmed death OR non-medically-confirmed death |
| | Neonatal death in a preterm live birth (gestational age ≥28to <37 weeks) |
| Level | Description |
| 1 | 1. Live born infant |
| | AND |
| | 2. Gestational age ≥28 and <37 weeks (Level of Certainty = 1) |
| | OR |
| | 3. Birth weight ≥1000 g but <2500 g |
| | AND |
| | 4. Death of infant in first 28 days of life |
| | AND |
| | 5. Medically-confirmed death |
| 2 | 1. Live born infant |
| | AND |
| | 2. Gestational age/size of newborn assesses as one or more of: |
| | a. Gestational age ≥28 and <37 weeks (GA Level of Certainty = 1 OR 2) |
| | b. Birth weight ≥1000 g but <2500 g |
| | AND |
| | 3. Death of infant in first 28 days of life |
| | AND |
| | 4. Medically-confirmed death OR non-medically-confirmed death |
| 3 | (MAY apply to LMIC- or may be non-viable in LMIC) |
| | 1. Live born infant |
| | AND |
| | 2. Gestational age ≥7 months but <9 months according to parent/family member/delivery attendant (GA |
| | Level of Certainty = 2 OR 3) |
| | AND 3. Dooth of infant in first 29 days of life |
| | 3. Death of infant in first 28 days of life AND |
| | 4. Medically-confirmed death OR non-medically-confirmed death |
| | Neonatal death in a term live birth |
| Level | Description |
| 1 | 1. Live born infant AND |
| ' | 2. Gestational age ≥37 weeks (GA Level of Certainty = 1) AND |
| | 3. Birth weight >2500 g |
| | OR |
| | 4. Documented intra-uterine growth retardation if ≤2500 g |
| | AND |
| | 5. Death of infant in first 28 days of life |
| | AND |
| | 6. Medically-confirmed death |
| L | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Neonatal death in a term live birth (continued) | |
|---|---|
| Level | Description |
| 2 | 1. Live born infant |
| | AND |
| | 2. Gestational age/size of newborn assesses as one or more of: |
| | a. Gestational age ≥37 weeks (GA Level of Certainty = 1 OR 2) |
| | b. Birth weight ≥2500 g |
| | AND |
| | 3. Death of infant in first 28 days of life |
| | AND |
| | 4. Medically-confirmed death OR non-medically-confirmed death which is confirmed by examination by |
| | (by at least) non-medically-trained attendant (e.g. undertaker, community member) |
| 3 | (apply to LowerMiddleIncomeCountries) |
| | 1. Live born infant AND 2. Gestational age ≥9 months according to parent/family member/delivery |
| | attendant (GA Level of Certainty = 2 OR 3) AND |
| | 3. Death of infant in first 28 days of life |
| | AND |
| | 4. Medically-confirmed death OR non-medically-confirmed death |

Reference: Pathirana J, Muñoz FM, Abbing-Karahagopian V, et al. Neonatal death: Case definition & guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2016;34(49):6027-6037.

## **Table 37** Neonatal Infections

Neonatal bacteraemia and sepsis (of early or late onset), meningitis, pneumonia and other respiratory infections such as bronchiolitis, caused by bacteria, parasites, viruses or fungi. Localised eye and ear infections, encephalitis, urinary tract infections and intestinal infections were excluded from these guidelines

| Neonatal invasive blood stream infections: bacterial/fungal/viral | |
|---|---|
| Level | Description |
| 1 | Recognised pathogen identified using a validated method and from a normally sterile site. |
| 2 | Not meeting Level 1 of evidence |
| | AND |
| | Meeting 3 or more of the following criteria: |
| | Temperature ≥37.5 °C or <35.5 °C |
| | Tachycardia or new or more frequent episodes of bradycardia |
| | •New or more frequent episodes of apnea or increased oxygen requirement or increased requirement for |
| | ventilatory support |
| | Lethargy or moving only when stimulated or hypotonia or irritability Difficulty in feeding or shadowing distances. |
| | <ul><li>Difficulty in feeding or abdominal distention</li><li>Pallor or poor perfusion or hypotension</li></ul> |
| | •Abnormal White Cell Count or I/T ratio >0.2 |
| | Abnormal platelet count |
| | •Increased inflammatory markers (CRP, procalcitonin) |
| | Metabolic acidosis as defined by a base excess |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| | Protocol Amendment 4 Fin |
|---|---|
| | Neonatal invasive blood stream infections: bacterial/fungal/viral (continued) |
| Level | Description |
| 3 | Not meeting Level 1 or 2 of evidence |
| | AND |
| | Meeting 2 or more of the following criteria: |
| | • Temperature ≥37.5 ∘C or <35.5 ∘C |
| | Tachypnea or severe chest in drawing or grunting or cyanosis |
| | Change in level of activity |
| | History of feeding difficulty |
| | • History of convulsions |
| Laval | Bacterial/fungal/viral meningitis |
| Level | Description |
| 1 | Recognised pathogen identified using a validated method from cerebrospinal fluid (CSF) |
| 2 | CSF pleocytosis OR positive IgM antibodies to a specific pathogen in the CSF |
| | AND |
| | Recognised pathogen identified using a validated method from a normally |
| | sterile site (other than CSF) AND |
| | Temperature ≥37.5 ∘C or <35.5 ∘C |
| | AND |
| | 1 or more criteria below: |
| | History of convulsions |
| | •Lethargy or irritability |
| | •Coma |
| | •Apnea |
| | •Bulging fontanel |
| | •Neck stiffness |
| 3a | CSF pleocytosis |
| | AND |
| | No pathogen identified using a validated method from a normally sterile site AND |
| | Temperature ≥37.5 ∘C or <35.5 ∘C |
| | AND |
| | 3 or more criteria below: |
| | History of convulsions |
| | Lethargy or irritability |
| | • Coma |
| | • Apnea |
| | Bulging fontanel |
| | Neck stiffness |
| 3b | No lumbar puncture done or no sample available |
| | AND |
| | Temperature ≥37.5 °C or <35.5 °C |
| | AND |
| | 4 or more criteria below: |
| | History of convulsions |
| | Lethargy or irritability |
| | • Coma |
| | • Apnea |
| | Bulging fontanel Neal of the search |
| | Neck stiffness |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Respiratory bacterial/fungal/viral infection Tel Description |
|---------------------------------------------------------------|
| or interlobar |
| e |
| or oxygen |
| or interlobar |

Reference: Vergnano S, Buttery J, Cailes B, et al. Neonatal infections: Case definition and guidelines for data collection, analysis, and presentation of immunisation safety data. Vaccine. 2016;34 (49):6038-6046

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# Table 38 Respiratory Distress in the Neonate

Constellation of clinical findings that support the presence of breathing difficulty in the neonate (0-28 days of life), independent from etiology or severity, and independent from the infant's gestational age or circumstances at the time of delivery

| Level | Description |
|---|---|
| 1 | Newborn 0 to 28 days of life |
| | AND |
| | Abnormal respiratory rate: |
| | Measurement of number of breaths per minute consistent with: |
| | Tachypnea = respiratory rate of more than 60 breaths per minute |
| OR | |
| | Bradypnea = respiratory rate of less than 30 breaths per minute |
| | OR |
| | Apnea = cessation of respiratory effort (no breaths) for at least 20 seconds |
| | AND |
| | Clinical symptoms consistent with labored breathing: |
| | Nasal flaring (dilatation of alae nasi) |
| | OR STATE OF THE ST |
| | Noisy respirations in the form of expiratory grunting, stridor, or wheeze |
| | OR |
| | <ul> <li>Retractions or increased chest in-drawings on respiration (subcostal, intercostal, sternal,</li> </ul> |
| | suprasternal notch) |
| | OŘ |
| | Central cyanosis (whole body, including lips and tongue) on room air |
| | OR |
| | <ul> <li>Low Apgar Score (&lt; 7 points) at 10 min, with respiration score &lt;2</li> </ul> |
| | AND |
| | Examination and documentation by qualified, trained, health care provider appropriate for the clinical |
| | setting. |
| 2 | Newborn 0 to 28 days of life |
| | AND |
| | Abnormal respiratory rate: |
| | Not measured, but reported as "rapid breathing", "slow breathing", having periods of "no breathing", or |
| | "abnormal breathing" |
| | AND |
| | Clinical symptoms consistent with labored breathing: |
| | Nasal flaring (dilatation of alae nasi) |
| | OR |
| | Noisy respirations in the form of expiratory grunting, stridor, or wheeze |
| | OR |
| | Retractions or increased chest in-drawings on respiration (subcostal, intercostal, sternal, |
| | suprasternal notch) or seesaw respirations |
| | OR |
| | Central cyanosis (whole body, including lips and tongue) on room air |
| | OR |
| | Low Apgar Score (< 7 points) at 10 min, with respiration score <2 |
| | AND No modical record decumentation, but reporting through either a non-modical observer (e.g. mother |
| | <ul> <li>No medical record documentation, but reporting through either a non-medical observer (e.g. mother, father, community worker) or via standard census mechanisms (e.g. Demographic and Health</li> </ul> |
| | Surveillance System) OR |
| | Collection of information from medical record review or billing codes. |
| 3 | · · |
| | No need for a level 3 per working group. Not enough information to ascertain case of respiratory distress. |
| 4 | |
| 5 | Not a case of respiratory distress in the neonate. |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Reference: Leigh R. Sweet, Cheryl Keech, Nicola P. Klein, et al. Respiratory distress in the neonate: Case definition & guidelines for data collection, analysis, and presentation of maternal immunization safety data. Vaccine. 2017; 35: 6506-6517.

## Table 39 Preterm Birth

Birth in less than 37 gestation-completed weeks (less than 259 days).

| Prematurity and assessment of gestational age | |
|---|---|
| Level | Description |
| 1 | Certain last menstrual period date (LMP) LMP or intrauterine insemination (IUI) date or embryo transfer (ET) date with confirmatory 1st trimester scan (≤13 <sup>6/7</sup> weeks). OR 1st trimester scan (≤13 <sup>6/7</sup> weeks) |
| 2a | Certain LMP* with 2nd trimester scan (14 <sup>0/7</sup> weeks to 27 <sup>6/7</sup> weeks). Note: If LMP and U/S do not correlate, default to U/S GA assessment. OR Certain LMP* with 1st trimester physical examination. |
| 2b | Uncertain LMP with 2nd trimester scan (14 <sup>0/7</sup> weeks to 27 <sup>6/7</sup> weeks). |
| 3a | Certain LMP with 3rd trimester scan ≥ 28 <sup>0/7</sup> weeks OR Certain LMP with confirmatory 2nd trimester Fundal Height (FH) OR Certain LMP with birth weight OR Uncertain LMP with 1st trimester physical examination. |
| 3b | Uncertain LMP with FH. OR Uncertain LMP with newborn physical assessment. OR Uncertain LMP with Birth weight |
| * | Definitions of LMP, birth weight and physical assessment in referenced article. |

Reference: Quinn JA, Munoz FM, Gonik B, et al. Preterm birth: Case definition & guidelines for data collection, analysis, and presentation of immunisation safety data. Vaccine. 2016;34(49):6047-6056.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

### Table 40 Failure to Thrive

Failure to Thrive (FTT) can be broadly defined as a faltering of growth from a previously established pattern of growth. It is universally established that a diagnosis of failure to thrive should be based on anthropometric data. However no consensus exits as to which measurements achieve the highest specificity and sensitivity. Weight is generally regarded is the indicator of choice, particularly a change in growth velocity, and as such has been selected as the standard for this case definition with a weight for age deceleration as the primary indicator of failure to thrive. The case definition should be applied when there is no clear alternative diagnosis for the reported event to account for the combination of symptoms.

| Level | Description |
|---|---|
| 1 | Infant age <sup>1</sup> determined by a documented birth date |
| | AND |
| | Weights obtained using an electronic scale AND |
| | AND At least 2 weights, measured at least 4 weeks apart |
| | AND |
| | Weight for age deceleration <sup>2</sup> through at least 2 centile spaces on growth chart <sup>3</sup> |
| 2a | Infant age determined by a documented birth date |
| | AND |
| | Weights obtained using a beam balance scale AND |
| | At least 2 weights, measured at least 4 weeks apart |
| | AND |
| | Weight for age deceleration through at least 2 centile spaces on |
| | growth chart |
| | OR |
| | Infants with an undocumented birth date, where age is determined |
| | based on Mothers recall to nearest month |
| | AND Weights obtained using electronic scale |
| | AND |
| | At least 2 weights, measured at least 4 weeks apart |
| | AND |
| | Weight for age deceleration through at least 2 centile spaces on |
| Oh | growth chart |
| 2b | Infant age determined by a documented birth date AND |
| | Weights obtained using a spring balance scale |
| | AND |
| | At least 2 weights, measured at least 4 weeks apart |
| | AND |
| | Weight for age deceleration through at least 2 centile spaces on |
| | growth chart |
| | OR |
| | Weight measured using electronic scale or beam balance scale |
| | AND Length taken using Infantometer |
| | AND |
| | Weight for length less than or equal to the 3rd centile on the |
| | appropriate growth chart |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Level | Description |
|---|---|
| 3a | Infants with an undocumented birth date, where age is determined based on Mothers recall to nearest month AND |
| | Weight obtain using either beam balance or spring balance scale AND |
| | At least 2 weights, measured as least 4 weeks apart AND |
| | Weight for age deceleration through at least 2 centile spaces on growth chart |
| 3b | Infants with no weight available AND |
| | Physical examination consistent with FTT <sup>4</sup> AND |
| | MUAC <sup>5</sup> indicative of severe wasting |

<sup>&</sup>lt;sup>1</sup>This case definition is limited to infants up to 12 months of age.

- Weight should be documented on the appropriate growth chart at the time of assessment. A fall through 2 centile spaces may be demonstrated at any point in the first 12 months of life, using any two weights as long as they are taken at least 4 weeks apart. Details of use of the weight balances allowable under this case definition and use of the Infantometer for length assessment are presented in the reference given below.
- <sup>3</sup> For infants born at 37 weeks gestation or above, the WHO growth charts should be applied. When using weight for age use the growth chart most accurate for the infants age. The birth to 6 months age range should be used where data is available for this range only, the birth to 2 years chart should be used where data is available beyond 6 months of life. When using weight for length, use the chart for birth to 2 years. For infants born less than 37 completed weeks gestation, the Intergrowth charts for postnatal growth standards in preterm infant should be used. All infants should be plotted on their respective growth chart using their corrected age. Links to relevant growth charts are presented in the reference given below.
- <sup>4</sup> Physical examination with signs of Failure to Thrive (must include at least 2 findings, with at least one major finding) Major findings: Reduced subcutaneous fat stores; poor muscle mass; loose skin folds; prominent ribs; thin limbs Other less specific signs include: sparse hair; rashes; pallor; miserable; lethargy/fatigue.
- Mid Upper Arm Circumference (MUAC): For infants 0–6 months, a MUAC of 6 110 mm is indicative of severe wasting. For infants 6–12 months, a MUAC of 6 115 mm is indicative of severe wasting. Instructions on performing MUAC are presented in the reference given below.

Reference: Ross E, Munoz F, Edem B et al. Failure to thrive: case definition and guidelines for data collection, analysis, and presentation of maternal immunization safety data. Vaccine. 2017; 35:6483-6491.

Table 41 Standard Definitions for Neonatal Events of interest not defined as events in GAIA

| Event of Interest | Definition |
|---|---|
| Large for gestational age | Birth weight > 90% for newborns of same gestational age in same population (>4000g |
| | at term). |
| Macrosomia | BW >4000 g (8 lb, 13 oz). |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# APPENDIX E AMENDMENTS AND ADMINISTRATIVE CHANGES TO THE PROTOCOL

| GlaxoSmithKline Biologicals | |
|-------------------------------------------|--------------------------|
| Vaccines R & D | |
| Protocol Amendment 1 | |
| eTrack study number and Abbreviated Title | 207636 (EPI-RSV-008 BOD) |
| Amendment number: | Amendment 1 |
| Amendment date: | 12-FEB-2018 |
| Co-ordinating author: | , Lead Science Writer |

## Rationale/background for changes:

The protocol has been amended to reflect the following changes and provide the following clarifications / corrections.

- A separate screening visit has been added.
- Evaluations of GBS rectovaginal colonization of pregnant women, and the occurrence of GBS bacteremia/septicemia in their newborn infants, have been removed as study objectives.
- The Study Procedures Table and Detailed Descriptions of Study procedures have been updated both for consistency with these changes, and for improved consistency with the content of the electronic Case Report Forms for the study.
- Parents / LARs/designates are to contact the study site whenever:
  - the infant has developed symptoms of respiratory tract infection (RTI),
  - the infant has developed symptoms of difficulty in breathing or wheezing,
  - the infant's RTI symptoms have worsened,
  - the parent(s)/LAR(s) (or their designate(s)) are concerned about the infant's RTI signs and/or symptoms (parental concern).
- Text describing the content and use of the maternal health memory aid and the infant health and RTI memory aid has been updated and clarified.
- Additional editorial changes have been made to ensure consistency with the modifications noted above, and typographical errors have been corrected.

Text that has been moved or added is presented in **bold italics** and deleted text in strikethrough in the following sections.

## **Contributing Authors:**

- PPD , Clinical Research and Development Lead
- PPD , PPD , PPD , Epidemiologists

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

### **List of Abbreviations**

**GBS Group B Streptococcus** 

**ICH** International Conference on Council for Harmonisation

Glossary

Level 2 ultrasound (or fetal morphology

ultrasound)

Definition is unchanged. Only the label has been

adjusted, as noted on the left.

Neonatal events of

interest

Events as described in Section 11.1 that occur from

birth through 28 days of age.

Pregnancy related events

of interest

Events as described in Section 11.1 that occur from post-

enrolment Visit 1 through Visit 6 (Day 42).

The International Conference on Council for

Harmonisation (ICH) ......

Respiratory tract infection

(RTI) with parental concern:

Protocol amendment:

Any RTI for which the parents/ LAR(s) have visited or

plan to visit a medical health care practitioner.

End of Study (Synonym of End of Trial) For studies without collection of human biological samples or imaging data, EoS is the Last Subject Last

Visit (LSLV).

# **Synopsis**

Number of subjects

UpApproximatey 4000 pregnant women (up to approximately 400 pregnant women  $\geq 24^{0/7}$  weeks and  $\leq 28^{0/7}$  weeks of gestation are planned to be enrolled per country.) Neonates of enrolled pregnant women who consent to the infant's continued study participation will also be enrolled.

**Sampling** schedule for neonates/infants

During the 1-year post-birth surveillance period, for each RTI with suspicion of difficulty in breathing, or wheezing, or with parental concern, a nasal swab will be collected at the LRTI study visit a

visit to assess potential LRTIs

Background and Rationale (Section 1.1 and Synopsis "Rationale for the Study and Study Design")

....... There are also a number of maternal vaccines in development that aim to protect neonates and infants from additional pathogens, including respiratory syncytial virus (RSV) and group B streptococcus (GBS). GlaxoSmithKline (GSK) will enter Phase II with its-is developing an-investigational vaccine for use in pregnant women, against RSV disease. GBS vaccines are also being developed by GSK. Of note, these vaccines are developed solely for immunization in pregnancy.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Maternal immunization is implemented worldwide and has the potential to make a major contribution to reducing RSV lower respiratory tract infections (LRTI) GBS and other disease burden in infants globally.

Whilst there is good documentation of the global burden of RSV disease, incidence of RSV-LRTI according to the World Health Organization (WHO) 2015 case definitions [Modjarrad, 2016] is lacking in the literature. Hence, this study will also estimate the incidence of infant RSV-LRTI using WHO case definitions across geographically distinct locations to support incidence rate assumptions for planning of future efficacy trials. There are limited data on the prevalence of GBS rectovaginal colonization in pregnant women, by serotype, in different global settings and this study will aim to address this gap.

To achieve these goals, GSK will be guided by the WHO recommendations on antenatal care for a positive pregnancy experience [WHO, 2016] and the Global Alignment of Immunization safety Assessment in pregnancy (GAIA) case definitions [Bonhoeffer, 2016]. Standardisation of surveillance methodology and case definitions (applicable to maternal immunization AEs) may support comparison of data across different countries [Jones , 2016 Bauwens 2016; Bonhoeffer 2016; Kochhar 2017].

## **Rationale for the Study Population (Section 1.1.1 and Synopsis)**

.......Regardless of enrolment location, healthy pregnant women aged 18 to 40 years with normal, uncomplicated, singleton pregnancies, who have had a second trimesterlevel 2 (fetal morphology) ultrasound without any significant findings will be eligible for possible study participation. Inclusion / exclusion criteria have been structured in a way that resembles those of Phase II/III exclusion criteria to ensure good comparability

Pregnant women will be enrolled starting at  $24^{0/7}$  and up to (but not including)  $28^{0/7}$  weeks of gestation will be enrolled, to ensure that they are followed as of the time of potential vaccination in a clinical trial.

# Rationale for the Surveillance System for the detection of pregnancy related events of interest (Section 1.1.2)

..... Study Information obtained from study-specific procedures and laboratory testing tests (e.g. blood sampling, vaginal swabs, urine dipstick) will be performed for epidemiological purposes only; the information obtained from these procedures and tests is not to be relied upon for clinical management of study subjects.

### Rationale for the inclusion of GBS scrotyping and surveillance

In addition to RSV, GSK is developing a GBS maternal vaccine. GBS is the leading cause of neonatal sepsis globally, and disease can occur from the time of birth through 3 months of age. There is a need to address some of the GBS knowledge gaps and if possible prepare sites to detect GBS invasive disease. Aligned with this strategy, this study may collect vaginal swabs and blood samples to assess GBS colonization and serotypes, and antibody levels in maternal and cord blood. Data regarding occurrence of GBS invasive disease (sepsis, pneumonia and meningitis) may be collected through 90 days after birth, if possible. In case of suspected neonatal sepsis, pneumonia or

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

meningitis, GBS culture results will be documented if performed by a local healthcare provider. Because GBS testing results from study vaginal swabs will be performed only for epidemiological purposes and will not be available in time to inform clinical management, the GBS portion of this protocol will only be implemented in settings that have ongoing routine implementation of risk based intrapartum antibiotic prophylaxis for GBS. Vaginal swabs will only be performed in settings that adhere to this risk based approach for intrapartum antibiotic prophylaxis.

# Rationale for the use of Global Alignment of Immunization safety Assessment in pregnancy (GAIA) case definitions (Section 1.1.3)

GAIA, a Brighton collaboration project, aims to develop standardized case definitions and criteria for diagnostic certainty of maternal and neonatal outcomes in the context of immunization trials [Bonhoeffer, 2016] Bauwens 2016, Bonhoeffer 2016, Kochhar 2017].

## **Risk Assessment (Section 2.1)**

| Vaginal Nasal swab sample collection from infant subjects may cause discomfort | Spontaneous<br>data | Sample collection will only be performed by appropriately trained personnel. |
|---|---|---|
| may cause disconnoit | | Sample collection will only performed if amniotic membranes are intact |
| | | Subjects Subjects' parent(s)/LAR(s) will be notified of this risk in the informed consent form. |

### **Benefit Assessment (Section 2.2)**

.... Data collected during the study may enhance understanding of the incidence of maternal events of interest in women with low risk pregnancies, neonatal events of interest, GBS colonization and serotype distribution in pregnant women, GBS invasive disease in neonates and infants, and lower respiratory tract infections associated with RSV infection in neonates and infants.

### Overall Benefit / Risk Conclusion (Section 2.3)

Potential risks to subjects participating in this study are limited to those associated with the collection of biological specimens for analysis by the sponsor.

### **Primary Objectives (Section 3.1 and Synopsis)**

In healthy pregnant women with uncomplicated pregnancies at the time as of enrolment *Visit 1*:

# **Secondary Objectives (Section 3.2 and Synopsis)**

In healthy pregnant women with uncomplicated pregnancies at the timeas of enrolment *Visit 1*:

## **Tertiary Objectives (Section 3.3 and Synopsis)**

• To exploredescribe the association of other respiratory viruses with the occurrence of RSV-LRTI in infants.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- To evaluatedescribe the association between RSV-LRTI in infants and the level of RSV neutralizing antibodies in cord blood.
- To describe the prevalence of GBS vaginal colonization and serotype distribution in pregnant women in the 2nd and 3rd trimester and at delivery (if possible).
- To describe GBS serotype specific antibody concentrations in pregnant women in the 2nd and 3rd pregnancy trimester and at delivery (if possible)
- To describe GBS serotype specific antibody concentrations in cord blood (if possible)
- To describe the occurrence of GBS invasive disease in infants (if possible).
- To describe occurrences of hospitalization and death due to GBS invasive disease (if possible).

### Study Design Figure 1 and accompanying footnotes (Section 4.0)

These have been adjusted to include a screening visit, to clarify that urine dipstick testing will be done at study site visits 1 through 4, to remove references to sample collection for GBS testing, and to remove the reference to oral glucose challenge/tolerance testing. Footnotes have been renumbered for consistency with these changes.



### **Study Design Footnotes**

D = day; M = month; V = visit; W = week; Y = year. NB = newborn; GA = Gestational age; BS = blood sample; US = urine sample *for dipstick testing*; IMM = immune response; HB = hematology/biochemistry; *RBC* = *red blood cell(s)*; *WBC* = *white blood cell(s)*; RSV = respiratory syncytial virus; RTI = respiratory tract infection; LRTI = lower respiratory tract infection;

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- <sup>1</sup>Visits may be replaced by V5 depending on the date of. If delivery occurs prematurely, skip to Visit 5 ("at delivery").
- <sup>2</sup> At Delivery, RSV-A antibody titers for all women
- <sup>3</sup>Red blood cells, white blood cells will be recorded when available. Record positive results of any urine culture(s), if performed.
- <sup>4</sup>Results of Oral glucose challenge / oral glucose tolerance test(s) should be recorded, if performed by local healthcare provider and available.
- <sup>53</sup> At V3, only hemoglobin testing.
- <sup>64</sup> Blood sample should be collected within 72 hours after delivery.
- 75 RSV-A antibodies in cord blood
- <sup>86</sup>Neonatal conditions of interest occur (by definition) between 0 and 28 days after birth. They will be reported once site staff become aware of them (whether this occurs during the first 28 days after birth, or at a later time).

# Study population (Section 4.0 and Synopsis)

- Study population (per country): Up to (approximately) 400 pregnant women ≥24<sup>0/7</sup> and < 28<sup>0/7</sup> weeks of gestation (at the first study visit) will be enrolled; neonates of consenting parent(s) / LAR(s) will be enrolled at birth. The study will be conducted in up to approximately 10 countries. Study population: The study will be conducted in multiple countries, in pregnant women and their neonates.
- Thus the total study population will consist of up to (approximately) 4000 pregnant women and their neonates.

 Table 1 and Synopsis Table 1
 Sampling schedule for pregnant women/mothers

| | | Visit | | | | |
|---|---|---|---|---|---|---|
| Sample | Parameter(s) evaluated | 1 | 2 | 3 | 4 | Delivery |
| Maternal | Hematology/ biochemistry <sup>1,4</sup> | Х | | X <sup>23</sup> | | |
| Blood | Antibody titer (RSV-A) | X | | X | | ≤ 72 hours after delivery <sup>35</sup> |
| | Antibody concentration (GBS) | <del>X</del> <sup>4</sup> | | <del>X</del> <sup>4</sup> | | ≤ 72 hours after delivery <sup>3</sup> |
| Cord | Antibody titer (RSV-A) | | | | | Х |
| Blood | | | | | | |
| | Antibody concentration (GBS) | | | | | × |
| Urine | Protein <del>, glucose</del> <b>glucose</b> , <b>RBC</b> , | Х | Χ | Χ | Χ | |
| | WBC 2, 4 | | | | | |
| <b>Vaginal</b> | GBS vaginal colonization and | <del>X</del> 4 | | <del>X</del> <sup>4</sup> | | Before rupture of membranes |
| swab | serotypes | | | | | |

Haematology/biochemistry and urine protein/glucose testing will To be performed preferentially by local healthcare providers The, as per local practice. To be performed by the investigator/study staff will collect biological samples ONLY if not done by the local healthcare provider as per local practice. When available, within 2 weeks before the study visit.

• Sampling schedule for **neonates/infants**: During the 1-year post-birth surveillance period, for each RTI with suspicion of difficulty in breathing, or wheezing, or with parental concern, a nasal swab will be collected at the LRTI study visit a visit to assess potential LRTIs.

<sup>&</sup>lt;sup>2</sup> The investigator/site staff will perform a urine dipstick results for red blood cells (RBC) and white blood cells (WBC) will also be collected test using supplies provided by GSK.

<sup>&</sup>lt;sup>23</sup> Haemoglobin only

<sup>&</sup>lt;sup>3</sup>This 4 If results are abnormal, subjects will be referred per local standard of care.

<sup>5</sup>This sample may also be collected as from start of labor (e.g. when the mother arrives at the hospital to deliver and an intravenous line is inserted).

<sup>4</sup> only in countries with routine implementation of risk based intrapartum antibiotic prophylaxis for GBS

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- Primary Completion Date (PCD): 42 days post-delivery/birth (i.e. Visit 6 for the mothers and Visit 2-NB for the infants) or last visit of Epoch +002.
- Duration of the study: Approximately 4.5 to 6 months for all-participating pregnant women-enrolled; approximately 1 year for all-participating infants-enrolled.
  - Epoch 001: *Screening*
  - Epoch 002: Primary starting at Visit 1 and ending 42 days post-delivery/birth (Visit 6 for the mothers and Visit 2-NB for the infants).\*
  - Epoch <del>002</del>003: Follow-up of infants starting 43 days post-delivery/birth and ending at Visit 5-NB (1 year post-birth).

 Table 2 and Synopsis Table 2
 Study groups and epochs foreseen in the study

| Study | Number of subjects | Age (Min/Max) | Epochs | | |
|---|---|---|---|---|---|
| Groups | enrolled | | Epoch 001 | Epoch 002 | Epoch 003 |
| Mothers | Up to ~ 400 ( <del>by</del> <b>per</b> | 18 years - 40 years | • | • | |
| | country) | | | | |
| Infants | Up to ∼ 400 ( <del>by</del> <b>per</b> | NA | | • | • |
| | country) | | | | |
| To achiev | ve the enrolment targets no | oted above, the number | of pregnant wor | men SCREENEL | ) in each |

- To achieve the enrolment targets noted above, the number of pregnant women SCREENED in each country may exceed 400
- Surveillance for pregnancy outcomes and pregnancy-related events of interest .....from enrolment *Visit 1* up to 42 days after delivery.
- Surveillance for neonatal events of interest ..... *that occur* from birth up to 28 days of age.
- Surveillance for GBS invasive disease (refer to Section 8.6) in infants, from birth through 90 days of age.

## **Case Definitions – Neonatal Events of Interest (Section 5.2)**

### Invasive GBS disease

GBS invasive disease is a serious bacterial infection that requires urgent referral to a hospital. A lack of prompt diagnosis and treatment may lead to infant death. Diagnosis of a case of GBS invasive disease requires routine collection of blood/cerebrospinal fluid for culture, and a subsequent GBS positive local laboratory result.

Signs and symptoms of potentially serious bacterial infection that may be caused by GBS and lead to the routine collection of blood/cerebrospinal fluid for culture may include:

- not able to feed since birth or stopped feeding well (confirmed by observation)
- convulsions
- fast breathing (60 breaths per minute or more) among infants less than 7 days old
- severe chest in-drawing
- fever (38°C or greater)

<sup>\*</sup>Any safety and disease surveillance data collected after Visit 2-NB will be collected in Epoch <del>002</del> **003**.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- low body temperature (less than 35.5 °C)
- movement only when stimulated or no movement at all.

# Case Definitions – Respiratory Tract Infection (RTI) / Lower respiratory tract infection (LRTI) (Section 5.3)

During the *data* analysis of the study data, cases of respiratory tract infection (RTI) identified from birth up to 1 year of age will be classified according to the case definitions in Table 3.

**Footnote to Table 3:**  $SpO_2 = blood$  oxygen saturation *by pulse oximetry*.

## Study Population - Number of Subjects / Centres (Section 6.1)

- Up The study will be conducted at multiple centres in multiple countries. The total enrolled study population will consist of up to (approximately) 4004000 pregnant women ≥ and their neonates.
- In each participating country, up to (approximately) 400 pregnant women  $\geq 24^{0/7}$  weeks and  $\leq 28^{0/7}$  weeks of gestation are planned to will be enrolled per country. Neonates of enrolled pregnant women who consent to their child's study participation will also be enrolled.

### **Inclusion Criteria for Enrolment (Section 6.2)**

## **Pregnant Women**

- Healthy pregnant women 18-40 years of age who are ≥ 24 0/7 weeks GA at screening and < 28 0/7 weeks GA at Visit 1, as established by ultrasound examination and/or last menstrual period (LMP) date
- Women whose pregnancy is considered low risk at the time of enrolment, based on medical history, obstetric history, and clinical findings during the current pregnancy
- Women who had no significant findings (such as abnormal fetal morphology, amniotic fluid levels, placenta, or umbilical cord) observed during a Level 2 ultrasound *(fetal morphology assessment)* after 18-<sup>0</sup>24<sup>0/7</sup> weeks and prior to enrolment.
- HIV uninfected women who have been tested within the past year and have documented HIV negative test results at the time of enrolment.
- Individuals (mother or mother and father) who, at the time of enrolment/their informed consent t, express willingness to enroll their infant in the study at the time of birth.
- Individuals who, at the time of enrolment, are in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator;
- Individuals who, in the opinion of the investigator at enrolment can and will comprehend and comply with all study procedures (e.g., return for study follow-up visits, be contactable and available on a regular basis for surveillance).

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

### **Exclusion Criteria for Enrolment (Section 6.3)**

## **Pregnant Women**

- Individuals determined at the time of enrolment to have one of the following conditions associated with increased risk for a serious obstetrical complication (specify any/all that apply in the eCRF)
  - Gestational diabetes uncontrolled by diet and exercise as per American College of Obstetricians and Gynecologists guidelines (ACOG Practice Bulletin 2013);
- Individuals determined to have (during the current pregnancy, prior to enrolment) one of the following infections or conditions associated with risk of adverse outcome (specify any/all that apply in the eCRF):
- Individuals who at the time of enrolment have any underlying condition or infection that would predispose them to increased risk for a serious obstetrical complication that is not mentioned above
- Individuals who at the time of enrolment have behavioral or cognitive impairment or
  psychiatric disease that, in the opinion of the investigator, could interfere with the
  subject's ability to participate in the study;
- Individuals *who* at the time of enrolment have known or suspected impairment of the immune system, an active autoimmune disorder that is not well-controlled, or who are receiving systemic immunosuppressive therapy;

# **Subject Identification (Section 8.1)**

Subject numbers for both-pregnant women (mothers) eonsenting who consent to participate in the study and will be assigned at screening. Subject numbers for their (yet to be born) neonates will be assigned at Visit 1. They Subject numbers will be assigned sequentially according to the range of subject numbers allocated to each study centre. Subject numbers of mother –infant pairs will be clearly linked.

## **General Study Aspects (Section 8.2)**

Supplementary study conduct information not mandated to be present in this protocol is provided in the accompanying Study Procedures Manual (SPM).

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# **Outline of Study Procedures (Section 8.3)**

Potential study participants (pregnant women) are to be screened at  $\geq 24$  Weeks gestational age. Pregnant women for whom eligibility has been confirmed are to complete Visit 1 not later than at 27 67 weeks gestational age.

**Table 4, List of Study Procedures** (a new column – for the screening visit was added, and text was adjusted. Both the original Table and the revised Table are reproduced below.)

List of study procedures for pregnant women/ mothers (original protocol)

| Gestational age | <del>24 <sup>0/7</sup> - 27 <sup>6/7</sup></del> | <del>28 <sup>0/7</sup> - 31 <sup>6/7</sup></del> | 32 <sup>0/7</sup> - 35 <sup>6/7</sup> | 36-0/7 - delivery | - | - | |
|---|---|---|---|---|---|---|---|
| Epoch | | | | | | | |
| Type of contact | Visit 1 | Visit 2 <sup>-1</sup> | Visit 3-1 | Visit 4-1 | Visit 5 | Visit 6 <sup>2,3</sup> | Additional antenatal/medical evaluations (external to study visits/procedures) |
| Timepoints | <del>Day 1</del> | Day 28 | Day 56 | Day 84 | At Delivery | Post-Delivery<br>Day 42 | |
| Eligibility Review and Confirmation | | | | | | | |
| Informed consent | • | | | | | | |
| Check inclusion/exclusion criteria | • | | | | | | |
| Assign subject study number (mother) | • | | | | | | |
| Assign subject study number (child) | 0 | | | | | | |
| Inform study paediatrician and/or staff of subject's participation | Φ | | | | 0 | | |
| | | Medical Histo | ory / Examination | n <del>s</del> | | | |
| Distribute maternal health card | θ | | | | | | |
| Record demographic and lifestyle characteristics data | • | | | | | | |
| Collect medical history | • | | | | | | |
| Collect obstetric history from current and past pregnancies | • | | | | | | |
| Travel history to, or living in, Zika virus endemic countries/regions | • | | | | | - | |
| Inquire whether mother would have agreed to take part in the study if an investigational vaccine were given | • | | | | | | |
| Record outcome of 2d trimester Level 2 ultrasound | • | | | | | | |

29-MAY-2020 143
207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Gestational age | <del>24 <sup>0/7</sup> - 27 <sup>6/7</sup></del> | <del>28 <sup>0/7</sup> - 31 <sup>6/7</sup></del> | <del>32 <sup>0/7</sup> - 35 <sup>6/7</sup></del> | 36 <sup>0/7</sup> - delivery | _ | _ | |
|---|---|---|---|---|---|---|---|
| Epoch | | | 02 00 | Epoch 001 | | | |
| Type of contact | Visit 1 | Visit 2 <sup>1</sup> | Visit 3-1 | Visit 4-1 | Visit 5 | Visit 6 <sup>2,3</sup> | Additional antenatal/medical evaluations (external to study visits/procedures) |
| Timepoints | <del>Day 1</del> | Day 28 | Day 56 | Day 84 | At Delivery | Post-Delivery<br>Day 42 | |
| Record outcome(s) of subsequent ultrasounds if performed | • | • | • | • | | | • |
| Record gestational age, expected date of delivery and method of EDD estimation | • | | | | | | |
| Record height | • | | | | | | |
| Record weight | • | • | • | • | | • | • |
| Record results of antenatal physical examination | • | • | • | • | • | • | • |
| Check and record medications, vaccinations, folate | | | | | | | |
| and/or iron (independently or included in a multivitamin) beginning the month before the estimated date of conception and while on study | • | • | • | • | • | • | • |
| Conception and write on study | Biolo | gical Specimens | : / Laboratory Te | et Posults | | | |
| Collect blood sample for antibody assessment by sponsor (~5 ml) | <b>₽</b> -5 | giour opcomient | <b>⊕</b> _5 | St Neound | • | | |
| Collect cord blood for antibody assessment by sponsor (~5 to 10 ml) | | | | | • | | |
| Collect vaginal swab to send to sponsor for analysis, where relevant | <u>_</u> 5 | | <b>_</b> 5 | | • | | • |
| Record results of blood sampling for local hematology/<br>biochemical analysis (~10 ml).4 | - | | _ <b>_</b> 6 | | | | • |
| Record results of urine dipstick to check for presence of proteins, glucose 4,7 | • | - | - | - | | | • |
| Record results of oral glucose tolerance test if performed by local healthcare provider and available | • | • | • | • | | | • |
| Record outcome of urine bacterial culture if performed by local healthcare provider and available | • | • | • | • | | | • |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Gestational age | 24 <sup>9/7</sup> - 27 <sup>6/7</sup> | 28 <sup>0/7</sup> - 31 <sup>6/7</sup> | <del>32 <sup>0/7</sup> - 35 <sup>6/7</sup></del> | 36 <sup>0/7</sup> - delivery | - | _ | |
|---|---|---|---|---|---|---|---|
| Epoch | | | | Epoch 001 | - | | |
| Type of contact | Visit 1 | <del>Visit 2</del> <sup>4</sup> | Visit 3-1 | <del>Visit 4 ¹</del> | <del>Visit 5</del> | Visit 6 <sup>2,3</sup> | Additional antenatal/medical evaluations (external to study visits/procedures) |
| Timepoints | Day 1 | Day 28 | <del>Day 56</del> | Day 84 | At Delivery | Post-Delivery<br>Day 42 | |
| Record results of any peri-natal laboratory tests | | | | | | | |
| pertinent to assess maternal safety if performed by | • | • | • | • | • | • | • |
| local healthcare provider and available | | | | | | | |
| | | <del>Labo</del> | <del>r / Delivery</del> | | | | |
| Record date and time of rupture of membranes | | | | | • | | |
| Record type of delivery | | | | | • | | |
| Record gestational age determined at delivery | | | | | • | | |
| | | Outcomes and | d Events of Inter | est | | | |
| Record Pregnancy/Delivery outcome(s) | | | | | • | | |
| Record pregnancy-related events of interest (and | | | | | | | |
| hospitalisations / other clinically significant events or | | • | • | • | • | • | • |
| diagnoses that could impact the pregnancy | | | | | | | |
| | | Serious A | Adverse Events | | | | |
| Record SAEs related to study participation | • | • | • | • | • | • | • |
| | Study Conclusion | | | | | | |
| Study conclusion | | | | | | • | |
| Investigator sign-off on eCRF before analysis | | | | | | • | |

eCRF = electronic case report form; SAE = serious adverse event; WHO = World Health Organization.

- is used to indicate a study procedure that requires documentation in the individual eCRF.
- o is used to indicate a study procedure that does not require documentation in the individual eCRF.

<sup>&</sup>lt;sup>1</sup>The visit may be replaced by Visit 5 depending on the date of delivery.

<sup>&</sup>lt;sup>2</sup>Visit 6 (Day 42) may take place in the subject's home or at the investigator's clinical facility as appropriate to the circumstances in the judgment of the investigator.

<sup>3-</sup>To coincide with Visit 2-NB (Day 42) for infants.

<sup>&</sup>lt;sup>4</sup>To be performed preferentially by local healthcare providers, in which case the information will be collected and recorded in the eCRF. The investigator/study staff will provide these procedures if not done by the local healthcare provider as per local practice. If abnormal, subjects will be referred per local standard of care.

<sup>5-</sup>Only in countries with routine implementation of risk based intrapartum antibiotic prophylaxis for GBS

<sup>&</sup>lt;sup>6</sup> At Visit 3, only hemoglobin testing.

<sup>7-</sup>When available, urine dipstick results for red blood cells (RBC) and white blood cells (WBC) will also be collected

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# List of study procedures for pregnant women/ mothers (Amended 12 February 2018)

| Gestational age | ≥ 24 <sup>0/7</sup> - 27 <sub>6/7</sub> | 24 <sup>0/7</sup> –<br>27 <sup>6/7</sup> | 28 <sup>0/7</sup> - 31 <sup>6/7</sup> | 32 <sup>0/7</sup> -<br>35 <sup>6/7</sup> | 36 <sup>0/7</sup> -<br>delivery | | | |
|---|---|---|---|---|---|---|---|---|
| Epoch | Epoch 001 | | • | | - | Epoch 002 | | |
| Type of contact | Screening | Visit 1 | Visit 2 1 | Visit 3 ¹ | Visit 4 ¹ | Visit 5 | Visit 6 2, 3 | Additional<br>antenatal/medical<br>evaluations (external to<br>study visits/procedures) 4 |
| Timepoints | | Day 1 | Day 28 | Day 56 | Day 84 | At<br>Delivery | Post-<br>Delivery<br>Day 42 | |
| Eligibility Review and Confirmation | | | | | | | | |
| Informed consent | • | | | | | | | |
| Check inclusion/exclusion criteria | • | 0 | | | | | | |
| Assign subject study number (mother) | • | | | | | | | |
| Assign subject study number (child) | | 0 | | | | | | |
| Inform study paediatrician and/or staff of subject's | | 0 | | | | 0 | | |
| participation | L | | | | | | | |
| Medical History / Examinations | I | | | | 0 | | I | |
| Distribute maternal health <i>memory aid</i> | | 0 | 0 | 0 | 0 | 0 | | |
| Record demographic data | • | _ | | | | | | |
| Record lifestyle characteristics Record outcome of Level 2 ultrasound (fetal morphology scan) 7 | • | • | | | | | | |
| Record outcome(s) of subsequent ultrasounds if clinically significant <sup>4</sup> | | 0 | 0 | 0 | 0 | 0 | | • |
| Review and collect medical history | 0 | • | | | | | | |
| Review and collect obstetric history from past pregnancies | • | | | | | | | |
| Review and collect obstetric history from current pregnancy, including: gestational age, expected date of delivery and method of EDD estimation | • | | | | | | | |
| Travel history to, or living in, Zika virus endemic countries/regions | 0 | • | | | | | | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Ocatational and | ≥ 24 <sup>0/7</sup> · 27 | <b>24</b> <sup>0/7</sup> – | 28 0/7 - | 32 0/7 - | 36 <sup>0/7</sup> - | | | |
|---|---|---|---|---|---|---|---|---|
| Gestational age | 6/7 | <b>27</b> 6/7 | 31 <sup>6/7</sup> | 35 <sup>6/7</sup> | delivery | | | |
| Epoch | Epoch 001 | | | | | Epoch 002 | | |
| Type of contact | Screening | Visit 1 | Visit 2 <sup>1</sup> | Visit 3 <sup>1</sup> | Visit 4 ¹ | Visit 5 | Visit 6 2, 3 | Additional<br>antenatal/medical<br>evaluations (external to<br>study visits/procedures) 4 |
| Timepoints | | Day 1 | Day 28 | Day 56 | Day 84 | At<br>Delivery | Post-<br>Delivery<br>Day 42 | |
| Where authorized by the local Ethics Committee, inquire whether mother would have agreed to take part in the study if an investigational vaccine were given | | • | | | | | | |
| Record outcome of HIV test 9 | • | | | | | | | |
| Record results of <b>General and Obstetric</b> examination <sup>10</sup> | • | • | • | • | • | | • | <b>●</b> 13 |
| Check and record prescription medications, vaccinations, folate and/or iron (independently or included in a multivitamin) 12 | | • | • | • | • | • | • | |
| Biological Specimens / Laboratory Test Results | | | | | | | | |
| Collect blood sample for antibody assessment by sponsor (~5 ml) | | | | | | • | | |
| Collect cord blood for antibody assessment by sponsor (~5 to 10 ml) | | | | | | • | | |
| Record results of local hematology/ biochemical analysis (up to 10 ml) <sup>5</sup> | | • | | • 8 | | | | • 13 |
| Record results of urine dipstick to check for presence of proteins, glucose, RBC, WBC <sup>6</sup> | | • | • | • | • | | | • 13 |
| Record results of oral glucose challenge / tolerance test(s) if performed by local healthcare provider and available <sup>4</sup> | • | 0 | 0 | 0 | 0 | | | • |
| Record results of any clinically significant abnormal laboratory tests (including positive urine culture) if performed by local healthcare provider and available <sup>4</sup> | | 0 | 0 | 0 | 0 | 0 | 0 | • |
| Labor / Delivery | | | | | | | | |
| Collect and record labor and delivery information <sup>11</sup> | | | | | | • | | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Gestational age | ≥ <b>24</b> <sup>0/7</sup> - <b>27</b> <sup>6/7</sup> | 24 <sup>0/7</sup> –<br>27 <sup>6/7</sup> | 28 <sup>0/7</sup> - 31 <sup>6/7</sup> | 32 <sup>0/7</sup> - 35 <sup>6/7</sup> | 36 <sup>0/7</sup> -<br>delivery | | | |
|---|---|---|---|---|---|---|---|---|
| Epoch | Epoch 001 | Z1 | J 31 " | 33 ·· | delivery | Epoch 002 | | |
| Type of contact | Screening | Visit 1 | Visit 2 <sup>1</sup> | Visit 3 ¹ | Visit 4 ¹ | Visit 5 | Visit 6 2, 3 | Additional<br>antenatal/medical<br>evaluations (external to<br>study visits/procedures) <sup>4</sup> |
| Timepoints | | Day 1 | Day 28 | Day 56 | Day 84 | At<br>Delivery | Post-<br>Delivery<br>Day 42 | |
| Outcomes and Events of Interest | | | | | | | | |
| Record Pregnancy/Delivery outcome(s) | | | | | | • | | |
| Record pregnancy-related events of interest and other clinically significant events or diagnoses that could impact the pregnancy | | • | • | • | • | • | • | |
| Record all hospitalizations (except hospitalization for delivery), and all extensions of hospitalizations (including extension of hospitalization for delivery). | | • | • | • | • | • | • | |
| Serious Adverse Events | | | | | | | | |
| Record SAEs related to study participation | | • | • | • | • | • | • | |
| Screening/Study Conclusion | | | | | | | | |
| Screening conclusion | • | | | | | | | |
| Study conclusion | | | | | | | • | |
| Investigator sign-off on eCRF before analysis | • | | | | | | • ( ODE) | |

SAE = serious adverse event; • is used to indicate a study procedure that requires documentation in the individual electronic case report form (eCRF)

 $<sup>\</sup>circ\,$  is used to indicate a study procedure that does not require documentation in the individual eCRF.

<sup>&</sup>lt;sup>1</sup> If delivery occurs prematurely, skip to Visit 5 ("at delivery").

<sup>&</sup>lt;sup>2</sup> Visit 6 (Day 42) may take place in the subject's home or at the investigator's clinical facility as appropriate to the circumstances in the judgment of the investigator.

<sup>&</sup>lt;sup>3</sup> To coincide with Visit 2-NB (Day 42) for infants.

<sup>&</sup>lt;sup>4</sup> Information from additional antenatal / medical evaluations (external to study visits/procedures) may be collected during, before or after a scheduled study visit but should only be recorded in the additional antenatal/medical evaluations eCRF.

<sup>&</sup>lt;sup>5</sup> To be performed preferentially by local healthcare providers **as per local practice**. **To be performed by** the investigator/site staff **ONLY** if not done by the local healthcare provider **within 2 weeks before the study visit. If results are abnormal, subjects will be referred per local standard of care.** 

<sup>&</sup>lt;sup>6</sup> The Investigator/ site staff will perform a urine dipstick test to detect the presence of proteins, glucose, RBC and WBC.

<sup>&</sup>lt;sup>7</sup> If ultrasound results are not available at time of screening, the ultrasound can be performed as a study procedure under certain conditions. Refer to SPM for further details. If abnormal, subjects will be referred per local standard of care. [Table 4 Footnotes continue on the next page]

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### **Table 4 Footnotes Continued**

- 8 At Visit 3, only hemoglobin testing.
- <sup>9</sup> If HIV test results are not available at time of screening, the HIV test can be performed as a study procedure under certain conditions. Refer to SPM for further details. If results are positive, subject will be referred per local standard of care.
- 10 Height at screening. Weight, vital signs, fetal heart tones, fetal movement, and fundal height at Screening and Visits 1 4. Vital signs at Visit 6.
- 11 Includes date and time of rupture of membranes, date and time of delivery, type of delivery, and other delivery information related to the health and safety of the mother and fetus.

**Table 5, List of Study Procedures** (both the table from the original protocol and the amended table are reproduced below). **List of study procedures for neonates/ infants (original protocol)** 

| Epoch | Epc | och 001 | Epoch 002 | Epoch 00 | 2 |
|---|---|---|---|---|---|
| Age | 0-10 days | 4 <del>2 Days</del> | 12 months | 0-12 montl | <del>1S</del> |
| Type of contact | Visit 1-NB | Visit 2-NB a | Visit 3-NB a | Contact for active/ passive surveillance b | LRTI Assessment |
| Timepoints | Birth | Day 42 | <del>Y1</del> | | |
| Check inclusion/exclusion criteria | • | | | | |
| Obtain informed consent of parent(s)/LAR(s) | • | | | | |
| Record infant's subject number | • | | | | |
| Record Apgar assessment | • | | | | |
| Record demographic and lifestyle characteristics data | | • | | | |
| Distribute child health card | 0 | | | | |
| Distribute RTI episode card (memory aid) to record | 0 | | | | Ð |
| disease symptoms | | | | | |
| Physical examination including weight, length and head circumference | • | • | • | | |
| Record medications / vaccinations / vitamins | • | • | • | | |
| Record neonatal events of interest | • | • | • | | |
| Nasal swab | | | | | • |
| Record occurrences of GBS invasive disease (sepsis, | • | • | • | • | |
| pneumonia and meningitis) | | | | | |
| Record outcome of GBS blood or cerebrospinal fluid | • | • | • | • | |
| testing, if performed by a local healthcare provider | | | | | |

<sup>&</sup>lt;sup>12</sup> Beginning the month before the estimated date of conception and while on study. (Routine concomitant medications administered during labor and delivery need not be collected.)

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Epoch | Epo | och 001 | Epoch 002 | Epoch 002 | |
|---|---|---|---|---|---|
| Age | 0-10 days | 42 Days | 12 months | 0-12 months | |
| Type of contact | Visit 1-NB | Visit 2-NB-a | Visit 3-NB-* | Contact for active/ passive surveillance b | LRTI Assessment |
| Timepoints | Birth | Day 42 | ¥1 | | |
| Record all hospitalizations and/or clinically significant | • | • | • | • | <b>⊕</b> _d |
| events | | | | | |
| Record SAEs related to study participation | • | • | • | • | • |
| Study conclusion | | | • | | |
| Investigator sign-off on eCRF before analysis | | • | • | | |

eCRF = electronic case report form; GBS = Group B Streptococcus; LAR = legally acceptable representative; LRTI = lower respiratory tract infection; M = month; NB = newborn; RTI = respiratory tract infection; SAE = serious adverse event; Y = year

Grey shaded columns represent study procedures to be performed for active/passive surveillance of RTIs which are applicable throughout the entire study period (from birth up to study end).

Note: The double-line borders indicate primary analyses.

- is used to indicate a study procedure that requires documentation in the individual eCRF.
- e is used to indicate a study procedure that does not require documentation in the individual eCRF.
- a-Visit 2-NB (Day 42), Visit 3-NB (Year 1) and LRTI assessment visits may take place in the subject's home or at the investigator's clinical facility as appropriate to the circumstances in the judgment of the investigator, and if the standard of care allows home visits
- b-Supplemental information about invasive GBS disease and hospitalization will be solicited during select RTI active surveillance contacts in order to capture GBS events that occur within the first 90 days of life. Relevant medical record abstraction should be performed for identified occurrences.
- <sup>e</sup> If an LRTI assessment visit is conducted, a nasal swab is collected, and the parents return for a follow up LRTI assessment visit at which symptoms have diminished / resolved, no additional nasal swab need be collected. If an LRTI assessment visit is conducted, a nasal swab is collected, and the parents return for a follow-up LRTI assessment visit because symptoms have worsened, an additional nasal swab may be collected at the discretion of the investigator.
- d If not previously communicated during a surveillance contact

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# List of study procedures for neonates/infants (Amended 12 February 2018)

| Epoch | Epo | ch 002 | Epoch 003 | Epoch 002 and | Epoch 003 |
|---|---|---|---|---|---|
| Age | 0-10 days | 42 Days | 12 months | 0-12 mo | nths |
| Type of contact | Visit 1-NB | Visit 2-NB <sup>a</sup> | Visit 3-NB <sup>a</sup> | Contact for active/<br>passive<br>surveillance | Visit to<br>assess<br>potential LRTI |
| Timepoints | Birth | Day 42 | Y1 | | |
| Check inclusion/exclusion criteria | • | | | | |
| Obtain informed consent of parent(s)/LAR(s) | • | | | | |
| Record infant's subject number | • | | | | |
| Record Apgar assessment | • | | | | |
| Record demographic data | • | | | | |
| Record lifestyle characteristics | | • | | | |
| Distribute infant health and RTI memory aid | 0 | 0 | | | 0 |
| Weight, length, head circumference, results of targeted medical history, and results of physical examination | • | • | • | | |
| Record <i>prescription</i> medications / vaccinations | • | • | • | | • |
| Record neonatal events of interest | • | • | • | | |
| Clinical evaluation of potential LRTI | | | | | • |
| Nasal swab <sup>b</sup> | | | | | • b |
| Record all hospitalizations and/or clinically significant events | • | • | • | • | • |
| Record SAEs related to study participation | • | • | • | • | • |
| Study conclusion | | | • | | |
| Investigator sign-off on eCRF before analysis | | • | • | | |

LAR = legally acceptable representative; LRTI = lower respiratory tract infection; NB = newborn; RTI = respiratory tract infection; SAE = serious adverse event; Y = year. Grey shaded columns represent study procedures to be performed for active/passive surveillance of RTIs/LRTIs which are applicable throughout the entire study period (from birth up to study end). Note: The double-line borders indicate primary analyses. Footnotes to Table 5 continue on the next page. Table 5 footnotes continued

<sup>•</sup> is used to indicate a study procedure that requires documentation in the individual electronic case report form (eCRF).

o is used to indicate a study procedure that does not require documentation in the individual eCRF.

<sup>&</sup>lt;sup>a</sup> Visit 2-NB (Day 42), Visit 3-NB (Year 1) and LRTI assessment visits may take place in the subject's home (*if the standard of care allows for home visits*), at the investigator's clinical facility *or at another facility* per the investigator's judgment.

b If more than one assessment visit is conducted to evaluate a potential LRTI episode, additional nasal swabs may be collected at the discretion of the Investigator.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## **Intervals Between Study Visits/Contacts (Section 8.4)**

Table 6: Intervals between study visits/contacts/observations

| Interval | Optimal interval*** | Allowed interval** |
|---------------------|---------------------|--------------------|
| Screening → Visit 1 | 1 days | 0 – 28 days |

<sup>\*\*</sup>If a subject returns for the visit outside the recommended allowed time interval, he/she will may still be considered for the analysis.

Investigators should make at least 3 documented attempts (through telephone call(s) or any other convenient procedure) to contact (as relevant) the pregnant woman/mother or the child's parents/ LAR(s) (or their designates) if they do not return for scheduled visits or follow-up. Additional details can be found in the SPM.

# **Eligibility Review and Confirmation (Section 8.5.1)**

- Check all applicable inclusion and exclusion criteria as described in Sections 6.2 and 6.3 before enrolment and record results<del>for each criterion in the eCRF</del>.
- Assign / record subject study number (motherpregnant woman)
- Assign subject study number (infant) *for eligible pregnant women who complete Visit 1.*
- Inform study paediatrician and/or staff of subject's the *pregnant woman's* participation
  - A copy of the informed consent should be forwarded to the study paediatrician and/or staff as soon as possible after the subject's a pregnant woman's enrolment to ensure the study paediatrician is informed in a timely manner of the approximate date of delivery and potential enrolment of the neonate.

## History and Examinations for pregnant women/mothers (Section 8.5.2)

- Distribute maternal health card the Maternal Health Memory Aid. It is intended to serve as a reference during study visits/contacts, to help the subject provide the investigator/study staff with protocol-specified data (and contact information for other healthcare providers, so medical records may be requested if required). (Refer to the SPM for details).
- Record demographic and lifestyle characteristics data. Demographic data, which may include (but is not limited to) information such as race, month and year of birth, ethnicity, and geographic location. Lifestyle characteristics (exposures) may include data on factors such as smoking status/exposures, household environment and other factors that could place subjects at risk of study outcomes.
- Record information about lifestyle characteristics (exposures), which may include (but are not limited to) data on highest level of education, factors such as smoking status/exposures, household environment, and other factors that could place subjects at risk of study outcomes.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- Record outcome of 2d trimester (Level 2 ultrasound (fetal morphology assessment). Please see GLOSSARY OF TERMS for description. If Level 2 ultrasound results are not available at screening, then the ultrasound can be performed as a study procedure under certain conditions. Refer to the SPM for further details.
- Record outcome(s) of any subsequent ultrasoundsultrasound(s) ONLY if clinically significant. Record gestational age along with GAIA level of certainty using priorities defined in APPENDIX C
- Record expected date of delivery (EDD) and method of estimation
- Record medical / obstetric history
  - Obtain the subject's medical history by interview and/or review of her medical records; record any pre-existing conditions or signs and/or symptoms present before participation in the study. Targeted questions may be asked about allergies, respiratory diseases (including asthma) and other conditions that may be related to study outcomes.
  - Obtain the subject's obstetric history by interview and/or review of her medical records<del>record any data from current</del> and-.
  - For past pregnancies, record:
    - o number of past pregnancies and their outcome(s),
    - o presence of caesarian section scars (if any).
  - For the current pregnancy, record:
    - number of prenatal visits attended up to the date of the study Screening visit,
    - o approximate date of first prenatal visit,
    - o results of any clinically significant, abnormal pregnancy screening laboratory tests,
    - o results of any procedures intended to screen for congenital anomalies.

Inquire Where authorized by the local Ethics Committee, inquire whether mother would have agreed to take part in the study if an investigational vaccine were given and record the answer

- Record results of antenatal General and Obstetric examination

Unless the study visit is performed concurrently with a routine antenatal care visit inat which the below data are collected, the investigator/study staff should perform an antenatal physical examination: General and Obstetric examinations as follows:

- All visits through Screening, Visits 1 4, and Visit 6 should include assessment of vital signs (systolic/diastolic blood pressure, heart rate and respiratory rate after at least 10 minutes of rest);
- All visits through Visit 5-Screening and Visits 1 4 should include assessment of fetal heart tones, fetal movement, and fundal height;

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- Visit 1 should include assessment of any scars from prior deliveries.
- If the Screening Visit and Visit 1 occur on the same day, only one General and Obstetric examination will be performed.
- Record medications / vaccinations / folate and iron supplements beginning the month before the estimated date of conception and while on study(this includes medications administered during labor and delivery).
  - ONLY medications that are NOT routine should be recorded during labor and delivery.

**Biological Specimens** / **Laboratory Data** *for pregnant women/mothers* (Section 8.5.3) Blood samples for assessment of antibody titers/concentrations: An overall volume of approximately 155 mL

- Vaginal Swabs:
- In countries with routine implementation of risk based intrapartum antibiotic prophylaxis for GBS, vaginal swabs should be collected at Visits 1, 3, and 5 (prior to rupture of membranes). In countries without routine implementation of risk based intrapartum antibiotic prophylaxis for GBS, vaginal swabs should ONLY be collected at Visit 5 (prior to rupture of membranes).
- WHO does not currently recommend the use of vaginal swabs to screen for GBS colonization.
- The vaginal swabs collected in this study will be used solely for epidemiological purposes. Samples will be analyzed by a central testing laboratory and results will not be available for diagnostic purposes. Thus, vaginal swabbing conducted as a study procedure is not intended to replace local standard of care practices or to inform clinical management.
- The Investigator/site staff will arrange for collection of maternal blood and cord blood samples at delivery.
- The Investigator/site staff will perform urine dipstick tests using supplies provided by GSK.
- If HIV test results are not available at time of screening, the HIV test can be performed as a study procedure under certain conditions. Refer to the SPM for further details. If results are positive, the subject will be referred per local standard of care.
- It is preferred that local healthcare providers perform haematology and biochemistry tests per local practice; the investigator/site staff will perform these procedures then collect and record the results. The investigator/site staff will only perform haematology/biochemistry tests if not done by the local healthcare provider as per local practice within 2 weeks before a study visit.
  - Perform dipstick test for presence of proteins and glucose in urine. When available, red blood cell (RBC) and white blood cell (WBC) results will also be collected.
  - Perform HIV test at Screening (to assess eligibility)

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- If performed record by local healthcare provider and available, the investigator/site staff will also:
  - **Record** oral glucose **challenge** / **oral glucose** tolerance test results
  - If performed, record Record any positive urine bacterial culture results
  - Record abnormal and clinically significant laboratory test results
  - Record results of any laboratory tests pertinent to assess maternal safety Group
     B Streptococcus screening test(s).

# **Labor and Delivery (Section 8.5.4)**

Record information related to labor and delivery; should include the following:, *including*:

- Medications administered during labor and delivery (if not routine)
- Gestational age as determined at delivery

# Additional antenatal/medical evaluations General and Obstetric examinations (Section 8.5.7)

For any additional antenatal/medical evaluations *General and Obstetric examinations* at which a pregnancy related event of interest is identified, record information that supports the diagnosis of the event.

Medications, Vaccinations, and Supplements for pregnant women/mothers (Section 8.5.5)

- Record medications / vaccinations / folate and iron supplements beginning the month before the estimated date of conception and while on study.
  - Folic acid and/or iron supplements should be reported when taken independently and/or when included in a multivitamin mineral supplement.
  - ONLY medications that are NOT routine should be recorded during labor and delivery.

# Surveillance for Outcomes and Events of Interest in pregnant women/mothers (Section 8.5.6)

- Maternal events of interest (including, but not limited to, those described in Section 11.1.1) occurring up to Visit 6 (Post-delivery Month 1.5) should be recorded in the eCRF along with additional details pertinent to the diagnosis, GAIA assessment and level of diagnostic certainty (Appendix D), when applicable.
- Record all hospitalizations and/or clinically significant events.
- Record all study participation related SAEs as specified in Section 9.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## **Eligibility Review and Confirmation** for Neonates / Infants (Section 8.6.1)

- Check all applicable inclusion and exclusion criteria as described in Sections 6.2 and 6.3. A pre-selected child A *neonate* who does not meet the eligibility criteria should be considered ineligible.
- Obtain informed consent from parent(s) / LAR(s) at Visit 1-NB, and update as per local requirements.

# **History and Examinations for Neonates / Infants (Section 8.6.2)**

- Record demographic data-and lifestyle characteristics at birth, and any changes in this information at subsequent visits: Data includes, including date of birth, gender, race and ethnicity; living environment and household composition, breastfeeding, passive smoking and day-care attendance
- Record lifestyle characteristics. Data may include (but are not limited to) passive smoking and day-care attendance.
- Record weight, length, -and head circumference at birth and at subsequent study visits.and results of age-targeted medical history, and results of physical examination(s).
- Record *prescription* medications/ vaccinations vitamins
- Record all hospitalizations and/or clinically significant events. For hospitalizations where an RSV infection is suspected, refer to Section 8.6.6.
- Distribute Child the Infant Health CardA child health card will be distributed and RTI Memory Aid to the parent(s)/LAR(s)/designate(s) at Visit 1 NB if one is not already provided by). Health and RTI Memory Aid to the parent(s)/LAR(s)/designate(s). The memory aid is intended to serve as a reference during study visits/contacts, to help parent(s)/LAR(s)/designate(s) provide the investigator/study staff with protocol-specified data (and contact information for other healthcare providers, so medical records may be requested if required). Refer to the healthcare provider. SPM for additional details.
- Record all hospitalizations and/or clinically significant events. For hospitalizations where an RSV infection is suspected, refer to Section 8.6.6.
- Record all study participation related SAEs (Section 9).

# Surveillance for Invasive GBS disease (Deleted Section)

• To ensure that all GBS cases are captured, data regarding occurrence of GBS invasive disease (sepsis, pneumonialifestyle characteristics and meningitis) will be collected within the first year of life, with a particular emphasis being placed on the first 90 days. Instructions will be given to mothers and local health care providers (through child health cards) to contact the study staff any subsequent changes in case of occurrence of GBS invasive disease. Information regarding GBS blood testing in the neonates/infants will be collected if performed by a local healthcare provider. In order to identify potential GBS cases that occur beyond Visit 2 NB,this information about potential GBS invasive disease in the first 90 days of life will be solicited during LRTI active surveillance contacts (described in Section 8.5.5).

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

During the initial months of LRTI surveillance, supplemental questions related to invasive GBS disease. Data includes living environment and household composition, breastfeeding, passive smoking and hospitalization will be included with the LRTI script.

• In case of suspected neonatal sepsis, pneumonia or meningitis, the outcome of blood or cerebrospinal fluid test results for GBS should be documented in the infant's eCRF if performed by a local healthcare provider day-care attendance.

# **Surveillance for Neonatal events of interest (Section 8.6.3)**

• Investigators should make at least 3 documented attempts (through telephone call(s) or any other convenient procedure) to contact the child's parents/ LAR(s) (or their designates) if they do not return for scheduled visits or follow-up. Additional details can be found in the SPM.

Surveillance for *episodes of potential Lower Respiratory Tract Infection (LRTI)* (Section 8.6.4)

# **Definitions (Section 8.6.4.1)**

- Symptoms of Respiratory Tract Infection (RTI) include:
  - regular bursts of cough,
  - nasal discharge running freely out of the infant's nose (runny nose), or
  - breathing through the mouth because the infant's nose is blocked (blocked nose).
- An episode of potential lower respiratory tract infection (LRTI) is one in which the infant has one or more of the RTI symptoms listed above AND at least one of the following:
  - Difficulty in breathing (fast breathing, poor feeding, working hard to breathe, or making unusual sounds when breathing);
  - Wheezing (a whistling sound when the infant breathes out);
  - Parental concern (the parent(s)/LAR(s) or their designate(s) are concerned about the infant's respiratory tract illness or general health and intend to seek medical care).
  - An RTI episode starts on the day when (per parental report) the first RTI symptom started.
  - An RTI episode ends on the day when (per parental report) the last RTI symptom resolved.
  - There must be at least 7 symptom-free days between 2 consecutive RTI episodes.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## Overview (Section 8.6.4.2)

It will be accomplished via two types of contact. Both may be made with/by either the Parent(s)/LAR(s), or a person designated by the parent(s)/LAR(s), such as grandparents or a nanny (as long as the parent(s)/LAR(s) have given approval).

- *In an* Active, wherein *contact*, site personnel contact the subject's parent(s) / LAR(s) *or their designate(s)*. Active contacts will occur at regular intervals and will be scripted.
- In a Passive, wherein contact, the subject's parent(s) / LAR(s) or their designate(s) notify site personnel. Site personnel will use a script to guide data collection once a passive contact has been made.

Active and passive surveillance contacts can also be made with/by a person designated by the parent(s)/LAR(s) (e.g. grandparents, nanny) as long as the parent(s)/LAR(s) have given approval.

Site staff will use information gathered during each active or passive surveillance contact to determine whether a visit to assess a potential LRTI .....should be scheduled.

For all interactions between parent(s)/LAR(s)/designates and study staff, the safety of the infant is paramount. For any reported illness, the investigator/study staff should assess the need for any intervention and provide this as part of regular healthcare or instruct/advise the parent(s) / LAR(s) where to obtain this seek care as necessary. This study is not intended to replace local standards of care.

# Figure 2

Two footnotes have been deleted, and 4 footnotes have been added to the figure. Revisions to the footnotes are presented on this page. The figure itself is presented on the next page. In the figure, the phrase "Perform assessment visit within 3 days" has been changed to read "Perform assessment visit ideally within 3 days."

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final



RR: Respiratory rate: SpO<sub>2</sub>: Blood oxygen saturation by pulse oximetry...

Refer to the GLOSSARY OF TERMS for a definition of RTI with parental concern.

<sup>&</sup>lt;sup>1</sup> Refer to the Study Procedures Manual (SPM) for signs and symwardhanptoms to be collected.

<sup>&</sup>lt;sup>1</sup>Details regarding Active and Passive Surveillance are provided in Sections 8.6.4.3, 8.6.4.4, and the SPM.

<sup>&</sup>lt;sup>2</sup>Cough, runny nose, blocked nose, difficulty in breathing, wheezing and parental concern are defined in Section 8.6.4.1.

<sup>&</sup>lt;sup>3</sup>Details regarding the assessment visit to evaluate a potential LRTI are provided in Section 8.6.5and the SPM.

<sup>&</sup>lt;sup>4</sup> Post-visit follow up is described in Section 8.6.6 and in the SPM.

<sup>&</sup>lt;sup>5</sup>If a follow-up assessment visit is conducted, collection of additional nasal swabs are at the Investigator's discretion.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## **Active surveillance (Section 8.6.4.3)**

The purpose of the contact is to check with the infant's parent(s)/LAR(s) or their designate(s) if, *as defined in Section 8.6.4.1:* 

- the infant has developed (new-RTI symptoms (cough, runny nose or blocked nose),
- the infant has developed new) symptoms of RTI, difficulty in breathing, or wheezing

the parent(s)/LAR(s) (or their designate(s)) are concerned about the infant's RTI signs and/or symptoms (there is parental concernDuring active surveillance contacts, Parent(s)/LAR(s) (or their designates) will be reminded to record RTI symptoms, their start and stop dates, and any medications taken, on the RTI episode card.

## Passive Surveillance (Section 8.6.4.4)

Infants' parents/LAR(s) or their designate(s) will be instructed to contact the site whenever:

- theirthe infant has developed (new) symptoms of RTI, difficulty in breathing, or wheezing as defined in Section 8.6.4.1,
- they (the parent(s) / LAR(s) or their designate(s)) are concerned about the infant's RTI signs and/or-symptoms worsen
- there is parental concern as defined in Section 8.6.4.1.
- During passive surveillance contacts, Parent(s) /LAR(s) (or their designates) will be reminded to record RTI symptoms, their start and stop dates, and any medications taken, on the RTI episode card.

# **Decision to conduct a** *visit to assess a potential LRTI* (Section 8.6.4.5) **If there is** NO suspicion of difficulty in breathing, nor wheezing, nor parental concern:

• No <del>LRTI</del> assessment visit will be conducted.

**If there** <u>IS</u> difficulty in breathing, or wheezing (both based on parental assessment), or there is parental concern:

- The parent(s)/LAR(s) will be informed that their infant potentially has a(n) (new) LRTL.
- AnLRTI assessment visit will be conducted as soon as possible, ideally within 3 calendar days after learning of the potential LRTI case (Section 8.6.5).

If it is not possible to perform the clinical evaluation and collect a nasal swab during an assessment visit (for example, if the child develops a potential LRTI while the family is travelling), then the LRTI assessment visit page of the eCRF should be filled in as completely as possible using available medical records.

Visit to assess a potential LRTI (Section 8.6.5)

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## **Overview (Section 8.6.5.1)**

The visit may take place in the subject's home *(if allowed per standard of care)*, the investigator's clinical facility or another medical facility, as appropriate to the circumstances in per the judgment of the investigator.

Note that if the reported symptoms are of a level of severity that warrantssevere enough to warrant urgent care, the parent(s)/LAR(s)/designates should be advised to seek urgent such care (e.g. Emergency Room).

## Clinical evaluation (Section 8.6.5.2)

The investigator/study staff will evaluate the clinical signs and symptoms of the RTI. Signs and symptoms *Data to be collected and* recorded in the eCRF will be listed in the Study Procedures Manual (SPM).include (but are not limited to):

- Temperature
- Respiratory rate
- Blood oxygen saturation (measured by pulse oximetry in room air, if feasible)
- Signs of difficulty in breathing (including wheezing, tachypnoea, nasal flaring, chest in-drawing and apnoea)

Refer to the Study Procedures Manual (SPM) for additional details.

## Nasal Swab (Section 8.6.5.3)

## Follow up assessment

A nasal swab will be collected *using sponsor-provided supplies and sent to the sponsor laboratory* for detection of RSV-A/B using quantitative RT-qPCR.

If an LRTI-more than one assessment visit is conducted to evaluate a nasal swab is collected, and the parents return for a follow-up LRTI assessment visit at which symptoms have diminished / resolved, nopotential LRTI episode, additional nasal swab need be collected.

If an LRTI assessment visit is conducted, a nasal swab is collected, and the parents return for a follow-up LRTI assessment visit because symptoms have worsened, an additional nasal swabs may be collected at the discretion of the investigator Investigator.

Note: If other nasal swabs are collected and tested locally as per routine standard of care, results will be entered into the eCRF. However, only the sponsor laboratory results will be used when applying the case definitions for data analysis in Table 3.

## Missed assessment visit (Section 8.6.5.4)

Note that the visit may be conducted, and a nasal swab collected, as long as symptoms are ongoing.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

If it is truly not possible to perform an assessment visit (for example, if the child develops a potential LRTI while the family is travelling, and all symptoms have resolved by the time the family returns), then the LRTI assessment visit page of the eCRF should be filled in as completely as possible using available medical records.

Follow-up after an assessment visit to evaluate a potential LRTI (Section 8.6.6) After an assessment visit (Section 8.6.5) the infant will be followed with at least weekly active surveillance contacts, until the RTI/LRTI episode has resolved. During these active contacts, worsening of symptoms will be assessed. Parent(s) / LAR(s) / designate(s) will be reminded to call/contact/visit the site if symptoms worsen.

If parent(s)/LAR(s)/designates report during an active or passive contact that symptoms have worsened, the site should perform a follow-up visit.

During the follow-up visit, collection of a nasal swab is at the Investigator's discretion. Additional details can be found in the SPM.

# **RSV Hospitalization (Section 8.6.7)**

- Study staff will collect *If possible*, a nasal swab will be collected from any subject who has been is hospitalized with a RTI (or soon after release, as long as symptoms are ongoing, per SPM specifications). The nasal swab should be collected using sponsor-provided supplies, for transmission to and testing by the sponsor laboratory.
- In order to establish a fast and accurate diagnosis, collection (using locally providedlocal supplies) of an additional nasal swab for testing at a local laboratory is recommended.
- If other specimens are collected and tested locally as per routine standard of care, results will be entered into the eCRF. However, only the sponsor laboratory results will be used when applying the case definitions for data analysis in Table 3.

## **Baseline Screening failures (Section 8.9)**

Baseline Screening failures are defined as subjects who withdraw or are withdrawn from the study after giving informed consent, but before study eligibility (presence of all inclusion and absence of all exclusion criteria) is confirmed. The Day 1 discovery Discovery during screening of any pregnancy related-event of interest or other condition that violates the requirements for study enrolmenteligibility should be considered to be a baseline screening failure. Discovery during Visit 1 of any condition that violates the requirements for study eligibility should also be considered a screening failure.

The subsequent development of such conditions (after DayVisit 1) aredoes not baseline failuresconstitute screening failure and should be captured on the eCRF, as applicable.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Limited data for screening failures will be reported to the eCRF. This limited data set is specified in the eCRF. for screening failures will be limited to:

- ICF information
- Demographic data
- Inclusion/Exclusion criteria
- Level II /Fetal Morphology Ultrasound
- Screening conclusion data
- Study conclusion data.

Medical history and OB/GYN physical assessment data (including height, weight and vital signs) do not need to be reported to the eCRF.

**Table 7 Biological samples** 

| Sample Type <sup>†</sup> | Quantity | Unit | Timepoint | Group |
|---|---|---|---|---|
| Sam | ples collected | by Inves | stigator / site staff | |
| Maternal Blood for antibody titers | ~-5 | ml | Visit 1 (Day 1) <sup>1</sup> 5 (Delivery) | All mothers in |
| | <del>~ 5</del> | ml | <del>Visit 3 (Day 56)</del> <sup>1</sup> | selected countries |
| | ~ 5 | ml | Visit 5 (Delivery) | All pregnant |
| | | | | women (mothers) |
| <del>Vaginal swab</del> | - | - | <del>Visit 1 (Day 1)¹</del> | All mothers in |
| | - | - | <del>Visit 3 (Day 56)¹</del> | selected countries |
| | - | - | <del>Visit 5 (Delivery) <sup>2</sup></del> | All mothers |
| <del>Nasal swab</del> | - | - | LRTI Assessment visit | All infants, event- |
| | | | | <del>driven</del> |
| Urine (dipstick)1 | - | - | Visit 1 (Day 1) | AII |
| | | | Visit 2 (Day 28) | pregnant women |
| | | | Visit 3 (Day 56) | (mothers) |
| | | | Visit 4 (Day 84) | |
| Cord blood | ~ 5 up to | ml | Visit 5 (Delivery) | All <b>pregnant</b> |
| | 10 | | | women (mothers) |
| | | | | (provides infant |
| | | | | antibody levels) |
| Nasal swab | - | - | LRTI Assessment visit | All infants, event- |
| | | | | driven |
| | collected by l | ocal hea | Ith care provider per local prac | tice <sup>1</sup> |
| Maternal Blood for haematology/ | Up to 10 | ml | Visit 1 (Day 1) | All <b>pregnant</b> |
| biochemistry | | | | women (mothers) |
| | Up to 10 | ml | Visit 3 (Day 56) <sup>2</sup> | |
| Urine (dipstick) | - | - | Visit 1 (Day 1) | All |
| , | | | <del>Visit 2 (Day 28)</del> | <del>(mothers)</del> |
| | | | <del>Visit 3 (Day 56)</del> | , , , |
| | | | <del>Visit 4 (Day 84)</del> | |
| | | | <del>Visit 5 (Delivery)</del> | |

<sup>&</sup>lt;sup>4</sup>Only in countries where routine implementation of risk based intrapartum antibiotic prophylaxis for GBS is the standard of care

<sup>&</sup>lt;sup>2</sup>Vaginal swab at delivery will only be collected prior to rupture of membranes.

<sup>&</sup>lt;sup>3</sup>Performed <sup>1</sup> To be performed preferentially by local healthcare providers, as per local practice. **To be performed by** the investigator/study staff **ONLY** if not done by the local healthcare provider **within 2 weeks before the study visit**.

<sup>&</sup>lt;sup>2</sup> Hemoglobin only

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## **Antibody determination (Section 8.10.3.1)**

 Testing for GBS antibody concentrations will be performed upon availability of assay.

Table 8 Humoral immunity (Antibody determination)

| System | Component | Method** | Kit / | Unit | Cut-off* | Laboratory** |
|---|---|---|---|---|---|---|
| | | | Manufacturer | | | |
| SERUM | Respiratory<br>Syncytial<br>Virus A Ab | NEUTRALISATION | In house | ED60 | To be defined | GSK Biologicals or GSK designated lab*** |
| SERUM | GBS | To be defined | To be defined | <del>To be</del> | To be | GSK Biologicals or GSK |
| | <del>antibody</del> | | | defined | defined | designated lab*** |

# **GBS** assessment of vaginal swabs

GBS vaginal colonization will be assessed by culture and/or molecular biology methodologies (GSK Biologicals or GSK designated laboratory) upon assay availability. If available, local laboratory results on GBS colonization will also be recorded in the eCRF.

The method that will be used to perform GBS serotyping remains to be determined (will be done at GSK Biologicals or by a GSK designated laboratory).

Table 10 GSB assessment of vaginal swabs\*

| Vaginal swab sampling timepoint Type of contact (timepoint) | Component | Method | Scale | Laboratory |
|---|---|---|---|---|
| Visit 1 (Day 1)*** Visit 3 (Day 56)*** Visit 5 (Delivery)** | <del>GBS</del> | To be determined | To be<br>determined | GSK Biologicals<br>or GSK<br>designated lab** |

<sup>\*</sup>Laboratory assays for GBS assessment of vaginal swabs to be confirmed (may be assessed by culture and/or molecular biology).

## Haematology, biochemistry and urinalysis (Section 8.10.3.3)

Haematology and biochemistry and urinalysis will tests are to be performed preferentially requested by local health carehealthcare providers. Information will, as per local practice. They are to be collected and recorded in the eCRF. If performed by the investigator/study staff ONLY if not done by the local healthcare provider as per local practice within 2 weeks before the investigator study staff visit.

The investigators will perform a urine dipstick test to detect for the tests specified in Table 10 presence of proteins, glucose, RBC and/or WBC.

<sup>\*\*</sup> Vaginal swab at delivery will only be collected prior to rupture of membranes.

<sup>\*\*\*</sup>Only in countries where routine implementation of risk based intrapartum antibiotic prophylaxis for GBS is the standard of care

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Table 10 Hematology, biochemistry, urine tests

| System | Discipline | Component | Time<br>point | Method | Scale | Laboratory |
|---|---|---|---|---|---|---|
| Whole<br>blood | Hematology | Hemoglobin | Visit 1 | As per local | Quantitative | Local laboratory |
| | | | Visit 3 | practice | | |
| | | Leukocytes (White Blood Cells) | Visit 1 | | | |
| | | Platelets | Visit 1 | | | |
| Serum | Biochemistry | Alanine<br>Aminotransferase<br>(ALT) | Visit 1 | As per local practice | ocal | Local<br>laboratory |
| | | Aspartate<br>Aminotransferase<br>(AST) | Visit 1 | | | |
| | | Creatinine | Visit 1 | | | |
| | | Urea Nitrogen | Visit 1 | | | |
| Urine | - | Protein | Visit 1 | As per | Ordinal | Local |
| | | | Visit 2 | local | | laboratory |
| | | | Visit 3 | practice, | | |
| | | | Visit 4 | dipsticks | | |
| | | Glucose | Visit 1 | provided | | |
| | | | Visit 2 | by GSK | | |
| | | | Visit 3 | Biologicals | | |
| | | | Visit 4 | | | |
| | | Hemoglobin | Visit 1 | | | |
| | | (RBC) | Visit 2 | | | |
| | | | Visit 3 | | | |
| | | | Visit 4 | | | |
| | | Leukocyte esterase | Visit 1 | | | |
| | | (WBC) | Visit 2 | | | |
| | | | Visit 3 | | | |
| | | | Visit 4 | | | |

<sup>&</sup>lt;sup>4</sup> When available, urine dipstick results for RBC and WBC will also be collected.

Table 11 Immunological read-outs

| Blood sampling timepoint | Group | | No. subjects | Component | Component priority rank |
|---|---|---|---|---|---|
| Type of contact and time point | | | | | |
| | | Materna | al Blood | | |
| Visit 1 (Day 1)** | All mothers in countrice | | ~400 maximum by country | GBS* | 1 |
| Visit 3 (Day 56)** | All mothers in selected countries | | ~400 maximum by country | GBS* | 1 |
| Visit 5 (Delivery) | | | | <del>GBS*</del> | 2 |
| | Cord Blood | | | | |
| Visit 5 (Delivery) | | · | | <del>GBS*</del> | <del>2</del> |

**GBS** = group B streptococcus; **RSV-A/B** = Respiratory syncytial virus subtype A/B.

<sup>&</sup>lt;sup>2</sup> Culture results will be obtained, if performed

<sup>\*</sup> Testing for GBS antibody concentrations will be performed upon availability of assay.

<sup>\*\*</sup>Only in countries where routine implementation of risk based intrapartum antibiotic prophylaxis for GBS is the standard of care

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

In case of insufficient blood sample volume to perform assays for all antibodies, the samples will be analysed according to the priority ranking provided in Table 11.

Table 12 Molecular biology for nasal swab specimen analysis

| Nasal swab sampling timepoint | | Crown | No aubicata |
|---|---|---|---|
| Type of contact (timepoint) | Sampling timepoint | Group | No. subjects |
| Visit to assess potential LRTI Assessment visit | Unscheduled | All infants* | Event-driven** |

Footnotes

## Table 13 Hematology/blood chemistry tests (footnotes only)

\* Number of subjects depending on country. Prenatal screening will Tests to be performed preferentially by local healthcare providers and information will be collected and recorded in the eCRF. The investigator/study staff will collect biological samples for prenatal screening the specified testing if not done by the local healthcare provider as per local practice.

# GBS assessment of vaginal swabs (Deleted Section)

Table 15 GSB assessment of vaginal swabs\*

| Vaginal swab sampling timepoint Type of contact (timepoint) | Group | No. subjects | Component |
|---|---|---|---|
| Visit 1 (Day 1)*** | All mothers, selected countries*** | ~400 maximum by country | <del>GBS*</del> |
| Visit 3 (Day 56)*** | All mothers, selected countries**** | ~400 maximum by country | <del>GBS*</del> |
| Visit 5 (Delivery)** | All mothers | ~400 maximum by country | GBS* |

<sup>\*</sup>Laboratory assays for GBS assessment of vaginal swabs to be confirmed (may be assessed by culture and/or molecular biology).

## **Event Identification (Section 9.2)**

Blood<del>, urine and vaginal swab</del>urine samples will be collected from pregnant women enrolled in the study. Nasal

## **Subject withdrawal (Section 10.2)**

Investigators will make an attempt at least 3 attempts to contact those subjects asubject who dodoes not return for a scheduled visits visit or follow-up as described in Section 8.4 and in the SPM.

A subject will be defined as lost to follow-up if there is no contact with the subject /subject's parent(s) / LAR(s) over a period of *at least 3 months after a planned visit* (see SPM for details). Efforts to contact the subject/subject's parents should be recorded in the

<sup>\*</sup>For each RTI with suspicion of difficulty in breathing, wheezing or parental concern reported during an active or passive surveillance contact a nasal swab will be collected. A nasal swab will also be collected at the examination visit performed in case parents/ LAR(s) come to the study site without previous surveillance contact (if RTI with suspicion of difficulty in breathing, wheezing or parental concern, and visit within 3 days after the start of symptoms).

<sup>\*</sup> Refer to Section 8.6.5.

<sup>\*\*</sup> Vaginal swab at delivery will only be collected prior to rupture of membranes.

<sup>\*\*\*</sup>Only in countries where routine implementation of risk based intrapartum antibiotic prophylaxis for GBS is the standard of care

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

source documents. The subject's data will be censored at the time of last contact once this definition is met.

Information relative *relevant* to the withdrawal will be documented in the eCRF. .....as well as which of the following possible reasons was responsible for withdrawal:

- Study procedure participation related SAE.
- Neonatal event of interest (specify). Note: includes death in infants *from* birth 28 days old
- Death in infants > 28 days old (specify cause). Note that death in neonates *from* birth -28 days old is captured as a neonatal event of interest).

Subjects who are withdrawn from the study because of *study participation related SAEs* must be clearly distinguished from subjects who are withdrawn for other reasons. Investigators will follow subjects who are withdrawn from the study as result of ana *study participation related* SAE until resolution of the event (see Section 9.6.2).

# Primary endpoints (Section 11.1.1), Primary Objectives Analysis (Section 11.6) and Synopsis

- Hypertensive disorders of pregnancy:
  - o gestational hypertension, and
  - o Pre-eclampsia, and
  - o Pre-eclampsia with severe features (including eclampsia),
- Neonatal Acute neonatal encephalopathy

# Secondary endpoints (Section 11.1.2), Secondary Objectives Analysis (Section 11.7) and Synopsis

Occurrence of nneonatal events of interest from birth through Day 28 days of age (as defined in primary endpoints) for each GAIA level of diagnostic certainty (where applicable and feasible)

# Tertiary endpoints (Section 11.1.3), Tertiary Objectives Analysis (Section 11.8) and Synopsis

- Human respiratory syncytial virus A (RSV A)
- Human respiratory syncytial virus B (RSV B)

# Exposed Set (ES) – pregnant women (mothers) (Section 11.3.1.1)

The ES will include all pregnant women (mothers) with a valid informed consent<del>form</del> who were enrolled in the study.

# Per Protocol Sets (PPS) – pregnant women (mothers) and Neonates/Infants (Sections 11.3.2)

The *maternal* PPS will include all pregnant women (mothers)

The *infant* PPS will include all enrolled neonates / infants

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## Derived and transformed data (Section 11.4)

Age of the *infant* subject at time of the LRTI case will be expressed in months and will be computed as the difference between the start date of the LRTI case and the date of birth

Age of the subject at time of blood sample collection will be expressed in months and will be computed as the difference between the sample collection date and the date of birth.

# Analysis of demographic and baseline characteristics (Section 11.5)

- For the ES and maternal PPS cohorts, the cohort, analyses of demographic analyses for pregnant women and baseline characteristics at Visit 1 will describe be described.
- For the infant PPS cohort, analyses of demographic characteristics of women at visit 1-nt Visit 1-NB will be described. Analyses of lifestyle characteristics will be described at Visit 2 NB.
- For the ES and PPS cohorts, the overall demographic analyses for neonate / infants will describe the demographic characteristics of the neonate / infants at visit 1-NB.
- For Screening Failures, reasons for non-eligibility will be described.

# Analysis of primary objectives (Section 11.6)

The primary objectives analyses will be performed on the PPS cohorts by country, and possibly by region or other relevant grouping are excluded from the PPS cohort then the analyses may be performed on the ES cohort.

## **Analysis of secondary objectives (Section 11.7)**

The secondary objectives analyses will be performed on the PPS cohorts (maternal or infant as applicable) overall by country and possibly by region or other relevant grouping. In case more than 5% of the subjects are excluded from the PPS cohort then the analyses may be performed on the ES cohort.

## **Analysis of tertiary objectives (Section 11.8)**

The following tertiary objectives analyses will be performed on infants within the PPS cohort overall by country, region, or other relevant grouping. In case more than 5% of the subjects are excluded from the PPS cohort then the analyses may be performed on the ES cohort:

The following tertiary objectives analyses will be performed on the PPS cohorts (maternal or infant as applicable) by country, region, or other relevant grouping. In case more than 5% of the subjects are excluded from the PPS cohort then the analyses may be performed on the ES cohort:

To describe GBS scrotype specific antibody concentrations in cord blood (if possible).

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- Geometric mean titers (GMTs) will be tabulated with 95% CI.
- Percentage of subjects above thresholds will be tabulated.

The following tertiary objectives analyses will be performed on pregnant women (mothers) within the PPS cohort overall by country, region, and/or other relevant grouping:

- To describe the prevalence of GBS vaginal colonization and serotypes
  distribution in pregnant women in the 2nd and 3rd trimester and at delivery (if
  possible).
  - The proportion of women colonized with GBS by serotype at each timepoint will be calculated. The proportion of colonized women will be calculated as the number of women having a positive result for GBS divided by the number of women for whom a vaginal swab has been taken. This will be presented overall and by serotype.
- To describe GBS scrotype specific antibody concentrations in pregnant women in the 2nd and 3rd trimester and at delivery (if possible).
  - For each serotype-specific GBS Concentration in serum of mothers and in cord blood the following analysis will be performed:
    - The proportion of women with serotype specific antibody concentrations above various thresholds will be calculated overall and by colonization status.
    - GMCs for each serotype will be calculated overall and by colonization status
    - Variation in colonization status and antibody titers will be calculate for each timepoint, when feasible.

The following tertiary objectives analyses will be performed on neonates / infants within the PPS cohort overall by country, region, or other relevant grouping:

- To describe the occurrence of GBS invasive disease in infants (if possible).
  - Incidence proportions will be calculated as the number of new invasive GBS disease cases occurring from birth up to 90 days of life (if feasible) divided by the number of infants included in the study.
  - Incidence proportions will be categorized as follows: early onset disease (during days 1-7) and late onset disease (during days 8-90) (if data available; i.e., depending on whether GBS blood and / or CSF testing is done as per local practice).
- To describe occurrences of hospitalization and death due to GBS invasive disease (if possible).
  - Incidence proportions will be calculated as the number of new hospitalizations due to GBS disease cases occurring from birth up to 1 year of life (if feasible) divided by the number of infants included in the study.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- Incidence proportions will be calculated as the number of new deaths due to GBS disease cases occurring from birth up to 1 year of life (if feasible) divided by the number of infants included in the study.
- Incidence proportion will categorized as follows: early onset disease (during days 1-7), late onset disease (during days 8-90), and post-late onset disease (≥91 days) (if data available; i.e., depending on whether GBS blood and / or CSF testing is done as per local practice).

# **Conduct of analyses (Section 11.11)**

Analyses will be performed in a stepwise manner after each country / group of countries / countries in a region have completed all study visits in Epoch 001 002 and again after completion of all study visits in Epoch 002 003.

Analyses of pregnancy outcomes, pregnancy related events of interest, and neonatal events of interest will be performed when all data up to 42 days post-delivery are available (Epoch 001002).

Final analyses will be performed when all data up to study end are available (Epoch 001002 and Epoch 002003).

Interim-Additional analyses may be performed if deemed necessary to inform the design or implementation of future clinical trials

## **References (Section 14)**

Barbas CF, Crowe JE, Cababa D, et al. Human monoclonal Fab fragments derived from a combinatorial library bind to respiratory syncytial virus F glycoprotein and neutralize infectivity. Proc Natl Acad Sci U S A. 1992;89(21):10164-8.

Bates JT, Keefer CJ, Slaughter JC, et al. Escape from neutralization by the respiratory syncytial virus-specific neutralizing monoclonal antibody palivizumab is driven by changes in on-rate of binding to the fusion protein. Virology. 2014; 454-455:139-144.

Bauwens J, Bonhoeffer J, Chen RT, editors. Harmonising Immunisation Safety Assessment in Pregnancy. Vaccine. 2016. 34 (49): 5991 – 6110.

DaSilva FT, Gonik B, McMillan M, et al. Stillbirth: Case definition and guidelines for data collection, analysis, and presentation of maternal immunization safety data. Vaccine. 2016;34(49):6057-6068.

DeSilva M, Munoz FM, Memillan M, et al. Congenital anomalies: Case definition and guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2016;34(49):6015-6026.

Gravett C, Eckert LO, Gravett MG, et al. Non-reassuring fetal status: Case definition & guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2016;34(49):6084-6092.

Harrison MS, Eckert LO, Cutland C, et al. Pathways to preterm birth: Case definition and guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2016;34(49):6093-6101.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Kochhar S, Bauwens J, Bonhoeffer J, editors. Harmonising Immunization Safety Assessment in Pregnancy – Part II. Vaccine. 2017. 35 (48): 6469-6582.

Kerr R, Eckert LO, Winikoff B, et al. Postpartum haemorrhage: Case definition and guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2016;34(49):6102-6109.

Pathirana J, Muñoz FM, Abbing-Karahagopian V, et al. Neonatal death: Case definition & guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2016;34(49):6027-6037.

Patwardhan M, Eckert LO, Spiegel H, et al. Maternal death: Case definition and guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2016;34(49):6077-6083.

Quinn JA, Munoz FM, Gonik B, et al. Preterm birth: Case definition & Samp; guidelines for data collection, analysis, and presentation of immunisation safety data. Vaccine. 2016;34(49):6047-6056.

Rouse CE, Eckert LO, Wylie BJ, et al. Hypertensive disorders of pregnancy: Case definitions & guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2016;34(49):6069-6076

Vergnano S, Buttery J, Cailes B, et al. Neonatal infections: Case definition and guidelines for data collection, analysis, and presentation of immunisation safety data. Vaccine. 2016;34(49):6038-6046

World Health Organization (WHO) WHO recommendations for prevention and treatment of maternal peripartum infections. Published in September 2015. Last accessed on 21 March 2017.

# APPENDIX D: Definitions Of Maternal, Fetal And Neonatal Events Of Interest As Per Gaia D

The 2 tables presented in the original protocol have been replaced with 21 separate tables (one for each of the 19 events of interest defined per GAIA, and two for events of interest – maternal and neonatal – not defined as such per GAIA). Definitions and levels of diagnostic certainty have been updated (where applicable) per the reference cited (beneath each table) for each event of interest.

The 2 tables in the original protocol, for reference, follow.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# Maternal events of interest – TABLE FROM PROTOCOL VERSION 01

| Maternal death The death of a woman while pregnant or within 42 days of termination of pregnancy, irrespective of the duration and site of the pregnancy, from any cause related to or aggravated by the pregnancy or its management but not from accidental or incidental causes. (As ICD-10 terminology). In the context of immunization: Level 1 Diagnosis of pregnancy established by any of the following documented criteria: a. Ultrasound examination b. Fetal heart tones c. Positive serum or urine human chorionic gonadotropin pregnancy test d. Delivery of a neonate or other products of conception (abortus, stillborn) And Death of the mother while pregnant or within 42 days of termination of pregnancy, irrespective of the duration and site of the pregnancy And Documentation of Cause of death as: | Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|---|
| "Death of a woman during pregnancy, childbirth and the puerperium that is closely related temporally to an immunization event of the mother which is likely the single or contributory cause" I be a large of the mother which is likely the single or contributory cause of the during pregnancy, childbirth and the puerperium: other or coincidental level 2 Diagnosis of pregnancy established by any of the following criteria in the absence of Level 1 criteria: a. LMP date b. Serial Symphysio Fundal Height examinations And Death of the mother while pregnant or within 42 days of termination of pregnancy, irrespective of the duration and site of the pregnancy And Documentation of Cause of death as: a. Direct: abortive outcome, hypertensive disorder, obstetric hemorrhage, pregnancy related infection, other obstetric complications, unanticipated complications b. Indirect: non-obstetric complications c. Death during pregnancy, childbirth and the puerperium: other or coincidental d. Unspecified: unknown or undetermined Level 3 Absence of Level 1 or 2 criteria for establishing diagnosis of pregnancy and: a. Unsure LMP b. No clinical examination documented And Death of the mother temporal to pregnancy, childbirth or the postpartum period when exact timing of death is unknown, And | | The death of a woman while pregnant or within 42 days of termination of pregnancy, irrespective of the duration and site of the pregnancy, from any cause related to or aggravated by the pregnancy or its management but not from accidental or incidental causes. (As ICD-10 terminology). In the context of immunization: "Death of a woman during pregnancy, childbirth and the puerperium that is closely related temporally to an immunization event of the mother which | Level 1 Diagnosis of pregnancy established by any of the following documented criteria: a. Ultrasound examination b. Fetal heart tones c. Positive serum or urine human chorionic gonadotropin pregnancy test d. Delivery of a neonate or other products of conception (abortus, stillborn) And Death of the mother while pregnant or within 42 days of termination of pregnancy, irrespective of the duration and site of the pregnancy And Documentation of Cause of death as: a. Direct: abortive outcome, hypertensive disorder, obstetric hemorrhage, pregnancy related infection, other obstetric com-plications, unanticipated complications b. Indirect: non obstetric complications c. Death during pregnancy, childbirth and the puerperium: other or coincidental Level 2 Diagnosis of pregnancy established by any of the following criteria in the absence of Level 1 criteria: a. LMP date b. Serial Symphysio Fundal Height examinations And Death of the mother while pregnant or within 42 days of termination of pregnancy, irrespective of the duration and site of the pregnancy And Documentation of Cause of death as: a. Direct: abortive outcome, hypertensive disorder, obstetric hemorrhage, pregnancy related infection, other obstetric complications, unanticipated complications b. Indirect: non-obstetric complications c. Death during pregnancy, childbirth and the puerperium: other or coincidental d. Unspecified: unknown or undetermined Level 3 Absence of Level 1 or 2 criteria for establishing diagnosis of pregnancy and: a. Unsure LMP b. No clinical examination documented And Death of the mother temporal to pregnancy, childbirth or the postpartum period when exact | [Patwardhan, |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | a. Direct: abortive outcome, hypertensive disorder, obstetric hemorrhage, pregnancy related | |
| | | infection, other obstetric com-plications, unanticipated complications | |
| | | b. Indirect: non-obstetric complications | |
| | | c. Death during pregnancy, childbirth and the puerperium: other or coincidental | |
| | | d. Unspecified: unknown or undetermined. | |
| Hypertensive | Gestational Hypertension is a clinical | <u>Preeclampsia</u> | [Rouse, 2016] |
| disorders of | syndrome characterized by pregnancy | For All Levels of Diagnostic Certainty | |
| pregnancy | ≥20 weeks AND new onset | Clinical syndrome characterized by pregnancy ≥20 weeks AND new onset hypertension | |
| Gestational | hypertension (systolic blood pressure | (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg) sustained on | |
| hypertension / | ≥140 mmHg and/or diastolic blood | two measurements over a minimum of 1 h AND new onset proteinuria | |
| Preeclampsia / | pressure ≥90 mmHg) sustained on two | Level 1 | |
| Eclampsia | measurements over a minimum of 1 h | proteinuria diagnosed with ≥300 mg of protein on 24 h urine collection OR≥0.3 on spot protein: | |
| | WITHOUT severe features (see | creatinine ratio | |
| | preeclampsia with severe features | Level 2 | |
| | category) and WITHOUT proteinuria | proteinuria diagnosed with ≥1+ protein on urine dipstick | |
| | Preeclampsia has conventionally been | Insufficient evidence blood pressure cannot be measured OR no proteinuria evaluation is | |
| | defined as the development of | available (note diagnosis of preeclampsia with severe features does not require proteinuria, | |
| | gestational hypertension and proteinuria | see definition below) | |
| | after 20 weeks gestation. | , and the second | |
| | Proteinuria can be quantified by 24 h | Preeclampsia with severe features | |
| | urine collection, a spot protein: | For All Levels of Diagnostic Certainty | |
| | creatinine ratio, or with urinary dipstick. | Clinical syndrome characterized by pregnancy ≥20 weeks AND new onset hypertension | |
| | Proteinuria of≥300 mg in a 24 h urine | (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg) sustained on | |
| | specimen (the gold standard for | two measurements over a minimum of 1 h AND At least one of the criteria for severe disease: | |
| | measurement of proteinuria), or ≥0.30 | Level 1 | |
| | on a spot protein: creatinine ratio, or | At least one of the following: | |
| | ≥1+ on a dipstick meets the criteria for | Systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥110mmHg, which is | |
| | preeclampsia. | confirmed after only minutes OR | |
| | Preeclampsia diagnose with severe | Development of severe, persistent headache OR | |
| | features | Development of visual changes OR | |
| | •Vascular: | Eclampsia OR | |
| | <ul> <li>Severely elevated blood pressures,</li> </ul> | New onset thrombocytopenia (platelets <100,000/L) OR | |
| | with systolic blood pressure≥160 mmHg | New onset unremitting epigastric pain ORAST and ALT elevated to twice upper limit of normal | |
| | and/or diastolic blood pressure ≥110 | OR | |
| | mmHg, which is confirmed after only | | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| Event of interest | minutes (to facilitate timely antihypertensive treatment) Neurologic: Development of a severe headache (which can be diffuse, frontal, temporal or occipital) that generally does not improve with over the counter pain medications (such as acetaminophen/paracetamol) Development of visual changes (including photopsia, scotomata,cortical blindness) Eclampsia, or new-onset grand mal seizures in a patient with pre-eclampsia, without other provoking factors (such as evidence of cerebral malaria or preexisting seizure disorder). Seizures are often preceded by headaches, visual changes or altered mental status Hematologic: New onset thrombocytopenia, with platelet count <100,000/L Gastrointestinal: New onset of nausea, vomiting, epigastric pain Transaminitis (AST and ALT elevated to twice the upper limit of normal) Liver capsular hemorrhage or liver rupture Renal: Worsening renal function, as evidenced by serum creatinine level greater than 1.1 mg/dL or a doubling of the serum creatinine(absent other renal disease) Oliguria (urine output <500 mL/24 h) | Evidence of liver capsular hematoma or liver rupture (diagnosed on clinical exam or with imaging) OR Worsening renal function, as evidenced by serum creatinine level greater than 1.1 mg/dL or a doubling of the serum creatinine (absent other renal disease) or oliguria (<500 cc/24 h) OR Pulmonary edema (confirmed on imaging with chest X-ray, or on clinical exam) Level 2 new onset nausea and vomiting Insufficient evidence blood pressure cannot be measured Gestational Hypertension For All Levels of Diagnostic Certainty Clinical syndrome characterized by pregnancy ≥20 weeks AND new onset hypertension (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg) sustained on two measurements over a minimum of 1 h WITHOUT severe features (see preeclampsia with severe features category) and WITHOUT proteinuria Level 1 of diagnostic certainty no proteinuria (as defined by 24 h urine collection < 300 mg, spot protein: creatinine ratio <0.3) Level 2 of diagnostic certainty no proteinuria (as defined by urine dipstick negative or trace) Insufficient evidence blood pressure cannot be measured OR no proteinuria evaluation is available | Reference |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | Respiratory: Pulmonary edema (confirmed on clinical exam or imaging) | | |
| Antenatal Bleeding | Antenatal bleeding is a clinical syndrome characterized by bleeding in the second or third trimester of pregnancy. Pathologic etiologies attributable to the pregnant state include placenta previa, morbidly adherent placenta, vasa previa, placental abruption, cesarean scar pregnancy, intra-abdominal pregnancy, and uterine rupture. For both levels of diagnostic certainty for each etiology of antenatal bleeding: Bleeding is either documented vaginally or suspected to be occurring intrauterine, intraperitoneally, or (rarely) retroperitoneally, based on clinical signs and symptoms. In the case of ultrasound-based diagnosis, transvaginal ultrasound is more specific than transabdominal ultrasound, and transvaginal ultrasound is recommended where available. | Placenta Previa Level 1 Second or third trimester ultrasound (and/or MRI) evidence of placental tissue overlying or abutting the internal cervical os. Level 2 Painless vaginal bleeding in the second or third trimester, AND a high presenting part or abnormal fetal lie. AND pelvic exam with fullness palpable in the fornices (avoiding digital cervical exam). Morbidly Adherent Placentation Level 1 Second- or third-trimester ultrasound or MRI evidence of placenta previa, AND one of the following ultrasound features: Greyscale: loss of the retroplacental sonolucent zone, irregular retroplacental sonolucent zone, thinning or disruption of the hyperechoic serosa—bladder interface, presence of focal exophytic masses invading the urinary bladder, abnormal placental lacunae Color Doppler: diffuse or focal lacunar flow, vascular lakes with turbulent flow (peak systolic velocity over 15 cm/s), hypervascularity of serosa—bladder interface, markedly dilated vessels over peripheral subplacental zone 3D Power Doppler: numerous coherent vessels involving the whole uterine serosa—bladder junction (basal view), hypervascularity (lateral view), inseparable cotyledonal and intervillous circulations, chaotic branching, detour vessels (lateral view) AND one of the risk factors: prior cesarean delivery, prior uterine surgery (including endometrial ablation) or cesarean scar pregnancy OR Morbidly adherent placentation found on histology in a hysterectomy or partial wedge resection specimen. Level 2 Ultrasound evidence of placenta previa, AND hypervascularity of the lower uterine segment, diagnosed at laparotomy. OR Difficulty with placental separation after delivery of the infant, at either a vaginal or cesarean delivery with resultant hemorrhage due to partial separation. | Prabhu M, Eckert LO, Belfort M, et al. Antenatal Bleeding: Case Definition & Guidelines for Data Collection, Analysis, and Presentation of Immunization Safety Data. Unpublished manuscript. |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | Vasa Previa Level 1 Second trimester ultrasound evidence of fetal vessels (vessel with fetal heart rate identified by color flow Doppler) running through the membranes and overlying the internal cervical os, AND post-delivery examination of the placental specimen with unsupported fetal vessels within the membranes. Level 2 Vaginal bleeding in the second or third trimester at the time of ruptured amniotic membranes, AND fetal heart rate changes ultimately resulting in sinusoidal rhythm/terminal bradycardia, AND delivery of a pale, anemic infant or recent stillbirth or neonatal death, AND post-delivery examination of the placental specimen with unsupported fetal vessels within the membranes. | |
| | | Placental Abruption Level 1 In the absence of placenta previa on ultrasound, vaginal bleeding in the second or third trimester, AND uterine irritability or labor, AND clinical signs of hypovolemic shock or coagulopathy. OR Placental pathology with histologic findings of a chronic abruption. Level 2 Vaginal bleeding in the second or third trimester, AND uterine irritability or labor, without clinical signs of hypovolemic shock or coagulopathy, OR Vaginal bleeding in the second or third trimester, AND clinical evidence of retroplacental clot or visually evident placental infarcts at the time of delivery. | |
| | | Cesarean Scar Pregnancy Level 1 Transvaginal ultrasound with the following characteristics: empty uterine cavity, AND empty cervical canal, without contact with the gestational sac, AND presence of gestational sac, +/- fetal pole, +/- cardiac activity, in the anterior uterine segment adjacent to the cesarean scar, AND absence or defect in myometrium between bladder and gestational sac, AND gestational sac well perfused on Doppler ultrasound (to differentiate from an expulsing, avascular gestational sac). | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | OR Hysterectomy specimen with evidence of pregnancy implanted into the cesarean scar. There is no Level 2 definition for this event. | |
| | | Intra-abdominal Pregnancy Level 1 At laparotomy, a fetus found within the abdominal cavity, without evidence of uterine rupture, and with placentation not within the uterine cavity. There is no Level 2 definition for this event. Uterine Rupture Level 1 Complete uterine disruption at the time of laparotomy in the context of vaginal or intra- | |
| | | abdominal bleeding. There is no Level 2 definition for this event. | |
| Postpartum<br>haemorrhage | Genital tract bleeding after delivery (up to 42 days) of a foetus or infant that leads to an adverse clinical outcome. Such as hypovolemia or anaemia e.g. exertional dyspnoea, postural presyncope, tiredness or reduced consciousness. At the furthest extreme uncorrected hypovolaemic shock can lead to organ-dysfunction and maternal death. ICD-10 definition: "heamorrhage after delivery of a foetus or infant" | Level 1 Genital bleeding after delivery leading to severe maternal out-come (maternal death or maternal near miss) as defined by WHO <sup>28</sup> . Level 2 Genital bleeding after delivery with at least one of the following: measured abnormal bleeding (1000 ml or more), or any bleeding leading to hypotension or blood transfusion. Level 3 Genital bleeding after delivery estimated at 1000 ml or more | [Kerr, 2016] |
| Fetal Growth<br>Restriction | A fetus with a sonographic estimation of fetal weight below the tenth percentile for a given gestational age with increasing specificity for adverse perinatal outcomes below the third percentile. | Level 1a Level 1 evidence of pregnancy dating AND Estimated fetal weight below 3% using locally-accepted growth curve OR Estimated fetal weight below 10% using locally-accepted growth curve AND Absent or reversed end-diastolic flow of the umbilical artery Doppler OR Oligohydramnios as defined by amniotic fluid index (AFI) < 8 or deepest vertical pocket (DVP) < 2. Level 1b Level 1 evidence of pregnancy dating AND Estimated fetal weight below 10%ile using locally-accepted growth curve AND | Easter SR, Eckert OL, Boghossian N, et al. Fetal Growth Restriction: Case Definition & Guidelines for Data Collection, Analysis, and |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | Lack of absent or reversed end-diastolic flow of the umbilical artery OR oligohydramnios as defined by AFI <8 or DVP <2. Level 2a Level 2 evidence of pregnancy dating AND Estimated fetal weight below 3% using locally-accepted growth curve OR Estimated fetal below 10% using locally-accepted growth curve AND Absent or reversed end-diastolic flow of the umbilical artery Doppler. OR Oligohydramnios as defined by AFI < 8 or DVP < 2. | Presentation of<br>Immunization<br>Safety Data.<br>Unpublished<br>manuscript. |
| | | Level 2b Level 2 evidence of pregnancy dating AND Estimated fetal weight below 10%ile using locally-accepted growth curve AND No findings of absent or reversed end-diastolic flow of the umbilical artery or oligohydramnios as defined by AFI <8 or DVP <2. OR Level 1 evidence of pregnancy dating AND Estimated fetal weight below 10% using locally-accepted growth curve with no findings of oligohydramnios as defined by AFI <8 or DVP <2 with inability to assess umbilical artery Doppler. Insufficient Evidence Absence of ultrasound for use in assessment of estimated fetal weight. | |
| Dysfunctional<br>Labor | Prolonged labor at or after 37 weeks and before 42 weeks of gestational age | First Stage of Labor For both levels of diagnostic the woman is in established labor defined by regular contractions and cervical dilation of at least 4cm. Level 1 Progress of less than 0.5 cm cervical dilation per hour, for at least 4 hours, in women in established labor (i.e. have regular contractions and cervical dilation of at least 4cm) and with confirmed ruptured membranes. Level 2 Progress of less than 0.5cm cervical dilation per hour in women, for at least 4 hours, with established labor, (i.e. that is, regular contractions and cervical dilation of at least 4cm) without certainty of ruptured membranes. Second Stage of Labor The definitions below are applicable in cases with or without regional analgesia. Level 1 Full dilation of the cervix AND onset of the active stage (active maternal effort (i.e. pushing) OR visible baby) AND | Boatin AA, Eckert LO, Boulvain M, et al. Dysfunctional Labor: Case Definition & Guidelines for Data Collection, Analysis, and Presentation of Immunization Safety Data. Unpublished manuscript. |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | greater than 2 hours of pushing in nulliparous women OR | |
| | | greater than 1 hour of pushing in multiparous women OR use of instrument OR | |
| | | caesarean delivery for the indication of dystocia. | |
| | | Level 2 | |
| | | Full dilation of the cervix in any phase of the second stage | |
| | | AND | |
| | | no delivery within 3 hours of full dilation in the nulliparous woman OR | |
| | | within 2 hours in multiparous women OR | |
| | | use of instrument OR | |
| | | caesarean delivery for the indication of dystocia. | |
| Gestational | Pregnancy induced hyperglycemia | For All Levels of Diagnostic Certainty | Kachikis A, |
| Diabetes Mellitus | i regramely madeca mypergry comma | Gestational diabetes mellitus (GDM) is a clinical syndrome characterized by | Eckert LO, |
| Diabotoo mointao | | the absence of pre-gestational diabetes diagnosis defined by | Walker C, et al. |
| | | Previous diagnosis of diabetes while not pregnant OR | Gestational |
| | | First trimester hemoglobin A1c level of ≥ 6.5% (47.5 mmol/mol) OR | Diabetes |
| | | First trimester fasting blood glucose 126 mg/dL / ≥ 7mmol/L AND | Mellitus: Case |
| | | Identification of sustained hyperglycemia during pregnancy not due to other known causes (i.e. | Definition & |
| | | corticosteroids, beta-mimetics, etc.) | Guidelines for |
| | | Level 1 | Data Collection, |
| | | Absence of pre gestational diabetes mellitus diagnosis in the first trimester as defined above | Analysis, and |
| | | with level 1-2 certainty for gestational age using GAIA definition for gestational age AND | Presentation of |
| | | Diagnosis of gestational diabetes based on a positive internationally recognized oral glucose | Immunization |
| | | tolerance test (see below "major criteria") using venous blood sample/samples | Safety Data. |
| | | Level 2 | Unpublished |
| | | Absence of pre gestational diabetes mellitus diagnosis in the first trimester as defined above | manuscript. |
| | | with at least level 3 certainty for gestational age using GAIA definition for gestational age AND | manasonpt. |
| | | Diagnosis of gestational diabetes based on positive internationally recognized oral glucose | |
| | | tolerance test (see below "major criteria") using capillary blood sample/samples | |
| | | Level 3 | |
| | | Absence of pregestational diabetes mellitus diagnosis in the first trimester as defined above | |
| | | with at least level 3 certainty for gestational age using GAIA definition for gestational age AND | |
| | | Diagnosis of gestational diabetes based on fasting plasma glucose of 5.1-6.9 mmol/l (92-125 | |
| | | mg/dL) using venous or capillary blood samples. | |
| | | Insufficient evidence for diagnosis | |
| | | Blood glucose cannot be measured OR | |
| | | Diodu giucose carriot de measureu OK | |
207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | Use of Hemoglobin A1c alone for the diagnosis of GDM without a diagnostic oral glucose tolerance test (OGTT) or elevated fasting plasma glucose level. OR Clinical and laboratory findings such as glucosuria, fundal height greater than dates, obesity, prior history of GDM or family history for the diagnosis of gestational diabetes mellitus without a diagnostic test. | |
| Non-reassuring fetal status | Indicator of underlying event resulting in temporary or permanent oxygen deprivation to the fetus which may lead to fetal hypoxia and metabolic acidosis | Level 1 Category III fetal heart rate tracings detected via continuous cardiotocography as defined by NICHD Absent baseline fetal heart rate variability AND any of the following: - recurrent late decelerations - recurrent variable deceleration - bradycardia (<110 bpm) OR Sinusoidal pattern AND Umbilical cord blood analysis consistent with metabolic acidosis (pH < 7.0 and Base deficit >12 mmol/L) Level 2 Category III fetal heart rate tracings detected via continuous cardiotocography as defined by NICHD Absent baseline fetal heart rate variability AND any of the following: - recurrent late decelerations - recurrent variable deceleration - bradycardia (<110 bpm)OR° Sinusoidal pattern Level 3 Fetal heart pattern detected via intermittent auscultation suggestive of fetal hypoxia Baseline FHR <110 bpm or >160 bpm Presence of repetitive or prolonged (>3 min) decelerations More than 5 contractions in a 10 min period | [Gravett, 2016] |
| Pathways to preterm birth | Premature preterm rupture of membranes Preterm labor Insufficient cervix Provider-initiated preterm birth | Premature preterm rupture of membranes All levels of certainty Patient is determined to be preterm as defined by GAIA On presentation, patient is determined to not be in preterm labor, having ≤4 contractions per hour documented clinically or on tocodynometer, with <2 cm cervical dilation (greater than 4 contractions per hour would qualify the patient as having preterm labor) Fluid can be noted to be clear, blood-tinged, meconium-tinged (fetal stool), purulent-tinged (yellowish, suggesting infection) Level 1 | [Harrison, 2016] |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | Clinical history of rupture of membranes AND | |
| | | Visible leakage of fluid on vaginal speculum exam AND | |
| | | Visible arborization (ferning) on microscopy of amniotic fluid OR | |
| | | Ultrasound with oligohydramnios (AFI <5 or MVP <2) AND | |
| | | Documented membrane rupture by a diagnostic test (one of the below options): | |
| | | Positive intra-amniotic dye-injection method | |
| | | Positive result on amniotic fluid alpha-fetoprotein test kit | |
| | | Amniotic fluid pH measurement (nitrazine paper test) | |
| | | Amniotic fluid placental alpha macroglobulin-1 protein assay (PAMG-1) test (AmniSure test) | |
| | | Amniotic fluid insulin-like growth factor binding protein(IGFBP-1) test (Actim PROM test) | |
| | | Level 2 | |
| | | Clinical history of rupture of membranes AND | |
| | | Visible leakage of fluid on vaginal speculum examination AND | |
| | | Visible arborization (ferning) on microscopy of amniotic fluid OR | |
| | | document membrane rupture by a diagnostic test (one of those listed above) OR Ultrasound | |
| | | with oligohydramnios (AFI <5 or MVP <2) | |
| | | Level 3 | |
| | | Clinical history of rupture of membranes AND | |
| | | Visible leakage of presumed amniotic fluid; this may be on vaginal speculum examination | |
| | | (pooling in vagina), on inspection of the perineum (wet perineum due to leakage of fluid from | |
| | | the vagina), or fluid soaked cloth/clothes/sanitary pad. | |
| | | Preterm labor | |
| | | For all levels of diagnostic certainty | |
| | | Patient is determined to be have delivered preterm as defined by the Brighton Collaboration | |
| | | definition | |
| | | Level 1 | |
| | | On presentation, >4 documented uterine contractions per hour as determined by a | |
| | | tocodynometer AND | |
| | | Documented change in length or dilation of cervix by physical examination or transvaginal | |
| | | ultrasound over a two hour period, with clinical criteria for documenting cervical change by | |
| | | exam including: | |
| | | a. Cervical dilation 2 cm or greater at the internal os by digital examination | |
| | | b. Cervical length of 1 cm or less by digital examination | |
| | | c. 50% or greater effacement by digital examination | |
| | | 3. 33 73 3. grouter endocriterit by digital examination | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | Level 2 Greater than 4 uterine contractions per hour as determined by a tocodynometer or clinical assessment AND Documented change in length or dilation of cervix by physical examination, with clinical criteria including: a. Cervical dilation 2 cm or greater at the internal os by digital examination b. Cervical length of 1 cm or less by digital examination c. 50% or greater effacement by digital examination Level 3 1. Greater than 4 documented uterine contractions per hour determined by clinical assessment AND 2. Documented change in cervical examination (change in dilation or effacement) over a two hour period | |
| | | Insufficient cervix For all levels of diagnostic certainty Patient is determined to be ≥16 weeks and <24 weeks gestation as defined by the Brighton Collaboration definitions of gestational age Patient is determined to have advanced cervical dilation (>2 cm) resulting in either treatment with a cerclage (cervical stitch) or preterm delivery Patient is determined to not be in preterm labor, having ≤4 con-tractions per hour documented clinically or on tocodynometer (with anything >4 contractions per hour falling into the category of preterm labor) Level 1 Internal cervical os dilation (>2 cm) with ≤4 contractions/h, as determined by transvaginal ultrasound AND digital examination | |
| | | Level 2 Internal cervical os dilation (>2 cm) with ≤4 contractions/h, as determined by digital examination Level 3 Patient reports fetal delivery without any painful contractions History excludes other causes of mid-trimester delivery Provider-initiated preterm birth For all levels of diagnostic certainty Patient is determined to be preterm as defined by the Brighton Collaboration definition | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | Level 1 | |
| | | Documentation in the healthcare record by a patient's delivering provider that there were no | |
| | | signs or symptoms of the spontaneous onset of preterm labor AND | |
| | | Documentation in the healthcare record by a patient's delivering provider that the patient | |
| | | needed to undergo induction of labor or cesarean delivery which led to the preterm delivery | |
| | | Level 2 | |
| | | From recall, delivering provider confirms that there was an absence of any signs or symptoms | |
| | | of the spontaneous onset of preterm labor AND | |
| | | Delivering provider reports from recall that he or she decided that the patient needed to | |
| | | undergo induction of labor or cesarean delivery | |
| | | Level 3 | |
| | | From recall, patient confirms that there was an absence of any signs or symptoms of the | |
| | | spontaneous onset of preterm labor AND | |
| | | Patient reports from recall that the healthcare provider indicated that she needed to undergo | |
| | | induction of labor or cesarean delivery | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# **Neonatal events of interest - TABLE FROM PROTOCOL VERSION 01**

| Event of interest | Description | Levels of diagnostic certainty (1 highest level to 4 lowest level of certainty) | Reference |
|---|---|---|---|
| Small for gestational age | Weight below 10th percentile for gestational age as assessed against a validated global, regional or local standard. | Level 1 Weight below 10th percentile for gestational age AND The following used in assessment of weight: Newborn weighed within 24 hours of birth Weight assessed using a calibrated electronic scale with 10 g resolution AND The following for assessment of gestational age: Certain LMP or IUI or embryo transfer date AND confirmatory ultrasound in first trimester OR The following for assessment of gestational age: First trimester ultrasound Level 2A Weight below 10th percentile for gestational age AND The following used in assessment of weight: Newborn weighed within 24 hours of birth on any scale with a < 50 g resolution, tared to zero and calibrated AND The following for assessment of gestational age: Certain LMP with first or second trimester ultrasound OR Certain LMP with first trimester physical exam2 Level 2B Weight below 10th percentile for gestational age AND The following used in assessment of weight: Newborn weighed within 24 hours of birth on any scale with a < 50 g resolution, tared to zero and calibrated AND The following assessment of gestational age: Uncertain LMP with second trimester ultrasound Level 3A Weight below 10th percentile for gestational age: Uncertain LMP with second trimester ultrasound Level 3A Weight below 10th percentile for gestational age AND The following assessment of gestational age: Uncertain LMP with the first 48 hours of life, Newborn weighed on any scale with a < 50 g resolution, tared to zero and calibrated AND The following assessment of gestational age: Certain LMP with third trimester ultrasound OR Certain LMP with third trimester ultrasound OR Certain LMP with third trimester ultrasound OR Certain LMP with confirmatory 2nd trimester fundal height OR Certain LMP with percentile for gestational age AND Weight below 10th percentile for gestational age AND | Schlaudecker EP, Munoz FM, Bardají A, et al. Small for Gestational Age: Case Definition & Guidelines for Data Collection, Analysis, and Presentation of Maternal Immunisation Safety Data. unpublished manuscript. |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | (1 highest level to 4 lowest level of certainty) | |
| | | The following used in assessment of weight: Infant weighed within the first 48 hours of life, | |
| | | Newborn weight assessed by measuring the difference between an adult holding the infant | |
| | | and the adult being weighed alone on any scale AND | |
| | | The following assessment of gestational age: | |
| | | Uncertain LMP with fundal height OR | |
| | | Uncertain LMP with newborn physical assessment OR | |
| | | Uncertain LMP with birthweight | |
| | | Level 4 | |
| | | Baby noted to be small, but no actual weight | |
| | | Baby with GA assessed only by infant examination | |
| | | Diagnosis extracted from billing codes or chart, with no documentation of actual birth weight | |
| | | or GA | |
| Low birth weight | LBW <2500 grams. Very low birth | Level 1 | Cutland CL, |
| (LBW) | weight (VLBW) <1500 grams and | 1. Newborn infant weighed within 24 hours of birth AND | Lackritz E, |
| | extremely low birth weight (ELBW) is | 2. Use electronic scale which is graduated to 10 grams AND | Alonso AB, et al. |
| | <1000grams. | 3. Scale is calibrated at least once a year AND | Low Birth |
| | | 4. Scale placed on level, hard surface AND | Weight: Case |
| | | 5. Scale tared to zero grams AND | Definition & |
| | | 6. Weight recorded as <2500 grams OR | Guidelines for |
| | | 7. Birth weight recorded as <2500 grams AND | Data Collection, |
| | | 8. Birth weight assessed as per health care facility's standard operating procedure, which | Analysis, and |
| | | fulfills criteria 1 to 5 | Presentation of |
| | | Level 2 | Maternal |
| | | 1. Newborn infant weighed within 24 hours of birth AND | Immunisation |
| | | 2. Scale (electronic/spring) is graduated to at least 50 grams AND | Safety Data. |
| | | 3. Scale is calibrated at least once a year, or more often if moved AND | Unpublished |
| | | 4. Scale tared to zero grams or 0.00kg AND | manuscript. |
| | | 5. Weight recorded as <2500 grams OR | · |
| | | 6. Birth weight recorded as <2500 grams AND | |
| | | 7. Birth weight assessed as per health care facility's standard operating procedure, which | |
| | | fulfills criteria 1 to 4 | |
| | | (Scale used could be electronic or spring scale, including colour-coded scale) | |
| | | Level 3 | |
| | | 1. Newborn infant weighed on day 1 or 2 of life (first 48 hours of life) AND | |
| | | 2. Weight measured using dial/spring/colour-coded scale AND | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| Acute Neonatal | Is a clinical syndrome presenting with | (1 highest level to 4 lowest level of certainty) 3. Weight assessed as <2500 grams Level 4 1. Newborn weight assessed between 3 and 7 days of age AND 2. Weight assessed using dial/ spring/ colour-coded scale OR 3. Proxy measure (Table 1 of reference) of birth weight used AND 4. Weight CATEGORY assessed as <2500 grams Level 1 | Sell E, Munoz |
| Encephalopathy | abnormal functioning of the central nervous system, in the earliest days of life in an infant born at or beyond 35 weeks of gestation, manifested by an abnormal level of alertness or seizures, and often accompanied by difficulty with initiating and maintaining respiration and depression of tone that may be due to a variety of etiologies including hypoxia/ischemia, metabolic disturbance, or infection. | Abnormal level of alertness AND Clinical Seizures with electroencephalographic correlation AND Difficulty with initiating and maintaining respiration AND Depression of tone Level 2 Abnormal level of alertness AND Clinical Seizures with or without electroencephalographic correlation AND Difficulty with initiating and maintaining respiration OR Depression of tone Level 3 Abnormal level of alertness AND Clinical Seizures OR Difficulty with initiating and maintaining respiration OR Depression of tone | FM, Soe A, et al. Acute Neonatal Encephalopathy: Case Definition & Guidelines for Data Collection, Analysis, and Presentation of Maternal Immunization Safety Data. Unpublished manuscript. |
| Congenital<br>Microcephaly | Congenital microcephaly, also referred to as primary microcephaly due to its presence in utero or at birth, is a descriptive term for a structural defect in which a fetus or infant's head (cranium) circumference is smaller than expected when compared to other fetuses or infants of the same gestational age, sex and ethnic background. | Postnatally diagnosed Congenital Microcephaly Case Definition Level 1 Live birth, stillbirth, or spontaneous or therapeutic abortion of at least 24 weeks of Gestational Age (GA) AND HC 2 SD below mean or <3% according to GA and gender, using appropriate standardized reference charts for the population (e.g., WHO growth reference charts if GA ≥37 weeks and Intergrowth-21st reference charts for GA 24–36 weeks) AND Measured between 24–36 hours after birth or end of pregnancy. Level 2A Live birth, stillbirth, or spontaneous or therapeutic abortion of at least 24 weeks of GA AND HC 2 SD below mean or <3% according to GA and gender, using appropriate standardized reference charts for the population (e.g., WHO growth reference charts if GA ≥37 weeks and Intergrowth-21st reference charts for GA 24–36 weeks) AND Measured within the first 24 hours OR | DeSilva M, Munoz FM, Sell E, et al. Congenital Microcephaly: Case Definition & Guidelines for Data Collection, Analysis, and Presentation of Safety Data after Maternal Immunisation. |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty (1 highest level to 4 lowest level of certainty) | Reference |
|---|---|---|---|
| | | Measured >36 hours and up to 6 weeks after birth or end of pregnancy with no apparent post- natal insult resulting in microcephaly Level 2B Live birth, stillbirth, or spontaneous or therapeutic abortion of at least 24 weeks of GA AND HC 2 SD below mean or <3% according to GA and gender, using appropriate standardized reference charts for the population (e.g., WHO growth reference charts if GA ≥37 weeks and Intergrowth-21st reference charts for GA 24–36 weeks) AND Measured within the first 24 hours OR Measured >36 hours and up to 6 weeks after birth or end of pregnancy with no apparent post- natal insult resulting in microcephaly Level 3 Live birth, stillbirth, or spontaneous or therapeutic abortion AND Case meets criteria for microcephaly using a validated algorithm: 1 inpatient diagnosis OR 2 outpatient diagnoses OR 1 outpatient diagnosis AND death in first year using the following diagnostic codes ICD-9-CM code 742.1 or ICD-10-CM code Q02 | Unpublished manuscript. |
| | | Level 4 Live birth, stillbirth, or spontaneous or therapeutic abortion AND Diagnosis of congenital microcephaly based on physical inspection without HC measurement OR Diagnosis of congenital microcephaly based on ICD-9-CM or ICD-10-CM code that does not meet validated algorithm criteria above. | |
| | | B. Prenatally diagnosed Congenital Microcephaly Case Definition Level 1A Fetus of at least 24 weeks GA based on certain LMP with confirmatory 1st trimester (<14 weeks) or 2nd trimester US scan IUI, or embryo transfer date AND HC 2 SD below mean or <3% according to fetal ultrasound (US) examination using appropriate standardized reference charts according to GA and gender for the population (eg. WHO growth reference charts if GA ≥37 weeks and Intergrowth-21st reference charts for GA 24–36 weeks) AND Confirmation of microcephaly (i.e., HC 2 SD below mean or <3%) in fetus by at least one additional US after 24 weeks and at least one week after first US OR Confirmation of microcephaly by HC measurement with standard tape measure at birth or autopsy | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | (1 highest level to 4 lowest level of certainty) | |
| | | Level 1B | |
| | | 1. Fetus of at least 24 weeks GA based on uncertain LMP with 2nd trimester US AND | |
| | | 2. HC 2 SD below mean or <3% according to fetal ultrasound (US) examination using | |
| | | appropriate standardized reference charts according to GA and gender for the population (eg. | |
| | | WHO growth reference charts if GA ≥37 weeks and Intergrowth-21st reference charts for GA | |
| | | 24–36 weeks) AND | |
| | | Confirmation of microcephaly (i.e., HC 2 SD below mean or <3%) in fetus by at least one | |
| | | additional US after 24 weeks and at least one week after first US OR | |
| | | Confirmation of microcephaly by HC measurement with standard tape measure at birth or | |
| | | autopsy | |
| | | Level 2 | |
| | | Fetus of at least 24 weeks GA based on LMP with fundal height and no confirmatory US scan | |
| | | AND | |
| | | HC 2 SD below mean or <3% according to fetal US examination using appropriate | |
| | | standardized reference charts according to GA and gender for the population (eg. WHO | |
| | | growth reference charts if GA ≥37 weeks and Intergrowth-21st reference charts for GA 24–36 | |
| | | weeks) AND | |
| | | Confirmation of microcephaly (i.e., HC 2 SD below mean or <3%) in fetus with at least one | |
| | | additional US after 24 weeks and at least one week after first US OR Confirmation of microcephaly by HC measurement with standard tape measure at birth or | |
| | | , , , | |
| | | autopsy<br>Level 3 | |
| | | Fetus of at least 24 weeks GA AND | |
| | | HC 2 SD below mean or <3% according to fetal US examination using appropriate | |
| | | standardized reference charts according to GA and gender for the population (eg. WHO | |
| | | growth reference charts if GA ≥37 weeks and Intergrowth-21st reference charts for GA 24–36 | |
| | | weeks) AND | |
| | | No confirmation of microcephaly with any additional US or by HC measurement at birth or | |
| | | autopsy | |
| | | Level 4 | |
| | | Fetus of at least 24 weeks GA AND | |
| | | No available measurement of HC in utero by US, but documentation on medical record review | |
| | | suggesting microcephaly based on US imaging AND | |
| | | No confirmation of microcephaly with any additional US or by HC measurement at birth or | |
| | | autopsy | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | (1 highest level to 4 lowest level of certainty) | |
| | | Level 5 | |
| | | Fetus of at least 24 weeks GA AND | |
| | | HC 2 SD below mean or <3% according to fetal US examination using appropriate | |
| | | standardized reference charts according to GA and gender for the population (eg. WHO | |
| | | growth reference charts if GA ≥37 weeks and Intergrowth-21st reference charts for GA 24–36 weeks) AND | |
| | | HC at birth or autopsy is in the normal range using appropriate standardized reference charts | |
| | | according to GA and gender for the population, which means that this is NOT a case of | |
| | | prenatally diagnosed congenital microcephaly | |
| Congenital | Congenital anomalies, also commonly | For all levels of diagnostic certainty | [DaSilva, 2016] |
| anomalies | referred to as birth defects, congenital | A major congenital anomaly is a structural or functional defect with the following three | [DaSilva, 2010] |
| anomanes | disorders, congenital malformations, or | characteristics: | |
| | con-genital abnormalities, are events of | 1. Of prenatal origin | |
| | prenatal origin that a represent at birth, | 2. Present at the time of live birth or fetal demise, or in utero | |
| | potentially impacting an infant's health, | 3. Affecting (or has the propensity to affect) the health, survival, or physical or cognitive | |
| | development and/or survival. | functioning of the individual | |
| | development and/or survival. | Major External Structural Defects | |
| | | Level 1 | |
| | | •Alterations in external anatomy visible at the time of <u>live birth</u> and persistent beyond the | |
| | | immediate peripartum period unless surgically repaired OR | |
| | | •Alterations in external anatomy visible in a <u>stillbirth</u> or in the products of conception of a | |
| | | spontaneous or therapeutic abortion AND | |
| | | •Confirmed by documentation of a diagnosis made by a clinician experienced in diagnosing | |
| | | congenital anomalies and with the highest level of morphology training for the specific setting | |
| | | Level 2 | |
| | | •Alterations in external anatomy visible at the time of live birth and persistent beyond the | |
| | | immediate peripartum period unless surgically repaired OR | |
| | | •Alterations in external anatomy visible in a stillbirth or in the products of conception of a | |
| | | spontaneous or therapeutic abortion AND | |
| | | •Confirmed by documentation of a diagnosis made by a clinician with some experience | |
| | | diagnosing congenital anomalies | |
| | | Level 3 | |
| | | •Alterations in external anatomy visible at the time of <u>live birth</u> and persistent beyond the | |
| | | immediate peripartum period unless surgically repaired OR | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | (1 highest level to 4 lowest level of certainty) | |
| | | •Alterations in external anatomy visible in a <u>stillbirth</u> or in the products of conception of a | |
| | | spontaneous or therapeutic abortion AND | |
| | | •Confirmed by documentation of a diagnosis made by a trained maternal or child health care | |
| | | provider with at least minimal experience diagnosing congenital anomalies OR | |
| | | •For live births, confirmed using individual (ICD-9/ICD-10) codes or as part of an ICD-9/ICD- | |
| | | 10 code based algorithm, where the outcome (individual code or algorithm) has been | |
| | | validated | |
| | | Level 4 (insufficient evidence to confirm) | |
| | | •Alterations in external anatomy visible at the time of live birth and persistent beyond the | |
| | | immediate peripartum period unless surgically repaired OR | |
| | | •Alterations in external anatomy visible in a stillbirth or in the products of conception of a | |
| | | spontaneous or therapeutic abortion AND | |
| | | •Confirmed by medical record review OR | |
| | | •Confirmed in claims data (ICD-9/ICD-10 diagnoses) | |
| | | Internal Structural Defects | |
| | | Level 1 | |
| | | •Alterations in internal anatomy present at the time of <u>live birth</u> and persistent beyond the | |
| | | immediate peripartum period unless surgically repaired AND | |
| | | •Confirmed by definitive imaging study or intraoperative diagnosis OR | |
| | | •Alterations in internal anatomy detected during autopsy for a stillbirth, spontaneous or | |
| | | therapeutic abortion confirmed by documentation by a pathologist or other relevant | |
| | | subspecialist | |
| | | Level 2 | |
| | | •Alterations in internal anatomy present at the time of <u>live birth</u> and persistent beyond the | |
| | | immediate peripartum period unless surgically repaired AND | |
| | | •Confirmed by documentation of a diagnosis made by a clinician experienced in diagnosing | |
| | | congenital anomalies and with the highest level of morphology training for the specific setting | |
| | | without definitive imaging or intraoperative evaluation OR | |
| | | •For stillbirth, spontaneous or therapeutic abortion, internal structural defect is visible by | |
| | | ultrasound or other imaging modality prenatally Level 3 | |
| | | •Alterations in internal anatomy present at the time of <u>live birth</u> and persistent beyond the immediate peripartum period unless surgically repaired AND | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | (1 highest level to 4 lowest level of certainty) | |
| | | Confirmed by documentation of a diagnosis made by a clinician with some experience diagnosing congenital anomalies OR Confirmed using individual (ICD-9/ICD-10) codes or as part of an ICD-9/ICD-10 code based algorithm, where the outcome (individual code or algorithm) has been validated Level 4 insufficient evidence to confirm Alterations in internal anatomy present at the time of live birth and persistent beyond the immediate peripartum period unless surgically repaired OR Alterations in internal anatomy present at time of stillbirth, spontaneous abortion, or induced abortion AND Confirmed through medical record review, with the medical record demonstrating that the anomaly was present at the time of live birth or time of fetal demise, and that the anomaly was diagnosed by a trained maternal or child health care provider with minimal experience diagnosing congenital anomalies OR Confirmed by claims data (ICD-9/ICD-10 diagnoses) | |
| | | Functional Defects Level 1 •For live births, alterations in functioning of one or more organs or body parts not due to a structural defect, present at the time of birth (or propensity to develop alteration present at live birth), and persistent beyond the immediate peripartum period, unless treated through gene therapy or stem cell transplantation OR •For stillbirths, spontaneous or therapeutic abortions, alterations in functioning of one or more organs or body parts, not due to a structural defect AND •Confirmed by definitive diagnostic study Level 2 •For live births, alterations in functioning of one or more organs or body parts not due to a structural defect, present at livebirth (or propensity to develop alteration present at live birth), and persistent beyond the immediate peripartum period, unless treated through gene therapy or stem cell transplantation OR •For stillbirths, spontaneous or therapeutic abortions, alterations in functioning of one or more organs or body parts, not due to a structural defect AND •Confirmed by documentation of a diagnosis made by a clinician experienced in diagnosing congenital anomalies and with the highest level of training in the diagnosis of functional defects for the specific setting | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | (1 highest level to 4 lowest level of certainty) | |
| | | •For live births, alterations in functioning of one or more organs or body parts not due to a | |
| | | structural defect, present at livebirth (or propensity to develop alteration present at live | |
| | | birth),and persistent beyond the immediate peripartum period, unless treated through gene | |
| | | therapy or stem cell transplantation OR | |
| | | •For stillbirths, spontaneous or therapeutic abortions, alterations in functioning of one or more | |
| | | organs or body parts, not due to a structural defect AND | |
| | | •Confirmed by documentation of a diagnosis made by a clinician with some experience | |
| | | diagnosing functional defects OR | |
| | | •Confirmed using individual (ICD-9/ICD-10) codes or as part of an ICD-9/ICD-10 code based | |
| | | algorithm, where the outcome(individual code or algorithm) has been validated | |
| | | Level 4 (insufficient evidence to confirm) | |
| | | •For live births, alterations in functioning of one or more organs or body parts not due to a | |
| | | structural defect, present at the time of live birth (or propensity to develop alteration present at | |
| | | livebirth), and persistent beyond the immediate peripartum period, unless treated through | |
| | | gene therapy or stem cell transplantation OR | |
| | | •For stillbirths, spontaneous or therapeutic abortions, alterations in functioning of one or more | |
| | | organs or body parts, not due to a structural defect AND | |
| | | •Confirmed through medical record review, with the medical record demonstrating that the | |
| | | anomaly was present at the time of live birth or time of fetal demise, and that the anomaly was | |
| | | diagnosed by a trained maternal or child healthcare provider who is not a qualified geneticist, | |
| | | neonatologist, pathologist, subspecialist, pediatrician, obstetrician, or family medicine | |
| | | practitioner OR | |
| | | •Confirmed by claims data (ICD-9/ICD-10 diagnoses) | |
| Neonatal death | Death of a live born infant regardless of | Neonatal death in a non-viable live birth | [Pathirana, 2016] |
| | gestational age at birth, within the first | Level 1 | |
| | 28 completed days of life. | 1. Live born infant AND | |
| | | 2. Gestational age <22 weeks (GA level of certainty = 1) OR | |
| | | 3. Birth weight <500 g AND | |
| | | 4. Death of infant in first 28 days of life AND | |
| | | 5. Medically-confirmed death | |
| | | Level 2 | |
| | | 1. Live born infant AND | |
| | | 2. Gestational age/size of newborn assessed as at least one of: | |
| | | a. Gestational age <22 weeks (GA Level of Certainty = 1 OR 2) | |
| | | b. Birth weight <500 g AND | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | (1 highest level to 4 lowest level of certainty) | |
| | | 3. Death of infant in first 28 days of life AND | |
| | | 4. Medically-confirmed death OR non-medically-confirmed death | |
| | | Level 3 | |
| | | 1. Live born infant AND | |
| | | 2. Gestational age <5 months according to parent/family member/delivery attendant (GA | |
| | | Level of Certainty = 2 OR 3) AND | |
| | | 3. Death of infant in first 28 days of life AND | |
| | | 4. Medically-confirmed death OR non-medically-confirmed death | |
| | | Neonatal death in an extremely preterm live birth | |
| | | Level 1 | |
| | | 1. Live born infant AND | |
| | | 2. Gestational age ≥22 and <28 weeks (GA Level of Certainty = 1) OR | |
| | | 3. Birth weight ≥500 g but <1000 g AND | |
| | | 4. Death of infant in first 28 days of life AND | |
| | | 5. Medically-confirmed death | |
| | | Level 2 | |
| | | 1. Live born infant AND | |
| | | 2. Gestational age/size of newborn assesses as one or more of: | |
| | | a. Gestational age ≥22 and <28 weeks (GA Level of Certainty = 1 OR 2) | |
| | | b. Birth weight ≥500 g but <1000 g AND | |
| | | 3. Death of infant in first 28 days of life AND | |
| | | 4. Medically-confirmed death OR non-medically-confirmed death | |
| | | Level 3 | |
| | | 1. Live born infant AND | |
| | | 2. Gestational age ≥5 months but <7 months according to neonate's parent | |
| | | (mother/father)/family member/delivery attendant (GA Level of Certainty = 2 OR 3) AND | |
| | | 3. Death of infant in first 28 days of life AND | |
| | | 4. Medically-confirmed death OR non-medically-confirmed death | |
| | | Neonatal death in a preterm live birth (gestational age ≥28to <37 weeks) | |
| | | Level 1 | |
| | | 1. Live born infant AND | |
| | | 2. Gestational age ≥28 and <37 weeks (Level of Certainty = 1)OR | |
| | | 3. Birth weight ≥1000 g but <2500 g AND | |
| | | 4. Death of infant in first 28 days of life AND | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | (1 highest level to 4 lowest level of certainty) | |
| | | 5. Medically-confirmed death | |
| | | Level 2 | |
| | | 1. Live born infant AND | |
| | | 2. Gestational age/size of newborn assesses as one or more of: | |
| | | a. Gestational age ≥28 and <37 weeks (GA Level of Certainty = 1 OR 2) | |
| | | b. Birth weight ≥1000 g but <2500 g AND | |
| | | 3. Death of infant in first 28 days of life AND | |
| | | 4. Medically-confirmed death OR non-medically-confirmed death | |
| | | Level 3 | |
| | | (MAY apply to LMIC- or may be non-viable in LMIC) | |
| | | 1. Live born infant AND | |
| | | 2. Gestational age ≥7 months but <9 months according to parent/family member/delivery | |
| | | attendant (GA Level of Certainty = 2 OR 3) AND | |
| | | 3. Death of infant in first 28 days of life AND | |
| | | 4. Medically-confirmed death OR non-medically-confirmed death | |
| | | Neonatal death in a term live birth | |
| | | Level 1 | |
| | | 1. Live born infant AND | |
| | | 2. Gestational age ≥37 weeks (GA Level of Certainty = 1) AND | |
| | | 3. Birth weight >2500 g OR | |
| | | 4. Documented intra-uterine growth retardation if ≤2500 g AND | |
| | | 5. Death of infant in first 28 days of life AND | |
| | | 6. Medically-confirmed death | |
| | | Level 2 | |
| | | 1. Live born infant AND | |
| | | 2. Gestational age/size of newborn assesses as one or more of: | |
| | | a. Gestational age ≥37 weeks (GA Level of Certainty = 1 OR 2) | |
| | | b. Birth weight ≥2500 g AND | |
| | | 3. Death of infant in first 28 days of life AND | |
| | | 4. Medically-confirmed death OR non-medically-confirmed death which is confirmed by | |
| | | examination by (by at least) non-medically-trained attendant (e.g. undertaker, community member) | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | (1 highest level to 4 lowest level of certainty) | |
| | | Level 3 (apply to LMIC) | |
| | | 1. Live born infant AND 2. Gestational age ≥9 months according to parent/family | |
| | | member/delivery attendant (GA Level of Certainty = 2 OR 3) AND | |
| | | 3. Death of infant in first 28 days of life AND | |
| | | 4. Medically-confirmed death OR non-medically-confirmed death | |
| Neonatal infections | Neonatal bacteraemia and sepsis (of | Neonatal invasive blood stream infections: bacterial/fungal/viral | [Vergnano, 2016] |
| | early or late onset), meningitis, | Level 1 | |
| | pneumonia and other respiratory | Recognised pathogen identified using a validated method and from a normally sterile site. | |
| | infections such as bronchiolitis, caused | Level 2 | |
| | by bacteria, parasites, viruses or fungi. | Not meeting Level 1 of evidence AND | |
| | Localised eye and ear infections, | 3 or more criteria: | |
| | encephalitis, urinary tract infections and | • Temperature ≥37.5 ∘C or <35.5 ∘C | |
| | intestinal infections were excluded from | Tachycardia or new or more frequent episodes of bradycardia | |
| | these guidelines. | •New or more frequent episodes of apnea or increased oxygen requirement or increased | |
| | | requirement for ventilatory support | |
| | | Lethargy or moving only when stimulated or hypotonia or irritability | |
| | | Difficulty in feeding or abdominal distention | |
| | | Pallor or poor perfusion or hypotension | |
| | | •Abnormal White Cell Count or I/T ratio >0.2 | |
| | | Abnormal platelet count | |
| | | •Increased inflammatory markers (CRP, procalcitonin) | |
| | | Metabolic acidosis as defined by a base excess | |
| | | Level 3 | |
| | | Not meeting Level 1 or 2 of evidence AND | |
| | | 2 or more of the following criteria: | |
| | | • Temperature ≥37.5 ∘C or <35.5 ∘C | |
| | | Tachypnea or severe chest in drawing or grunting or cyanosis | |
| | | Change in level of activity | |
| | | History of feeding difficulty | |
| | | History of convulsions | |
| | | Bacterial/fungal/viral meningitis | |
| | | Level 1 | |
| | | Recognised pathogen identified using a validated method from cerebrospinal fluid (CSF) | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | (1 highest level to 4 lowest level of certainty) | |
| | | Level 2 | |
| | | CSF pleocytosis OR | |
| | | positive IgM antibodies to a specific pathogen in the CSF AND | |
| | | Recognised pathogen identified using a validated method from a normally | |
| | | sterile site (other than CSF) AND | |
| | | Temperature ≥37.5 °C or <35.5 °C AND | |
| | | 1 or more criteria: | |
| | | History of convulsions | |
| | | •Lethargy or irritability | |
| | | •Coma | |
| | | •Apnea | |
| | | •Bulging fontanel | |
| | | •Neck stiffness | |
| | | Level 3a | |
| | | CSF pleocytosis AND | |
| | | No pathogen identified using a validated method from a normally sterile site AND | |
| | | Temperature ≥37.5 °C or <35.5 °C AND | |
| | | 3 or more criteria: | |
| | | History of convulsions | |
| | | Lethargy or irritability | |
| | | • Coma | |
| | | • Apnea | |
| | | Bulging fontanel | |
| | | Neck stiffness | |
| | | Level 3b | |
| | | No lumbar puncture done or no sample available AND | |
| | | Temperature ≥37.5 °C or <35.5 °C AND | |
| | | 4 or more criteria: | |
| | | History of convulsions I otherwy or irritability | |
| | | Lethargy or irritability Coma | |
| | | Apnea Pulsing fentanel | |
| | | Bulging fontanel Neals of ffree and the second se | |
| | | Neck stiffness Particular to a toric life or and triple of a time. | |
| | | Respiratory bacterial/fungal/viral infection | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | (1 highest level to 4 lowest level of certainty) | |
| | | Level 1 | |
| | | New or progressive or persistent infiltrate or shadowing or fluid in the intrapleural cavity or | |
| | | interlobar fissure on chest X-ray AND | |
| | | Recognised virus identified using a validated assay from an upper respiratory sample OR | |
| | | Recognised pathogen identified using a validated method and from a normally sterile site | |
| | | AND | |
| | | 3 or more criteria: | |
| | | • Temperature ≥37.5 °C or <35.5 °C | |
| | | Tachypnea or Nasal flaring or Chest in-drawing or Grunting | |
| | | <ul> <li>Desaturations or increased oxygen requirements or increased ventilator requirements or</li> </ul> | |
| | | oxygen saturation <95% | |
| | | • Apneas | |
| | | <ul> <li>Increased respiratory secretions or Increased suctioning requirements</li> </ul> | |
| | | Cough or wheeze or crepitations | |
| | | Increased CRP or procalcitonin | |
| | | Level 2 | |
| | | New or progressive or persistent infiltrate or shadowing or fluid in the intrapleural cavity or | |
| | | interlobar fissure on chest X-ray AND | |
| | | 4 or more criteria: | |
| | | • Temperature ≥37.5 ∘C or <35.5 ∘C | |
| | | Tachypnea or Nasal flaring or Chest in-drawing or Grunting | |
| | | <ul> <li>Desaturations or increased oxygen requirements or increased ventilator</li> </ul> | |
| | | requirements or oxygen saturation <95% | |
| | | • Apneas | |
| | | <ul> <li>Increased respiratory secretions or Increased suctioning requirements</li> </ul> | |
| | | Cough or wheeze or crepitations | |
| | | Increased CRP or procalcitonin | |
| | | Level 3 | |
| | | 2 or more criteria: | |
| | | Difficulty in breathing/Tachypnea | |
| | | Severe chest in-drawing | |
| | | Nasal flaring | |
| | | • Grunting | |
| | | Wheezing | |
| | | • Stridor | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | (1 highest level to 4 lowest level of certainty) | |
| | | • Fever | |
| Respiratory distress | Constellation of clinical findings that | Level 1 | Sweet LR, Keech |
| in the neonate | support the presence of breathing | Newborn 0 to 28 days of life AND | C, Klein NP, et |
| | difficulty in the neonate. | Abnormal respiratory rate: | al. Respiratory |
| | | Measurement of number of breaths per minute consistent with: | Distress in the |
| | | Tachypnea = respiratory rate of more than 60 breaths per minute OR | Neonate: Case |
| | | Bradypnea = respiratory rate of less than 30 breaths per minute OR | Definition & |
| | | Apnea = cessation of respiratory effort (no breaths) for at least 20 seconds | Guidelines for |
| | | AND | Data Collection, |
| | | Clinical symptoms consistent with labored breathing | Analysis, and |
| | | Nasal flaring (dilatation of alae nasi) OR | Presentation of |
| | | Noisy respirations in the form of expiratory grunting, stridor, or wheeze OR | Maternal |
| | | Retractions or increased chest in-drawings on respiration (subcostal, intercostal, sternal, | Immunization |
| | | suprasternal notch) OR | Safety Data. |
| | | Central cyanosis (whole body, including lips and tongue) on room air OR | Unpublished |
| | | Low Apgar Score (< 7 points) at 10 min, with respiration score <2 AND | manuscript. |
| | | Examination and documentation by qualified, trained, health care provider appropriate for the | |
| | | clinical setting. | |
| | | Level 2 | |
| | | Newborn 0 to 28 days of life AND | |
| | | Abnormal respiratory rate: | |
| | | Not measured, but reported as "rapid breathing", "slow breathing", having periods of "no | |
| | | breathing", or "abnormal breathing" AND | |
| | | Clinical symptoms consistent with labored breathing | |
| | | Nasal flaring (dilatation of alae nasi) OR | |
| | | Noisy respirations in the form of expiratory grunting, stridor, or wheeze OR | |
| | | Retractions or increased chest in-drawings on respiration (subcostal, intercostal, sternal, | |
| | | suprasternal notch) or seesaw respirations OR | |
| | | Central cyanosis (whole body, including lips and tongue) on room air OR | |
| | | Low Apgar Score (< 7 points) at 10 min, with respiration score <2 AND | |
| | | No medical record documentation, but reporting through either a non-medical observer (e.g. | |
| | | mother, father, community worker) or via standard census mechanisms (e.g. Demographic | |
| | | and Health Surveillance System) OR | |
| | | Collection of information from medical record review or billing codes. | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | (1 highest level to 4 lowest level of certainty) | |
| | | Level 3 | |
| | | No need for a level 3 per working group. | |
| | | Level 4 | |
| | | Not enough information to ascertain case of respiratory distress. | |
| Stillbirth | Fetal death occurring before birth after | Antepartum Stillbirth | [DaSilva, 2016] |
| | a 20 to 28 weeks of gestation (variation | Fetal death occurs prior to the evidence of labor. | |
| | due to country definitions). | Level 1 | |
| | | •Delivery of an infant with no of signs of life at birth (No spontaneous movements, no umbilical | |
| | | cord pulse, no heartbeat, no respirations, Apgar score of 0 at 1 and 5 min) determined by | |
| | | physical examination after delivery (with or without electronic monitoring of heart rate, | |
| | | respiratory rate, and pulse oximetry). AND | |
| | | Prenatal ultrasound examination documenting lack of fetal cardiac activity or movement | |
| | | before the onset of labor. OR | |
| | | •Auscultation for fetal heart tones (using electronic devices or non-electronic devices) | |
| | | documenting lack of fetal heartbeat. AND | |
| | | •Maternal report of lack of fetal movement for 24 h or more. OR | |
| | | •Maternal physical examination confirming lack of fetal movement. OR | |
| | | •Radiology findings consistent with intrauterine fetal death. AND | |
| | | •Attended delivery followed by fetal physical examination afterbirth consistent with antepartum | |
| | | death, by obstetrician, neonatologist, pediatrician, maternal-fetal medicine specialist, or | |
| | | pathologist. In the setting where access to a specialist is not feasible, diagnosis by a health | |
| | | care provider trained or experienced to make the diagnosis is acceptable (e.g. general | |
| | | practice physician, mid-wife, nurse practitioner, a physician's assistant or other qualified | |
| | | trained practitioner). OR | |
| | | •Fetal/placental pathology report consistent with antepartum death. AND | |
| | | Gestational age within pre-defined range for selected stillbirth definition as assessed by | |
| | | maternal and/or fetal parameters (Level1 or 2 in GA assessment algorithm). | |
| | | Level 2 | |
| | | •Delivery of an infant with no of signs of life at birth (No spontaneous movements, no umbilical | |
| | | cord pulse, no heartbeat, no respirations, Apgar score of 0 at 1 and 5 min) determined | |
| | | physical examination after delivery. AND | |
| | | •Maternal report of lack of fetal movement for 24 h or more. OR | |
| | | •Maternal physical examination confirming lack of fetal movement. OR | |
| | | •Auscultation for fetal heart tones (using electronic or non-electronic devices) documenting | |
| | | lack of fetal heartbeat. AND | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty (1 highest level to 4 lowest level of certainty) | Reference |
|---|---|---|---|
| | | Attended delivery followed by physical examination after birth consistent with antepartum death, by specialist or qualified trained practitioner appropriate to the health care setting. OR Fetal/placental pathology report consistent with antepartum death. AND Gestational age within pre-defined range for selected stillbirth definition as assessed by maternal and/or fetal parameters (Level1–2 in GA assessment algorithm). Level 3 Delivery of an infant reported to have no of signs of life at birth(No spontaneous movements, no umbilical cord pulse, no heart-beat, no cry or spontaneous respirations, no chest movement, and whole body cyanosis). AND Maternal report of lack of fetal movement for 24 h or more prior to delivery. OR Report of auscultation for fetal heart tones (using electronic or non-electronic devices) documenting lack of fetal heartbeat. AND Non-attended delivery followed by physical examination of the fetus after birth consistent with antepartum death by a healthcare professional appropriate to the level of standard of care in the health care setting. OR Verbal history by a trained health care provider, non-medical witness or the mother of a fetus born with no signs of life or unresponsive to resuscitation efforts immediately after birth and with physical features consistent with antepartum death. AND Gestational age within pre-defined range for selected stillbirth definition as assessed by maternal and/or fetal parameters (Level2–3 in GA assessment algorithm). Level 4•Report of stillbirth but fetus is not available for physical examination after birth (no objective assessment can be made) Maternal information insufficient to assess gestational age | |
| | | Intrapartum stillbirth Fetal death occurs during labor and before delivery Level 1 •Delivery of an infant with no of signs of life at birth, including: No spontaneous movements, no umbilical cord pulse, no heartbeat, no respirations, and Apgar score of 0 at 1 and 5 min •Determination of the absence of signs of life is made by physical examination after delivery, with or without electronic monitoring of heart rate, respiratory rate, and pulse oximetry. AND •Evidence of live fetus prior to onset of labor (documentation of fetal movement and of fetal heart tones by ultrasound prior to onset of labor) (Note: in the absence of evidence of a live fetus prior to the onset of labor, the fetal death should be reported as a stillbirth or an antepartum stillbirth).AND | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | (1 highest level to 4 lowest level of certainty) | |
| | | •Attended delivery followed by physical examination afterbirth consistent with intrapartum | |
| | | death by obstetrician, neonatologist, pediatrician, maternal-fetal medicine specialist, | |
| | | pathologist. In the setting where access to a specialist is not feasible, diagnosis by a health | |
| | | care provider trained or experienced to make the diagnosis is acceptable (e.g. general | |
| | | practice physician, midwife, or other qualified trained practitioner).AND | |
| | | •Gestational age within pre-defined range for selected stillbirth definition as assessed by | |
| | | maternal and/or fetal-neonatal parameters (Level 1 in GA assessment algorithm) | |
| | | Level 2 | |
| | | •Delivery of an infant with no of signs of life at birth, including: No spontaneous movements, | |
| | | no umbilical cord pulse, no heartbeat, no respirations, and Apgar score of 0 at 1 and 5 min. | |
| | | •Determination of the absence of signs of life is made by physical examination after delivery, | |
| | | with or without electronic monitoring of heart rate, respiratory rate, and pulse oximetry OR | |
| | | documentation of lack of response to resuscitation efforts. AND | |
| | | •Evidence of live fetus prior to onset of labor (maternal report of fetal movement prior to onset | |
| | | of labor and documentation of fetal heart tones by auscultation or hand held Doppler) (Note: | |
| | | in the absence of evidence of a live fetus prior to the onset of labor, the fetal death should be | |
| | | reported as a stillbirth or an antepartum stillbirth). AND | |
| | | •Attended delivery followed by physical examination after birth consistent with intrapartum | |
| | | death by a health care professional appropriate to the level of standard of care in the health | |
| | | care setting. AND | |
| | | •Gestational age within pre-defined range for selected stillbirth definition as assessed by | |
| | | maternal and/or fetal parameters (Level1–2 in GA assessment algorithm). | |
| | | Level 3 | |
| | | •Delivery of an infant reported to have no of signs of life at birth, including: No spontaneous | |
| | | movements, no umbilical cord pulse, no heartbeat, no cry, no spontaneous respirations or | |
| | | chest movement, and whole body cyanosis. AND | |
| | | •Evidence of live fetus prior to onset of labor (maternal report of fetal movement prior to onset | |
| | | of labor OR auscultation of fetal heart tones) (Note: in the absence of evidence of a live fetus | |
| | | prior to the onset of labor, the fetal death should be reported as a stillbirth or an antepartum | |
| | | stillbirth). AND | |
| | | •Non-attended delivery followed by physical examination of the fetus after birth consistent with | |
| | | intrapartum death by a healthcare professional appropriate to the level of standard of care in | |
| | | the health care setting OR verbal history by a trained health care provider, non-medical | |
| | | witness or the mother of a fetus born with no signs of life or unresponsive to resuscitation | |
| | | efforts immediately after birth. AND | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Event of interest | Description | Levels of diagnostic certainty | Reference |
|---|---|---|---|
| | | (1 highest level to 4 lowest level of certainty) | |
| | | •Gestational age within pre-defined range for selected stillbirth definition as assessed by maternal and/or fetal parameters (Level2–3 in GA assessment algorithm). Level 4 | |
| | | •Report of stillbirth but fetus is not available for physical examination after birth (no objective assessment can be made). •Maternal information insufficient to assess gestational age. | |
| Preterm birth | Birth in less than 37 gestation completed weeks (less than 259 days). | Prematurity and assessment of gestational age Level 1 Certain LMP or intrauterine insemination (IUI) date or embryo transfer (ET) date with confirmatory 1st trimester scan (≤13 6/7 weeks). OR 1st trimester scan (≤13 6/7 weeks) Level 2A Certain LMP* with 2nd trimester scan (14 0/7 weeks to 27 6/7weeks). If LMP and U/S do not correlate, default to U/S GAassessment.OR2. Certain LMP* with 1st trimester physical examination. Level 2B Uncertain LMP with 2nd trimester scan (14 0/7 weeks to 276/7 weeks). Level 3A Certain LMP with 3rd trimester scan – 28 0/7 weeks + OR Certain LMP with confirmatory 2nd trimester FH OR Certain LMP with birth weight OR Uncertain LMP with 1st trimester physical examination. Level 3B Uncertain LMP with FH. OR Uncertain LMP with newborn physical assessment. OR Uncertain LMP with Birth weight Definitions of LMP, birth weight and physical assessment in article. | [Quinn, 2016] |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| GlaxoSmithKline Biologicals | |
|---|---|
| Vaccines R & D | |
| Protocol Ameno | dment 2 |
| eTrack study number and Abbreviated Title | 207636 (EPI-RSV-008 BOD) |
| Amendment number: | Amendment 2 |
| Amendment date: 03-JUL-2018 | |
| Co-ordinating author: | , Lead Science Writer |

### Rationale/background for changes:

The protocol has been amended to reflect the following changes and provide the following clarifications / corrections.

- The title and detailed title have been re-phrased in an effort to improve their clarity.
- The Glossary of terms has been updated.
- Objectives and endpoints have been re-phrased for improved consistency with epidemiological terminology.
- In the inclusion criteria for pregnant women, language regarding informed consent has been clarified.
- Language describing inclusion criteria for infants has been clarified.
- For infants, a Month 6 visit has been added.
- Memory aids have been replaced with Diary cards.
- Subject cards have been added.
- An interim analysis has been added.
- Laboratory assays described in Appendix B have been updated.
- Laboratory addresses in Appendix B have been updated.
- Additional editorial changes have been made to ensure consistency with the modifications noted above, and typographical errors have been corrected.

Text that has been moved or added is presented in bold italics and deleted text in strikethrough in the following sections.

## Global changes:

Global additions/replacements are displayed in boldface italics in the document but are not enumerated word by word here.

US spellings replace UK spellings of terms such as hospitaliszation, paediatric, haematology, enrol*l*ment, labour, and tit*e*re.

"Maternal/fetal" has been replaced throughout with the term "maternal."

"Difficulty breathing" has been replaced with "Difficulty *in* breathing."

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Where reference is made to specifically to the first 28 days of life, the term "neonate/infant" has been replaced with the term "neonate."

### Title:

A <u>Prospective Epidemiological</u> prospective epidemiological study of <u>Outcomes</u> pregnancy outcomes and of events of interest in pregnant women, <u>Neonates</u> neonates and <u>Infants</u> infants (PE**P**NI)

### **Detailed Title:**

A prospective epidemiological study of women as of between 24-27 weeks of pregnancyand their infants up to 1 year of age, to describe maternal, fetal and neonatal pregnancy outcomes, pregnancy-related and /infant and events of interest and in the occurrence mother and neonate, as well as determine incidence in neonates-infants of RSV LRTI and RSV hospitalization.

## **Contributing Authors:**

Two lists are now provided. The first is a list of authors who contributed to Amendment 2. The second is a list of authors who contributed to previous versions of the document. Persons who appear as contributing authors for the first time are:

| • PPD | , Clinical Research and Development Lead |
|----------|------------------------------------------|
| • PPD | , Expert Epidemiology Biostatistician |
| • PPD | , Clinical Trial Supply manager |
| • PPD | , Clinical Read-Out Team Leader |
| • PPD | , Safety Physician |
| • PPD | , Study Delivery Lead |
| PPD | replaces PPD as the CEPL. |
| Classamy | |

## Glossary

Child A young human being below the legal age of majority (generally  $\leq$  < 18 years of age).

204

Enrollment

Pregnant woman who meet all eligibility criteria at the Screening visit and return to the study site for Visit 1 are considered enrolled. Live born neonates who meet all eligibility criteria and complete Visit 1-NB are considered enrolled.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

**GAIA** 

Global Alignment of Immunization Safety Assessment in pregnancy. A project that aims to improve the quality of outcome data from clinical vaccine trials in pregnant women with a specific focus on the needs and requirements for safety monitoring in low to middle income countries.

Local healthcare provider

A healthcare provider who provides subjects with medical care per local standards. This individual may or may not be a member of the study staff.

Neonatal events of interest

Events as described in Clinically significant events that

occur from birth through 28 days of age and may be

considered adverse events if they occur after

vaccination. They are listed in Section 11.1 that occur from birth through 28 days of age.and described in detail

in APPENDIX D.

Parental concern

The parent(s) / Legally Acceptable Representative(s) or their designates are concerned about the infant's respiratory tract illness or general health and intend to seek medical care

Pregnancy related events

of interest

Events as described in Section 11.1 that occur from Visit 1 through Visit 6 (Day 42). Clinically significant events that occur up to 42 days after delivery and may be considered adverse events if they occur after vaccination. They are listed in Section 11.1 and described in detail in APPENDIX D.

## **Synopsis:**

### **Rationale for the study:**

This multi-country study will enroll pregnant women  $\geq 24^{0/7}$  weeks and  $\leq 28^{0/7}$  weeks gestational age (GA). Study procedures in this protocol are defined to ensure that maternal and neonatal events of interest are captured. They are not intended to replace procedures performed by local healthcare providers as part of standard care. Prenatal screening and care will be provided by local healthcare providers as much as possible and information will be collected and recorded in this study's electronic case report form (eCRF (in accordance with local standards).

- End of Study (EoS): ... samples collected up to *Visit* 3 *4-NB.*..
- Epoch 003: ... ending at *Visit* 3 *4-NB* (1 year post-birth).

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# Background and Rationale (Section 1.1 and Synopsis "Rationale for the Study and Study Design")

...Several marketed vaccines are already recommended for and routinely administered to pregnant women, including influenza, tetanus and Tdap vaccines (MMWR 2013, ACIP 2012). CDC 2013a, CDC 2013b). There are also a number of maternal vaccines in development that aim to protect neonates and infants from additional pathogensineluding in addition to respiratory syncytial virus (RSV). GlaxoSmithKline (GSK) is developing an investigational vaccine for use in pregnant women, against RSV disease. Of note these vaccines are this vaccine is developed solely for immunization in pregnancy.

Maternal immunization is implemented worldwide and has the potential to make a major contribution to reducing RSV lower respiratory tract infections (LRTI) and other disease the burden of other diseases in infants globally.... GSK is proactively addressing potential challenges of conducting clinical trials in pregnant women in low- and middle income countries (LMIC).

Understanding Before conducting clinical trials it is important to understand the frequency of pregnancy outcomes and the maternal, and neonatal outcomes and events of interest (i.e. clinically significant events that may be considered adverse events if they occur after vaccination) in each setting prior to conducting where clinical trials is critical may be conducted for better interpretation of safety data. Also, to ensure safety of the participating women, and to characterize the safety profile of the product, adverse events (AEs) in pregnancy should be appropriately detected and managed. This study addresses gaps in understanding of anticipated rates of pregnancy outcomes and as well as events of interestFurtherin pregnant women and neonates. Furthermore, this study will be conducted at potential sites for future maternal immunization trials and will help assure the capacity of sites to detect and manage clinically significant events of interest in pregnant women and their neonates. It will also establish surveillance mechanisms for infections and events of interest.

**Secondarily, the study** will establish surveillance mechanisms for RSV infections *in the neonate/infant(through the first 12 months of life.* Whilst there is good documentation of the global burden of RSV disease, incidence of RSV-LRTI according to the World Health Organization (WHO) 2015 case definitions [Modjarrad, 2016] is lacking *limited* in the literature, *particularly in many LMIC settings*. Hence, this study will also estimate the incidence of infant RSV-LRTI using WHO case definitions across geographically distinct locations to support incidence rate assumptions for planning of future efficacy trials.

Section 1.1 only: Standardization of surveillance methodology and case definitions (applicable to maternal immunization AEs) may support comparison of data across different countries [Jones, 2016].

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

### **Rationale for the Study Population (Section 1.1.1 and Synopsis)**

The intention of this trial epidemiological study is to obtain an estimate of the background rate of adverse pregnancy outcomes and events that will may be seen in future vaccine trial populations and, separately, to assess whether sites are suitable for Phase II/III vaccine trials.

# Rationale for the Surveillance System for the detection of pregnancy related events of interest (Section 1.3)

There are particular challenges in conducting clinical trials in pregnant women, among them limited data on background rates of *pregnancy outcomes as well as what may be observed in clinical trials as* maternal and neonatal outcomes and adverse events.

This study is not intended to provide comprehensive antenatal care or to replace local antenatal standard of care, but rather to leverage the data (e.g., clinical findings, diagnoses, laboratory results) captured in local antenatal standard of care. *Information obtained from s*tudy specific procedures and laboratory *tests* (e.g. blood sampling, urine dipstick) is not to be relied upon for clinical management of study subjects.

To achieve these goals, GSK will be guided by the WHO recommendations on antenatal care for a positive pregnancy experience [WHO, 2016] and the Global Alignment of Immunization Safety Assessment in pregnancy (GAIA) case definitions [Bonhoeffer, 2016; Bauwens, 2016; Kochhar, 2017]. Standardization of surveillance methodology and case definitions (applicable to maternal immunization AEs) may support comparison of data across different countries [Jones, 2016].

The number and timing of study visits was informed by WHO recommendations on antenatal care [WHO, 2016]. However, local standards of care differ *from* country-by-to country. Women should follow the local standard of care. Study visits *data* will be used to collect and record *collected*, *in part, from records of* the data obtained during the locally recommended antenatal care visits.

In this study, best efforts will be made to work with local healthcare providers to collect the key data on maternal, fetal-and, neonatal *and infant* health from routine health records to avoid duplication and an undue burden on the trial subjects.

# Rationale for the use of Global Alignment of Immunization safety Assessment in pregnancy (GAIA) case definitions (Section 1.4)

GAIA, a Brighton collaboration project, aims to develop standardized case definitions and criteria for diagnostic certainty of maternal *outcomes and events of interest* and neonatal *outcomes events of interest* in the context of immunization trials [Bauwens 2016, Bonhoeffer 2016, Kochhar 2017].

Rationale for the active and passive surveillance for RSV associated respiratory tract infections (RTI) with suspicion of difficulty in breathing/wheezing or with parental concern in neonates/ infants (Section 1.5)

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

As part The implementation of the RSV maternal program, this study aims to set up the surveillance will also assist in establishing robust infrastructure and processes for RSV-LRTI and RSV hospitalization detection, for site preparedness in future vaccine trials.

### **Benefit Assessment (Section 2.2)**

Study procedures aim to ensure adequate-surveillance for maternal and neonatal outcomes of pregnancy and events of interest and neonatal events of interest. The attention to adequate surveillance of these events may enhance the ability to detect these safety events and to refer subjects for management according to local standard of care. The protocol also includes procedures that may enhance surveillance for RSV, and possibly other lower respiratory tract infections, in neonates and infants. Thus, the procedures described in this protocol may enhance the ability to detect these events or infections and to refer subjects for management according to local standard of care.

Data collected during the study may enhance understanding of the incidence *frequency* of maternal events of interest in women with low risk pregnancies, neonatal events of interest, and *RSV-associated* lower respiratory tract infections associated with RSV infection in neonates and infants.

## **Overall Benefit: Risk Conclusion (Section 2.3)**

......and by the knowledge gained about the incidence *frequency* of medical events of interest.

# **Primary Objectives (Section 3.1 and Synopsis)**

- *To determine the frequencies* of *Visit 1*: To detect and describe pregnancy outcomes.
- To detect and describe determine the frequencies of pregnancy related events of interest
  - from enrollment (Visit 1) through 42 days after delivery (Visit 6).
  - (Although pregnancy related events of interest occur within the first 42 days after delivery they may only be detected later, and are to be reported throughout the study.)
- To detect and describe determine the frequencies of neonatal events of interest.

Neonatal AEs of interest occur within the first 28 days after birth, but may only be detected later and are to be reported throughout the study.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## **Secondary Objectives (Section 3.2 and Synopsis)**

In healthy pregnant women with uncomplicated pregnancies as of Visit 1 at enrollment:

- To detect and describe determine frequencies of pregnancy related events of interest according (where these are specified) to GAIA levels of diagnostic certainty (where these are specified) (APPENDIX D) from enrollment (Visit 1) through 42 days after delivery (Visit 6). (Although pregnancy related events of interest occur within the first 42 days after delivery they may only be detected later, and are to be reported throughout the study.)
- To describe *the distribution of* RSV-A antibody titers in maternal blood at delivery
- To detect and describe determine frequencies of neonatal events of interest according (where these are specified) to GAIA levels of diagnostic certainty (where these are specified). (APPENDIX D).

  Neonatal AEs of interest occur within the first 28 days after birth, but may only be detected later and are to be reported throughout the study.
- To describe *the distribution of* RSV-A antibody titers in cord blood *at delivery*.
- To describe occurrences of determine the incidence of all, of severe, and of very severe RSV-lower respiratory tract infections (LRTIs).
- To describe occurrences determine the incidence of RSV hospitalization.
- Refer to the GLOSSARY OF TERMS for the definition of enrollment.

### **Tertiary Objectives (Section 3.3 and Synopsis)**

- To *describe* the association *co-infections* of *RSV-LRTI* with other respiratory viruses with the occurrence of RSV-LRTI in infants.
- To describe estimate the association between of RSV-LRTI in neonates/infants and the level of RSV neutralizing antibodies in cord blood.
- To describe determine risk factors for pregnancy-related and neonatal events of interest
- If deemed necessary, to further characterize the immune responses to the diseases under study RSV and other infections in pregnant women/mothers and infants, and/or to explore further parameters in pregnant women (mothers) or their infants.(based on maternal serum and cord blood).

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## Study Design Figure 1 and accompanying footnotes (Section 4.0)

The design figure has been adjusted to add a 6-month visit in infants and to indicate that an interim analysis will be performed. The entire figure is reproduced below.



### **Study Design Footnotes**

Refer to Section 11.11 for additional information about the analyses indicated above.

### Study population (Section 4.0 and Synopsis)

• Study population: The study will be conducted in multiple countries, in pregnant women and their neonates in fants.

<sup>&</sup>lt;sup>4</sup> Blood Allowed interval for blood sample should be collected within collection begins with start of labor (e.g. when the mother arrives at the hospital to deliver and an intravenous line is inserted) and ends 72 hours after delivery.

<sup>&</sup>lt;sup>6</sup>Neonatal conditions events of interest occur (by definition) between 0 and 28 days after birth. They will be reported once site staff become aware of them (whether this occurs during the first 28 days after birth, or at a later time).

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# Sampling schedule for pregnant women/mothers, Table 1 and Synopsis Table 1, footnote 5:

<sup>5</sup>This sample may be collected <del>as</del> from start of labour (e.g. when the mother arrives at the hospital to deliver and an intravenous line is inserted) ) *through 72 hours after delivery*.

- Sampling schedule for **neonates/infants**: Surveillance for RSV LRTI will be conducted in infants through the 12 month study period. During the this 1-year post-birth surveillance period, for each RTI with suspicion of difficulty in breathing, or wheezing, or with parental concern, a nasal swab will be collected at a visit to assess potential RSV associated RTIs/LRTIs.
- Epoch 003: Follow-up of infants starting 43 days post-delivery/birth and ending at Visit 3-4-NB (1 year post-birth).
- Surveillance for pregnancy outcomes and pregnancy-related events of interest (Section 8.5.8) *that occur* from Visit 1 up to 42 days after delivery (*Visit 6*).

### **Footnotes to Table 3:**

## Pregnancy related events of interest (Section 5.1)

Pregnancy related events of interest are *briefly defined in the GLOSSARY OF TERMS* ......

## **Neonatal events of interest (Section 5.2)**

Neonatal events of interest are *briefly defined in the GLOSSARY OF TERMS*...

<sup>&</sup>lt;sup>2</sup> For blood oxygen saturation (SpO<sub>2</sub>), the lowest value monitored will be used. *In high altitudes (>2500m), SpO*<sub>2</sub> <92% for LRTI, <90% for severe LRTI, <87% for very severe LRTI.

<sup>&</sup>lt;sup>5</sup> RSV sampling and testing is based on medical judgment of medical practitioner or driven by algorithm.

<sup>6</sup> Hospitalization is defined as a medical decision that the child requires admission for observation or treatment based on the judgement of a health care provider.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

### **Inclusion Criteria for Enrolment (Section 6.2)**

## **Pregnant Women (Section 6.2.1)**

- Individuals who gave give written or witnessed/thumb printed informed consent after the study had has been explained according to local regulatory requirements. Informed
  - The informed consent given at screening should either include consent for study both the mother's participation and participation of the mother should be obtained from the mother or infant after the infant's birth (if consistent with local regulations/guidelines), or consent for the mother's participation and expressed willingness to consider permitting the infant to take part after the infant has been born (if local regulations/guidelines require parent(s) to provide an additional informed consent after the infant's birth).
  - Both mother and father, as applicable by local law, prior to performance of any study specific procedures; should consent if local regulations/guidelines require it.
- Individuals (mother or mother and father) who, at the time of their informed consent, express willingness to enroll their infant in the study at the time of birth.

## Infants (Section 6.2.2):

- Infants live born to enrolled women that resulted from the enrolled pregnancy Infants who were *in utero at the time maternal (and paternal, if required)* informed consent *was given, and* who are live-born.
- If local law requires it: Written or witnessed/thumb printed informed consent for study participation of the infant obtained from the infant's mother and/or father, as applicable by local law, or parent(s)/LAR(s) within 10 days of birth.

## **General Study Aspects (Section 8.2)**

Supplementary Critical study conduct information not mandated to be present in this protocol is provided in the Study Procedures Manual (SPM). As such, the SPM should be viewed as a companion document that should be read carefully to fully understand the study protocol. The SPM provides the investigator and the site personnel with administrative and detailed technical operational information that is essential for correct study execution and does not impact the safety of the subjects.

Study *visits and* procedures in this protocol are defined to ensure that maternal, fetal and neonatal events of interest, *as well as RSV-associated LRTIs and RSV hospitalization in infants*, are captured. Prenatal screening and care will be provided by local healthcare providers and information will be collected and recorded in the eCRF. (in accordance with local standards).

Study visits are not intended to replace local standard of care antenatal visits. If local standard of care recommends additional visits/medical evaluations during pregnancy, women participating in this study should comply with their regular antenatal care visit schedules, per local recommendations.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Study procedures are not intended to replace procedures performed by local healthcare providers as part of standard care.

# **Outline of Study Procedures (Section 8.3)**

# **Table 4, List of Study Procedures**.

No columns were added with this amendment. Only rows where changes were made have been presented. Only footnotes where changes were made have been presented.

| Gestational age | ≥ 24 <sup>0/7</sup> - 27 <sup>6/7</sup> | 24<br>0/7 _<br>27<br>6/7 | 28 <sup>0/7</sup><br>-<br>31 <sup>6/7</sup> | 32 <sup>0/7</sup><br>-<br>35 <sup>6/7</sup> | 36 <sup>0/7</sup> -<br>delivery | | | |
|---|---|---|---|---|---|---|---|---|
| Epoch | Epoch<br>001 | Epoch 002 | | | | | | |
| Type of contact | Screening | Visit<br>1 | Visit 2 2 | Visit 3 <sup>2</sup> | Visit 4 <sup>2</sup> | Visit 5 | Visit 6 | Additional antenatal/medical evaluations (external to study visits/procedures)4 |
| Timepoints | | Day<br>1 | Day<br>28 | Day<br>56 | Day 84 | At<br>Delivery | Post-<br>Delivery<br>Day 42 | |
| Eligibility Review and Confirmation | | | | | | | | |
| Informed consent 1 | • | | | | | | | |
| Inform study paediatrician and/or staff of | | | | | | | | |
| subject's participation Ensure that site study physicians | | 0 | | | | 0 | | |
| (both obstetrician(s) and pediatrician(s)) are informed | | | | | | | | |
| Medical History / Examinations | | | | | | | | |
| Distribute<br>Maternal Subject<br>Card | | o | | | | | | |
| Distribute maternal health memory aid diary card | | 0 | 0 | 0 | 0 | 0 | 0 | |
| Review and collect maternal diary card | | | 0 | 0 | 0 | 0 | 0 | |
| Transcribe applicable diary card data to the eCRF | | | • | • | • | • | • | |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| | | | | | | | 1 1010001 | Amendment 4 mile |
|---|---|---|---|---|---|---|---|---|
| Gestational age | ≥ 24 <sup>0/7</sup> - 27 <sup>6/7</sup> | 24<br>0/7 _<br>27<br>6/7 | 28 <sup>0/7</sup><br>-<br>31 <sup>6/7</sup> | 32 <sup>0/7</sup><br>-<br>35 <sup>6/7</sup> | 36 <sup>0/7</sup> -<br>delivery | | | |
| Epoch | Epoch<br>001 | Epoch 002 | | | | | | |
| Type of contact | Screening | Visit<br>1 | Visit 22 | Visit | Visit 4 <sup>2</sup> | Visit 5 | Visit 6 | Additional antenatal/medical evaluations (external to study visits/procedures)4 |
| Timepoints | | Day<br>1 | Day<br>28 | Day<br>56 | Day 84 | At<br>Delivery | Post-<br>Delivery<br>Day 42 | |
| Travel history to, or living in, Zika virus endemic countries/regions with Zika virus transmission | 0 | • | | | | | | |
| Record results of<br>General and<br>Obstetric<br>examination <sup>10</sup> | • | • | • | • | • | | • | • 13 |
| Check and record prescription medications, vaccinations, folate and/or iron (independently or included in a multivitamin) 12 | • | • | • | • | • | • | • | • |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| | | | | | | | 1 1010001 | Amenament 4 rin |
|---|---|---|---|---|---|---|---|---|
| 0.445 | ≥ <b>24</b> <sup>0/7</sup> - | 24<br>0/7 _ | 28 0/7 | 32 0/7 | 36 <sup>0/7</sup> - | | | |
| Gestational age | <b>27</b> 6/7 | <b>27</b> 6/7 | 31 <sup>6/7</sup> | 35 <sup>6/7</sup> | delivery | | | |
| Epoch | Epoch<br>001 | | | l . | E | Epoch 002 | | |
| Type of contact | Screening | Visit<br>1 | Visit 2 <sup>2</sup> | Visit | Visit 4 <sup>2</sup> | Visit 5 | Visit 6 | Additional antenatal/medical evaluations (external to study visits/procedures)4 |
| Timepoints | | Day<br>1 | Day<br>28 | Day<br>56 | Day 84 | At<br>Delivery | Post-<br>Delivery<br>Day 42 | |
| Biological<br>Specimens /<br>Laboratory Test<br>Results | | | | | | | | |
| Record results of local hematology/biochemical analysis ( <i>up to</i> 10 <i>Visit</i> 1~5.5 ml; <i>Visit</i> 3~2 ml – hemoglobin only) | | • | | • | | | | ●13 |
| Record results of<br>urine dipstick to<br>check for<br>presence of<br>proteins, glucose,<br>RBC, WBC <sup>7</sup> | | • | • | • | • | | | ●13 |
| Record results of any clinically significant abnormal laboratory tests (including positive urine culture) if performed by local healthcare provider and available <sup>5</sup> | | 0 | 0 | 0 | 0 | 0 | 0 | • |
| Outcomes and<br>Events of Interest | | | | | | | | |
| Record pregnancy-related events of interest and other clinically significant events or diagnoses that could impact the pregnancy | | • | • | • | • | • | • | • |

<sup>&</sup>lt;sup>1</sup> Refer to Section 6.2.1, fifth bullet.

<sup>&</sup>lt;sup>8</sup>-At Visit 3, only hemoglobin testing.
207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### **Table 5, List of Study Procedures**

One column was added to account for the 6 month visit. Because a column was added, the amended table has been presented in its entirety. All footnotes (since only 1 was unchanged) have also been provided.

| Epoch | Еро | ch 002 | Ерос | h 003 | Epoch 002 a | nd Epoch 003 |
|---|---|---|---|---|---|---|
| Ago | 0-10 | 42 | 6 | 12 | 0.12 n | nonths |
| Age | days | Days | Months | months | | iioiitiis |
| Type of contact | Visit<br>1-NB | Visit 2-<br>NB <sup>b</sup> | Visit 3-<br>NB <sup>b</sup> | Visit 4-<br>NB <sup>b</sup> | Contact for active/ passive surveillance | Visit to assess potential LRTI |
| Timepoints | Birth | Day 42 | | Y1 | | |
| Check inclusion/exclusion criteria | • | | | | | |
| Obtain <b>post-delivery</b> informed consent of <b>from</b> parent(s)/LAR(s) <b>if required per local regulations</b> | • a | | | | | |
| Record infant's subject number | • | | | | | |
| Record Apgar assessment | • | | | | | |
| Record demographic data | • | | | | | |
| Record lifestyle characteristics | | • | | | | |
| Distribute Infant's Subject Card | 0 | | | | | |
| Distribute <i>infant</i> health and RTI memory aiddiary card <sup>d</sup> | 0 | 0 | 0 | | | 0 |
| Review infant diary card | | 0 | 0 | 0 | | 0 |
| Collect infant diary card ef | | 0 | 0 | 0 | | 0 |
| Transcribe applicable infant diary card data to eCRF | | • | • | • | | • |
| Weight, length, head circumference, results of targeted medical history, and results of physical examination | • | • | • | • | | |
| Record prescription medications / vaccinations | • | • | • | • | • | • |
| Record neonatal events of interest | • | • | • | • | | |
| Clinical evaluation of potential LRTI | | | | | | • |
| Nasal swab <sup>b</sup> | | | | | | ● c |
| Record all hospitalizations and clinically significant events | • | • | • | • | • | • |
| Record SAEs related to study | • | • | • | • | • | |
| participation | | | | | | • |
| Study conclusion | | | | • | | |
| Investigator sign-off on eCRF before analysis | | • | • g | • | | |

a If local regulations require that confirmation of consent for the infant's participation be obtained at birth.

<sup>&</sup>lt;sup>13</sup> Beginning the month before the estimated date of conception and while on study. (Routine <del>concomitant medications</del> administered during labor and delivery need not be collected.)

<sup>14</sup> Record If-clinically significant abnormal results

b Visits 2-, 3-, and 4-NB Visit 2-NB (Day 42), Visit 3-NB (Year 1) and LRTI assessment visits may take place in the subject's home (if the standard of care allows for home visits), at the investigator's clinical facility or at another facility per the investigator's judgment.

<sup>&</sup>lt;sup>c</sup> If more than one assessment visit is conducted to evaluate a potential LRTI episode, additional nasal swabs may be collected at the discretion of the Investigator.

<sup>&</sup>lt;sup>d</sup> Distribute at V1-NB: Distribute additional diary cards at subsequent visits as needed.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Table 6: Intervals between study visits/contacts/observations

| Interval | Optimal interval *** | Allowed interval** |
|---|---|---|
| Birth → Visit 3-NB | 180 days | 166 -194 days |
| Birth → Visit 3 4-NB | 365 days | 351 <del>– 407</del> - 379 days |

#### **Eligibility Review and Confirmation (Section 8.5.1)**

- Obtain informed consent as The signed/witnessed/thumb printed informed consent of the subject must be obtained before study participation. Refer to Section 7.1 for the requirements on how to obtain informed consent, as appropriate. The father of the unborn child should also sign the mother's ICF, if required by the local regulations/guidelines/described in Sections 6.2.1 and 7.1.
- Inform-For eligible pregnant women who complete visit 1 (are enrolled): ensure that site study paediatrician physicians (both obstetrician(s)) and pediatrician(s)) are informed. In particular, the study pediatrician and/or staff of the pregnant woman's participation copy of the informed consent should be forwarded to the study paediatrician and/or staff notified as soon as possible after a pregnant woman's enrolment to ensure the study pediatrician is informed in a timely manner of the approximate date of delivery and potential enrolment of the neonate.

#### History and Examinations for pregnant women/mothers (Section 8.5.2)

- Distribute the Maternal Health Memory Aid. It is intended to serve as a reference during study visits/contacts, to help the subject provide the investigator/ study staff with protocol-specified data (and contact information for other healthcare providers, so medical records may be requested if required). (Refer to the SPM for details).
- Distribute *the Maternal Subject Card* (Section 9.3).
- Distribute the Maternal Diary Card to the subject (Section 8.5.4).
- Record demographic data, which may include (but is not limited to) information such as race, month and year of birth, *and* ethnicity *and geographic location*.
- Record information about whether the subject has travelled to / is living in Zika virus endemiccountries / regions with Zika virus transmission.

#### Maternal Diary Card (Section 8.5.3)

A maternal diary card will be provided to each subject at visit 1, then collected and replenished throughout the study as needed. It will document any prescription medications, folate and/or iron (independently or included in a multivitamin) taken, any vaccinations received during pregnancy and after delivery, and any additional visits the subject may make to a healthcare provider not affiliated with the study.

Collect diary cards that are fully filled out and / or document (L)RTI episodes that have ended (as defined in Section 8.6.5.1). Provide new diary cards as needed.

f Collect all diary cards for potential RTIs that are considered resolved. Collect the diary card for the current potential LRTI once the episode has ended (as defined in Section 8.6.5.1).

g After at least 50% of infants have completed Visit 3-NB, an interim analysis on data that is as clean as possible will be performed.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

The diary card will be reviewed with the subject during study visits. If review indicates that the subject visited a healthcare provider not affiliated with the study, study staff should (if permitted by local regulation) contact that healthcare provider to obtain the medical record(s) for the visit.

Refer to the SPM for additional details.

## Biological Specimens / Laboratory Data for pregnant women/mothers (Section 8.5.4)

• If performed by local healthcare provider and *results are* available, the investigator/site staff will also......

#### **Labor and Delivery (Section 8.5.4)**

 Medications Any medications administered during labor and delivery as per standard of care if not considered routine

Concomitant medications Medications, vaccinations, and supplements for administered to pregnant women/mothers as per standard of care (Section 8.5.6)

See Section 8.5.6 for medications administered during labor and delivery

#### Outcomes and Events of Interest in pregnant women/mothers (Section 8.5.7)

- If there is no live birth, all study visits and procedures related to the maternal subject should *still* be followed up to study end.
- Maternal events of interest (including, but not limited to, those described in Section 11.1.1) occurring up to Visit 6 (Post-delivery Month 1.5Day 42) should be recorded in the eCRF

## Additional Antenatal / medical evaluations external to study visits / procedures (Section 8.6.8)

For any additional antenatal / medical evaluations at which a pregnancy related event of interest is identified, record information that supports the diagnosis of the event, *if* available.

#### Eligibility Review and Confirmation for Neonates (Section 8.6.1)

- Check all applicable inclusion and exclusion criteria *as described in Sections 6.2.2* and 6.3.2. A neonate who does not meet the eligibility criteria should be considered ineligible.
- Obtain informed consent from parent(s) / LAR(s) at Visit 1-NB, as per local requirements.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### **History and Examinations for Neonates / Infants (Section 8.6.2)**

- Record lifestyle characteristics. Data may include (but are not limited to) passive smoking and day-care attendance contact with young children under 6 years of age.
- Distribute *the Infant* Health and RTI Memory Aid Subject Card to the parent(s)/LAR(s)/designate(s). The memory aid is intended to serve as a reference during study visits/contacts, to help (Section 9.3).
- **Distribute the Infant Diary Card** to the parent(s)/LAR(s)/designate(s) provide the investigator/ study staff with protocol-specified data (and contact information for other healthcare providers, so medical records may be requested if required). (Section 8.6.3).

#### Infant Diary Cards (Section 8.6.3)

[Note that numbering for all subsections that follow this *new* section was incremented, and the adjustments are reflected in updated cross references].

Infant diary cards will be provided at the infant Visit 1 NB. They should be completed by the Parent(s)/LAR(s)/designate(s) of the infant subject.

The infant diary cards will be used to document:

- RTI symptoms experienced by the infant, including start and end dates for those symptoms, and
- Additional visits to a pediatric healthcare provider not affiliated with the study, as well as prescription medications (including those taken to treat an RTI) and vaccinations administered to the infant. (If the infant subject was taken to a healthcare provider not affiliated with the study, the study staff should (if permitted by local regulation) contact that healthcare provider to obtain the medical record(s) for the visit.)

Documentation of RTI episodes (Section 8.6.3.1):

One diary card should be completed for each RTI episode whether or not an Assessment Visit (Section 8.6.6) takes place. An RTI episode has "ended" if it satisfies the criteria in Section 8.6.5.1.

At each study visit (including any assessment visits), RTI episode(s) may have ended or may be ongoing.

For any RTI episode(s) that has/have ended by the time of a study visit:

• Study staff should collect the Diary card(s), and replenish the parent(s)/LAR(s)/designate(s) supply of blank cards as needed.

For any RTI episode that is ongoing at the time of a study visit (including any assessment visit):

• Study staff should review the diary card, make a photocopy of it, and return it to the parent(s)/LAR(s)/designate(s) so information can continue to be collected until the episode has ended.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

• Once the episode has ended, study staff must collect the completed diary card by a site visit, home visit., or postal mail, whichever is most effective based on local practice. The site should make every effort to collect completed diary cards as soon after the end of an episode as possible. If diary card collection occurs during a visit to the study site or to the subject's home, a brief clinical evaluation may be performed to confirm that the episode has ended.

Refer to the SPM for additional details.

#### **Surveillance for Neonatal events of interest (Section 8.6.4)**

In addition, the investigator or study staff will perform (if not performed by local healthcare provider) a minimum of 2 clinical examinations: one at birth (or up to 72 hours after birth), and another at approximately 42 days of age.

## Surveillance for episodes of potential Lower Respiratory Tract Infection (Section 8.6.5)

#### **Definitions (Section 8.6.5.1)**

- snot nasal discharge running freely out of the infant's nose (runny nose), or
- An RTI episode starts on the day when (per parental report, as written in the Diary Card and/or provided verbally during an assessment visit) the first RTI symptom started.
- An RTI episode ends on the day when (per parental report, as written in the last RTI symptom-Diary Card and/or provided verbally during an assessment visit) either cough or difficulty in breathing has resolved, whichever resolves later.
- There must be at least 7 symptom-free days between 2 consecutive RTI episodes; the only exception is runny nose, which is a symptom that can persist during that minimum 7-day period that would distinguish one episode from a new episode.

#### Active surveillance (Section 8.6.5.3)

Three attempts should be made to contact the infant's parents/ LAR(s) (or their designates) within the week of a scheduled contact-before it is abandoned. If these attempts are unsuccessful, that active contact is considered a missed contact. The next active contact will be made according to schedule.

#### Decision to conduct a visit to assess a potential LRTI (Section 8.6.6)

An assessment visit will be conducted as soon as possible, ideally within 3 calendar days after learning of the potential LRTI case. *Note that the visit may be conducted, and a nasal swab collected, even if beyond the ideal 3-day window as long as symptoms are ongoing.* 

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### Nasal Swab (Section 8.6.7.3)

A nasal swab will be collected using sponsor-provided supplies and sent to the sponsor *(or sponsor-designated)* laboratory for detection of RSV-A/B using quantitative RT-aPCR.

If more than one assessment visit is conducted to evaluate a potential LRTI episode, additional nasal swabs may be collected (using sponsor-provided supplies and sent to the sponsor laboratory) at the discretion of the Investigator.

Note: Only the results generated by the sponsor (or sponsor-designated) laboratory (analyzing nasal swabs collected using sponsor-provided supplies) will be used when applying the case definitions for data analysis in Table 3. If other nasal swabs are collected and tested locally as per routine standard of care, results will be required to be entered into the eCRF. However, only the sponsor laboratory results however this will be used when applying thenot form part of the sponsor's application of case definitions for data analysis in Table 3...

Therefore where mandated by the protocol every effort should please be made to obtain samples for analysis by the sponsor (or sponsor-designated) laboratory.

#### Missed assessment visit (Section 8.6.7.4)

Note that If the criteria for an assessment visit may be conducted, and a nasal swab collected, as long ashave been met, but the visit cannot take place while symptoms are ongoing, it is a missed assessment visit.

If it is truly not possible to perform an assessment visit (for example, if the child develops a potential LRTI while the family is travelling, and all symptoms have resolved by the time the family returns), then the LRTI assessment visit page of the eCRF should be filled in as completely as possible using available medical *history and medical* records.

#### Follow-up after an assessment visit to evaluate a potential LRTI (Section 8.6.8)

Additional After an RTI episode that resulted in one or more assessment visits has ended (Section 8.6.5.1), site staff will ensure that the diary card for that episode is returned to the site via site visit, home visit, or postal mail (depending on the most effective local best practice for prompt retrieval of the completed infant diary card following the end of an RTI episode).

*Important* details ean be found are provided in the SPM.

#### Biological sample handling and analysis (Section 8.10)

• .... to allow GSK or a contracted partner use of the samples for future research .....

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### **Table 7 Biological Samples**

| Sample Type <sup>†</sup> | Quantity | Unit | Timepoint | Group |
|---|---|---|---|---|
| Samples preferen | Samples preferentially collected by local health care provider per local practice <sup>1</sup> | | | |
| Maternal Blood for hematology/<br>biochemistry <sup>1</sup> | Up to<br>105.5 | ml | Visit 1 (Day 1) | All Pregnant women (mothers) |
| Maternal Blood for hemoglobin | Up to <del>10-</del> 2 | ml | Visit 3 (Day 56) <sup>2</sup> | |

<sup>&</sup>lt;sup>2</sup>Hemoglobin only

#### Table 8 Humoral immunity (Antibody determination

| System | Component | Method**** | Kit /<br>Manufacturer | Unit | Cut-off | Laboratory*** |
|---|---|---|---|---|---|---|
| SERUM | Respiratory<br>Syncytial<br>Virus A Ab | NEUTRALISATION | In house | ED60 | To be defined | GSK Biologicals***** or GSK designated lab******** |

**Ab** = antibody; **ED60** = serum dilution inducing 60% inhibition in plague forming units.

#### **Table 9 Molecular Biology**

For Multiplex real time PCR of nasal swabs, Allplex<sup>TM</sup> Respiratory Panel *(Seegene)* or equivalent\*\* \* has been added as the kit manufacturer

#### Haematology, biochemistry and urinalysis (Section 8.10.3.3)

The investigators will perform a urine dipstick tests to detect for the presence of proteins, glucose, RBCs and/or WBCs. These tests do not replace those performed by local healthcare practitioners, per local practice, for clinical management of study subjects.

Table 10 Hematology, biochemistry, urine tests: neutrophils, lymphocytes, monocytes, basophils, and eosinophils have been added as components.

#### Additional tests (Section 8.10.3.4)

Additional exploratory testing on the disease under study and/or other respiratory tract infections or infections of relevance to pregnant women and their newborns may be .....

29-MAY-2020 222

<sup>\*</sup> Assay cut-off and unit might be subject to change during the course of the study (e.g. in case of requalification, revalidation or standardization). In this case, this will be documented in the study report.

<sup>\*\*\*</sup> Refer to APPENDIX B for the laboratory addresses.

<sup>\*\*\*\*\*\*\*</sup> GSK Biologicals laboratory refers to the Clinical Laboratory Sciences (CLS) in Rixensart, Belgium; Wavre, Belgium.

<sup>\*\*\*\*\*</sup> Testing may possibly be outsourced to a laboratory designated by GSK. In this case, the method and unit may be different than the one indicated in this table.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

**Table 11 Immunological read-outs** 

| Blood sampling timepoint Type of contact and time point | Group | No. subjects | Component | Component priority rank |
|---|---|---|---|---|
| | | Maternal Bloo | d | |
| Visit 5 (Delivery) All pregnant women (mothers) | | ~400 <del>maximum</del><br>by country | Respiratory Syncytial Virus A Ab (RSV-A neutralising antibody) | 1 |
| | | Cord Blood | | |
| Visit 5 (Delivery) | All pregnant women<br>(mothers) (provides<br>infant antibody levels) | ~400 <del>maximum</del><br>by country | Respiratory Syncytial Virus A Ab (RSV-A neutralising antibody) | 1 |

RSV-A/B = Respiratory syncytial virus subtype A/B.

Table 13 Hematology/blood chemistry

| Blood sampling timepoint Type of contact (timepoint) | Group | No. subjects | Component |
|---|---|---|---|
| Visit 1 (Day 1) | All pregnant women (mothers) | ~400 <del>maximum</del> by country* | Hematology (Leukocytes, Hemoglobin,<br>Platelets)<br>Biochemistry (ALT, AST, Creatinine,<br>blood urea nitrogen) |
| Visit 3 (Day 56) | All pregnant women (mothers) | ~400 <del>maximum</del> by country* | Hematology (Hemoglobin) |

#### Subject Cards (Section 9.3)

Study subjects/parents/LARs must be provided with the address and telephone number of the main contact for information about the clinical study. The investigator (or designate) must therefore provide subjects/parents/LARs with a "subject card."

For this study, a subject card will be provided to each pregnant woman who enrolls. A second subject card will be provided for each infant who is enrolled.

In an emergency situation these cards serve to inform the responsible attending physician(s) that the subject is in a clinical study and that relevant information may be obtained by contacting the investigator.

In a non-emergency situation, if subjects visit a local healthcare provider not affiliated with the study, these cards serve to inform the responsible local healthcare provider that the subject is in a clinical study and that relevant information may be obtained by contacting the investigator. Further, subject will have information on the card to contact the study site at any time.

Subjects/parents/LARs must be instructed to keep the subject cards in their possession at all times during the study.

GSK Contact information, GSK Reporting Timeframes, and Regulatory reporting requirements (Section 9.4)

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

GSK Biologicals has a legal responsibility to promptly notify, as appropriate, both the local regulatory authority and other regulatory agencies *(as applicable, per country)* about the event

## Primary endpoints (Section 11.1.1), Primary Objectives Analysis (Section 11.6) and Synopsis

- Pregnancy Occurrence of pregnancy related events of interest from Visit 1 through Visit 6. (Although pregnancy related events of interest occur within the first 42 days after delivery they may only be detected later, and are to be reported throughout the study.) They These
- Neonatal Occurrence of neonatal events of interest from birth through 28 days of age.. Neonatal AEs of interest occur within the first 28 days after birth, but may only be detected later and are to be reported throughout the study. They. These include...

## Secondary endpoints (Section 11.1.2), Secondary Objectives Analysis (Section 11.7) and Synopsis

- **Pregnancy** Occurrence of pregnancy related events of interest from Visit 1 through Visit 6 (as defined in primary endpoints) for each GAIA level of diagnostic certainty (where applicable and feasible)
- *Neonatal*Occurrence of neonatal events of interest from birth through 28 days of age (as defined in primary endpoints) for each GAIA level of diagnostic certainty (where applicable and feasible)
- Maternal RSV-A neutralizing antibody titertiters in maternal blood at delivery
- Titers of RSV-A neutralizing antibodies antibody titers in cord blood at delivery.
- *Episode(s)* Occurrence of RSV-LRTI from birth up to 1 year of age.
- *Episode(s)* of Occurrence RSV hospitalization from birth up to 1 year of age.

## Tertiary endpoints (Section 11.1.3), Tertiary Objectives Analysis (Section 11.8) and Synopsis

- **Co-infections**Occurrence of RSV-LRTI associated with other respiratory viruses **in infants**, confirmed by PCR of nasal swabs in infants from birth up to 1 year of age:
- **Potential**Occurrence of potential risk factors for maternal, fetal pregnancy related and neonatal events of interest.
- Any further exploratory immunology to detect disease-related characterization of immune responses, such as but not limited to RSV B neutralizing antibody titers.and/or other respiratory tract infections or infections of relevance to pregnant women and their newborns (based on maternal serum and cord blood).

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### Derived and transformed data (Section 11.4)

Duration of the study for each subject will be computed as the difference between the date of last contact (i.e., active or passive surveillance contact or the date of the censoring) and the date of enrollment (date when ICF was first signed by *the subject* / subject's parent[s]/LAR[s]).

#### Analysis of primary objectives (Section 11.6)

- To detect and describe determine the frequencies of pregnancy outcomes.
  - The number and percentage (with exact 95% CI) of women presenting the following events of interest *outcomes*: live birth, fetal death/still birth, and elective/therapeutic termination will be reported for each event by presence or absence of congenital anomalies.
- To detect and describe determine the frequencies of pregnancy related events of interest
- To detect and describe determine the frequencies of neonatal related events of interest.

#### **Analysis of secondary objectives (Section 11.7)**

- To detect and describe determine frequencies of pregnancy related events of interest according (where these are specified) to GAIA levels of diagnostic certainty (where these are specified) (APPENDIX D)
- To describe the distribution of RSV-A antibody titers in maternal blood collected at delivery.
- To detect and describe determine frequencies of neonatal events of interest according (where these are specified) to GAIA levels of diagnostic certainty (where these are specified). (APPENDIX D)
- To describe *the distribution of* RSV-A antibody titers in cord blood *at delivery*.
- To describe occurrences of determine the incidence of all, of severe, and of very severe RSV-lower respiratory tract infections (LRTIs).
  - from visit 1-NB to visit 3 4-NB......
  - Incidence rates of LRTI infections will be calculated, with exact 95% CI, taking into account all LRTI events reported in the study during the first year of life.
     The period at risk would be the whole follow-up time of the subjects during the study.
- To describe occurrences determine the incidence of RSV hospitalization.
  - ... from visit 1-NB to visit 3 4-NB...
  - Incidence rates of RSV hospitalizations will be calculated, with exact 95% CI, taking into account all RSV hospitalisations reported in the study during the first year of life. The period at risk would be the whole follow-up time of the subjects during the study.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### **Analysis of tertiary objectives (Section 11.8)**

- To explore the association of describe co-infections of RSV-LRTI with other respiratory viruses with the occurrence of RSV-LRTI in infants.
  - ... from visit 1-NB to visit 34-NB......
- To evaluate estimate the association between of RSV-LRTI in neonates/infants and the level of RSV neutralizing antibodies in cord blood.
- To describe determine risk factors for maternal, fetal and neonatal pregnancy-related and neonatal events of interest.
  - ... (such as multiple logistic regression for binary outcomes and multiple Poisson/negative binomial *and/or other appropriate* models for count outcomes) ....
- If deemed necessary, to further characterize the immune responses to the disease under study in mothers/infants, or to explore RSV and other parameters infections in pregnant women/mothers or their and infants (based on maternal serum and cord blood).

#### Statistical considerations for interim analyses (Section 11.11.1)

All analyses are descriptive. Therefore, the conduct of interim analyses has no impact on interpretation of study results.

#### Interim analysis for RSV LRTIs

An interim analysis will be performed on RSV surveillance data as part of the secondary objective of determining incidence of RSV LRTI. This interim analysis will be performed to obtain preliminary information on the performance of the case definitions used for RSV LRTI, severe LRTI, and very severe LRTI (Table 3). The interim analysis will occur after the database freeze at the time point when at least 50% of infants will have completed 6 months of follow up during the surveillance period following birth. Data cleaning plans will be scheduled as needed to supply data for interim analyses in a timely manner. This interim analysis will be performed on data that is as clean as possible. Preliminary results will be made available in a timely manner for use in the potential adjustment of the RSV LRTI case definitions to be used in pivotal clinical trials scheduled to begin shortly thereafter. The results pertaining to this analysis will be purely descriptive, with no adjustment of type I error, and will be reported in an interim statistical report.

#### **References (Section 14)**

Centers for Disease Control and Prevention (CDC). Updated recommendations for use of tetanus toxoid, reduced diphtheria toxoid, and acellular pertussis vaccine (Tdap) in pregnant women. Advisory Committee on Immunization Practices (ACIP) - 2012. MMWR. 2013a; 62 (7):131-135.

Centers for Disease Control and Prevention (CDC). Influenza Vaccination Coerage Among Pregnant Women — United States, 2012–13 Influenza Season. MMWR. 2013b; 62 (38): 787–792.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### **Appendix A Laboratory Assays**

#### Neutralization assay

First, virus Virus neutralization is performed by incubating a fixed amount of RSV-A long strain (Long, ATCC No. VR-26) or RSV-B strain (18537, ATCC No. VR-1580) with serial dilutions of the test serum. Then, the The serum-virus mixture is then transferred onto a monolayer of Vero cells (African Green Monkey, kidney, Cercopitheus aethiops, ATCC CCL-81) and incubated for three days to allow infection of the Vero cells by non-neutralized viruses virus and the formation of plaques in the cell monolayer. Following the a fixation period step, RSV-infected cells are detected using a primary antibody directed against RSV (anti-RSV IgG) and a secondary antibody conjugated with fluorescein isothiocyanateto horse-radish peroxidase (HRP), allowing the visualization of plaques by immunofluorescence after coloration with TrueBlueTM peroxidase substrate.

- Quantitative *RT*-PCR able to discriminate RSV-A and RSV-B subtypes:
- Qualitative multiplex *RT*-PCR for detection of a panel of viruses.

A qualitative *RT*-PCR multiplex assay is used ...:

**Table 18** Outsourced laboratories

| Laboratory | Address |
|---------------------------|-----------------------|
| DDL Diagnostic Laboratory | Fonteijnenburghlaan 7 |
| B.V. | Voorburg |
| | Netherland |
| | Headquarters |
| | Visseringlaan, 25 |
| | 2288 ER Rijswijk - NL |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

# GlaxoSmithKline Biologicals Vaccines R & D Protocol Amendment 3 eTrack study number and Abbreviated Title 207636 (EPI-RSV-008 BOD) Amendment number: Amendment 3 Amendment date: 18-FEB-2019 Co-ordinating author: PPD , Lead Science Writer

The protocol has been amended to reflect the following changes and provide the following clarifications / corrections.

- The overall sample size has been reduced from 4,000 to 2,300, as the original number of subjects will no longer be required to move the RSV Maternal immunization program to the next stage of development.
- The terms respiratory tract infection and lower respiratory tract infection have been replaced with the terms respiratory tract illness and lower respiratory tract illness to improve consistency with World Health Organization terminology.
- The phrase "pregnant women (mothers)" has been replaced with the term "maternal subjects."
- The List of Abbreviations and Glossary of terms have been updated.
- Language describing mitigation of the risks associated with venipuncture has been clarified.
- The reference to nasal obstruction in Footnote 1 of Table 3 has been removed.
- Eligible maternal subjects may now be up to 45 years of age and must now have a pre-pregnancy body mass index within the range specified in the inclusion criteria.
- "Geographic ancestry (race)" replaces the word "race."
- A footnote has been added to Table 4 to indicate that if results of an oral glucose challenge / tolerance test are not available, then fasting blood glucose or haemoglobin A1C test results may be used as described in Table 26.
- Language has been added to clarify that "parental concern" as described in Sections 8.6.4 through 8.6.8 occurs in the context of a respiratory tract illness.
- Instructions for infant diary completion and for collection of RTI/LRTI symptom start and stop dates have been re-written in an effort to improve clarity.
- A definition for respiratory tract illness/lower respiratory tract illness symptom "worsening" has been added.
- Objectives, endpoints and the text of Appendix D have been adjusted to improve consistency with GAIA criteria.
- References to country and/or region-specific analyses have been removed from Section 11 10
- Assessment of blood oxygen saturation (by pulse oximetry) in maternal subjects has been added.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- Text has been added to clarify that levels of RSV-A neutralising antibody in maternal and cord blood at delivery will be assessed during the interim analysis.
- Text that addresses study / site closure has been added.
- Laboratory addresses in Appendix B have been updated.

Additional editorial changes have been made to ensure consistency with the modifications noted above, and typographical errors have been corrected

Text that has been moved or added is presented in **bold italics** and deleted text in strikethrough in the following sections.

#### **Global changes:**

- "Pregnant women (mothers)" has been replaced with *maternal subjects*
- Age 18 40 has been replaced with 18-45
- $<28^{9/7}$  has been replaced with  $\le 27^{6/7}$  weeks gestational age (GA)
- Number of subjects enrolled has changed from 4000 to 2300 ("up to 400" to "200-300" per country)
- "Respiratory tract infections" has been replaced with respiratory tract illnesses
- "Race" has been replaced with "geographic ancestry (race)"

#### List of contributing authors:

| • | PPD | , Lead PPD Epidemiologist |
|---|---|---|
| • | PPD | , Clinical Research and Development Lead |
| • | PPD | , Expert Epidemiology Biostatistician, PPD , Lead Epi |
| | Statistician | |
| • | PPD | , PPD , Study Delivery |
| | Leads | |
| • | PPD | , Clinical Trial Supply manager |
| • | PPD | , Clinical Read-Out Team Leader |
| • | PPD | , Safety Physician |
| • | PPD | , Oversight Data Manager |
| • | PPD | Study Data Manager (Tata Consultancy Services for GSK Biologicals) |
| • | PPD | , Regulatory Affairs Representative |

#### Authors who contributed to previous versions of the protocol

- PPD , Study Delivery Leads
- PPD , Safety Physician

#### **Synopsis and Secondary Objectives**

Neonatal *events* AEs of interest occur within the first 28 days after birth, but may only be detected later and are to be reported throughout the study

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### **Synopsis and Introduction**

4<sup>th</sup> pargraph: Secondarily, the study will establish surveillance mechanisms for RSV *associated illnesses* infections

 $7^{\text{th}}$  paragraph: Pregnant women  $24^{0/7}$  up to **and** but not including  $27^628^{0/7}$  weeks of gestation

#### **Section 1.5, Introduction:**

RSV infects 50-70% of infants in their first year of life, and practically all children have experienced RSV infection *and/or illness* 

#### Synopsis Table 2 and Table 2

#### Study groups and epochs foreseen in the study

| Study Groups | Number of | Age (Min/Max) | Epochs | | |
|---|---|---|---|---|---|
| | subjects enrolled | | Epoch 001 | Epoch 002 | Epoch 003 |
| Maternal subjects | Up to ~ <b>2300</b> 400 | 18 years – <b>45</b> 40 | X | Х | |
| Pregnant women | (per country) | years | | | |
| (mothers) | , | - | | | |
| Infants | Up to ~ <b>2300</b> 400 | NA | | Х | Х |
| | <del>per country)</del> | | | | |

Approximately 200 to 300 subjects per country. To achieve the enrollment targets noted above, the number of pregnant women SCREENED in each country may exceed the country-specific enrollment target. 400

#### Synopsis and Section 11.1, Primary Endpoints

- Pregnancy outcomes. Of note, fetal death/stillbirth has multiple subcategories. For example, fetal death/stillbirth with no congenital anomalies is an outcome with two subcategories that include: 1) antepartum stillbirth; 2) intrapartum stillbirth. For each outcome, the investigator should select the applicable sub-category.
  - Fetal death/stillbirth (loss at or after 22 weeks of gestation) with no congenital anomalies:
    - o Antepartum stillbirth
    - Intrapartum stillbirth
  - Fetal death/stillbirth (loss at or after 22 weeks of gestation) with congenital anomalies:
    - Antepartum stillbirth
    - Intrapartum stillbirth
  - Pregnancy related events of interest from Visit 1 through Visit 6..... They are listed below. Of note, some events of interest fall under a single category but have multiple subcategories. For example, hypertensive disorders of pregnancy is an event with three subcategories that include: 1) gestational hypertension; 2) pre-eclampsia; and 3) pre-eclampsia with severe features

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

(including eclampsia). For each event, the investigator should identify the event and select the applicable sub-category.

- Antenatal bleeding:
  - Morbidly adherent placenta
  - o Placental abruption
  - o Cesarean Scar Pregnancy
  - o Uterine rupture
- Dysfunctional labor
  - o first stage of labor
  - o second stage of labor
- Gestational Liver Disease:
  - o Intrahepatic Cholestasis of Pregnancy (ICP)
  - o Acute Fatty Liver of Pregnancy
- Maternal Sepsis

Neonatal events of interest from birth through 28 days of age. Neonatal *events* AEs of interest......

- Congenital microcephaly,
  - o Postnatally diagnosed
  - o Prenatally diagnosed
- Congenital anomalies
  - Major external structural defects
  - Internal structural defects
  - Functional defects
- Neonatal death,
  - $\circ$  Neonatal death in a preterm live birth (gestational age>=28 to < 37 weeks)
  - Neonatal death in a term live birth
- Neonatal infections,
  - Blood stream infections
  - Meningitis
  - o Respiratory infection
- Failure to thrive,

Any other neonatal event considered by the investigator to be of concern (specify, *e.g. neurodevelopment delay*).

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Section 11.1.1 (Primary Endpoints – pregnancy outcomes and pregnancy related events of interest; text does not appear in Synopsis):

Section 11.1.1.2: For events of interest that include subcategories, the frequency of the main event of interest and of each event subcategory will be included in the analysis. The overall frequency will include mothers who present at least one of the subcategory events.

Section 11.1.1.3: For events of interest that include subcategories, the frequency of the main event of interest and of each event subcategory will be included in the analysis. The overall frequency will include infants who present at least one of the subcategory events.

#### **Synopsis and Secondary Endpoints**

Of note, some events of interest fall under a single category but have multiple subcategories. For each event, the investigator should identify the event and select the applicable sub-category and the GAIA level of diagnostic certainty.

#### **List of Abbreviations**

---

| Body mass index |
|---|
| Lower Respiratory Tract Illness Infection |
| Respiratory Tract Illness Infection |
| A key index for relating weight to height. Calculated as follows: Weight (kg) / (Height (m)) $^2$ |
| The parent(s) / Legally Acceptable Representative(s) or their designates are concerned about the infant's respiratory tract illness, or general health <i>in the context of the respiratory tract illness</i> , and intend to seek medical care |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### Section 2.1, Risk Assessment

| Important Potential/Identified Risk | Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Study Procedures | | |
| Blood sample collection- While giving blood the subject may feel faint, or | Spontaneous data | Sample collection will only be performed by appropriately trained study personnel. |
| locally experience mild pain, bruising, irritation or redness. | | All Subjects will remain under observation, post venipuncture, through completion of the applicable study visit be observed for at least 30 minutes after blood sample collection. |
| | | Subjects will be notified of this risk in the informed consent form. |

#### Section 4, Study Design Overview

Figure 1 has been replaced. The current Figure, followed by the Figure as presented in Amendment 2, follow.





- Primary Completion Date (PCD): 42 days post-delivery/birth (i.e. Visit 6 for *maternal subjects* the mothers and Visit 2-NB for *infant subjects* the infants) or last visit of Epoch 002.
- Duration of the study: Approximately 4.5 to 6 months for *maternal subjects* participating pregnant women; approximately 1 year for *infant subjects* participating infants.
- Epoch 002: Primary starting at Visit 1 and ending 42 days post-delivery/birth (Visit 6 for *maternal subjects* and Visit 2-NB for *infant subjects* ).\*

#### **Section 5.4, Case Definitions, Table 3:**

**Footnote 1:** Based on history reported by parents/LARs and includes difficulty in breathing (e.g. showing signs of wheezing or stridor, tachypnoea, flaring [of nostrils], chest in-drawing, apnoea) associated with nasal obstruction.

**Footnote 5:** RSV sampling and testing is *described in Sections 8.6.7, 8.6.8 and 8.6.9.* based on judgment of medical practitioner or driven by algorithm.

#### Section 6.2.1, Inclusion criteria for maternal subjects

- \* The level of diagnostic certainty of the gestational age should be established by using the GAIA gestational age assessment *form* tool (provided in APPENDIX C).
- Women with pre-pregnancy body mass index (BMI)  $\geq$ 18.5 and  $\leq$  39.9 kg/m<sup>2</sup>.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### 6.3, Exclusion criteria for enrollment in maternal subjects:

The following criteria should be checked at the *screening visit and at Visit 1.*time of study entry.

• primary *genital* herpes simplex infection

#### **Section 8, Detailed Study Procedures**

#### Table 4

| Review and collect obstetric history from current pregnancy, including: gestational age, expected date of delivery and method of EDD estimation <i>including pre-pregnancy weight</i> | 0 | • | | | | | |
|---|---|---|---|---|---|---|---|
| Travel history to, or living in, countries/regions with Zika virus transmission (during the current pregnancy) | 0 | • | 0 | 0 | 0 | 0 | • |

Footnote 7: If results of an oral glucose challenge / tolerance test are not available to confirm that the subject does not have Gestational Diabetes at screening, then fasting blood glucose or hemoglobin A1C test results (if performed by local healthcare provider and available) may be used as described in Table 27.

Footnote 10: In the Philippines, where If HIV test results are testing is not available at time part of the standard of care for pregnant women, the screening the HIV test can be performed locally as a study procedure under certain conditions. Refer to SPM for further details. If results are positive, subject will be referred per local standard of care.

Footnote 11: Height, weight during the month before the subject became pregnant, and pre-pregnancy BMI at screening. Weight, temperature, systolic/diastolic blood pressure, heart rate and respiratory rate after at least 10 minutes of rest, blood oxygen saturation by pulse oximetry vital signs, fetal heart tones, fetal movement, and fundal height at Screening and Visits 1 – 4. Temperature, systolic/diastolic blood pressure, heart rate and respiratory rate after at least 10 minutes of rest, and blood oxygen saturation by pulse oximetry Vital signs at Visit 6.

#### Table 5 footnotes

- <sup>a</sup> If local regulations require that **written consent** / confirmation of consent for the infant's participation be obtained at birth.
- c If more than one assessment visit is conducted to evaluate a potential LRTI<del>episode</del>, additional nasal swabs may be collected at the discretion of the Investigator.
- Collect diary cards that are fully filled out and / or document (L)RTI episodes-symptoms that have ended-(as defined in Section 8.6.5.1). Provide new diary cards as needed.
- <sup>f</sup> Collect all diary cards for potential RTIs that are considered resolved. Collect the diary card for the current potential LRTI once the episode-*LRTI symptoms have* has ended (as defined in Section 8.6.5.1).
- <sup>9</sup> When approximately 50% of infants have completed up to Visit 3-NB, an interim analysis will be conducted to assess the accumulated RSV LRTI cases and the distribution of maternal and cord blood serum RSV A Ab.

### Section 8.5.2, History for *Maternal subjects* and Examinations for pregnant women/mothers

Record demographic data, which may include (but *are* is not limited to) information such as *geographic ancestry* (race), month and year of birth, *and* ethnicity.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Record information about whether *(during the current pregnancy)* the subject has travelled to / is living in countries / regions with Zika virus

Record the subject's pre-pregnancy weight (i.e., weight during the months before the subject became pregnant) at screening. This information can be obtained either via medical record review or subject interview and should be recorded in the subject's eCRF.

Confirm that the subject's pre-pregnancy BMI is within the range specified in Section 6.2.1. This information can be obtained from the medical record, or, if unavailable, may be calculated based on the subject's height and reported pre-pregnancy weight.

Obtain the subject's medical *and obstetric* history by interview and/or .....

Obtain the subject's obstetric history by interview and/or review of her medical records

#### Section 8.5.3: Examinations of maternal subjects

Record height at screening and Weight at screening and Visits 1-4.

- Screening and Visits 1 4 should include assessment of *weight*, fetal heart tones, fetal movement, and fundal height;
- Screening, Visits 1 to 4, and Visit 6 should include assessment of *temperature*, vital signs systolic/diastolic blood pressure, heart rate and respiratory rate after at least 10 minutes of rest) and *blood oxygen saturation by pulse oximetry*.

#### Section 8.5.8, Outcomes and Events of Interest

- Record delivery and pregnancy outcomes. Of note, fetal death/stillbirth has multiple subcategories. For example, fetal death/stillbirth with no Record Delivery and Pregnancy Outcomes congenital anomalies is an outcome with two subcategories that include: 1) antepartum stillbirth; 2) intrapartum stillbirth. For each outcome, the investigator should select the applicable subcategory.
- Maternal events of interest (including, but not limited to, those described in Section 11.1.1) occurring up to Visit 6 (Post-delivery *Day 42*) should be recorded in the eCRF along with additional details pertinent to the diagnosis, GAIA assessment and level of diagnostic certainty (APPENDIX D), when applicable. Of note, some events of interest fall under a single category but have multiple subcategories. For example, hypertensive disorders of pregnancy is an event with three subcategories that include: 1) gestational hypertension; 2) pre-eclampsia; and 3) pre-eclampsia with severe features (including eclampsia). For each event, the investigator should identify the event and select the applicable sub-category.
- Information about maternal *hospitalizations*, hospitalization and clinically significant events, *and* diagnoses that could impact the pregnancy will be recorded.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### Section 8.6, Description of Study Procedures for Neonates/Infants

Note that the investigator or study staff will perform (if not performed by local healthcare provider) a minimum of 2 clinical examinations: one at birth (or up to 10 days after birth), and another at approximately 42 days of age.

#### Section 8.6.2, History and Examinations for Neonates/Infants

• Record demographic data including month and year of birth, gender, *geographic* ancestry (race) and ethnicity.

#### Section 8.6.3, Infant Diary Cards

#### 8.6.3.1 Documentation of RTI episodes:

One diary card should be completed for each RTI episode whether or not an Assessment Visit (Section 8.6.6) takes place. An RTI episode has "ended" if it satisfies the criteria in Section 8.6.5.1.

At each study visit (including any assessment visits), RTI *symptoms episode(s)* may have ended or may be ongoing.

If blocked nose, cough and symptoms of difficulty in breathing (including wheezing) For any RTI episode(s) that has/have ended by the time of a study visit:

 Study staff should collect the Diary card(s), and replenish the parent(s)/LAR(s)/designate(s) supply of blank cards as needed.

For any RTI episode that is If blocked nose, cough or symptoms of difficulty in breathing (including wheezing) are ongoing at the time of a study visit (including any assessment visit):

- Study staff should review the diary card, make a photocopy of it, and return it to the parent(s)/LAR(s)/designate(s) so information can continue to be collected until the episode has the symptoms have ended.
- As soon as possible after Once the episode these symptoms have has ended, study staff must collect the completed diary card by a site visit, home visit, or postal mail, whichever is most effective based on local practice. The site should make every effort to collect completed diary cards as soon after the end of an episode symptoms have ended as possible. If diary card collection occurs during a visit to the study site or to the subject's home, a brief clinical evaluation may be performed to confirm that the episode symptoms have has ended.

## **8.6.4, Surveillance for** episodes of potential Lower Respiratory Tract *Illness* Infection (LRTI)

• A An episode of potential lower respiratory tract *illness* infection (LRTI) is one in which the infant has one or more of the RTI symptoms listed above AND at least one of the following:

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- Wheezing (a whistling sound when the infant breathes out) (another sign of difficulty in breathing);
- Parental concern (the parent(s)/LAR(s) or their designate(s) are concerned about the infant's respiratory tract illness, or general health in the context of the respiratory tract illness, and intend to seek medical care).

Worsening means any clinically observed/diagnosed symptoms and signs that are reported during the same respiratory tract illness and reflect a deterioration in the child's respiratory tract functions.

- An RTI episode starts on the day when (per parental report, as written in the Diary Card and stop dates will be collected inor provided verbally during an assessment visit) the diary card for first RTI symptom started
- An RTI episode ends on the day when (per parental report, as written in the Diary Card and/or provided verbally during an assessment visit) either cough, runny nose, blocked nose, wheezing and difficulty in breathing has resolved, whichever resolves later.
- Start and stop dates will be collected in the diary card for cough, runny nose, blocked nose, wheezing and difficulty in breathing.
- Start dates for all symptoms will also be recorded in the eCRF.
- Only stop dates for cough and difficulty in breathing will be recorded in the eCRF so that GSK may later define the end of each LRTI episode (Section 5.4)
- There must be at least 7 symptom-free days between 2 consecutive RTI episodes; the only exception is runny nose, which is a symptom that can persist during that minimum 7-day period that would distinguish one episode

#### Figure 5 footnote

Worsening is defined in Section 8.6.5.1

#### 8.6.5.3 Active Surveillance

• there is parental concern as defined in Section 8.6.5.1

#### 8.6.5.4 Passive Surveillance

• the infant's symptoms worsen as defined in Section 8.6.5.1

#### 8.6.6 Decision to conduct a Visit to assess.....

If there is <u>NO</u> suspicion of difficulty in breathing, nor wheezing, nor parental concern *in* the context of the RTI:

**If there** <u>IS</u> difficulty in breathing, or wheezing (both based on parental assessment), or there is parental concern *in the context of the RTI*:

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### **8.6.7.3** Nasal swabs

.....If more than one assessment visit is conducted to evaluate a potential LRTI<del>episode</del>

#### 8.6.8 Follow up after an assessment.....

After an assessment visit (Section 8.6.7) the child will be followed with at least weekly active surveillance contacts, until the RTI/LRTI episode has resolved. During these active contacts, worsening of symptoms (clinically observed/diagnosed symptoms and signs that are reported during the same respiratory tract illness and reflect a deterioration in the child's respiratory tract functions; for example, onset of additional symptoms or an increase in the intensity of a previously reported symptom) will be assessed. Parent(s) / LAR(s) / designate(s) will be reminded to call/contact/visit the site if symptoms worsen.

After symptoms an RTI episode that resulted in one or more assessment visits have has ended (Section 8.6.5.1), site staff will ensure that the diary card for those symptoms that episode is returned to the site via site visit, home visit, or postal mail (depending on the most effective local best practice for prompt retrieval of the completed infant diary card following the end of the symptoms an RTI episode).

Table 7, Biological samples

| Sample Type <sup>†</sup> | Quantity | Unit | Timepoint | Group |
|---|---|---|---|---|
| Samples preferentially collected by local health care provider per local practice <sup>1</sup> | | | | |
| Maternal Blood for Hematocrit | Up to 2 | ml | Visit 3 (Day 56) | |
| Hemoglobin | | | , , , | |

#### **Table 8, Humoral Immunity, footnote**

#### Table 9, Molecular Biology, footnote

\*\* GSK Biologicals laboratory refers to the Clinical Laboratory Sciences (CLS) in Rixensart, Belgium; Wavre, Belgium. *Marburg, Germany* 

#### **Section 11.2 Determination of Sample size**

Assuming a drop-out rate of about 10% during the course of follow-up, there will be up to approximately 180 to 270 360 evaluable subjects by country.

Considering a sample size of up to approximately **180** to **270** 360 evaluable subjects by country, Table 16 illustrates the precision (exact 95% confidence interval [CI]) one can get on the percentage of subjects with maternal, fetal and neonatal events of interest.

Precision (exact 95% CI) has also been computed for a sample size of 270, **180** and 100 evaluable subjects for estimate by study site.

<sup>\*\*</sup> GSK Biologicals laboratory refers to the Clinical Laboratory Sciences (CLS) in Rixensart, Belgium; Wavre, Belgium. *Marburg, Germany* 

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Table 16: Precision (exact 95% confidence interval) on the percentage of subjects with maternal, fetal and neonatal events of interest for sample size of 360 270, 180 and 100 subjects

| | 360 subjects | | | 270 subjects | | | | 180 subje | ects | 100 subjects | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| % | N | Lower<br>limit | Upper<br>limit | N | Lower<br>limit | Upper<br>limit | N | Lower<br>limit | Upper<br>limit | N | Lower<br>limit | Upper<br>limit |
| 35 | <del>126</del> | <del>30.1</del> | 40.2 | 94.5 | 29.3 | 41.0 | 63 | 28.1 | 42.4 | 35 | 25.7 | 45.2 |
| 30 | <del>108</del> | <del>25.3</del> | <del>35.0</del> | 81 | 24.6 | 35.8 | 54 | 23.4 | 37.3 | 30 | 21.2 | 40.0 |
| 25 | 90 | <del>20.6</del> | <del>29.8</del> | 67.5 | 19.9 | 30.6 | 45 | 18.9 | 32 | 25 | 16.9 | 34.7 |
| 20 | <del>72</del> | <del>16.0</del> | <del>24.5</del> | 54 | 15.4 | 25.3 | 36 | 14.4 | 26.6 | 20 | 12.7 | 29.2 |
| 15 | <del>54</del> | <del>11.5</del> | <del>19.1</del> | 40.5 | 11.0 | 19.8 | 27 | 10.1 | 21.1 | 15 | 8.6 | 23.5 |
| 10 | <del>36</del> | <del>7.1</del> | <del>13.6</del> | 27 | 6.7 | 14.2 | 18 | 6 | 15.3 | 10 | 4.9 | 17.6 |
| 5 | <del>18</del> | 3.0 | <del>7.8</del> | 13.5 | 2.7 | 8.3 | 9 | 2.3 | 9.3 | 5 | 1.6 | 11.3 |
| 3 | <del>10.8</del> | <del>1.5</del> | <del>5.3</del> | 8.1 | 1.3 | 5.8 | 5.4 | 1 | 6.8 | 3 | 0.6 | 8.5 |
| 1 | <del>3.6</del> | 0.2 | <del>2.7</del> | 2.7 | 0.2 | 3.0 | 1.8 | 0.1 | 3.9 | 1 | 0 | 5.4 |
| 0 | 0 | 0 | 4 | 0 | 0 | 1.4 | 0 | 0 | 2 | 0 | 0 | 3.6 |

#### Section 11.6, Analysis of primary objectives

The primary objectives analyses will be performed on the PPS cohorts overall by country, and possibly by region or other relevant grouping.

The number and percentage (with exact 95% CI) of women presenting the following outcomes: live birth, fetal death/*stillbirth* (*antepartum or intrapartum*), and elective/therapeutic termination will be reported for each event by presence or absence of congenital anomalies.

## • To determine the frequencies of pregnancy related events of interest as specified in Section 11.1.1.2.

The number and percentage (with exact 95% CI) of pregnant women presenting with the following events of interest *specified in Section 11.1.1.2*. The number and percentage (with exact 95% CI) of pregnant women presenting with the following events of interest *specified in Section 11.1.1.2* will be tabulated for each event within appropriate time windows to be specified in the statistical analysis plan (SAP).

#### The events are:

- Hypertensive disorders of pregnancy:
  - o gestational hypertension, and
  - Pre-eclampsia, and
  - Pre-eclampsia with severe features (including eclampsia)
- Antenatal bleeding
- Fetal growth restriction
- Non reassuring fetal status

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- Pathways to preterm birth:

   premature preterm rupture of membranes,
   preterm labor, and
   provider initiated preterm birth

   Postpartum hemorrhage
   Chorioamnionitis
   Oligohydramnios
   Polyhydramnios
- To determine the frequencies of neonatal events of interest as specified in Section 11.1.1.3.

The number and percentage (with exact 95% CI) of neonates presenting the following events of interest *specified in Section 11.1.1.3....* 

- All of the following events of interest.
  - Small for gestational age
  - Low birth weight including very low birth weight
  - Large for gestational age
  - Macrosomia

Maternal death

- Preterm birth
- Neonatal encephalopathy
- Respiratory distress in the neonate
- Neonatal infections
- Congenital microcephaly
- Congenital anomalies

#### **Section 11.7** Analysis of Secondary objectives

The secondary objectives analyses will be performed on the PPS cohorts (maternal or infant as applicable) overall by country *and possibly* by region or other relevant grouping.

#### **Section 11.8 Analysis of Tertiary objectives**

The following tertiary objectives analyses will be performed on infants within the PPS cohort overall *and possibly* by country region or other relevant grouping.

• To describe co-infections of RSV-LRTI with other respiratory viruses in infants.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Considering all infants followed from visit 1-NB to visit 4-NB, the percentage of subjects with the occurrence of RSV-LRTI and having other respiratory viral co- infection or colonized with another viral etiology identified

#### Section 11.11, Conduct of analyses

Analyses will be performed in a stepwise manner after *all subjects in all* each country / group of countries / countries in a region have completed all study visits in Epoch 002 and again after completion of all study visits in Epoch 003.

... For these analyses a statistical report *but no CSR* will be prepared. for each country/group of countries / countries in a region. No CSRs will be prepared.

Final analyses will be performed when all data up to study end are available (Epoch 002 and Epoch 003). One or more *An* integrated *CSR* elinical study reports (bycounty / group of countries / countries in a region).......

#### **Section 11.11.1 Statistical considerations for interim analysis**

This interim analysis will be performed to obtain preliminary information on the performance of the case definitions used for RSV LRTI, severe LRTI, and very severe LRTI (Table 3) and to assess levels of RSV-A neutralising antibody in maternal and cord blood at delivery. The interim analysis will occur after the database freeze at the time point when approximately 50% of infants will have completed up to 6 months of follow up during the surveillance period following birth (up to Visit 3-NB). No CSR will be prepared.

#### Section 12.1, Electronic case report form instructions

Once the database is archived and the clinical study report is complete and approved by all parties, each participating investigator will be provided with a CD-ROM of the final version of the data generated at his/her investigational site.

#### Section 12.3, Study and site closure has been added.

GSK or its designee reserves the right to close the study site or terminate the study at any time for any reason at the sole discretion of GSK, provided there is sufficient notice given to account for patient's safe exit from study participation. Study sites regular closure will be upon study completion. A study site is considered closed when all required data/documents and study supplies have been collected and a study-site closure visit has been performed.

The investigator may initiate study-site closure at any time, provided there is reasonable cause and sufficient notice is given in advance of the intended termination.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

Reasons for the early closure of a study site by the sponsor or investigator may include but are not limited to:

- Failure of the investigator to comply with the protocol, the requirements of the IRB/IEC or local health authorities, the sponsor's procedures, or GCP guidelines
- Inadequate recruitment of subjects by the investigator
- Discontinuation of further study treatment development

#### Appendix B, Clinical Laboratories, table 17

| GSK Vaccines GmbH | Emil-von-Behring-Str. 76 |
|-------------------------------|--------------------------|
| Clinical Laboratory Sciences, | 35041 Marburg |
| Marburg, Germany | Germany |

#### Appendix B, Clinical Laboratories, Table 18

| NÉOMED-LABS Inc. | 525, Cartier Ouest Laval, |
|------------------|---------------------------|
| | Québec |
| | Canada H7V 3S8 |

## Appendix D, Definitions of maternal, fetal and neonatal events of interest as per GAIA

The order of the tables has been adjusted for consistency with the order in which endpoints are presented in the body of the protocol. Stillbirth (now Table 19) is presented as a pregnancy outcome rather than as a neonatal event of interest.

#### Table 29 has been updated to include the following events:

| Gestational | Intrahepatic cholestasis also called obstetric cholestasis should be suspected when |
|---|---|
| liver disease | pruritis develops during pregnancy in the absence of a rash. Lab evidence of |
| (Intrahepatic | cholestasis includes elevated bile acids (Glyco and Taurochenodeoxycholic Acid )(> 10 |
| Cholestasis of | umol/L). Up to 60% of patients will have elevated transaminases and 20% of patients will |
| Pregnancy or | have increased direct bilirubin levels. |
| ICP)1 | Jaundice may or may not be present. ICP typically is transient and resolves after |
| | delivery. Women that had ICP in previous pregnancy have higher risk to developing ICP |
| | in the following pregnancies or other hepatobiliary disorders in later life. ICP is |
| | associated with adverse fetal outcome like meconium-stained liquor, fetal asphyxia, |
| | spontaneous preterm delivery and intrauterine death. |
| Gestational | Acute fatty liver of pregnancy (AFLP) is a rare, potentially fatal complication that occurs |
| liver disease | in the third trimester or early postpartum period. AFLP is characterized by |
| (Acute Fatty | microvesicular fatty infiltration of hepatocytes without any inflammation or necrosis. |
| Liver of | Most frequent signs and symptoms are the following: |
| Pregnancy) <sup>2</sup> | Jaundice |
| | Abdominal Pain (usually right upper quadrat, midepigastric or radiating to back) |
| | Central nervous system (altered sensorium, confusion, disorientation, psychosis, |
| | restlessness, seizures or even coma) |
| | Disseminated intravascular coagulation |
| | Nausea and vomiting |
| | Gastrointestinal bleeding |
| | Acute renal failure |
| | Oliguria |
| | Tachycardia |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| | Late onset pyrexia Hypoglycemia ALT<500 U/L Hyperbilirubinemia, elevated ammonia, leukocytosis, hypofibrinogenemia Ultrasound examination and computed tomography may demonstrate fatty infiltration of the liver but are not sufficient for diagnosis | | | | | |
|---|---|---|---|---|---|---|
| Maternal<br>Sepsis³ | Maternal sepsis is a life-threatening condition defined as organ dysfunction resulting from infection during pregnancy, child-birth, post-abortion, or post-partum period. Organ dysfunction can be identified as an acute change in total SOFA score ≥2 points consequent to the infection. The baseline SOFA score can be assumed to be zero in patients not known to have preexisting organ dysfunction. A SOFA score ≥2 reflects an overall mortality risk of approximately 10% in a general hospital population with suspected infection. Even patients presenting with modest dysfunction can deteriorate further, emphasizing the seriousness of this condition and the need for prompt and appropriate intervention, if not already being instituted. | | | | | |
| | Table 1. Sequential [Sep | sis-Related] Organ Fai | lure Assessment Score <sup>a</sup> | | | |
| | | Score | | | | |
| | System | 0 | 1 | 2 | 3 | 4 |
| | Respiration | | | | | |
| | Pao <sub>2</sub> /Fio <sub>2</sub> , mm Hg<br>(kPa) | ≥400 (53.3) | <400 (53.3) | <300 (40) | <200 (26.7) with respiratory support | <100 (13.3) with respiratory support |
| | Coagulation | | | | | |
| | Platelets, ×10 <sup>3</sup> /μL | ≥150 | <150 | <100 | <50 | <20 |
| | Liver | | | | | |
| | Bilirubin, mg/dL<br>(µmol/L) | <1.2 (20) | 1.2-1.9 (20-32) | 2.0-5.9 (33-101) | 6.0-11.9 (102-204) | >12.0 (204) |
| | Cardiovascular | MAP ≥70 mm Hg | MAP < 70 mm Hg | Dopamine <5 or<br>dobutamine (any dose) <sup>b</sup> | Dopamine 5.1-15<br>or epinephrine ≤0.1<br>or norepinephrine ≤0.1 <sup>b</sup> | Dopamine >15 or<br>epinephrine >0.1<br>or norepinephrine >0.1 <sup>b</sup> |
| | Central nervous system | | | | | |
| | Glasgow Coma Scale<br>score <sup>c</sup> | 15 | 13-14 | 10-12 | 6-9 | <6 |
| | Renal | | | | | |
| | Creatinine, mg/dL<br>(µmol/L) | <1.2 (110) | 1.2-1.9 (110-170) | 2.0-3.4 (171-299) | 3.5-4.9 (300-440) | >5.0 (440) |
| | Urine output, mL/d | | | | <500 | <200 |
| | | | AP, mean arterial pressure; | | are given as µg/kg/min for at | |
| | Pao <sub>2</sub> , partial pressure of o | | | <sup>c</sup> Glasgow Coma Scale scores range from 3-15; higher score indicates better neurological function. | | |
| | MAP = mean a<br>related] Organ | | ıre; qSOFA = qu<br>essment | ick SOFA; SOFA | A = Sequential | [Sepsis- |

References:

- 1 Geenes V et al . Intrahepatic cholestasis of pregnancy
- 2 Can J Gastroenterol Vol 20 26 No 1 January 2006
- 3 Bonet et al. Reproductive Health (2017) 14:67

Table 39, Failure to Thrive, has been added.

Failure to Thrive (FTT) can be broadly defined as a faltering of growth from a previously established pattern of growth. It is universally established that a diagnosis of failure to thrive should be based on anthropometric data. However no consensus exits as to which measurements achieve the highest specificity and sensitivity. Weight is generally regarded is the indicator of choice, particularly a change in growth velocity, and as such has been selected as the standard for this case definition with a weight for

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

age deceleration as the primary indicator of failure to thrive. The case definition should be applied when there is no clear alternative diagnosis for the reported event to account for the combination of symptoms.

| Level | Description |
|---|---|
| 1 | Infant age¹ determined by a documented birth date AND |
| | Weights obtained using an electronic scale AND |
| | At least 2 weights, measured at least 4 weeks apart |
| | Weight for age deceleration <sup>2</sup> through at least 2 centile spaces on growth chart <sup>3</sup> |
| 2a | Infant age determined by a documented birth date AND |
| | Weights obtained using a beam balance scale AND |
| | At least 2 weights, measured at least 4 weeks apart AND |
| | Weight for age deceleration through at least 2 centile spaces on growth chart |
| | OR |
| | Infants with an undocumented birth date, where age is determined based on Mothers recall to nearest month AND |
| | Weights obtained using electronic scale AND |
| | At least 2 weights, measured at least 4 weeks apart AND |
| | Weight for age deceleration through at least 2 centile spaces on growth chart |
| 2b | Infant age determined by a documented birth date AND |
| | Weights obtained using a spring balance scale AND |
| | At least 2 weights, measured at least 4 weeks apart AND |
| | Weight for age deceleration through at least 2 centile spaces on growth chart |
| | OR |
| | Weight measured using electronic scale or beam balance scale AND |
| | Length taken using Infantometer AND |
| | Weight for length less than or equal to the 3rd centile on the appropriate growth chart |
| 3a | Infants with an undocumented birth date, where age is determined based on Mothers recall to nearest month |
| | AND Weight obtain using either beam balance or spring balance |
| | scale<br>AND |
| | At least 2 weights, measured as least 4 weeks apart AND |
| | Weight for age deceleration through at least 2 centile spaces on |

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

| Level | Description |
|-------|-------------------------------------------------------|
| | growth chart |
| 3b | Infants with no weight available |
| | AND |
| | Physical examination consistent with FTT <sup>4</sup> |
| | AND |
| | MUAC <sup>5</sup> indicative of severe wasting |

<sup>&</sup>lt;sup>1</sup>This case definition is limited to infants up to 12 months of age.

- <sup>2</sup> Weight should be documented on the appropriate growth chart at the time of assessment. A fall through 2 centile spaces may be demonstrated at any point in the first 12 months of life, using any two weights as long as they are taken at least 4 weeks apart. Details of use of the weight balances allowable under this case definition and use of the Infantometer for length assessment are presented in the reference given below.
- <sup>3</sup> For infants born at 37 weeks gestation or above, the WHO growth charts should be applied. When using weight for age use the growth chart most accurate for the infants age. The birth to 6 months age range should be used where data is available for this range only, the birth to 2 years chart should be used where data is available beyond 6 months of life. When using weight for length, use the chart for birth to 2 years. For infants born less than 37 completed weeks gestation, the Intergrowth charts for postnatal growth standards in preterm infant should be used. All infants should be plotted on their respective growth chart using their corrected age. Links to relevant growth charts are presented in the reference given below.
- <sup>4</sup> Physical examination with signs of Failure to Thrive (must include at least 2 findings, with at least one major finding) Major findings: Reduced subcutaneous fat stores; poor muscle mass; loose skin folds; prominent ribs; thin limbsOther less specific signs include: sparse hair; rashes; pallor; miserable; lethargy/fatique.
- <sup>5</sup> Mid Upper Arm Circumference (MUAC): For infants 0–6 months, a MUAC of 6 110 mm is indicative of severe wasting. For infants 6–12 months, a MUAC of 6 115 mm is indicative of severe wasting. Instructions on performing MUAC are presented in the reference given below.
- Reference: Ross E, Munoz F, Edem B et al. Failure to thrive: case definition and guidelines for data collection, analysis, and presentation of maternal immunization safety data. Vaccine. 2017; 35:6483-6491.

#### Table 40, macrosomia definition has been corrected

| Macrosomia | BW >4000 g (8 <i>lb</i> , 13 <i>oz</i> \(\frac{1}{10}\)). |
|------------|-----------------------------------------------------------|
|------------|-----------------------------------------------------------|

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

, Lead Science Writer

## GlaxoSmithKline Biologicals Vaccines R & D Protocol Amendment 4 eTrack study number and Abbreviated Title 207636 (EPI-RSV-008 BOD) Amendment number: Amendment 4 Amendment date: 29-MAY-2020

PPD

#### Rationale/background for changes:

This amendment outlines measures that may be applicable during special circumstances (e.g., COVID-19 pandemic). The primary purpose of the amendment is to protect the subject's welfare, and as far as possible ensure the potential benefit to the subject and promote data integrity. Several additional modifications and clarifications have also been made.

Changes are outlined below.

Co-ordinating author:

- Globally:
  - Intervals between study visits/contacts/observations: the window for the first infant subject visit has been extended from 0-10 to 0-21 days to provide site personnel with additional time to obtain and document post-delivery/birth informed consent (where this is required).
  - References to Gestational Age Range at maternal Visits 2, 3 and 4 have been removed as their inclusion was only intended as a guide and was not intended to further restrict allowed intervals between study visits.
- Synopsis, Section 3.3, Tertiary Objectives, and Section 11.1.3, Tertiary Endpoints, have been updated to indicate that the incidence of LRTIs/ Severe LRTIs (using alternative case definitions) will also be evaluated.
- Synopsis and Section 11.1.3, Tertiary Endpoints, has been updated to clarify that
  further exploratory characterization of immune responses to RSV and/or other
  respiratory tract infections or infections of relevance to pregnant women and their
  newborns (based on maternal serum and cord blood) includes, for example, levels
  of RSV-B neutralizing antibodies.
- The List of Abbreviations has been updated to include a reference to COVID-19.
- Section 2.3, Overall Benefit: Risk Conclusion has been updated.
- Section 4, Figure 1: A note has been added to indicate that COVID-19 cases identified within the surveillance framework of the study will be captured to the eCRF.
- Section 5.4, Table 4, Alternative LRTI/Severe LRTI Case Definitions, has been added. All subsequent Table numbers therefore increase by one.
- Section 8.2.1, Study procedures during special circumstances, has been added.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- Section 8.3, Tables 5 and 6, List of study procedures for maternal subjects, and List of study procedures for neonates/infants, have been clarified to indicate that COVID-19 cases are considered clinically significant events and will be recorded as such in the eCRF.
- Sections 8.5.8, 8.6.2, 8.6.7 have been modified to reference the collection of COVID-19 case information.
- Section 8.6.5.2 has been modified to clarify that RTI surveillance in infants cannot begin before additional consent for the infant's participation (where required) has been supplied.
- Section 8.7, Reporting COVID-19 cases, has been added.
- Section 11.3 has been modified to introduce definitions for the Enrolled set, and to clarify definitions for the Exposed and Per Protocol sets for analysis.
- Sections 11.6, 11.7 and 11.8 have been modified for consistency with the changes in Section 11.3.
- Section 11.11.1, Statistical considerations for interim analysis, has been modified to indicate that an interim analysis for RSV LRTIs may be performed if deemed necessary.
- Section 14 has been updated to include a reference to the WHO Guidance for surveillance of COVID-19.
- Additional editorial clarifications have been made and typographic errors have been corrected.

Text that has been moved or added is presented in **bold italics** and deleted text in strikethrough in the following sections.

#### Contributing Authors:

- PPD , Expert *Epidemiology* Biostatistician, PPD PPD Lead Epidemiology Statistician *Biostatistician*
- •—PPD , Clinical Trial Supply manager
- PPD , Clinical Laboratory Sciences Study Manager, Business & Decision Life Sciences Contractor for GSK Biologicals
- PPD , Oversight Data Manager
- PPD Study Data Manager (Tata Consultancy Services for GSK Biologicals)

#### Synopsis and Section 3.3, Tertiary objectives:

• To determine the incidence of LRTIs/ Severe LRTIs (using alternative case definitions)

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### **Synopsis and Section 11.1.3, Tertiary endpoints:**

• Episodes of LRTIs/Severe LRTIs up to one year of age - using alternative case definitions

Any further exploratory characterization of immune responses to RSV and/or other respiratory tract infections or infections of relevance to pregnant women and their newborns (based on maternal serum and cord blood). (*For example, levels of RSV-B neutralizing antibodies*).

#### List of Abbreviations:

COVID-19 Corona Virus Disease 2019

#### Section 2.3, Overall Benefit: Risk Conclusion:

This is an epidemiologic study that describes the prevalence of pregnancy outcomes and maternal/neonatal events of interest. The study does not include the administration of any investigational vaccine. It is not expected that the participation of pregnant women and their babies in the study would create any further risk to study participants. The study includes the establishment of a surveillance system for lower respiratory tract infections (LRTI) which may facilitate detection of respiratory tract infections, including COVID-19 cases, that might be diagnosed in children enrolled in the study.

#### Section 4, Figure 1, Study Design:

References to GA in the original figure have been removed and a footnote specifically referencing COVID-19 has been added. The previous figure and the current figure are presented in full below.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### Previous:



NOTE: Covid-19 cases identified within the surveillance framework of the study in maternal and infant subjects will also be recorded.

Epoch 003

Child: V3-NB

Epoch 002

Mother: V1 through V6

Child: V1-NB through V2-NB

Epoch 001

Screening

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### Section 5.4, Table 4, Alternative LRTI / Severe LRTI Case Definitions:

| | RSV<br>confirmed | Documented physical examination (PE) findings indicating lower respiratory tract involvement (at least one symptom) | Objective measures of clinical severity (at least one symptom) |
|---|---|---|---|
| LRTI | Confirmed | Rhonchi <sup>1</sup> | Increased respiratory rate (bpm) |
| | RSV infection | Rales <sup>1</sup> | ≥ 60 for < 2 mo |
| | | Crackles | ≥ 50 for 2-6 mo |
| | | Wheeze | Нурохетіа: |
| | | | SpO2 <95% at ≤1800 meters |
| | | | SpO2 <92% at > 1800 meters |
| | | | New onset apnea |
| | | | Nasal flaring |
| | | | Retractions <sup>2</sup> |
| | | | Grunting |
| Severe<br>LRTI | Confirmed<br>RSV infection | Rhonchi <sup>1</sup> | Нурохетіа |
| | | Rales <sup>1</sup> | SpO2 <93% at ≤1800 meters |
| | | Crackles | SpO2 <90% at > 1800 meters |
| | | Wheeze | Acute hypoxic or ventilatory failure <sup>3</sup> |
| | | | Dehydration due to respiratory distress |
| | | | requiring IV hydration⁴ |
| | | | Failure to respond or unconscious |

<sup>&</sup>lt;sup>1</sup>Term not listed in the eCRF page in this study.

#### Section 6.1, Number of subjects / centers:

The study will be conducted at multiple eentres centers.....

#### Section 6.2.2, Inclusion criteria for enrollment; infants:

• If local law requires it: Written or witnessed/thumb printed informed consent for study participation of the infant obtained from parent(s)/LAR(s) within 10 21 days of birth.

#### Section 8.2.1, Study procedures during special circumstances:

During special circumstances (e.g., the COVID-19 pandemic), the specific guidance from local public health and other competent authorities regarding the protection of individuals' welfare must be applied.

For the duration of such special circumstances, the following measures may be implemented for enrolled subjects if deemed feasible by the investigator.

<sup>&</sup>lt;sup>2</sup> Intercostal recession or chest wall indrawing are considered synonymous with and will be used as alternatives to the term "retractions," which is not listed in the eCRF page for this study.

<sup>&</sup>lt;sup>3</sup> Acute hypoxic or ventilatory failure is not listed in the eCRF page for this study. Instead, the presence of either respiratory support excluding mechanical ventilation OR requirement for mechanical ventilation or both will be used.

<sup>&</sup>lt;sup>4</sup> Dehydration due to respiratory distress requiring IV hydration is not listed in the eCRF page for this study. Skin turgor > 2 seconds or administration of IV fluid therapy will be used instead.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- If it is not possible to conduct a protocol-specified, scheduled or event-driven (e.g., LRTI assessment) visit as described in Section 8.3, the visit may be replaced with a contact conducted by telephone, videotelephony or telemedicine. SMS and email are not allowed.
- Biological samples may be collected at a different location\* other than the study site, or at-the subject's home. Biological samples should not be collected if they cannot be obtained within the visit interval (Section 8.4), processed in a timely manner or appropriately stored until the intended use.
- Nasal swabs should only be collected using centrally provided supplies.
- Cord Blood for assessment of immune response may be collected locally but must be retrieved, processed and stored in accordance with the Investigator Laboratory Manual.
- Additional blood samples for assessment of immune response should only be collected using centrally provided supplies.
- Diary cards may be transmitted from and to the site by electronic mail, and / or conventional mail.

Impact on the per protocol sets for analysis will be determined on a case by case basis.

Any impact of the above mentioned measures on the study results will be described in the clinical study report.

\* It is the investigator's responsibility to identify an alternate location. The investigator should ensure that this alternate location meets ICH GCP requirements, such as adequate facilities to perform study procedures, appropriate training of the staff and documented delegation of responsibilities in this location. This alternate location should be covered by proper insurance for the conduct of study on participants by investigator and staff at a site other than the designated study site. Refer to EMA Guidance on the Management of Clinical Trials during the COVID-19 (Coronavirus) pandemic (version 2, 27 March, 2020) for more details.

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

## Section 8.3, Outline of Study Procedures, Table 5, list of study procedures for maternal subjects:

| Gestational age | 24<br>0/7<br>-<br>27<br>6/7 | 24<br>0/7 _<br>27<br>6/7 | 28- <sup>9/7</sup><br>-<br>31- <sup>6/7</sup> | 32- <sup>9/7</sup><br>-<br>35- <sup>6/7</sup> | 36- <sup>97</sup><br><del>delivery</del> | | | |
|---|---|---|---|---|---|---|---|---|
| Timepoints | | Day<br>1 | Day<br>28 | Day<br>56 | Day 84 | At<br>Delivery | Post-<br>Delivery<br>Day 42 | |
| Record pregnancy-<br>related events of<br>interest. Record other<br>clinically significant<br>events or diagnoses <sup>15</sup> | | • | • | • | • | • | • | • |

<sup>&</sup>lt;sup>1</sup> Refer to Section 6.2.1. fifth sixth bullet.

## Section 8.3, Outline of study procedures, Table 6, list of study procedures for neonates/Infants:

| Age | 0- <del>10</del> <i>21</i> days | 42<br>Days | 6<br>Months | 12<br>months | _ | 12<br>nths |
|---|---|---|---|---|---|---|
| Timepoints | Birth | Day<br>42 | М6 | Y1 | | |
| Record all hospitalizations and clinically significant events h | • | • | • | • | • | • |
| Investigator<br>sign-off on<br>eCRF before<br>analysis | | • | | • | | |

LAR = legally acceptable representative; LRTI = lower respiratory tract illness; NB = newborn; RTI = respiratory tract illness; SAE = serious adverse event; *M=month*; Y = year.

#### Section 8.4, Intervals between study visits, Table 7:

| Interval | Optimal interval | Allowed interval** |
|--------------------|------------------|----------------------------------|
| Birth → Visit 1-NB | 0 davs | 0 – <del>10</del> <b>21</b> davs |

<sup>&</sup>lt;sup>10</sup> In the Philippines Where HIV testing is not part of the standard of care for pregnant women, the screening HIV test can be performed locally as a study procedure. Refer to SPM for further details. If results are positive, subject will be referred per local standard of care.

<sup>&</sup>lt;sup>15</sup>Includes events or diagnoses that could impact the pregnancy including COVID-19 cases

<sup>&</sup>lt;sup>9</sup>When approximately 50% of infants have completed up to Visit 3-NB, an interim analysis will *may* be conducted to assess the accumulated RSV LRTI cases and the distribution of maternal and cord blood serum RSV A Ab.

<sup>&</sup>lt;sup>h</sup> Includes COVID-19 cases

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### Section 8.5.8, Outcomes and Events of Interest in maternal subjects:

- Any events of interest in mother or fetus detected by surveillance will be referred to and managed by the routine health services as locally appropriate.
- Record all hospitalizations and/or clinically significant events, *including COVID-19* cases.

#### **Section 8.6, Description of study procedures for Neonates / Infants:**

Note that the investigator or study staff will perform (if not performed by local healthcare provider) a minimum of 2 clinical examinations: one at birth (or up to 10 21 days after birth), and another at approximately 42 days of age.

#### **Section 8.6.2, History and Examinations for Neonates / Infants:**

Record all hospitalizations and/or clinically significant events, *including COVID-19* cases.

## Section 8.6.5.2, Surveillance for potential Lower Respiratory Tract Illness (LRTI); Overview:

Surveillance for potential LRTIs begins at birth (or after additional consent, has been provided for the infant's participation in the study, if required,) and ends with the Year 1 study visit.

#### Section 8.6.7.1, Visit to assess a potential LRTI; Overview:

The appropriately qualified person will also evaluate whether the LRTI might be related to COVID19. The appropriately qualified person must follow the local standard of care regarding the reporting, and management of COVID-19 cases (suspected, probable or confirmed COVID-10 case), and complete both the COVID-19 form and LRTI form in the CRF. Refer to Section 8.7.

#### Section 8.6.7.2, Visit to assess a potential LRTI; Clinical Evaluation:

• Possible presence of COVID-19 infection (Section 8.7). As noted above, both the LRTI and COVID-19 eCRFs are to be completed (whether or not the investigator/study staff consider the LRTI to be due to COVID-19.

#### Section 8.7, Reporting Covid-19 Cases – Maternal and Infant subjects:

In addition to satisfying local reporting requirements for COVID-19 cases, maternal and infant COVID-19 cases identified within the existing framework of the study will be captured and reported on the COVID-19 eCRF for the study.

COVID-19 cases should be reported in the eCRF according to the WHO Case Definition [WHO, 2020] using one of the following terms:

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

- Suspected COVID-19 infection
- Probable COVID-19 infection
- Confirmed COVID-19 infection

#### Section 8.11.3.1, Antibody determination, Table 9:

| System | Component | Method | Kit /<br>Manu-<br>facturer | Unit | Cut-off | Laboratory* |
|---|---|---|---|---|---|---|
| SERUM | Respiratory<br>Syncytial<br>Virus A Ab | NEUTRALISATION | In house | ED60<br>and/or<br>IU/ML | ED60: 18;<br>IU/ml: 56 | GSK Biologicals**<br>or GSK designated<br>lab*** |

Ab = antibody; ED60 = serum dilution inducing 60% inhibition in plaque forming units; *IU/mL: International Unit/milliliter* 

#### Section 9.7, Follow-up of SAEs related to study participation:

The investigator will follow-up subjects with SAEs related to study participation until the event has resolved, subsided, stabilised stabilised .....

#### Section 9.7.2, Follow-up after the subject is discharged from the study:

The investigator is obliged to assist. If a subject dies during participation in the study or during a recognised recognized.....

#### Section 11.1.3, Tertiary endpoints:

- Any further exploratory characterization of immune responses to RSV and/or other respiratory tract infections or infections of relevance to pregnant women and their newborns (based on maternal serum and cord blood) (*For example, levels of RSV-B neutralizing antibodies.*)
- Episode(s) of RSV-LRTI/severe LRTI based on alternative case definitions, from birth up to 1 year of age.

#### Section 11.3.1.1, Exposed Sets, Pregnant women (mothers):

The ES will include all pregnant women (mothers) *who signed a valid* informed consent *form*.

#### Section 11.3.1.2, Exposed Sets, Neonates/Infants:

Not applicable.

#### Section 11.3.2.1, Enrolled Sets, Pregnant women (mothers):

The enrolled set will include all pregnant women (mothers) with a valid informed consent who completed Visit 1.

255

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

#### Section 11.3.2.2, Enrolled Sets, Neonates/infants:

The ESE nrolled Set will include all study eligible neonates/infants with

- born to pregnant women in the enrolled set, and
- *Who have* a valid ICF signed by the mother/ parent(s) /LAR(s) (as appropriate per local regulations).

#### 11.3.3, Per Protocol Sets (PPS), Pregnant women (mothers):

• The maternal PPS will include all pregnant women (mothers) meeting in the enrolled set who meet.....

#### 11.3.3.2, Per Protocol Sets (PPS), Neonates/infants:

The infant PPS will include all enrolled neonates / infants meeting

- born to pregnant women in the PPS and
- *who* meet.....

Sections 11.6, Analysis of primary objectives and 11.7, Analysis of Secondary Objectives:

If there is a difference of 5% or more between the number of participants in the enrolled set and the PPS, primary objectives analyses on the enrolled set will also be performed.

#### Section 11.8, Analysis of tertiary objectives:

If there is a difference of 5% or more between the number of participants in the enrolled set and the PPS, primary objectives analyses on the enrolled set will also be performed.

- To determine the incidence of LRTIs/Severe LRTIs (using alternative case definitions)
- If deemed necessary, to further characterize the immune responses to RSV and other infections in maternal subjects and infants (based on maternal serum and cord blood).
  - For example, for levels of neutralizing antibodies such as but not limited to RSV-B:

#### Section 11.11.1, Statistical considerations for interim analysis:

If deemed necessary, an interim analysis will may be performed on RSV surveillance data as part of the secondary objective of determining incidence of RSV LRTI. This interim analysis will may be performed to obtain preliminary information on the performance of the case definitions used for RSV LRTI, severe LRTI, and very severe LRTI (Table 3) and to assess levels of RSVA neutralising antibody in maternal and cord blood at delivery. The interim analysis willmay occur after the database freeze at the time

207636 (EPI-RSV-008 BOD) Protocol Amendment 4 Final

point when approximately 50% of infants will have completed up to 6 months of follow up during the surveillance period following birth (up to Visit 3-NB). *If an interim analysis is performed*, data cleaning plans will be scheduled as needed to supply data for interim analyses in a timely manner. This interim analysis will may be performed on data that is as clean as possible. Preliminary results will be made available in a timely manner for use in the potential adjustment of the RSV LRTI case definitions to be used in pivotal clinical trials scheduled to begin shortly thereafter. The results pertaining to this analysis *(if performed)* will be purely descriptive, with no adjustment of type I error, and will be reported in an interim statistical report. No CSR will be prepared.

#### **Section 14, References:**

World Health Organization [WHO]. Global Surveillance for COVID-19 caused by human infection with COVID-19 virus: Interim Guidance. March 2020. Available at: https://apps.who.int/iris/rest/bitstreams/1272502/retrieve. Accessed 8 May 2020.